Clinical Study Report Appendix 16.1.9

Drug Substance MEDI7352

Study Code D5680C00002

# Appendix 16.1.9 Documentation of Statistical Methods and Supporting Statistical Analysis

| Document Name | Edition/Version No. | Edition/Version Date |
|---|---|---|
| NRS Pain/PK/ADA/Total NGF Analysis Plan<br>(Interim Analyses) | 1.0 | 10 February 2023 |
| Statistical Analysis Plan | 1.0 | 12 July 2023 |
| Statistical Analysis Plan | 1.1 | 31 August 2023 |
| Table, Listing, and Figure Shells | 1.0 | 12 July 2023 |
| Table, Listing, and Figure Shells | 1.1 | 31 August 2023 |
| Table, Listing, and Figure Shells | 1.2 | 04 October 2023 |

#### NRS pain/PK/ADA/Total NGF Analysis Plan

Drug Substance MEDI7352

Study Code D5680C00002

Edition Number 1.0

Date 10/February/2023

# NRS pain/PK/ADA/Total NGF Analysis Plan (Interim Analyses) Study D5680C00002

A Randomised, Double-Blind, Placebo-Controlled, Dose-Response Study of the Efficacy and Safety of MEDI7352 in Subjects with Painful Diabetic Neuropathy

#### **TABLE OF CONTENTS**

| TITLE P. | AGE | |
|---|---|---|
| TABLE ( | OF CONTENTS | 2 |
| INTERIN | M ANALYSIS SAP SIGNATURE PAGE | 4 |
| 1 | INTRODUCTION | 5 |
| 2 | EFFICACY OBJECTIVES | |
| 3 | PKCCI AND IMMUNOGENICITY OBJECTIVES | |
| 4 | PK <sup>CCI</sup> AND IMMUNOGENICITY ASSESSMENTS | |
| 5 | PROCESS & DATA FLOWPREMIER-SUPPLIED ANALYSES | |
| <ul><li>5.1</li><li>5.2</li></ul> | INTIQUAN-SUPPLIED ANALYSESINTIQUAN-SUPPLIED ANALYSES | |
| 6 | STATISTICAL METHODS | |
| 6.1<br>6.1.1 | NRS Pain Data Conventions for Statistical Analysis of ePRO Pain Diary Data | |
| 6.1.2 | Handling of Missing Diary Data | |
| 6.1.3 | Derivation of Endpoints | |
| 6.1.4 | Descriptive Statistics | 11 |
| 6.1.5 | Statistical Analysis | |
| 6.1.6 | Updated Statistical Power Calculation | 13 |
| 6.2 | PK | 13 |
| 6.3 | Total NGF | 14 |
| 6.4 | Anti-drug Antibody | 14 |
| 6.5 | Individual Subject Profiles | 14 |
| 6.6 | Other Data | 15 |
| 6.6.1 | Subject Disposition and eligibility for statistical analysis | |
| 6.6.2 | Demographic data | 15 |
| 7 | SOFTWARE DETAILS | 16 |
| 8 | STATISTICAL APPENDIX | 16 |
| 9 | REPORTING | 18 |
| 10 | OUTPUT SHELLS EXAMPLES | 21 |
| LIST O | OF TABLES | |
| | | 10 |
| Table 1 | Planned Tables | |
| Table 2 | Planned Figures | 19 |

#### LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation or special term | Description |
|---|---|
| ADA | Anti-drug antibody |
| ADaM | Analysis Data Model |
| AZ | AstraZeneca |
| BLQ | Below the limit of quantification |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence interval |
| CPQP | Clinical Pharmacology and Quantitative Pharmacology |
| CTX-II | C-terminal cross-linked telopeptide of type II collagen |
| CXCL13 | Chemokine C-X-C motif ligand 13 |
| IA | Interim analysis |
| IARC | Interim Analysis Review Committee |
| ID | Identification |
| IP | Investigational product |
| NONMEM | Non-linear mixed effect modelling |
| NGF | Nerve growth factor |
| MAD | Multiple-ascending dose |
| PDN | Painful Diabetic Neuropathy |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| CCI | |
| SAD | Single-ascending dose |
| SDTM | Study Data Tabulation Model |
| TNFα | Tumour necrosis factor alpha |
| VPC | Visual predictive check |

#### INTERIM ANALYSIS SAP SIGNATURE PAGE

This document has been reviewed and approved by the signatories listed below:

| | PPD |
|--------------------------------------------------|-------------|
| PPD | |
| Author and Statistical Consultant to AstraZeneca | |
| Neuroscience | |
| | Date<br>PPD |
| PPD | |
| PPD | |
| AstraZeneca Neuroscience | |
| | Date |
| | nnn - |
| PPD | PPD |
| PPD Clinical Pharmacology and | |
| Quantitative Pharmacology | |
| AstraZeneca | |
| | Date |
| | PPD |
| PPD | |
| Biostatistician (Blinded) | |
| Premier Research, Spain | |
| ⁄ <b>1</b> | |
| | Date |
| PPD | PPD |
| Biostatistician (Unblinded) | |
| Premier Research, UK | |
| | Date |

#### 1 INTRODUCTION

MEDI7352 is a new modality bispecific fusion protein targeting both nerve growth factor (NGF) and tumour necrosis factor alpha (TNF $\alpha$ ) that is being developed to treat chronic pain. Both the anti-NGF and anti-TNF $\alpha$  pathways are precedented. This data analysis plan document provides a high-level description of the dataflow that will be followed and the outputs to be generated for the NRS pain scores, PK, ADA and total NGF variables in support of the interim analysis(es) for the Phase 2 dose response study D5680C00002 conducted with MEDI7352 in subjects with painful diabetic neuropathy. Full details of the study design can be found in the Clinical Study Protocol version 7.0 (13<sup>th</sup> April 2022).

#### **Study Description Overview**

- Phase of development: Phase 2.
- Patient population: Participants with painful diabetic neuropathy.
- Study size: Approximately 272 eligible subjects will be randomly assigned to double-blind treatment with one of 4 dose levels of MEDI7352 (dependent upon stage of the study) or placebo to ensure that approximately 236 subjects are evaluable for the efficacy analysis of stages 2-4 combined.
- General design: This is a multicentre, multinational, randomised, double-blind, placebo-controlled, parallel-group study.
- Route of administration: intravenous.
- Doses investigated: CCI . Each subject will receive 6 doses, 1 dose every 2 weeks (Days 1, 14, 28, 42, 56, and 70), administered IV over a 60-minute period. Note: only CCI and CCI doses are included in the Interim Analysis (from stages 2 and 3).
- Development objectives: proof of efficacy.

#### 2 EFFICACY OBJECTIVES

The primary objective is to assess the efficacy of MEDI7352 versus placebo on chronic pain in subjects with PDN currently taking standard of care medication for their PDN pain. A secondary objective is to characterise the dose-response relationship of MEDI7352 on chronic pain in subjects with PDN. However, this interim analysis plan will not cover the latter objective.

# AND IMMUNOGENICITY OBJECTIVES The Pharmacokinetics, pharmacodynamic (total NGF) and immunogenicity of MEDI7352 are secondary objectives/endpoints in the study. CCI A description of these objectives/endpoints is provided below.

Secondary objectives:

To assess the PK, PD, and immunogenicity of MEDI7352 in subjects with PDN

Exploratory objectives:



# 4 PK AND IMMUNOGENICITY ASSESSMENTS

Blood samples for determination of serum MEDI7352 concentrations and serum total NGF concentrations are collected at the following time-points:

Day 1 (pre-treatment), Day 14, Day 28, Day 42, Day 56, Day 70 (pre-dose, end of infusion, and 8 h), Day 71, Day 77, Day 84 and Early termination (if relevant).

Blood samples for determination of presence of anti MEDI7352 antibodies (ADA) are collected at the following time-points:

Baseline, Day 14, Day 28, Day 56, Day 70, Day 84 and Week 18.

Note: on dosing days, blood samples are taken prior to IP administration.

#### 5 PROCESS & DATA FLOW

Prior to the interim database lock, it is expected that data within scope of the Interim Analysis will be cleaned and have no outstanding edit checks.

#### 5.1 PREMIER-SUPPLIED ANALYSES

Prior to the interim analysis, a dummy run will be performed on a blinded data transfer using dummy randomization codes. This blinded analysis step will also be used by the sponsor blinded statistician to perform the sponsor QC of the primary analysis. Premier will perform their own QC as per standard operating procedures. The unblinded interim analysis will be performed by the unblinded Premier statistician. Both the blinded Premier statistician and blinded Sponsor statistician will be prohibited from access to the unblinded interim analysis.

#### 5.2 INTIQUAN-SUPPLIED ANALYSES

Data Management and Biostatistics at PREMIER will generate datasets containing the PK, ADA (immunogenicity) and total NGF data with additional study variables (i.e. baseline weight; dosing time; treatment allocation; PK, ADA and total NGF sampling time), and a dataset containing the efficacy data (i.e. NRS scores) for the purpose of generating individual profile plots (generated by IntiQuan) in support of the main efficacy data analysis conducted by PREMIER Biostatistics. The data structure and transfer process from Premier to AZ will be detailed in a separate Data Transfer Guideline document, and control of blinding will be described in MEDI7352 Study D5680C00002 Interim Analysis Review Committee Charter.

#### 6 STATISTICAL METHODS

#### Handling of missing or unquantifiable data:

Except for specific NRS pain analyses (described in section 6.1) missing data will not be imputed. PK and Total NGF data below the limit of quantification will be handled using a left censoring approach (i.e. values BLQ are defined as >=0 and <BLQ). ADA titre reported as <30 (below the minimum required dilution) is a negative result for the presence of ADA and will be treated as missing in the calculation of ADA titre summary statistics.

#### Populations for analysis:

Details of the populations for analysis as described in the CSP are presented below:

- Modified intent-to-treat (mITT): all randomised subjects who receive at least 1 dose of double-blind study medication and have at least 1 post-baseline NRS assessment. If a subject is randomised incorrectly or is administered the incorrect IP, analyses of the mITT population will be based on the IWRS-assigned treatment. In addition, for the purposes of the efficacy interim analysis of weekly average NRS pain score, it is also required that subjects have an evaluable 'Average Week 12 Pain NRS (LOCF)'score, which is defined as having completed two doses of IP and recorded sufficient pain NRS data for at least 2 weeks to enable the week 2 average calculation as described in section 6.1.
- Safety set: The safety population will include all subjects who receive at least 1 dose of double-blind study medication.
- PK set: all subjects for whom a PK sample was obtained and analysed.

In addition, a "Completers" set will be analysed for efficacy, defined as the subset of the mITT population who have a week 12 average NRS score.

A further subset of the mITT population "Week 6 LOCF" may be used to for efficacy analyses if the number of subjects with week 6 to week 11 NRS weekly averages (but no week 12 weekly average) is at least 20% the size of those with complete week 12 NRS averages.

For the purposes of the IA 'all PK and PD data available by the data cut-off date for the IA' will be included in the population PK and population PKPD analyses.

For the Safety set data presentations, The following clarifies how to handle the situation where a participant receives a treatment other than that to which the participant was randomised:

- If a participant randomised to placebo receives at least one dose of MEDI7352 XX µg/kg during the entire double-blind treatment period then the actual treatment arm = MEDI7352 XX, where XX corresponds to the lowest dose of MEDI7352 that the participant received during the double-blind treatment period.
- If a participant took only MEDI7352 XX μg/kg treatment during the entire double-blind treatment period, then the actual treatment arm = MEDI7352 XX, where XX corresponds to the dose of MEDI7352 that the participant took during the entire double-blind treatment period, regardless of what treatment the participant was randomized to.
- If a participant took a mix of MEDI7352 XX μg/kg treatments during the entire double-blind treatment period, then the actual treatment arm = MEDI7352 XX, where XX corresponds to the lowest dose of MEDI7352 that the participant received during the double-blind treatment period, regardless of what treatment the participant was randomized to.

#### 6.1 NRS Pain

For all outputs the placebo group will include subjects pooled across stages 2 and 3.

#### 6.1.1 Data Conventions for Statistical Analysis of ePRO Pain Diary Data

- 'Baseline' period: is defined as the seven day period prior to randomization i.e. Day -7 to Day -1, inclusive. A subject is considered to have a valid Baseline Pain score at study entry if there are at least 5 days of recorded diary pain scores in the 7 day period. This is consistent with the protocol inclusion criterion 9. However, for the purposes of inclusion in the statistical analysis of ePRO Pain Diary data, a subject is considered to have an evaluable baseline if they have at least 4 days out of 7 have recorded diary pain scores.
- 'Week 12' period: is defined for each subject as the seven day period ending within the protocol stipulated window (day 84 ± 3), where at least 4 days out of 7 have recorded diary pain scores. Where several such windows exist the one ending closest to day 84 will be selected. If there are two such windows that are equidistant from day 84 then the one with the largest number of diary entries will take precedence. If they have the same number of entries then the later of the two end dates will be chosen. If no such window exists then week 12 will be considered missing for the purposes of weekly average scoring. For example:

| Day | 77 | 78 | 79 | 80 | 81 | 82 | 83 | 84 | 85 | Number non missing |
|---|---|---|---|---|---|---|---|---|---|---|
| 7-day Window 85 | Y | N | Y | Y | N | N | Y | Ν | Y | 4 |
| 7-day Window 84 | Y | N | Y | Y | N | N | Y | N | Y | 3 (So technically Missing) |
| 7-day Window 83 | Y | N | Y | Y | N | N | Y | N | Y | 4 |

In the example above, the 7 day window ending at day 84 has only 3 days of entries, so cannot be used as week 12 average. However Day 83 and day 85 have exactly 4 entries in their 7 day windows. These are equidistant from the ideal day 84, so the algorithm chooses day 85 to take the average i.e. the later of the two.

The same approach as for week 12 will be taken for weeks 2,4,6,8 and 10, but using the corresponding nominal study days and the  $\pm 3$  days visit windows as described in the protocol, as follows:

- 'Week 2' period: is defined for each subject as the seven day period ending within the protocol stipulated window (day 14 ± 3), where at least 4 days out of 7 have recorded diary pain scores.
- 'Week 4' period: is defined for each subject as the seven day period ending within the protocol stipulated window (day 28 ± 3), where at least 4 days out of 7 have recorded diary pain scores.
- 'Week 6' period: is defined for each subject as the seven day period ending within the protocol stipulated window (day 42 ± 3), where at least 4 days out of 7 have recorded diary pain scores.
- 'Week 8' period: is defined for each subject as the seven day period ending within the protocol stipulated window (day  $56 \pm 3$ ), where at least 4 days out of 7 have recorded diary pain scores.
- 'Week 10' period: is defined for each subject as the seven day period ending within the protocol stipulated window (day 70 ± 3), where at least 4 days out of 7 have recorded diary pain scores.

#### 6.1.2 Handling of Missing Diary Data

- '<u>Missing Baseline</u>': Subjects with missing baseline data (i.e. zero or 1-3 days of diary pain scores will not be included in the Interim Analysis because the primary analysis is change-from-baseline.
- 'Missing Week 12': If a subject has zero or ≤ 3 days of diary pain data in each of the possible seven day periods ending within the protocol definition of week 12 (day 84 + 3), then an imputed 'week 12 LOCF' will be calculated from the latest

7 'non-missing' entries of the subject's diary closest to their nominal week 12 visit (i.e. the latest 7 day period containing at least 4 NRS values), provided that this would qualify as at least 'week 2' according to the windowing definition above. Otherwise, the week 12 LOCF weekly average NRS pain score will be set to missing.

#### **6.1.3** Derivation of Endpoints

- 'Average Baseline Pain NRS': is defined as the arithmetic average of the 'non-missing' daily pain scores within the baseline period defined above. For example, if a subject has 4 days of non-missing pain scores their average will be calculated over 4 days, not the full 7 day baseline period.
- 'Average Week 12 Pain NRS': is defined as the arithmetic average of the 'non-missing' daily pain scores within each subject's specific week 12 period defined above.
- 'Average Week 12 Pain NRS (LOCF)': is defined as the arithmetic average of the 'non-missing' daily pain scores within each subject's specific week 12 period or according to the imputed 'week 12 LOCF' approach described above.
- 'Change from Baseline to Week 12 Pain NRS': is defined for each subject as 'Average Week 12 Pain NRS' minus 'Average Baseline Pain NRS'.
- 'Change from Baseline to Week 12 Pain NRS (LOCF)': is defined for each subject as 'Average Week 12 Pain NRS (LOCF)' minus 'Average Baseline Pain NRS'.

#### **6.1.4** Descriptive Statistics

Tables of arithmetic mean, standard deviation, minimum, maximum, median, 1st and 3rd quartiles and N, will be provided by treatment group and total, for the following NRS endpoints:

- Baseline weekly average pain NRS
- Weekly average pain NRS for weeks 2, 4, 6, 8, 10 and 12
- Change from Baseline Pain NRS to weeks 2, 4, 6, 8, 10 and 12
- Week 12 LOCF: Weekly average pain NRS and Change from Baseline

In addition, the following plots will be produced:

 Mountain plots (also known as folded empirical distribution plots) and boxplots, by treatment group, of Weekly Average and 'Change from Baseline to Week 12 Pain NRS (LOCF)' will be presented.

- Line plots of the observed Weekly Average and Change from baseline in mean Daily NRS scores for each treatment group from baseline through to the day 87 (the upper limit of the week 12 visit window), with Week 12 LOCF as an additional plotting point.
- Spaghetti/Connected line time plot of individual subjects for observed Weekly Average (these will be presented as individual profiles as in section 6.5) and Change from Baseline to week 12.

#### 6.1.5 Statistical Analysis

#### ANCOVA of 'Change from Baseline to Week 12 Pain NRS (LOCF)':

The linear model will be an analysis of covariance (ANCOVA) with dependent variable 'Change from Baseline to Week 12 Pain NRS (LOCF)', and independent variables will be dose group (as a factor, with placebo group as the reference level), and 'Baseline weekly average pain NRS' as the continuous covariate. The random error is assumed to be normally and independently distributed with constant variance. The following outputs from the fitted model will be tabulated:

- Parameter estimates of the difference between each dose group and placebo, t-value, degrees of freedom, standard error, conventional 95% 2-sided and also 'Lalonde-type' asymmetric confidence intervals (i.e. lower limit of 1-sided 90% CI and upper limit of 1-sided 80% CI), and model residual standard deviation (RMSE).
- Least squares means estimates of change from baseline to week 12 for column and Placebo groups, with 95% 2-sided confidence intervals. The least squares mean is a model estimate using fitted group parameter and the baseline weekly average pain NRS parameter evaluated at the grand mean over both groups.
- As a sensitivity analysis, an estimate of the treatment effect at week 12, together with 95 % 2-sided confidence intervals and also 'Lalonde-type' asymmetric confidence intervals (i.e. lower limit of 1-sided 90% CI and upper limit of 1-sided 80% CI), will also be obtained from a "Mixed Effects Repeated Measures model", which assumes a Multivariate Normal distribution across visits within patient, with a fully parameterized unstructured covariance matrix and contains treatment, baseline NRS, visit and treatment-by-visit interaction as fixed effects, using all available data (but not LOCF). If there are convergence issues then a simpler covariance structure, such as AR1 will be implemented.
- Bayesian posterior probabilities that the 'Reduction' in Week 12 Pain NRS (LOCF) of versus Placebo is (a) Greater than zero i.e. the probability of a non-zero treatment effect. (b) Greater than the target 1.25-point reduction treatment effect. Superimpose the above values on a plot of Bayesian posterior probability versus reduction on a grid ranging from zero to 2. The Bayesian

linear model will be fitted using the bfitmod function within the R Dosefinding package. Further details are included in the appendix.

#### **6.1.6** Updated Statistical Power Calculation

The original power calculation will be re-visited using knowledge about the observed residual standard deviation (RMSE) from the column and columns placebo ANCOVA analysis, and the observed effects of column versus placebo. The eMax dose response curve used for any power simulations of stage 4 data will be based upon the ED50 required to fit the observed effect of column at the IA and two scenarios of the columns assumed effect size: 1) the Protocol assumed effect size of 1.25 versus placebo, and 2) the observed effect of column versus placebo at the IA. If the estimated ED50 is negative, then linear interpolation will be used instead of an Emax approach.

Revised power calculation will be performed as follows:

<u>Conditional Power of Test of Dose Response Curve under original stage 4</u> sample size and dose allocation

The conditional power of the pre-planned final test of the dose response curve will be simulated under the above two assumptions regarding the true maximum treatment effect for octaon for data accruing after the interim analysis with sample sizes per group as per protocol and using the observed data in stage 2 and 3 combined. Further details are given in the programming appendix.

The above analyses will be performed by Premier.

#### 6.2 PK

Pharmacokinetic data from this phase 2 study conducted in subjects with PDN will be appended to the existing PK data from other MEDI7352 studies conducted in subjects with painful osteoarthritis of the knee. Data will subsequently be analysed by population methods using nonlinear mixed-effects modelling. The existing 1-compartment population PK model with time-dependent clearance reflecting ADA-mediated elimination of the drug developed based on the SAD/MAD and phase 2B OA study data will be used as a starting point and updated as required based on the emerging new data. The analysis will be carried out using appropriate software (e.g., NONMEM, MONOLIX). The impact of prospectively selected covariates (i.e. weight), if available, on MEDI7352 exposure (e.g. clearance, volumes) will be evaluated. Population PK parameter estimates (e.g., clearance, volume, rate of absorption and bioavailability) with 95% CI from the final model will be tabulated. The uncertainty in the parameter estimates in the final model will be assessed (e.g. from the standard error estimates provided by NONMEM or from the 95% CI estimates provided by other appropriate analysis conducted using other software). Finally, the final model performance will be investigated

using a set of goodness of fit plots as well as Visual Predictive Check (VPC) method. Other evaluation methods may be used (e.g., bootstrapping) if deemed appropriate.

The above analyses will be performed by IntiQuan. Premier will supply the Serum MEDI7352 concentration dataset and ancillary variables as described in the Data Transfer Guidelines document.

#### 6.3 Total NGF

Total NGF data collected in this phase 2 study conducted in subjects with PDN will be appended to the existing total NGF data from other MEDI7352 studies and will subsequently be analysed by population methods using nonlinear mixed-effects modelling.

The existing semi-mechanistic drug-target binding population PKPD model developed based on the SAD/MAD and phase 2B OA study data will be used as a starting point and updated as required based on the emerging new data. The analysis will be carried out using appropriate software (e.g., NONMEM, MONOLIX). The impact of potential covariates (if available) on the PD parameters (e.g. maximum effect) will be evaluated, if deemed appropriate. The population PD parameter estimates with 95% CI from the final model will be tabulated. The uncertainty in the parameter estimates in the final model will be assessed (e.g. from the standard error estimates provided by NONMEM or from the 95% CI estimates provided by other appropriate analysis conducted using other software). Finally, the final model performance will be investigated using a set of goodness of fit plots as well as Visual Predictive Check (VPC) method. Other evaluation methods may be used (e.g., bootstrapping) if deemed appropriate.

The above analyses will be performed by IntiQuan.

### 6.4 Anti-drug Antibody

Anti-Drug Antibody response during the entire study period and at each study assessment will be summarised according to prevalence, incidence and titre value for the Safety Set.

The above analyses will be performed by Premier.

#### 6.5 Individual Subject Profiles

Individual subject trellis-type plots presenting observed PK (concentration), ADA titre, total NGF concentration and predicted free NGF concentration profiles over time as well as individual observed daily and weekly averaged NRS score (six plots on 1 page per subject) will be generated by IntiQuan in support of the interpretation of the main efficacy data analysis conducted by PREMIER.

The time axis of each sub-plot will be in weeks. The Y-axis of each of the 6 sub-plots will be as follows:

- a) Serum MEDI7352 Concentration (ng/mL) on log10 scale, with a separate plot symbol for BLOQ values.
- b) ADA Titre on log scale, with a red symbol for ADA positive values and green symbol for ADA negative values
- c) Serum free NGF % change from baseline (predicted) on linear scale
- d) Serum total NGF concentration on log10 scale
- e) NRS Daily score, values connected by lines. Reference lines for baseline average daily score and minimum daily score post-baseline.
- f) Average weekly NRS score, values connected by lines. Weekly value taken from efficacy analysis approach. Reference lines for baseline average Weekly score and minimum Weekly score post-baseline.

#### 6.6 Other Data

#### 6.6.1 Subject Disposition and eligibility for statistical analysis

A table will be produced to show for stage 2 and 3 of the study the number of subjects:

- Screened
- Enrolled

For Total and by dose group the number of subjects:

- Randomized
- Included in the mITT population
  - Evaluable Week 12 efficacy
  - Evaluable LOCF efficacy
- Not efficacy evaluable
- Completed study
- Reasons for withdrawal

#### 6.6.2 Demographic data

A table of arithmetic mean, standard deviation, minimum, maximum, median, 1st and 3rd quartiles and N (observed and missing), will be provided by treatment

group and total, for age. And frequency tables by treatment group and total for gender and race.

The above analyses will be performed by Premier.

#### 7 SOFTWARE DETAILS

Efficacy: SAS version 9.4 and R version 4.2.1 will be used to create the D5680C00002 interim analysis outputs, as appropriate.

Monolix version 2019R1 (Lixoft) will be used for conducting the cross-study population analyses and R version 3.6.3 (R-project, www.r-project.org) will be used for generation of the associated outputs.

#### 8 STATISTICAL APPENDIX

- A1. <u>Bayesian linear model to calculate posterior probabilities of the maximum treatment effect (CCI versus Placebo data)</u> using **bFitMod** function within **DoseFinding** package
  - Calculate the Least Squares Means for each dose group and their variancecovariance matrix (using package 'emmeans')
  - Create indicator variable for dose: 0=Placebo and 1=CC
  - Execute **bFitMod** with:
    - a. model as "linear"
    - b. Independent Gaussian Priors for intercept and slope parameters: N(0,100). With starting values of 0.
    - c. Lsmean Estimates and Variance-Covariance for placebo and column as inputs from the ANCOVA described in section 6.1.5, and
    - d. simulate 100,000 draws from the posterior distribution, with seed = 301020 (to allow for independent replication).
    - e. Process the saved **bFitMod** object as follows:
      - Select the 'samples' element from the saved bFitMod object
      - The 'delta' variable within the 'samples' element is the posterior value of the treatment difference between CCI and placebo
  - Estimate the posterior probabilities that the treatment effect is
    - a. Greater than zero

b. Greater than a 1.25-point reduction from the posterior sample of the slope parameter.

by computing the proportion of posterior 'delta' values less than zero and -1.25, respectively.

# A2. Simulation of Conditional Power of the Dose Response Curve test under original stage 4 sample size and dose allocation

- There is no formula available to compute conditional power of the dose response test, therefore a simulation approach will be taken as follows:
- Calculate the residual standard deviation (RMSE) from the ANCOVA model fitted to the interim data.
- Simulate the stage 4 data for each of the four dose groups from an emax model with an appropriate ED50 and random error = residual standard deviation.

The parameters for the emax model, from which to simulate from, will be calculated (fixed) as follows:

```
ED50 = 450*(Y_{IA}-Y_{450})/(Y_{450}-450*Y_{IA}/150) and 
emax = Y_{450}*(ED_{50}+450)/450
```

where  $Y_{IA}$ = observed effect of CCI versus placebo,  $Y_{450}$  = one of the two scenarios of the CCI effect versus placebo.

If the estimated ED50 is negative then the data are not consistent with an Emax model therefore linear interpolation between zero and CCI will be used instead of an Emax approach for estimating the effect of the CCI dose in stage 4 as follows: Lsmean for CCI versus placebo = (CCI )\*Lsmean CCI versus placebo .

The 'intercept'  $(E_0)$  of the Emax model is set to the 'intercept plus the regression term for baseline value evaluated at the average of the baseline values' from the ANCOVA model of the interim analysis. The maximum effect over placebo at the highest dose studied in stage 4 (currently planned to be CCI is set at values as specified in section 6.1.6.

The algorithm for simulating Change-from-baseline and baseline values for each subject is as follows:

- Simulate 10,000 stage 4 datasets. Each simulation consists of:
  - For each dose group, select a sample of baseline values of size as per protocol with replacement from the combined distribution of baseline values in the interim dataset.
  - For each dose group, simulate a change-from-baseline value for each subject from the simulation model conditional upon the subject's baseline value

- Combine stage 2 and 3 observed data and stage 4 simulated data and analyze using the **MCTtest** function of the **R Dosefinding** package, with the candidate models as specified in the protocol and options type="normal", alternative="one.sided", alpha=0.025 and addCovars = baseline.
- Output the minimum adjusted p-value of the multiplicity adjusted test
- Calculate conditional Power of the dose response test as 100\*(number of minimum p-values < 0.025 / number of simulations)</li>
- Repeat for each column effect scenario. If the estimated ED50 is negative then linear interpolation will be used instead of an Emax approach scenario.

#### 9 REPORTING

In support of the interim analysis which have for primary focus efficacy, Tables and Figures will be created. In addition, results from the PK, ADA and total NGF data analysis may also be summarised in a PowerPoint presentation created by AZ CPQP/IntiQuan.

Tables and figures listed in Table 1 and Table 2, respectively, will be generated, as data permits.

Table 1 Planned Tables

| Number | Description | Producer |
|---|---|---|
| Table 1.1.1 | Demography | PREMIER |
| Table 1.1.2 | Subject Disposition | PREMIER |
| Table 1.2.1 | Descriptive Statistics of Weekly Average Pain NRS from Baseline and all visits to Week 12: Observed Values and Week 12 LOCF: mITT Population | PREMIER |
| Table 1.2.2 | Descriptive Statistics of Weekly Average Pain NRS from Baseline and all visits to Week 12: Observed Values: mITT Population with week 12 NRS Weekly Averages | PREMIER |
| Table 1.2.3 | Statistical Analysis of Change from Baseline to Week 12 Pain NRS (LOCF): ANCOVA: mITT Population | PREMIER |
| Table 1.2.4 | Statistical Analysis of Change from Baseline to Week 12 Pain NRS:<br>ANCOVA: mITT Population with week 12 NRS Weekly Averages | PREMIER |
| Table 1.2.5 | Statistical Analysis of Change from Baseline to Week 12 Pain NRS: MMRM: mITT Population | PREMIER |
| Table A1.1 | Population PK parameter estimates with 95% CI from the final PK model | IntiQuan |
| Table A1.2 | Population PD parameter estimates with 95% CI from the final PKPD model | IntiQuan |
| Table A1.3 | Summary of Anti-Drug Antibody responses during the study | PREMIER |

Table 1Planned Tables

| Number | Description | Producer |
|---|---|---|
| Table A1.4 | Anti-Drug Antibody results and titre summary by timepoint | PREMIER |
| Table A1.5 | Predicted average % change from baseline in serum free NGF concentration following intravenous administration of MEDI7352 and tanezumab 2.5 and 5 mg SC | IntiQuan |

#### Table 2Planned Figures

| Number | Description | |
|---|---|---|
| Figure 1.1 | Mountain plot of Weekly Average to Week 12 Pain NRS (LOCF) by treatment group | PREMIER |
| Figure 1.2 | Mountain plot of Change from Baseline to Week 12 Pain NRS (LOCF) by treatment group | PREMIER |
| Figure 1.3 | Boxplot of Weekly Average to Week 12 Pain NRS (LOCF) by treatment group | PREMIER |
| Figure 1.4 | Boxplot of 'Change from Baseline to Week 12 Pain NRS (LOCF) | PREMIER |
| Figure 1.5 | Mean Weekly Average Pain NRS from Baseline to Week 12 (including Week 12 LOCF) | PREMIER |
| Figure 1.6 | Mean Change from Baseline Pain NRS from Week 1 to Week 12 (including Week 12 LOCF) | PREMIER |
| Figure 1.7 | Individual Spaghetti plot of Mean Weekly Average Pain NRS from Baseline to Week 12 | PREMIER |
| Figure 1.8 | Individual Spaghetti plot Change from Baseline Pain NRS from Week 1 to Week 12 | PREMIER |
| Figure 1.9 | Bayesian Predicted Probabilities of Effect Size versus Placebo | PREMIER |
| Figure 1.10 | Conditional Power of MCP-MOD test | PREMIER |
| Figure A1.1 | Model goodness of fit plots (population PK analysis) | IntiQuan |
| Figure A1.2 | Visual predictive check (population PK analysis) | IntiQuan |
| Figure A1.3 | Observed/predicted serum MEDI7352 concentration-time profiles (by participant) (population PK analysis) | IntiQuan |
| Figure A1.4 | Observed serum MEDI7352 concentration-time profiles by ADA status (by treatment) | IntiQuan |
| Figure A1.5 | Population mean (95% CI) serum MEDI7352 concentration-time profiles by treatment | IntiQuan |
| Figure A1.6 | Population mean (95% CI) serum MEDI7352 concentration-time profiles by ADA status and by treatment | IntiQuan |
| Figure A1.7 | Model goodness of fit plots (population PKPD analysis) | IntiQuan |
| Figure A1.8 | Visual predictive check (population PKPD analysis) | IntiQuan |

Table 2Planned Figures

| Number | Description | |
|---|---|---|
| Figure A1.9 | Observed/predicted serum total NGF concentration-time profiles (by participant) (population PKPD analysis) | IntiQuan |
| Figure A1.10 | Predicted serum free NGF concentration-time profiles (by participant) (population PKPD analysis) | IntiQuan |
| Figure<br>A1.11 | Observed serum total NGF concentration-time profiles by ADA status (by treatment) | IntiQuan |
| Figure A1.12 | Predicted serum free NGF concentration-time profiles by ADA status (by treatment) | IntiQuan |
| Figure A1.13 | Predicted median % change from baseline serum free NGF concentration-time profiles by treatment | IntiQuan |
| Figure<br>A1.14 | Predicted median % change from baseline serum free NGF concentration-time profiles by ADA status and by treatment | IntiQuan |
| Figure A1.15 | Predicted median % change from baseline serum free NGF concentration-time profiles following intravenous administration of MEDI7352 and tanezumab 2.5 and 5 mg SC | IntiQuan |
| Figure<br>A1.16 | Individual observed serum MEDI7352 concentration, ADA titre and serum total NGF concentration profiles over time, observed daily as well as weekly averaged NRS pain scores as well as predicted serum free NGF concentration -time profiles (6 plots per participant) | IntiQuan |

#### 10 OUTPUT SHELLS EXAMPLES

The format of selected tables and figures created by Premier is described in separate documents

# Statistical Analysis Plan



| Sponsor | AstraZeneca |
|---|---|
| Protocol Title: | A Randomised, Double-Blind, Placebo-Controlled, Dose-<br>Response Study of the Efficacy and Safety of MEDI7352 in<br>Subjects with Painful Diabetic Neuropathy |
| Development Phase | 2 |
| Protocol Number: | D5680C00002 |
| Premier Research PCN: | MEDU177093 |
| Document Version: | Final Version 1.0 |
| Document Date: | 12-Jul-2023 |



#### **Approvals**

| Role | Signatures |
|-----------------|-----------------------------------------------------|
| Piostotisticion | Print Name: PPD Biostatistician, Premier Research |
| Biostatistician | Sign Name: PPD |
| Peer Reviewer | Print Name: PPD PPD Biostatistics, Premier Research |
| Peer Reviewer | Sign Name: PPD |



| Role | Signatures | |
|-----------------|----------------------------------------------|------------|
| AstraZeneca | Print Name:PPD Statistical Consultant to As | straZeneca |
| Biostatistician | Sign Name: | PPD |
| AstraZeneca | Print Name: PPD PPD AstraZeneca Neuroscience | |
| Representative | Sign Name: | PPD |





## **Document History**

| Version | Date | Author | Description |
|---------|-------------|--------|---------------|
| 0.1 | 27-Mar-2019 | PPD | Draft Version |
| 0.2 | 16-Apr-2021 | PPD | Draft Version |
| 0.3 | 25-Jun-2021 | PPD | Draft Version |
| 0.4 | 24-Mar-2023 | PPD | Draft Version |
| 0.5 | 21-Apr-2023 | PPD | Draft Version |
| 0.6 | 24-May-2023 | PPD | Draft Version |
| 0.7 | 20-Jun-2023 | PPD | Draft Version |






#### **Table of Contents**

| Approvais | |
|-----------------------------------------------|-------------|
| Document History | 4 |
| Table of Contents | 5 |
| List of Tables | 7 |
| List of Figures | 7 |
| List of Abbreviations | 8 |
| 1. Overview | 12 |
| 2. Study Objectives and Endpoints | |
| 2.1. Study Objectives | 12 |
| 2.1.1. Primary Objective | 12 |
| 2.1.2. Secondary Objectives | 12 |
| 2.1.3. Exploratory Objectives | |
| 2.2. Study Endpoints | 13 |
| 2.2.1. Efficacy Endpoints | |
| 2.2.2. Safety Endpoints | 14 |
| 2.2.3. Pharmacokinetic/Pharmacodynamic Varia | ble(s)14 |
| 2.2.4. Other Endpoints | 15 |
| 3. Overall Study Design and Plan | 15 |
| 3.1. Overall Design | 15 |
| 3.2. Sample Size and Power | 15 |
| 3.3. Study Population | 16 |
| 3.4. Treatments Administered | 17 |
| 3.5. Method of Assigning Subjects to Treatmen | nt Groups17 |
| 3.6. Blinding and Unblinding | 17 |
| 3.7. Schedule of Events | |
| 4. Statistical Analysis and Reporting | 18 |
| 4.1. Introduction | 18 |
| 4.2. Interim Analysis and Data Monitoring | 19 |
| 5. Analysis Populations | 19 |
| 6. General Issues for Statistical Analysis | 20 |
| 6.1. Statistical Definitions and Algorithms | 20 |
| 6.1.1. Baseline | 20 |
| 6.1.2. Adjustments for Covariates | 20 |
| AD-ST-33.06 Effective date: 12-Nov-2020 | |




| | 6.1.3. | Multiple Comparisons | 20 |
|---|---|---|---|
| | | Handling of Dropouts or Missing Data | |
| | | Analysis Visit Windows | |
| | | Pooling of Sites | |
| | 6.1.7. | Efficacy Variables | 22 |
| | 6.1.8. | Derived Variables. | 23 |
| | 6.1.9. | Data Adjustments/Handling/Conventions | 25 |
| 7. | | dy Patients/Subjects and Demographics | |
| | 7.1. | Disposition of Patients/Subjects and Withdrawals | 26 |
| | 7.2. | Protocol Deviations | 27 |
| | 7.3. | Demographics and Other Baseline Characteristics | 27 |
| | 7.4. | Exposure | |
| 8. | Eff | icacy Analysis | 28 |
| | 8.1. | Primary Efficacy Analysis | 28 |
| | 8.1.1. | Sensitivity Analyses of the Primary Efficacy Endpoint | 30 |
| | 8.2. | Secondary Efficacy Analysis | 30 |
| | 8.3. | Exploratory Efficacy Analysis. | 31 |
| 9. | Sa | fety and Tolerability Analysis | 31 |
| | 9.1. | Adverse Events | 33 |
| | 9.1.1. | Adverse Events Leading to Discontinuation of IP | 33 |
| | 9.1.2. | Deaths and Serious Adverse Events. | 34 |
| | 9.1.3. | Drug-Induced Liver Injury | 34 |
| | 9.1.4. | Infection Risk | 34 |
| | 9.2. | COVID-19 Vaccination and Screening | 34 |
| | 9.3. | Clinical Laboratory Evaluations | 34 |
| | 9.4. | Vital Signs | 35 |
| | 9.5. | Electrocardiograms | 35 |
| | 9.6. | Physical and Neurological Examination | 36 |
| | 9.7. | Total Neuropathy Score-Nurse. | 36 |
| | 9.8. | Motor and Sensory Nerve Conduction Studies | 36 |
| | 9.9. | Strength and Deep Tendon Reflexes. | 36 |
| | 9.10. | Hypersensitivity/Anaphylactic Reactions, Injection Site or Infusion Reactions | 36 |
| | 9.11. | Prior and Concomitant Medication and Procedures | 37 |
| 10. | Ch | anges from Planned Analysis | 38 |
| 11. | Ot | ner Planned Analysis | 38 |
| AD. | -ST-33.0 | 6 Effective date: 12-Nov-2020 | |





| 11.1. Biomarkers. | 38 |
|-------------------------------------------------------------|----|
| 11.2. Immunogenicity | 39 |
| 11.3. Pharmacokinetic Analysis | 39 |
| 12. References | 40 |
| 13. Tables, Listings, and Figures | 41 |
| 13.1. Demographic Data | 41 |
| 13.2. Efficacy Data | 42 |
| 13.3. Safety Data | 43 |
| 13.4. Pharmacokinetic/Pharmacodynamic Data | 46 |
| 13.5. Planned Listing Descriptions | 46 |
| 13.6. Planned Figure Descriptions | 48 |
| 14. Tables, Listing and Figure Shells | 50 |
| 14.1. Standard Layout for all Tables, Listings, and Figures | 50 |
| 15. Appendix: Calculation of Dose to achieve target effects | 52 |
| List of Tables | |
| Table 1: Demographic Data Summary Tables and Figures | 41 |
| Table 2: Efficacy Data | 42 |
| Table 3: Safety Data | 43 |
| Table 4: Pharmacokinetic/Pharmacodynamic Data | 46 |
| Table 5: Planned Listings | 46 |
| Table 6: Planned Figures | 49 |
| List of Figures | |
| Figure 1: Standardized Layout | 51 |





## **List of Abbreviations**

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| ADA | Anti-Drug Antibody |
| AE | Adverse Event |
| AIC | Akaike Information Criterion |
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| BOCF | Baseline Observation Carried Forward |
| CI | Confidence Interval |
| СМН | Cochran-Mantel-Haenszel |
| COVID-19 | Coronavirus Disease 2019 |
| CSR | Clinical Study Report |
| DSIS | Daily Sleep Interference Scale |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| ED50, ED90 | The Dose to achieve 50%, 90% of the Maximum Effect. |
| EMA | European Medicines Agency |

AD-ST-33.06 Effective date: 12-Nov-2020





| Abbreviation | Definition |
|--------------|---------------------------------------------------------|
| Emax | The Model-Based Maximum Treatment Effect Versus Placebo |
| ePRO | Electronic Patient-Reported Outcome System |
| FDA | Food and Drug Administration |
| gCV% | Geometric Coefficient of Variation |
| GEE | Generalized Estimating Equation |
| gmean | Geometric Mean |
| gSD | Geometric Standard Deviation |
| HL | Hy's Law |
| HR | Heart Rate |
| ICH | International Council for Harmonization |
| IP | Investigational Product |
| IV | Intravenous |
| IWRS | Interactive Web Response System |
| LLOQ | Lower Limit of Quantification |
| LOCF | Last Observation Carried Forward |
| LS | Least Squares |
| MCP-mod | Multiple Comparison Procedure Modelling |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-Treat |





| Abbreviation | Definition |
|--------------|----------------------------------------|
| MMRM | Mixed Effects Models Repeated Measures |
| NC | Not Calculable |
| NCA | Noncompartmental Analysis |
| NPS | Neuropathic Pain Scale |
| NQ | Not Quantifiable |
| NRS | Numeric Rating Scale |
| PD | Pharmacodynamics |
| PDN | Painful Diabetic Neuropathy |
| PGIC | Patient Global Impression of Change |
| CCI | |
| PHT | Potential Hy's Law |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| QTcF | QT Fridericia's Correction |
| CCI | |
| RPOA | Rapidly Progressive Osteoarthritis |
| SAE | Serious Adverse Event |
| SAF | Safety |
| SAP | Statistical Analysis Plan |





| Abbreviation | Definition |
|--------------|------------------------------------------|
| SAS® | a Software System Used for Data Analysis |
| SDTM | Study Data Tabulation Model |
| SF-36 | 36-Item Short Form Health Survey |
| SiAP | Statistical Interim Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TBL | Total Bilirubin |
| TEAE | Treatment-Emergent Adverse Event |
| tNGF | Total Nerve Growth Factor |
| TNSn | Total Neuropathy Score-Nurse |
| ULN | Upper Limit of Normal |
| ULOQ | Upper Limit of Quantification |





#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for AstraZeneca protocol number D5680C00002 (A Randomised, Double-Blind, Placebo-Controlled, Dose-Response Study of the Efficacy and Safety of MEDI7352 in Subjects with Painful Diabetic Neuropathy), dated 13-Apr-2022 version 7.0. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials (ICH, 1998). All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association (ASA, 2018) and the Royal Statistical Society (RSS, 2014), for ethical statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts.

The statistical plan described hereafter has been developed by blinded study team members prior to the Interim Analysis but after the Administrative Analysis has been conducted. It will be approved before final unblind, performing inferential or descriptive analysis of hard-locked data from AstraZeneca's study D5680C00002.

#### 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

#### 2.1.1. Primary Objective

The primary objective is to assess the efficacy of MEDI7352 versus placebo on chronic pain in subjects with painful diabetic neuropathy (PDN) currently taking standard of care medication for their PDN pain.

#### 2.1.2. Secondary Objectives

The secondary objectives are:

- To assess the safety and tolerability of MEDI7352 in subjects with PDN
- To assess the pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of MEDI7352 in subjects with PDN





• To characterise the dose-response relationship of MEDI7352 on chronic pain in subjects with PDN

#### 2.1.3. Exploratory Objectives



#### 2.2. Study Endpoints

#### 2.2.1. Efficacy Endpoints

#### 2.2.1.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is the change in the weekly average of the average daily pain scores from the baseline week to Week 12 of MEDI7352 compared to placebo, as measured on an 11-point (0-10) numeric rating scale (NRS).

The target population is the entire patient population, i.e., the collection of all patients eligible to be included in the randomized clinical trial based on prespecified (and duly justified) inclusion/exclusion criteria.

The study was not designed using the Estimand framework. However, the following general aspects of an Estimand can be inferred: the Estimand can be generically defined as the true between-treatment difference in the target population endpoint means for the change from baseline for the Pain NRS at Week 12, while-on-treatment and regardless of prohibited or rescue medication use.

#### 2.2.1.2. Secondary Efficacy Endpoint(s)

The secondary efficacy endpoints of this study include the following:

- Change in the weekly average of the average daily pain score, as measured on an 11-point (0-10) NRS, from baseline to Weeks 2, 4, 6, 8, and 10 of treatment and the week before the follow-up visit.
- Percentage of subjects who have achieved ≥30% and ≥50% reductions in the weekly average of the average daily pain score from baseline during Weeks 4, 8, and 12 of treatment and the week before follow-up.


- Change in Galer Neuropathic Pain Scale (NPS) from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in Daily Sleep Interference Scale (DSIS) from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Proportion of subjects who have 'improved', 'much improved,' or 'very much improved' relative to baseline on the Patient Global Impression of Change (PGIC) on Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in the 36-item Short-Form Health Survey (SF-36) from baseline to Day 84 of treatment.
- Usage of rescue medication (yes/no) from baseline to Week 12 of treatment.

## 2.2.1.3. Exploratory Efficacy Endpoint(s)



#### 2.2.2. Safety Endpoints

The safety endpoints of this study include the following:

- Adverse events (AEs) and serious adverse events (SAEs)
- Physical and neurological examinations
- Neuropathy assessments Total Neuropathy Score-Nurse (TNSn) S
- Strength (dorsiflexion), and deep tendon reflex (knee and ankle) assessments
- Vital signs
- 12 lead digital electrocardiogram (ECGs)
- Clinical laboratory testing (hematology, chemistry, coagulation, and immunology)
- Motor and sensory nerve conduction studies
- Concomitant medications and therapies
- Injection site reactions and infusion reactions

## 2.2.3. Pharmacokinetic/Pharmacodynamic Variable(s)

The pharmacokinetic (PK) endpoints of the study include the MEDI7352 concentrations measurements in serum/plasma.

The pharmacodynamic (PD) endpoints of the study include total nerve growth factor (tNGF) measurements in serum/plasma.





## 2.2.4. Other Endpoints

The following endpoints will be assessed:

- Change in the weekly average of the average daily pain scores from the baseline week to Week 12, as measured on an 11-point (0-10) NRS, versus dose.
- Immunogenicity (ADA) assessments.

#### 3. Overall Study Design and Plan

This is a randomised, double-blind, placebo-controlled study of MEDI7352 in subjects with moderate to severe chronic PDN persistent for 6 months or longer, not adequately controlled by standard of care treatments, caused by type 1 or type 2 diabetes mellitus. The study incorporates a screening period of up to 45 days and a 12-week double-blind treatment period during which MEDI7352 or placebo will be administered intravenously (IV) on 6 occasions, with each dose separated by 14 days. There will be a 6-week follow-up period.

## 3.1. Overall Design

## 3.2. Sample Size and Power

There is no formal sample size calculation for stage 1; 10 subjects in stage 1 are considered sufficient for the initial assessment of safety. The sample size for stages 2-4 combined was determined by a formal power calculation (see below) and the size of stage 3 was defined to enable decision making for the stage 4 sample size and dose allocation ratio.

This study is powered at greater than 80% to detect a statistically significant (1-sided alpha = 0.025) dose-response relationship when the true Week 12 placebo-corrected change from baseline difference at the column dose is 1.25 on the 11-point NRS scale (MEDI7352-placebo treatment) and the true dose-response follows a hyperbolic Emax relationship, with ED50 within the range column. This calculation also assumes:

AD-ST-33.06 Effective date: 12-Nov-2020



- The true standard deviation (SD) is 2.4, which is based on other studies undertaken with pregabalin in PDN (Satoh et al. 2011, Lesser et al. 2004, Rosenstock et al. 2004, Tölle et al. 2008).
- The data from stages 2, 3, and 4 are combined so that the number of subjects for the dose-response analysis is 236 with the total number evaluable for placebo, column doses equal to 81, 37, 51, and 67, respectively. This is comprised of, assuming an overall 10% non-evaluability rate:
  - o 28 out of 30 randomised in stage 2; 14 per arm
  - o 60 out of 67 randomised in stage 3; 30 per arm, and
  - o 148 out of 165 randomised in stage 4; 37 per arm
- The dose-response hypothesis test is multiplicity adjusted as described by Pinheiro et al. 2006 in order to control the type 1-error.

The above calculations were performed using the software R and the R-package 'DoseFinding' [https://cran.r-project.org/web/packages/DoseFinding/DoseFinding.pdf] with the following parameters:

- Population SD (of change from baseline to week 12) = 2.4
- Placebo effect = 1 point reduction in NRS and CCl effect = 2.25 reduction from baseline, ie, delta= 1.25
- Linear contrasts were determined from 5 'candidate dose' response models which are all  $E_{max}$  models with decreasing potency/increasing ED50: 7.5, 15, 30, 60, 750 µg/kg. The 5th case is essentially linear in dose.  $E_{max}$  models were chosen following the recommendations in a recent meta-analysis of dose response studies by Thomas et al., 2014.
- Power was assessed across 16 alternative true dose response curves, 12 E<sub>max</sub> with ED50 ranging from 0.375 to 750 μg/kg, 3 logistic and 1 quadratic, all having a Week 12 placebo-corrected change from baseline difference at the column dose of 1.25.

The overall withdrawal rate is anticipated to be approximately 10%. However, since the primary analysis will use Last Observation Carried Forward (LOCF) for withdrawn subjects, and the SD estimate is taken from studies which also used the LOCF approach, the only additional subjects recruited will be to account for withdrawals in stages 2, 3, and 4 if withdrawal occurs at, or prior to, the Week 2 visit.

The number of subjects who will agree to participate in the genetic research is unknown. It is therefore not possible to establish whether sufficient data will be collected to allow a formal statistical evaluation or whether only descriptive statistics will be generated.

### 3.3. Study Population

Male or female (postmenopausal or surgically sterile) subjects aged ≥18 to ≤80 years with





chronic PDN persistent for 6 months or longer, not adequately controlled by standard of care treatments.

#### 3.4. Treatments Administered

Once randomized, subjects will be dosed with either MEDI7352 or placebo on Day 1, Day 14, Day 28, Day 42, Day 56, and Day 70. MEDI7352 or placebo will be administered IV over a 60-minute period. To maintain the blind, a placebo volume equivalent to the MEDI7352 volume will be administered for each dosing.

## 3.5. Method of Assigning Subjects to Treatment Groups

The randomisation schedule will be computer generated using a permuted block algorithm appropriate to the treatment groups included in each stage and will randomly allocate investigational product (IP) to randomisation numbers. The randomisation numbers will be assigned sequentially through a central interactive web response system (IWRS) as subjects are entered into the study. The randomisation schedule will not be stratified, and study centre will not be a blocking factor in the randomisation schedule.

The randomisation schedule has been prepared by Premier Research before the start of the study. No one involved in the study performance will have access to the randomisation schedule before official unblinding of treatment assignment. No subject will be randomised into this study more than once.

## 3.6. Blinding and Unblinding

All subjects, investigators, and study personnel involved in the conduct of the study, including data management, will be blinded to treatment assignment with the exception of a specified unblinded statistician and programmer from Premier Research who will have access to the randomization code, unblinded site monitors and clinical manager from Premier Research, and the unblinded pharmacist at each study site. The unblinded study personnel will not participate in study procedures or data analysis prior to unblinding of the study data to all study related personnel. Unblinded personnel who are not otherwise involved in the study will prepare data for review and interim analysis.

Study personnel will make every effort to safeguard the integrity of the study blind to minimize bias in the conduct of the study. Treatment unblinding is discouraged if knowledge of the treatment assignment will not materially change the planned management of a medical emergency. Unblinding will be permitted in a medical emergency that requires immediate knowledge of the subject's treatment assignment.

Unblinding should be discussed in advance with the medical monitor if possible. For emergency unblinding, study personnel will use the IWRS. Only authorized users will have access to the unblinding function in the IWRS, and the IWRS will reveal the treatment information for the selected subject only. If the investigator is not able to discuss treatment unblinding in advance, then he/she must notify the medical monitor as soon as possible about the unblinding incident without revealing the subject's treatment assignment. The IWRS will also send a blinded notification to the clinical team alerting them that a break blind occurred.





The investigator or designee must record the date and reason for treatment unblinding on the appropriate electronic case report form (eCRF) for that subject. In all cases that are not emergencies, the investigator must discuss the event with the medical monitor prior to unblinding the subject's treatment assignment.

If treatment assignment is unblinded for an individual subject, study personnel will be notified of that subject's treatment assignment without unblinding the treatment assignments for the remaining subjects in the study. Thus, the overall study blind will not be compromised. If a subject's treatment assignment is unblinded, he/she will be asked to withdraw from the study. The investigator will make this decision after consultation with the medical monitor.

Overall unblinding will take place at the end of the study only after database lock has been achieved.

#### 3.7. Schedule of Events

Please see the protocol Tables 2-1, 2-2 for a detailed schedule of events.

## 4. Statistical Analysis and Reporting

All efficacy and safety statistical analysis will be based on data from stages 1, 2, 3 and 4 combined, unless specified otherwise.

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will primarily use SAS (release 9.4 or higher). The multiple comparison and modelling (MCP-Mod) analysis will be performed using R (release 4.2.1 or higher) and the DoseFinding package (version 1.0-3 or higher). If a use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, the number of missing values, arithmetic mean, SD, median, 1<sup>st</sup>, and 3<sup>rd</sup> quartiles (where applicable), minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment group, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population with non-missing data at each visit, unless otherwise specified.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be





reported to 1 degree of precision more than the observed data and measures of spread will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified.

Unless otherwise indicated, all statistical tests will be conducted at the 0.025 significance level using 1-tailed tests, and *P* values will be reported. For estimation purposes, 2-sided 95% confidence intervals (CI) will be presented.

Total NGF and PK concentration data will be summarized by dose as per the quantitative variables and presenting the number (n) of non-missing observations, and the n < lower limit of quantification (LLOQ). PD and PK parameters will be summarized by dose and will include the arithmetic mean, SD, geometric mean (gmean), gmean  $\pm$  geometric SD, geometric coefficient of variation (gCV%), median, minimum and maximum.

## 4.2. Interim Analysis and Data Monitoring

Details of the interim analysis have been included in the Statistical Interim Analysis Plan (SiAP) version 1.0 dated 10-Feb-2023.

## 5. Analysis Populations

The following analysis populations are planned for this study:

- Screening Population (Screened): All subjects who provide informed consent and/or assent and provide demographic and/or baseline screening assessments, regardless of the subject's randomisation and treatment status in the study. The Screening Set will be analysed as randomised, according to planned treatment.
- Safety Population (SAF): The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication. The Safety Set will be analysed according to actual treatment.
- Modified Intent-To-Treat Population (mITT): The modified intent-to-treat population will be used for all efficacy analyses and will include all randomised subjects who receive at least 1 dose of double-blind study medication and have at least 1 daily NRS assessment while receiving double-blind treatment. The mITT Set will be analysed as randomised, according to planned treatment.
- Pharmacokinetic Population (PK): The PK Population will include all subjects for who a PK sample was obtained and analysed. The PK Set will be analysed according to actual treatment.

Assignment of subjects to populations will be confirmed at a blinded data review meeting to be held before the study database is locked.





If a subject is randomised incorrectly or is administered the incorrect IP, analyses of the mITT population will be based on the IWRS-assigned treatment whereas all other analyses will be based on the actual treatment.

## 6. General Issues for Statistical Analysis

### 6.1. Statistical Definitions and Algorithms

### 6.1.1. Baseline

For all safety endpoints, the last observation recorded prior to the first dose of treatment will be used as the baseline observation for calculations of change from baseline.

For pain diary data the baseline period is defined as the seven-day period prior to randomization, i.e., Day -7 to Day -1, inclusive. A subject is considered to have an evaluable baseline pain score if there are at least 4 days of recorded diary pain scores in the 7-day period.

## 6.1.2. Adjustments for Covariates

In addition to treatment group, the baseline value of the variable undergoing analysis and the co-medication type (Anticonvulsant versus Antidepressant) will be included in the analysis of covariance (ANCOVA) model as additive covariates. Co-medication type will be determined by blinded clinical review of each subject's medication record at baseline.

Covariates in the mixed effects models repeated measures (MMRM) and generalized estimating equations (GEE) analyses include those specified for the ANCOVA analyses, together with time and its interaction with dose group.

The crossing of co-medication type and median baseline pain score will be used as strata in the Cochran-Mantel-Haenszel (CMH) model tests. Assuming two co-medication types, the strata will be:

- 1) Anticonvulsant (Baseline NRS < Median),
- 2) Anticonvulsant (Baseline NRS > Median),
- 3) Antidepressant (Baseline NRS < Median),
- 4) Antidepressant (Baseline NRS > Median).

Where the median baseline NRS is calculated over all subjects.

### **6.1.3.** Multiple Comparisons

A multiple comparison procedure modelling approach (MCP-Mod) on LOCF data will be used for primary efficacy endpoints.

No adjustments will be made for multiple comparisons outside the MCP-Mod approach.

AD-ST-33.06 Effective date: 12-Nov-2020





## 6.1.4. Handling of Dropouts or Missing Data

For the analyses of the primary efficacy endpoints based on the mITT Population, a variety of methods will be used to deal with missing data, including:

- Primary Method: LOCF.
- Observed cases analysis.
- Baseline observation carried forward (BOCF)

Subjects with missing weekly average NRS baseline data (i.e., zero or 1-3 days of diary pain scores) will not be included in the efficacy analysis because the primary analysis is change-from-baseline. If a subject has zero or  $\leq 3$  days of diary pain data in each of the possible post-baseline seven day periods ending within the protocol definition of week 12 (day  $84 \pm 3$ ), then an imputed 'week 12 LOCF' weekly average NRS pain score will be calculated from the latest 7 'non-missing' entries of the subject's diary closest to their nominal week 12 visit (i.e., the latest 7 day period containing at least 4 NRS values), provided that this would qualify as at least 'week 2' according to the windowing outlined in Section 6.1.5. Otherwise, the week 12 LOCF weekly average NRS pain score will be set to missing.

## 6.1.5. Analysis Visit Windows

Statistical analyses will be based on scheduled visits and windows as per Protocol Table 2-1: Schedule of Events. If an assessment falls between 2 windows, then the closest visit will be used only if an assessment result is not provided within that window. All other visits will be listed only as unscheduled visits. For presentation purposes these will be mapped to the visit prior and labeled, e.g., Unscheduled Visit 3.1, if Visit 3 was the closest date prior.

For pain diary data the following analysis periods will be defined:

• Week X<sub>i</sub>: the 7-day period ending within the protocol window Day Y<sub>i</sub>±3 where at least 4 days out of 7 have recorded diary pain scores. Where several such windows exist the one ending closest to day Y<sub>i</sub> will be selected. If there are two such windows that are equidistant from day Y<sub>i</sub>, then the one with the largest number of diary entries will take precedence. If they have the same number of entries, then the later of the two end dates will be chosen. If no such window exists, then week X<sub>i</sub> will be considered missing for the purposes of weekly average scoring.

Where:

- $X_1=2, Y_1=14$
- $X_2=4, Y_2=28$
- $X_3=6, Y_3=42$
- $X_4=8, Y_4=56$

AD-ST-33.06 Effective date: 12-Nov-2020



- $X_5=10, Y_5=70$
- $X_6=12, Y_6=84$
- The week before follow-up is defined as the 7-day period prior to the last day of pain diary data for subjects completing the study (i.e., entering in the Week 18) where at least 4 days out of 7 have recorded diary pain scores.

## **6.1.6.** Pooling of Sites

Analysis by investigative site will not be conducted.

## 6.1.7. Efficacy Variables

## 6.1.7.1. Pain Numerical Rating Scale

Subjects will assess their perceived average neuropathic pain over the previous 24 hours using an 11-point NRS, with 0 representing no pain and 10 representing the worst pain imaginable. Subjects will be instructed to assess their average daily pain at approximately the same time every morning, and to record their response in a subject diary (ePRO).

## 6.1.7.2. Neuropathic Pain Scale

Subjects will assess their neuropathic pain using the Galer NPS. The NPS includes 2 descriptors of pain, including intensity and unpleasantness, and 8 descriptors that assess specific qualities of neuropathic pain: sharp, hot, dull, cold, sensitive, itchy, deep, and surface pain. Each of these 10 dimensions has a 0 to 10 NRS in which 0 is equal to no pain and 10 equals the most intense pain. There is an additional descriptor about duration and frequency of pain, which has a 1 to 3 NRS. In which 1 = I feel a background pain all the time and occasional flare-ups (breakthrough pain) some of the time, 2 = I feel a single type of pain all the time, and 3 = I feel a single type of pain only sometimes. Other times, I am pain free.

## 6.1.7.3. Daily Sleep Interference Scale

Subjects will assess how their neuropathic pain interferes with their sleep using the DSIS. The DSIS is an 11-point Likert scale, with 0 indicating that pain did not interfere with sleep and 10 indicating that pain completely interfered with sleep. The DSIS is completed by subjects once a day (upon awakening) to accurately capture variability in sleep interference due to pain on a daily basis, thus minimizing recall bias.

### 6.1.7.4. Patient Global Impression of Change

Subjects will rate their overall improvement in health status using the PGIC. The PGIC consists of a 7-point scale where 1 = "very much improved" and 7 = "very much worse." Subjects will be asked the following question: "How would you rate your overall improvement with treatment during the clinical study?" The response options include the following:

AD-ST-33.06 Effective date: 12-Nov-2020





- Very Much Improved 1
- Much Improved 2
- Minimally Improved 3
- No Change 4
- Minimally Worse 5
- Much Worse 6
- Very Much Worse 7

## 6.1.7.5. Short-Form Health Survey

The subject's health status and quality of life will be assessed using the SF-36. The SF-36 assesses 8 health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. The items use Likert-type scales with either 5 or 6 points, or 2 or 3 points. Scores will be derived by the validated built-in scoring tool. Higher SF-36 scores indicate a better state of health.

### 6.1.7.6. Rescue Medication Use

Subjects will record all rescue medications they take for neuropathic pain in a paper diary. This will be transcribed in to the eCRF collecting usage, date and time of rescue medication, medication administered, dose, frequency and route.

Subjects will be grouped by the following for rescue medication use:

- Compliant with protocol guidance on permitted therapies
- Non-compliant with protocol guidance on permitted therapies

A review of medications will be conducted at a blinded data review meeting to be held before the study database is locked.



#### 6.1.8. Derived Variables

• Change from baseline = value at current time point – value at baseline.

AD-ST-33.06 Effective date: 12-Nov-2020

Version 1.0 | Date 12-Jul-2023 | AD-PR-109.02 Effective date: 17-Aug-2020




- Reference End Date = Date of completion/discontinuation.
- Study duration = Reference end date date of first dose of treatment + 1
- Duration of exposure (days) = min(date of last dose of treatment + 14 days or date of death) date of first dose of treatment + 1.
- Treatment-emergent AEs (TEAEs) are defined as:
  - o AEs with onset at the time of or following the start of treatment with IP and not more than 30 days after the last administration of IP, or
  - AEs starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with IP and not more than 30 days after the last administration of IP.
- Average Baseline Pain NRS = the arithmetic average of the 'non-missing' daily pain scores within the baseline period defined in Section 6.1.1. For example, if a subject has 5 days of non-missing pain scores their average will be calculated over 5 days, not the full 7-day baseline period.
- Average Week X Pain NRS = the arithmetic average of the 'non-missing' daily pain scores within each subject's specific week X period defined in Section 6.1.5.
- Average Week 12 Pain NRS (LOCF) = the arithmetic average of the 'non-missing' daily pain scores within each subject's specific week 12 period or according to the imputed LOCF/BOCF approach defined in Section 6.1.4.
- Change from Baseline to Week X Pain NRS = for each subject 'Average Week X Pain NRS' minus 'Average Baseline Pain NRS'.
- Change from Baseline to Week 12 Pain NRS (LOCF/BOCF) = for each subject 'Average Week 12 Pain NRS (LOCF)' minus 'Average Baseline Pain NRS'.
- Galer NPS Total Score (ranges from 0 to 100): sum of Pain Intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, and Surface Pain Intensity (All in an 11-point NRS).
- Change from Baseline to Week X Galer NPS Total Score = for each subject 'Galer NPS Total Score' minus 'Baseline Galer NPS Total Score'.
- Total number of days rescue medication was used = End Date of Medication Start Date of medication + 1. Each day on which rescue medication was used at least once is counted.





- Cumulative consumption (mg) of paracetamol rescue medication use = Total dose of rescue medication (mg) consumed during the days in which paracetamol was used.
- Average daily dose (mg) of paracetamol rescue medication use = Cumulative consumption of paracetamol rescue medication (mg) /total number of days paracetamol rescue medication was used.

## 6.1.9. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

All P values will be displayed in four decimals and rounded using standard scientific notation (e.g., 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as <0.0001.

AEs and medical histories will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) thesaurus available at time of programming.

If partial dates of AEs occur, the convention for replacing missing dates for the purpose of TEAE is as follows: if just day is missing then the day assigned is the first day of the month or the date of first dose (if in the same month), whichever is later; if just month is missing then the month assigned is the month of the first dose, unless that results in a date prior to the first dose in which case the month after the first dose is used; and if both month and day are missing then the month assigned is the month of the first dose and the day assigned is either the first day of the month or the first dose date, whichever is later.

If partial times occur, the convention is as follows: if the missing time occurs on the day of the first dose and both the hour and minute are missing then the time assigned is the time of the first dose, otherwise if both the hour and minute are missing and the date is not the date of first dose the time assigned is 12:00; if the date is the same as the date of the first dose and only hour is missing the hour assigned is 12 or the hour of first dose, whichever is later, and if the date is the same as the date of first dose and only the minute is missing the minute assigned is 30 or the minute of first dose, whichever is later. Otherwise the hour assigned is 12 if the hour is missing and the date is not the same as the date of first dose and the minute assigned is 30 is the the date is not the same as the date of first dose.

These conventions will be applied only to AE onset dates and times with the following precaution: if the missing date and time reflect the date and time of onset of an AE, the modified date and time will be constructed to match the first documented date/time post drug administration while preserving the order in which the AE was reported in the eCRF.

In general, for quantitative laboratory values reported as '<X' or ' $\le$ X', the LLOQ will be used for analysis (i.e., the value of X will be used in the analysis for lab values reported as '<X' or ' $\le$ X'). Similarly, for quantitative laboratory values reported as '>X' or ' $\ge$ X', the upper limit of





quantification (ULOQ) will be used for analysis (i.e., the value of X will be used in the analysis for lab values reported as '>X' or ' $\geq$ X').

For analysis purposes, repeat laboratory test results will not be used unless the original laboratory value is missing or indicated as invalid, in which case the first non-missing repeated laboratory value will be used for data analysis.

ADA titre reported as <30 (below the minimum required dilution) is a negative result for the presence of ADA.

For descriptive statistics of serum concentration summaries:

- At a time-point where less than or equal to 50% of the values are not quantifiable (NQ, below LLOQ), all NQ values will be set to the LLOQ, and all descriptive statistics will be calculated accordingly.
- If more than 50%, but not all, of the concentrations are NQ, the geometric mean, geometric mean ± geometric SD and gCV% will be reported as not calculable (NC). The maximum value is reported from the individual data, and the minimum and median are set as NQ.
- If all concentrations are NQ at a time-point, the geometric mean, minimum, median and maximum are reported as NQ and the gCV% and geometric mean ± geometric SD as NC.

# 7. Study Patients/Subjects and Demographics

#### 7.1. Disposition of Patients/Subjects and Withdrawals

The total number of subjects for each of the following analysis populations will be presented for the Screening Population by randomized treatment group and overall:

- Screening Population
- Safety Population
- mITT Population
- Included in the mITT population
  - Evaluable Week 12 efficacy
  - Evaluable LOCF efficacy
- Not efficacy evaluable
- PK Population

For the Screening Population, disposition will include tabulation of:

- the number of screened subjects
- the number of re-screened subjects
- the number of enrolled subjects

The output will be further presented by treatment group and overall summarising:

• the number of randomized subjects

AD-ST-33.06 Effective date: 12-Nov-2020





- the number of subjects who completed study treatment
- the number of completed subjects
- the number of subjects withdrawing (discontinued)
- the reasons for discontinuation from study treatment and withdrawal from the study.

For all categories of subjects by treatment group, percentages will be calculated using the number of subjects randomized as the denominator.

#### 7.2. Protocol Deviations

Major protocol deviations, as determined by a Sponsor blinded review of the data prior to database lock and unblinding of the study will be reported in listings.

The Sponsor or designee will be responsible for producing the final deviation file. This file will be finalized prior to database lock, and all information will be included in the SDTM.DV domain (deviations domain).

All protocol deviations will be presented in a data listing, with a flag to indicate if a deviation was considered major.

A summary table by treatment group and overall will be generated based on protocol deviation severity (minor/major) and the classification of protocol using the following categories:

- o Inclusion
- Exclusion
- Study drug
- o Assessment safety
- Assessment– efficacy
- Lab/endpoint data
- Visit window
- Informed consent
- o Prohibited co-medication
- o Overdose/misuse
- o Other

## 7.3. Demographics and Other Baseline Characteristics

Descriptive summaries of the demographic and other baseline characteristics will be presented for all analysis populations. All demographic and baseline characteristics will be presented both overall and by treatment group.

The following demographic and baseline data will be presented in tables:

• Demographics: age, gender, ethnicity, race, height, weight, and body mass index (BMI)





- For female the number and percentage of women surgically sterile and postmenopausal will be described.
- Diagnosis of osteoarthritis: number of subjects with osteoarthritis diagnosis and area affected, clinical significance, radiological investigations, radiological significance, Kellgren-Lawrence score.

The number and percent of subjects reporting various medical histories, grouped by MedDRA system organ class (SOC) and preferred term (PT), will be tabulated by treatment group.

This analysis will be conducted for the Safety Population.

## 7.4. Exposure

The following parameters of study drug exposure and compliance will be summarized by treatment group for the Safety Population:

- Maximum number of doses administered
- Total duration of exposure
- Total (cumulative) dose infused

In addition, any incomplete infusions will be listed.

## 8. Efficacy Analysis

All efficacy variables will be summarized descriptively including number of observations, number of missing values, mean, SD, minimum, median, and maximum for continuous variables, and frequency of observations in each category and percentage for categorical variables.

Primary and secondary endpoint efficacy data will be tabulated according to the observed cases, LOCF, and BOCF approaches.

### 8.1. Primary Efficacy Analysis

The primary efficacy endpoint of this study is the change in the weekly average of the average daily pain scores from the baseline week to Week 12 measured on an 11-point (0-10) NRS.

MCP-Mod approach. The main statistical analysis of the primary efficacy endpoint will use the MCP-Mod approach on LOCF data, which is a well-established statistical methodology for establishing both the existence of a dose response and modelling the underlying dose-response relationship. The modelling step ('MOD' step) from the MCP-MOD approach will only be conducted if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

There are two steps to MCP-Mod:





- 1. The 'MCP' step is a rigorous method to establish presence of a dose response while protecting the type I error and, if the dose-response relationship is statistically significant, then
- 2. The 'MOD' step estimates the dose response function and associated model parameters.

The MCP test will use linear contrasts corresponding to the five candidate models described in Section 3.2. The test will use pre-specified model parameters and optimal contrasts for each will be generated. The hypotheses are as follows:

Null hypothesis (H<sub>0</sub>): Optimal contrasts  $\mu \ge 0$  for all models

Alternative hypothesis (H<sub>A</sub>): Optimal contrasts  $\mu$  <0 for at least one model

where  $\mu$  is the true event rate.

The underlying model will be an ANCOVA with dependent variable 'change from baseline to Week 12 (LOCF)', and independent variables will include:

- dose group as a factor variable with the placebo group as the reference level
- baseline score, i.e., baseline weekly average pain (NRS), as a continuous variable
- co-medication type.

The random error is assumed to be normally and independently distributed with constant variance. The parameter estimates of the difference between each dose group and placebo, least square (LS) Means estimates of change from baseline to Week 12 for each dose, standard errors, 95% unadjusted, 'Lalonde-type' asymmetric CI (i.e., lower limit of 1-sided 90% CI and upper limit of 1-sided 80% CI), and *P* values will be presented.

If the MCP test is statistically significant, then the MOD step will select the most appropriate model from hyperbolic  $E_{max}$ , sigmoidal  $E_{max}$  or linear using the ' $E_{maxlin}$ ' approach as described by Kirby et al (2011). From this model (including the same covariates as the ANCOVA model), various estimates will be derived (together with CI) of parameters of interest such as ED50, effective dose to achieve 90% of maximum effect (ED90), dose to achieve selected target effects, and model estimates of the treatment effect at doses studied (see Appendix in Section 15).

**MMRM:** In addition, changes from baseline in continuous endpoints will be compared between treatment groups using mixed models repeated measures including terms for:

- co-medication type (as a factor)
- treatment (as a factor)
- time (as a factor)
- the interaction between treatment and time point
- and the baseline value of the variable undergoing analysis

The mixed model for repeated measure will use average of average daily pain score of observed data at week 2, 4, 6, 8, 10, and 12. An unstructured covariance matrix will be used to model the

AD-ST-33.06 Effective date: 12-Nov-2020





within-subject errors. The Kenwards-Roger method will be used to estimate degrees of freedom. If this analysis fails to converge, a simpler structure (e.g., first-order ante-dependent or heterogeneous compound symmetry structures) will be found using Akaike information criterion (AIC).

The results will be presented using LS Means estimates, corresponding 95% CI for each treatment group and timepoint, along with the LS Means of differences with Placebo, standard error, 95% CI and p-values.

The primary efficacy analysis will be based on the mITT population.

## 8.1.1. Sensitivity Analyses of the Primary Efficacy Endpoint

To complement the MCP-MOD outputs, estimates and CI of each pairwise comparison versus placebo from the ANCOVA model described in the MCP step will be produced.

## 8.2. Secondary Efficacy Analysis

The MMRM model outlined in Section 8.1 will be applied for secondary endpoints using observed cases:

- Change in Galer NPS total score from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in DSIS from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in the eight SF-36 parameters from baseline to Day 84 of treatment.

A GEE approach for binary data will be used for the following dichotomous endpoints:

- Percentage of subjects who have achieved ≥30% reductions in the weekly average of the average daily pain score from baseline during Weeks 4, 8, and 12 of treatment and the week before follow-up.
- Percentage of subjects who have achieved ≥50% reductions in the weekly average of the average daily pain score from baseline during Weeks 4, 8, and 12 of treatment and the week before follow-up.

The GEE model specification will include a binomial distribution, a logit link function, and an unstructured covariance matrix. If this analysis fails to converge, a simpler structure (e.g. first-order autoregressive or compound symmetry structures) will be found using AIC. The model will include terms for:

- co-medication type (as a factor)
- treatment (as a factor)
- time (as a factor)
- the interaction between treatment and time





A CMH test stratified by the crossing of co-medication subgroup and median baseline pain score will also be carried out for the above dichotomous endpoints. The CMH risk difference at Week 12 will be estimated between the treatment group and placebo. The number and percentage of subjects meeting the reduction response will be displayed, along with the risk difference, 95% CI and *P* value.

The proportion of subjects who have 'improved', 'much improved,' or 'very much improved' relative to baseline on the PGIC on Days 28, 56, and 84 of treatment and the follow-up visit will be tested using a CMH statistics.

The efficacy analysis of secondary endpoints will be based on the observed cases and on the mITT population.

Usage of rescue medication (yes/no) will be summarized by dose group for each visit from baseline to Week 12 of treatment and over the whole treatment period. The following additional variables will be derived and summarised:

- Total number of days rescue medication was used.
  - Each day on which rescue medication was used at least once is counted.
- Cumulative consumption (mg) of paracetamol rescue medication use.
  - Calculated as the total dose of rescue medication (mg).
- Average daily dose (mg) of paracetamol rescue medication use.
  - Calculated as: cumulative consumption of rescue medication (mg)/total number of days rescue medication was used.

#### 8.3. Exploratory Efficacy Analysis



#### 9. Safety and Tolerability Analysis

All safety analyses will be performed on the Safety Population using descriptive statistics. Descriptive summaries by treatment group and overall will be produced. No inferential statistical tests will be performed.

AD-ST-33.06 Effective date: 12-Nov-2020





The analysis of safety assessments in this study will include summaries of the following categories of safety and tolerability data collected for each patient:

- Adverse events
  - o TEAEs
  - o SAEs
  - Significant AEs
    - TEAEs leading to discontinuation of IP
  - AEs of Special Interest
    - Positively-adjudicated possible or probable rapidly progressive osteoarthritis (RPOA), subchondral insufficiency fractures, primary osteonecrosis, or pathological fracture
    - Infections that meet SAE and/or severe AE criteria
    - Anaphylactic reactions or infusion-related reactions that lead to permanent discontinuation of administration of IP
  - o TEAEs associated with abnormal liver
  - o Any deaths

Drug induced liver injury Clinical laboratory investigations

- Vital signs
- Electrocardiograms (ECG)
- COVID-19 screening
- Physical and neurological examination
- Total neuropathy score-nurse
- Motor and sensory nerve conduction studies
- Strength and deep tendon reflexes
- Hypersensitivity / Anaphylactic reactions
- Injection site or infusion reactions
- Liver diagnostic investigations, risk factors, signs and symptoms.
- Infection diagnostic investigations, risk factors, signs and symptoms.
- Prior and concomitant medications and therapies





#### 9.1. Adverse Events

A summary table by treatment group will present the number and percent of subjects reporting:

- Any AEs
- Non-serious AEs occurring in more than 5% of subjects
- Any TEAEs
- Any SAEs
- Any TEAEs possibley related to study drug
- Any TEAEs leading to discontinuation of IP
- Any SAEs possibley related to study drug
- Life-threatenings SAEs
- SAEs resulting in death

Summaries of the incidence of TEAEs will be displayed by treatment group, by ADA status, by severity and by:

- SOC and PT
- SOC, PT, and maximum severity (mild, moderate, severe)
- SOC, PT, and maximum causality (not related, possibly related) to the study drug

In the summaries showing severity and relationship to study drug the event with the maximum severity or strongest relationship will be reported. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = related).

In the case of multiple occurrences of the same AE within the same subject, each subject will only be counted once for each level of summarization.

All AEs will be presented in a by-treatment and by-subject listing, detailing the verbatim term given by the Investigator, the PT, SOC, onset date and time, end date and time, severity, outcome, relationship to study drug, action taken with study drug, other action taken, seriousness, and criteria for seriousness.

## 9.1.1. Adverse Events Leading to Discontinuation of IP

A summary of incidence rates (frequencies and percentages) of TEAEs leading to discontinuation of IP, by treatment group, SOC, and PT will be prepared. The table will also be produced separately by maximum severity and maximum causality.





A data listing of TEAEs leading to discontinuation of IP will also be provided, displaying details of the event(s) captured on the rCRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study and serious adverse events will be listed.

A summary of incidence rates (frequencies and percentages) of SAEs by treatment group, SOC, and PT will be prepared. The table will also be produced separately for life-threatening SAEs, for SAEs with outcome death and for SAEs by relationship to study medication.

## 9.1.3. Drug-Induced Liver Injury

A summary of incidence rates of TEAEs associated with abnormal liver by treatment group, SOC, and PT will be prepared.

The type and the results of the liver diagnostic investigation performed will be tabulated by treatment group.

The number and percentage of subjects within each type of liver risk factors and style events will be tabulated by treatment group. Liver signs and symptoms will be presented in the same way.

#### 9.1.4. Infection Risk

A summary of incidence rates of infections that meet SAE or severe AE criteria by treatment group, SOC, and PT will be prepared.

The type and the results of infection diagnostic investigation performed will be tabulated by treatment group.

The number and percentage of subjects within each type of infection risk factors and style events will be tabulated by treatment group. Infection signs and symptoms will be presented in the same way.

### 9.2. COVID-19 Vaccination and Screening

The number and percentage of fully vaccinated subjects at baseline will be summarized by treatment group.

The symptoms, tests, and results from coronavirus disease 2019 (COVID-19) screening will be tabulated for each visit by treatment group.

COVID-19 vaccination, signs, symptoms and impact will be presented in listings.

## 9.3. Clinical Laboratory Evaluations

Absolute values and changes from baseline will be summarized using descriptive statistics by





treatment group and visit for chemistry, hematology, coagulation, and urinalysis tests.

The number of subjects with clinical laboratory values (chemistry, hematology, coagulation, and urinalysis) categorized as below, within, or above normal ranges (or as either normal or abnormal for urinalysis variables that do not have quantitative ranges) and whether they are clinically significant or not will be tabulated for each clinical laboratory analyte by treatment group and visit. A shift table showing change from baseline in range categories for each clinical laboratory analyte will be produced by treatment group and by visit.

The number of subjects with values for Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)  $\geq 3 \times \text{upper limit of normal (ULN)}$ , and with values for total bilirubin (TBL)  $\geq 2 \times \text{ULN}$  will be summarized in AST, ALT vs. TBL shift tables to identify Potential Hy's Law (PHL) and Hy's Law (HL) cases by treatment group.

Diagnostic immunology, urine pregnancy, and urine drug tests will be presented in by-subject listings only.

All laboratory values will be displayed in the data listings and those that are outside the normal range will be flagged, along with corresponding normal ranges.

## 9.4. Vital Signs

Descriptive summaries of actual values and changes from baseline by treatment group, visit and time point will be presented for:

- Supine heart rate
- Supine systolic blood pressure
- Supine diastolic blood pressure
- Respiratory rate
- Body temperature
- Standing heart rate
- Standing systolic blood pressure
- Standing diastolic blood pressure

Height, weight, and BMI will be presented at baseline only.

#### 9.5. Electrocardiograms

The number and percentage of subjects with normal, abnormal not clinically significant, and abnormal clinically significant ECG results will be summarized by treatment group and by visit.

If applicable (digital ECGs), descriptive summaries will be presented by treatment group, visit and time point (for Day 1 only) for ECG measures of PR, QRS, QT, RR intervals and for the calculated variables QTcF and HR for each treatment group and time point.

Heart rate (HR) and Fridericia's correction (QTcF) will be derived as follows:





Heart Rate (HR) 
$$HR = 10^{3} \frac{60}{RR_{msec}}$$
Fridericia's Correction 
$$QTc_{f} = \frac{QT_{msec}}{\sqrt[3]{RR}}$$
Sec.

# 9.6. Physical and Neurological Examination

The physical and neurological examination findings will be presented in listings.

## 9.7. Total Neuropathy Score-Nurse

Descriptive summaries of the TNSn will be presented by treatment groups and by visit. Additionally, the number and percentage of subjects within each category (0, 1, 2, 3, and 4) for each sub-score (sensory symptom, motor symptom, autonomic symptom, pin sensibility, vibration sensibility) will be summarized by treatment group and by visit.

## 9.8. Motor and Sensory Nerve Conduction Studies

Amplitude, peak latency, conduction velocity, and duration of nerve action potentials will be summarized by treatment group and visit for each location and evaluation type. The number of subjects with normal and abnormal evaluation will be tabulated by treatment group and by visit.

## 9.9. Strength and Deep Tendon Reflexes

The number and percentage of subjects within each category of the ankle dorsiflexion strength and the deep tendon reflexes will be tabulated by treatment group and by visit.

#### 9.10. Hypersensitivity/Anaphylactic Reactions, Injection Site or Infusion Reactions

The type and symptoms of hypersensitivity/ anaphylactic reactions will be tabulated by treatment group.

Injection site reactions will be tabulated describing the severity of pain, tenderness, erythema/redness, and induration/swelling by treatment group and by visit.

Anaphylactic reactions and infusion related reactions will be summarized in line with AEs, displayed by treatment group and by:

- SOC and PT
- SOC, PT, and maximum severity (mild, moderate, severe)

Hypersensitivity/anaphylactic and infusion related reactions will also be presented in a by-

AD-ST-33.06 Effective date: 12-Nov-2020





treatment and by-subject listings, detailing type of reaction, severity grade for symptom with highest severity and onset time for hypersensitivity/anaphylactic reactions, and assessment result for injection site or infusion related reactions.

#### 9.11. Prior and Concomitant Medication and Procedures

Prior medications will be presented separately from concomitant medications.

Medications will be coded using the latest version of the WHO Drug Dictionary.

Medications that started before first dose of study medication will be considered prior, whether they were stopped before first dose of study medication or not.

A concomitant medication is defined as any medication continuing or starting after first dose of study medication. This includes medications which start before first dose of study medication and continue while on-treatment, and medications that started after first dose of study medication.

The frequency and percentage of concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) class 2 and preferred name by treatment groups, unless otherwise specified.

In listings, all medications will be displayed.

If the start/stop dates of a medication are partially or completely missing, then the medication will be assumed to be concomitant if it cannot be definitely shown from the start/stop dates that it was not administered while on-treatment. Missing dates will not be replaced.

Thus, the following approach will be taken for exclusion from concomitant medications because of discontinuation before start of treatment:

- If the stop day is missing but the month is complete, then the medication will be excluded from concomitant medications only if the stop month is before the month of the first dose of study medication.
- If the stop day and month are missing but the year is complete, then the medication will be excluded from concomitant medications only if the stop year is before the year of the first dose of study medication.
- If the stop date is completely missing, then the medication will not be excluded.

For concomitant medication exclusion (because of the late start after the end of the treatment period):

• If the start day is missing but the month is complete, then the medication will be excluded from concomitant medications only if the start month is after the last month of the treatment period.





- If the start day and month are missing but the year is complete, then the medication will be excluded from concomitant medications only if the start year is after the year of the treatment period.
- If the start date is completely missing, then the medication will not be excluded.

A similar approach will be used for summarizing concomitant procedures.

## 10. Changes from Planned Analysis



The PK endpoints involving derivation of PK parameters for each dose and for each subject will be conducted by a population PK analysis of the data as part of a pooled data analysis instead of by a noncompartmental analysis (NCA). This will be documented in the CSR as a change in planned analysis. The pooled data analysis will be described in a separate modelling analysis plan. As a result, description of TLFs related to PK parameters are removed from this SAP.

Additional analyses with pooled site as a covariate are not going to be conducted and as such, they are removed from this SAP.

It was planned to have a supplementary analysis to the primary using an adaptive MCP-MOD method. In this analysis, stages 2+3 and stage 4 were going to be analysed separately and the results combined using an inverse-normal *P* value combination function (with weights related to the original planned sample sizes). This supplementary analysis is removed from this SAP.

The Cochran-Mantel-Haenszel test for the non-binary categorical endpoints has been extended to include the secondary endpoint of pain response.

### 11. Other Planned Analysis





AD-ST-33.06 Effective date: 12-Nov-2020





## 11.2. Immunogenicity

Blood samples will be collected for assessment of ADA levels. Anti-Drug Antibody response during the entire study period and at each study assessment will be summarised according to ADA category and titre value for the Safety population with evaluable ADA results. A listing of the ADA test results will be produced.

For immunogenicity analysis, the presence of detectable (i.e., positive) ADAs against MEDI7352 will be reported. ADA results from each sample are reported as either positive or negative. In addition, the ADA titer result will be reported for samples confirmed positive for the presence of ADAs. A participant is defined as being ADA-positive if a positive ADA result is available at any time, including baseline and all post-baseline measurements, otherwise ADA negative.

The following ADA categories will be determined:

- ADA positive if a collected sample is tested positive at any time during the study, including baseline and/or post-baseline. (The percentage of these participants in a population is known as ADA prevalence).
- Treatment-emergent ADA positive (TE-ADA+): A positive post-baseline result and either of the following statements holds:
  - o Baseline is ADA negative and at least one post-baseline assessment is ADA positive. This is called treatment-induced ADA positive.
  - o Baseline is ADA positive, and the baseline titre is boosted by greater than the variability of the assay (i.e., ≥X-fold increase, commonly 4-fold) at ≥1 post-baseline timepoint. This is called treatment-boosted ADA positive.

(The percentage of these participants in a population is known as ADA incidence)

- Only baseline positive if a collected sample is tested positive at baseline.
- Non-Treatment-emergent ADA positive (non-TE-ADA+): Participants who are ADA positive but not fulfilling the conditions for TE-ADA+.
- Treatment-emergent Persistently ADA positive: ADA negative at baseline and having at least 2 post-baseline ADA positive measurements with ≥16 weeks (112 days) between first and last positive, or an ADA positive result at the last available post-baseline assessment.
- Treatment-emergent Transiently ADA positive: ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive
- ADA positive post-baseline and positive at baseline.

### 11.3. Pharmacokinetic Analysis

Pharmacokinetic concentration data will be summarized using descriptive statistics by dose and treatment visit overall and by ADA status (positive/negative) presenting the number (n) of non-





missing observations, and the n < LLOQ. A figure of geometric mean (with and without gSD) serum MEDI7352 concentration over time by treatment group will be generated (overall and by ADA status (positive/negative)). Additionally, pharmacokinetic concentration data will be listed and presented graphically as spaghetti plots of individual participant profiles by treatment group and ADA status (positive/negative).

#### 12. References

- 1. ICH (1998) ICH Harmonised Tripartite Guideline. Statistical Principles for Clinical Trials E9; 1998. https://database.ich.org/sites/default/files/E9 Guideline.pdf
- 2. ASA. (2018) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2018. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 4. Satoh J, Yagihashi S, Baba M, Suzuki M, Arakawa A, Yoshiyama T. Efficacy and safety evaluation of pregabalin treatment over 52 weeks in patients with diabetic neuropathic pain extended after a double-blind placebo-controlled trial. *J Diabetes Investig*. 2011;2(6):457-463. Doi: 10.1111/j.2040-1124.2011.00122.x.
- 5. Lesser H, Sharma U, LaMoreaux L, Poole RM. Pregabalin relieves symptoms of painful diabetic neuropathy: a randomized controlled trial. *Neurology*. 2004;63(11):2104-2110.
- 6. Rosenstock J, Tuchman M, LaMoreaux L, Sharma U. Pregabalin for the treatment of painful diabetic peripheral neuropathy: a double-blind, placebo-controlled trial. *Pain*. 2004;110(3):628-638.
- 7. Tölle T, Freynhagen R, Versavel M, Trostmann U, Young JP Jr. Pregabalin for relief of neuropathic pain associated with diabetic neuropathy: a randomized, double-blind study. *Eur J Pain*. 2008;12(2):203-213.
- 8. Pinheiro J, Bornkamp B, Bretz F. Design and analysis of dose-finding studies combining multiple comparisons and modelling procedures. *J Biopharm Stat.* 2006;16(5):639-656. Doi: 10.1080/10543400600860428.
- 9. Thomas N, Sweeney K, Somayaji V. Meta-analysis of clinical dose–response in a large drug development portfolio. *Stat Biopharm Res.* 2014;6(4):302-317. Doi: 10.1080/19466315.2014.924876.
- 10. Kirby S, Brain P, Jones B. Fitting E(max) models to clinical trial dose-response data. Pharma Stat. 2011;10(2):143-149. Doi: 10.1002/pst.432.





# 13. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (eCRF page or listing number).

The following are planned summary tables for protocol number D5680C00002. The table numbers and page numbers are place holders only and will be determined when the tables are produced.

### 13.1. Demographic Data

Table 1: Demographic Data Summary Tables and Figures

| - I | | • |
|---|---|---|
| Table Number | Population | Table Title/Summary |
| Table 14.1.2 | Screening | Subject Disposition |
| Table 14.1.3 | Screen Failure | Summary of Reasons for Screening Failure |
| Table 14.1.4.1 | Screening | Demographics and Baseline Characteristics |
| Table 14.1.4.2 | Safety | Demographics and Baseline Characteristics |
| Table 14.1.4.3 | mITT | Demographics and Baseline Characteristics |
| Table 14.1.4.4 | PK | Demographics and Baseline Characteristics |
| Table 14.1.5.1 | Screening | Osteoarthritis Characteristics |
| Table 14.1.5.2 | Safety | Osteoarthritis Characteristics |
| Table 14.1.5.3 | mITT | Osteoarthritis Characteristics |
| Table 14.1.5.4 | PK | Osteoarthritis Characteristics |
| Table 14.1.6 | Safety | Medical History by System Organ Class and Preferred Term |
| Table 14.1.7 | Safety | Prior Medications by ATC Class and Preferred Name |
| Table 14.1.8 | Safety | Protocol Deviations |
| Table 14.1.9 | Safety | Overall Study Drug Exposure |

AD-ST-33.06 Effective date: 12-Nov-2020



# 13.2. Efficacy Data

**Table 2: Efficacy Data** 

| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.2.1.1.1 | mITT | Daily Pain NRS: Summary Statistics (Observed Cases) |
| Table 14.2.1.1.2 | mITT | Daily Pain NRS: Summary Statistics (LOCF) |
| Table 14.2.1.1.3 | mITT | Daily Pain NRS: Summary Statistics (BOCF) |
| Table 14.2.1.2.1 | mITT | Daily Pain NRS: Primary MCP-Mod Analysis (LOCF) |
| Table 14.2.1.2.2 | mITT | Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) |
| Table 14.2.1.3.1 | mITT | Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) |
| Table 14.2.1.3.2 | mITT | Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) |
| Table 14.2.2.1 | mITT | Galer NPS: Summary Statistics (Observed Cases) |
| Table 14.2.2.2 | mITT | Galer NPS: MMRM Analysis (Observed Cases) |
| Table 14.2.3.1 | mITT | DSIS: Summary Statistics (Observed Cases) |
| Table 14.2.3.2 | mITT | DSIS: MMRM Analysis (Observed Cases) |
| Table 14.2.4.1 | mITT | SF-36: Summary Statistics (Observed Cases) |
| Table 14.2.4.2 | mITT | SF-36: MMRM Analysis (Observed Cases) |
| Table 14.2.5.1 | mITT | Rescue Medication Use: Summary Statistics |
| Table 14.2.6.1 | mITT | Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel-Haenszel (Observed Cases) |
| Table 14.2.6.2 | mITT | Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) |
| Table 14.2.7.1 | mITT | Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel-Haenszel (Observed Cases) |
| Table 14.2.7.2 | mITT | Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) |
| Table 14.2.8.1 | mITT | Patient Global Impression of Change: Summary Statistics |
| Table 14.2.8.2 | mITT | Patient Global Impression of Change: Cochran-Mantel-Haenszel |
| CCI | | |



# 13.3. Safety Data

**Table 3: Safety Data** 

| Table Number | Population | Table Title / Summary |
|---|---|---|
| 14.3.1 Displays | 14.3.1 Displays of Adverse Events | |
| Table 14.3.1.1 | Safety | Summary of Overall Adverse Events |
| Table 14.3.1.2 | Safety | Treatment Emergent Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.1.3 | Safety | Treatment Emergent Adverse Events by Severity, System Organ Class and Preferred Term |
| Table 14.3.1.4 | Safety | Treatment Emergent Adverse Events by Relationship to Study<br>Medication, System Organ Class and Preferred Term |
| Table 14.3.1.5 | Safety | Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term |
| Table 14.3.1.6 | Safety | Treatment Emergent Adverse Events Leading to Discontinuation of Study drug by System Organ Class and Preferred Term |
| Table 14.3.1.7 | Safety | Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term |
| Table 14.3.1.8 | Safety | Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term |
| Table 14.3.1.9 | Safety | Treatment Emergent Adverse Events by Preferred Term |
| 14.3.2 Summary | of Deaths, Other Ser | rious and Significant Adverse Events |
| Table 14.3.2.1.1 | Safety | Serious Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.2.1.2 | Safety | Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.2.1.3 | Safety | Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term |
| Table 14.3.2.1.4 | Safety | Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term |
| 14.3.2.2 Displays of Significant Adverse Events and Adverse Events of Special Interest | | |
| Table 14.3.2.2.1 | Safety | Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term |
| Table 14.3.2.2.2 | Safety | Potential Joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term |
| Table 14.3.2.2.3 | Safety | Serious and/or severe Infections by System Organ Class and Preferred<br>Term |

AD-ST-33.06 Effective date: 12-Nov-2020

Version 1.0 | Date 12-Jul-2023 | AD-PR-109.02 Effective date: 17-Aug-2020




| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.3.2.2.4 | Safety | Ana phylactic Reactions, Hypersensitivity or Infusion-Related Reactions<br>Leading to Discontinuation of IP by System Organ Class and Preferred<br>Term |
| 14.3.3 Narrative | s of Deaths and Oth | er Serious Adverse Events |
| Table 14.3.3.1 | Safety | Listing of Serious Adverse Events |
| Table 14.3.3.2 | Safety | Listing of Deaths |
| 14.3.4 Laborator | y Data Summary T | ables |
| Table 14.3.4.1 | Safety | Descriptive Summary of Clinical Chemistry |
| Table 14.3.4.2 | Safety | Shift Table of Clinical Chemistry Results |
| Table 14.3.4.3 | Safety | Descriptive Summary of Hematology |
| Table 14.3.4.4 | Safety | Shift Table of Hematology Results |
| Table 14.3.4.5 | Safety | Descriptive Summary of Coagulation |
| Table 14.3.4.6 | Safety | Shift Table of Coagulation Results |
| Table 14.3.4.7 | Safety | Descriptive Summary of Urinalysis |
| Table 14.3.4.8 | Safety | Shift Table of Urinalysis Results |
| Table 14.3.4.9 | Safety | Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin |
| 14.3.6 Other Saf | ety Data Summary T | Γables |
| Table 14.3.5.1 | Safety | Descriptive Summary of Vital Signs |
| Table 14.3.5.2 | Safety | Descriptive Summary of ECG Data |
| Table 14.3.5.3 | Safety | Summary of Overall Evaluation of safety ECG Data |
| Table 14.3.5.4 | Safety | Covid-19 Screening |
| Table 14.3.5.5 | Safety | Summary of Sub-Scores for Total Neuropathy Score-Nurse |
| Table 14.3.5.6 | Safety | Descriptive Summary of Total Neuropathy Score-Nurse |
| Table 14.3.5.7 | Safety | Summary of Motor and Sensory Nerve Conduction Studies |
| Table 14.3.5.8 | Safety | Summary of Strength and Deep Tendon Reflexes |
| Table 14.3.5.9 | Safety | Summary of Local Injection Site Reactions |
| Table 14.3.5.10 | Safety | Summary of Anaphylactic Reactions |
| Table 14.3.5.11 | Safety | Summary of Liver Diagnostic Investigations |
| Table 14.3.5.12 | Safety | Summary of Liver Risk Factors and Lifestyle Events |
| Table 14.3.5.13 | Safety | Summary of Liver Signs and Symptoms |

AD-ST-33.06 Effective date: 12-Nov-2020



| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.3.5.14 | Safety | Summary of Infection Diagnostic Investigations |
| Table 14.3.5.15 | Safety | Summary of Infection Risk Factors and Lifestyle Events |
| Table 14.3.5.16 | Safety | Summary of Infection Signs and Symptoms |
| Table 14.3.5.17 | Safety | Summary of Concomitant Medications by ATC Level 2 and Preferred Term |
| Table 14.3.5.18 | Safety | Summary of Concomitant Procedures |
| Table 14.3.5.19 | Safety | Anti-Drug Antibody Results and Titre Summary by Timepoint |
| Table 14.3.5.20 | Safety | Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories |



## 13.4. Pharmacokinetic/Pharmacodynamic Data

Table 4: Pharmacokinetic/Pharmacodynamic Data

| Table Number | Population | Table Title / Summary |
|---|---|---|
| 14.4 Pharmacokinetic and Pharmacodynamic Data Summary Tables | | |
| Table 14.4.1 | e 14.4.1 PK Summary of Serum MEDI7352 Concentrations | |
| Table 14.4.2 | Safety | Summary of Serum total NGF Concentrations |

## 13.5. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number D5680C00002.

In general, one listing will be produced per eCRF domain. All listings will be sorted by treatment, site, and subject number. All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 5: Planned Listings** 

| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data Listin | 16.2 Subject Data Listings | |
| 16.2.1 Subject Discontin | nuations/Completion | as |
| Listing 16.2.1.1 | Screening | Subject Disposition |
| Listing 16.2.1.2 | Screening | Assignment to Analysis Populations |
| Listing 16.2.1.3 | Safety | Reason for IP Discontinuation and Withdrawal from the Study |
| Listing 16.2.1.4 | Screen Failure | List of Reasons for Screening Failure |
| Listing 16.2.1.5 | Screening | Visits List and COVID-19 Impact |
| 16.2.2 Protocol Deviation | 16.2.2 Protocol Deviations | |
| Listing 16.2.2.1 | Screening | Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria |
| Listing 16.2.2.2 | Safety | Protocol Deviations Protocol Deviations |
| 16.2.3 Randomization | 16.2.3 Randomization | |
| Listing 16.2.3 | Safety | Randomization and Treatment Group |

AD-ST-33.06 Effective date: 12-Nov-2020

Version 1.0 | Date 12-Jul-2023 | AD-PR-109.02 Effective date: 17-Aug-2020




| Data Listing Number | Population | Data Listing Title/Summary |
|---|---|---|
| 16.2 Subject Data Listin | igs | |
| 16.2.4 Demographic Date | ta and Other Baselir | ne Characteristics |
| Listing 16.2.4.1 | Screening | Demographic and Baseline Characteristics |
| Listing 16.2.4.2 | Safety | MedicalHistory |
| Listing 16.2.4.3 | Screening | Osteoarthritis Characteristics |
| 16.2.5 Compliance and/o | or Drug Concentrati | ion Data |
| Listing 16.2.5.1 | Safety | Study Drug Administration: Individual Doses |
| 16.2.6 Individual Effica | cy Response Data | |
| Listing 16.2.6.1 | mITT | Daily Pain NRS |
| Listing 16.2.6.2 | mITT | Ga ler NPS |
| Listing 16.2.6.3 | mITT | DSIS |
| Listing 16.2.6.4 | mITT | SF-36 |
| Listing 16.2.6.5 | mITT | Rescue Medication Usage |
| Listing 16.2.6.6 | mITT | Patient Global Impression of Change |
| CCI | | |
| 16.2.7 Adverse Event Li | stings (by Patient/S | ubject) |
| Listing 16.2.7.1 | Safety | Adverse Events |
| Listing 16.2.7.2 | Safety | Treatment Emergent Adverse Events Leading to Study Drug<br>Discontinuation |
| Listing 16.2.7.3 | Safety | Treatment Emergent Adverse Events Associated with Abnormal Liver |
| Listing 16.2.7.4 | Safety | Joint Related Adverse Events of Special Interest |
| Listing 16.2.7.5 | Safety | Serious and/or Severe Infections |
| Listing 16.2.7.6 | Safety | Anaphylactic Reactions, Hypersensitivity or Infusion-Related<br>Reactions Leading to Discontinuation of Study Drug |
| 16.2.8 Laboratory Values (by Patient/Subject) | | |
| Listing 16.2.8.1 | Safety | Clinical Chemistry Laboratory Evaluations |
| Listing 16.2.8.2 | Safety | Hematology Laboratory Evaluations |
| Listing 16.2.8.3 | Safety | Coagulation Laboratory Evaluations |
| Listing 16.2.8.4 | Safety | Urina ly sis La boratory Evaluations |
| Listing 16.2.8.5 | Safety | Serology Laboratory Evaluations |
| Listing 16.2.8.6 | Safety | Pregnancy Test Results |

AD-ST-33.06 Effective date: 12-Nov-2020



| Data Listing Number | Population | Data Listing Title/Summary |
|---|---|---|
| 16.2 Subject Data Listin | | |
| Listing 16.2.8.7 | Safety | Drug Test Results |
| Listing 16.2.8.8 | Safety | COVID-19 Screening |
| 16.2.9 Other Clinical Ol | oservations and Mea | asurements (by Patient/Subject) |
| Listing 16.2.9.1 | Safety | Vital Signs Measurements |
| Listing 16.2.9.2 | Safety | ECGResults |
| Listing 16.2.9.3 | Safety | Physical Examination Results |
| Listing 16.2.9.4 | Safety | Neurological Examination Results |
| Listing 16.2.9.5 | Safety | Total Neuropathy Score-Nurse |
| Listing 16.2.9.6 | Safety | Motor and Sensory Nerve Conduction Studies |
| Listing 16.2.9.7 | Safety | Strength and Deep Tendon Reflexes |
| Listing 16.2.9.8 | Safety | Injection Site Reactions |
| Listing 16.2.9.9 | Safety | Anaphylactic Reactions |
| Listing 16.2.9.10 | Safety | Liver Diagnostic Investigations |
| Listing 16.2.9.11 | Safety | Liver Risk Factors and Lifestyle Events |
| Listing 16.2.9.12 | Safety | Liver Signs and Symptoms |
| Listing 16.2.9.13 | Safety | Infection Diagnostic Investigations |
| Listing 16.2.9.14 | Safety | Infection Risk Factors and Lifestyle Events |
| Listing 16.2.9.15 | Safety | Infection Signs and Symptoms |
| Listing 16.2.9.16 | Safety | Prior and Concomitant Medications |
| Listing 16.2.9.17 | Safety | Prohibited Concomitant Medications |
| Listing 16.2.9.18 | Safety | Concomitant Procedures |
| Listing 16.2.9.19 | Safety | Anti-drug Antibody Test Results |
| 16.2.10 Pharmacokineti | c/Pharmacodynami | c Measurements |
| Listing 16.2.10.1 | PK | Serum MEDI7352 Concentrations |
| Listing 16.2.10.2 | Safety | Serum total NGF Concentrations |

# 13.6. Planned Figure Descriptions

The following are planned summary figures for protocol number D5680C00002. The figure numbers and page numbers are place holders only and will be determined when the figures are produced.

AD-ST-33.06 Effective date: 12-Nov-2020





**Table 6: Planned Figures** 

| Figure Number | Population | Figure Title/Summary |
|---|---|---|
| Figure 14.2.1.1 | mITT | Daily Pain NRS: MCP-Mod Dose Response Model |
| Figure 14.2.1.2 | mITT | Daily Pain NRS: Boxplots at Week 12 by Treatment<br>Group and Missing Data Handling |
| Figure 14.2.1.3 | mITT | Daily Pain NRS: Boxplots at Week 12 by Treatment<br>Group and Co-Medication Subgroup |
| Figure 14.2.1.4 | mITT | Daily Pain NRS: MMRMLS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases) |
| Figure 14.3.6.1.1 | Safety | Vital Sign Profiles: Mean (±SD) Systolic Blood Pressure over time |
| Figure 14.3.6.1.2 | Safety | Vital Sign Profiles: Mean (±SD) Dia stolic Blood<br>Pressure over time |
| Figure 14.3.6.1.3 | Safety | Vital Sign Profiles: Mean (±SD) Heart Rate over time |
| Figure 14.3.6.1.4 | Safety | Vital Sign Profiles: Mean (±SD) Respiratory Rate over time |
| Figure 14.3.6.1.5 | Safety | Vital Sign Profiles: Mean (±SD) Temperature over time |
| Figure 14.4.1.1 | PK | Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 over time |
| Figure 14.4.1.2 | PK | Pharmacokinetics: Individual Plot of Serum MEDI7352<br>Concentrations over time |
| Figure 14.4.2.1 | Safety | Pharmacodynamics: Line Plot of Geometric Mean (with and without gSD) Serum total NGF over time |
| Figure 14.4.2.2 | Safety | Pharmacodynamics: Individual Plot of Serum total NGF over time |




## 14. Tables, Listing and Figure Shells

## 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all Tables, Listings, and Figures in support of this study. Note that programming notes may be added if appropriate after each table, listing and figure shell. All shells will be provided as a separate document.





## Figure 1: Standardized Layout

| Astra Zeneca | | Page xx of xx |
|---|---|---|
| Protocol: D5680C00002 | | Version |
| | Table Listing Figures vv v | |
| | <table, figure="" listing,=""> xx.x.x</table,> | |
| | Title of Table, Listing or Figure | |
| Stud | ly Population and if applicable subgroup Description | |
| | Body of Table, Listing or Figure | |
| | Body of Table, Eisting of Figure | |
| Note: If directly Applicable | | |
| Footnote 1 | | |
| Footnote 2 | | |
| Footnote n | | |
| Footnote n+1 SAS program path and name | e Executed on ddmmmyyyy at hh:mm on data from ddmmmyy | уу |



## 15. Appendix: Calculation of Dose to achieve target effects

Although only one dose-response model type (Emax) is pre-specified in the protocol for the primary analysis,

Let us assume the R® *DoseFinding* package original parametrization for these two dose-response model functions below:

Journal of Statistical Software

9

| Name | $f(d, oldsymbol{	heta})$ | $f^0(d,oldsymbol{	heta^*})$ | (*) | (#) |
|---|---|---|---|---|
| linear | $E_0 + \delta d$ | d | | |
| linlog | $E_0 + \delta \log(d+c)$ | $\log(d+c)$ | | c |
| quadratic | $E_0 + \beta_1 d + \beta_2 d^2$ | $d + \delta d^2$ if $\beta_2 < 0$ | δ | |
| emax | $E_0 + E_{\rm max} d / (ED_{50} + d)$ | $d/(ED_{50} + d)$ | $ED_{50}$ | |
| logistic | $E_0 + E_{\text{max}} / \{1 + \exp[(ED_{50} - d)/\delta]\}$ | $1/\{1 + \exp[(ED_{50} - d)/\delta]\}$ | $(ED_{50}, \delta)^{\top}$ | |
| exponential | $E_0 + E_1(\exp(d/\delta) - 1)$ | $\exp(d/\delta) - 1$ | δ | |
| sigEmax | $E_0 + E_{\text{max}} d^h / (ED_{50}^h + d^h)$ | $d^h/(ED_{50}^h + d^h)$ | $(ED_{50},h)^{\top}$ | |
| betaMod | $E_0 + E_{\text{max}} B(\delta_1, \delta_2) (d/D)^{\delta_1} (1 - d/D)^{\delta_2}$ | $B(\delta_1, \delta_2)(d/D)^{\delta_1}(1 - d/D)^{\delta_2}$ | $(\delta_1, \delta_2)^{\top}$ | D |

Table 1: Dose-response models implemented in the MCPMod package. Column (\*) lists for

1. Equations for Target Dose  $D_{\Delta}$  to achieve a Delta ( $\Delta$ ) versus placebo

Emax:  $TD_{\Lambda} = ED_{50}/((E_{max}/\Delta) - 1)$ , where  $ED_{50}$  and  $E_{max}$  are estimated from the fitted Emax model

Exponential:  $TD_{\Delta} = \delta * \log((\Delta/E_1) + 1)$ , where  $\delta$  and  $E_1$  are estimated from the fitted exponential model

(The function TD from the DoseFinding package will be used for the above)

2. Equations for Dose (ED<sub>P</sub>) to achieve a certain proportion P of the effect of the maximum dose studied versus placebo (See DoseFinding manual page 51 where ED is 'Effective Dose')





Emax: 
$$ED_P = (P * ED_{50}*max(doses))/(ED_{50}+(1-P)*max(doses)) = (P * ED_{50}*150)/(ED_{50}+(1-P)*150)$$
  
Exponential:  $ED_P = \delta *log((P*exp(max(doses)/\delta) + 1-P)) = \delta *log((P*exp(150/\delta) + 1-P))$   
(The function ED from the DoseFinding package will be used for the above)

3. Equation for Dose (asym  $ED_{\underline{P}}$ ) to achieve a certain proportion P of the asymptotic maximum effect ( $E_{max}$ ) versus placebo

Emax: asymptotic  $ED_P = (P*ED_{50})/(1-P)$ 

Simulation-based CI will be created for each of the above quantities from the mean and covariance matrix of the model parameters, assuming multivariate normality. Therefore 10,000 samples from the multivariate distribution will be taken, and for each simulation the TD and ED estimates calculated. The 2.5% and 97.5% percentiles will then form the appropriate 95% two-sided CI.

# Statistical Analysis Plan



| Sponsor | AstraZeneca |
|---|---|
| Protocol Title: | A Randomised, Double-Blind, Placebo-Controlled, Dose-<br>Response Study of the Efficacy and Safety of MEDI7352 in<br>Subjects with Painful Diabetic Neuropathy |
| Development Phase | 2 |
| Protocol Number: | D5680C00002 |
| Premier Research PCN: | MEDU177093 |
| Document Version: | Final Version 1.1 |
| Document Date: | 31-Aug-2023 |

## Approvals

| Role | Signatures |
|-----------------|------------------------------------------------------|
| Biostatistician | Print Name: PPD Biostatistician, Premier Research |
| | Sign Name: PPD |
| | Print Name: PPD PPD Biostatistics, Premier Research |
| Peer Reviewer | Sign Name: PPD |



| Role | Signatures |
|---|---|
| | Print Name: PPD Statistical Consultant to AstraZeneca |
| AstraZeneca<br>Biostatistician | Sign Name: PPD |
| | Print Name: PPD |
| | AstraZeneca Neuroscience |
| AstraZeneca<br>Representative | Sign Name: PPD |





## **Document History**

| Version | Date | Author | Description |
|---------|-------------|--------|---------------|
| 0.1 | 27-Mar-2019 | PPD | Draft Version |
| 0.2 | 16-Apr-2021 | PPD | Draft Version |
| 0.3 | 25-Jun-2021 | PPD | Draft Version |
| 0.4 | 24-Mar-2023 | PPD | Draft Version |
| 0.5 | 21-Apr-2023 | PPD | Draft Version |
| 0.6 | 24-May-2023 | PPD | Draft Version |
| 1.0 | 12-Jul-2023 | PPD | Final Version |
| 1.1 | 31-Jul-2023 | PPD | Final Version |






## **Table of Contents**

| Approvals | 1 |
|-------------------------------------------------------|-----|
| Document History | 3 |
| Table of Contents | 4 |
| List of Tables | 6 |
| List of Figures | 6 |
| List of Abbreviations. | 7 |
| 1. Overview | 11 |
| 2. Study Objectives and Endpoints | 11 |
| 2.1. Study Objectives | 11 |
| 2.1.1. Primary Objective | 11 |
| 2.1.2. Secondary Objectives | 11 |
| 2.1.3. Exploratory Objectives | 12 |
| 2.2. Study Endpoints | .12 |
| 2.2.1. Efficacy Endpoints | 12 |
| 2.2.2. Safety Endpoints | 13 |
| 2.2.3. Pharmacokinetic/Pharmacodynamic Variable(s) | 13 |
| 2.2.4. Other Endpoints | 14 |
| 3. Overall Study Design and Plan | 14 |
| 3.1. Overall Design | 14 |
| 3.2. Sample Size and Power | 14 |
| 3.3. Study Population | 15 |
| 3.4. Treatments Administered | 16 |
| 3.5. Method of Assigning Subjects to Treatment Groups | 16 |
| 3.6. Blinding and Unblinding | 16 |
| 3.7. Schedule of Events | 17 |
| 4. Statistical Analysis and Reporting. | 17 |
| 4.1. Introduction. | 17 |
| 4.2. Interim Analysis and Data Monitoring | 18 |
| 5. Analysis Populations | 18 |
| 6. General Issues for Statistical Analysis | 19 |
| 6.1. Statistical Definitions and Algorithms | 19 |
| 6.1.1. Baseline | 19 |
| 6.1.2. Adjustments for Covariates | 19 |
| AD-ST-33.06 Effective date: 12-Nov-2020 | |



| | 6.1.3. | Multiple Comparisons | 19 |
|---|---|---|---|
| | 6.1.4. | Handling of Dropouts or Missing Data | 20 |
| | 6.1.5. | Analysis Visit Windows | 20 |
| | 6.1.6. | Pooling of Sites | 21 |
| | 6.1.7. | Efficacy Variables | 21 |
| | 6.1.8. | Derived Variables. | 23 |
| | 6.1.9. | Data Adjustments/Handling/Conventions | 24 |
| 7. | | dy Patients/Subjects and Demographics | |
| | 7.1. | Disposition of Patients/Subjects and Withdrawals | 25 |
| | 7.2. | Protocol Deviations | 26 |
| | 7.3. | Demographics and Other Baseline Characteristics | 26 |
| | 7.4. | Exposure | 27 |
| 8. | Eff | icacy Analysis | 27 |
| | 8.1. | Primary Efficacy Analysis | 27 |
| | 8.1.1. | Sensitivity Analyses of the Primary Efficacy Endpoint | 29 |
| | 8.2. | Secondary Efficacy Analysis | 29 |
| | 8.3. | Exploratory Efficacy Analysis | 30 |
| 9. | Sat | fety and Tolerability Analysis | 30 |
| | 9.1. | Adverse Events | 32 |
| | 9.1.1. | Adverse Events Leading to Discontinuation of IP | 32 |
| | 9.1.2. | Deaths and Serious Adverse Events. | 33 |
| | 9.1.3. | Drug-Induced Liver Injury | 33 |
| | 9.1.4. | Infection Risk | 33 |
| | 9.2. | COVID-19 Vaccination and Screening | 33 |
| | 9.3. | Clinical Laboratory Evaluations | 33 |
| | 9.4. | Vital Signs | 34 |
| | 9.5. | Electrocardiograms | 34 |
| | 9.6. | Physical and Neurological Examination | 35 |
| | 9.7. | Total Neuropathy Score-Nurse. | 35 |
| | 9.8. | Motor and Sensory Nerve Conduction Studies | 35 |
| | 9.9. | Strength and Deep Tendon Reflexes. | 35 |
| | 9.10. | Hypersensitivity/Anaphylactic Reactions, Injection Site or Infusion Reactions | 35 |
| | 9.11. | Prior and Concomitant Medication and Procedures | 36 |
| 10 | . Ch | anges from Planned Analysis | 37 |
| 11 | . Otl | her Planned Analysis | 37 |
| 4 17 | OT 22 C | 00 Effective date: 12 Nov. 2020 | |
| | | 06 Effective date: 12-Nov-2020 | 27: |
| Vei | rsion 1.1 | Date 31-Aug-2023 AD-PR-109.02 Effective date: 17-Aug-2020 Page 5 | ot 54 |





| 11.1. Biomarkers | 37 |
|-------------------------------------------------------------|----|
| 11.2. Immunogenicity | 38 |
| 11.3. Pharmacokinetic Analysis | 39 |
| 12. References | 39 |
| 13. Tables, Listings, and Figures | 41 |
| 13.1. Demographic Data | 41 |
| 13.2. Efficacy Data | 42 |
| 13.3. Safety Data | 43 |
| 13.4. Pharmacokinetic/Pharmacodynamic Data | 46 |
| 13.5. Planned Listing Descriptions | 46 |
| 13.6. Planned Figure Descriptions | 49 |
| 14. Tables, Listing and Figure Shells | 51 |
| 14.1. Standard Layout for all Tables, Listings, and Figures | 51 |
| 15. Appendix: Calculation of Dose to achieve target effects | 53 |
| List of Tables | |
| Table 1: Demographic Data Summary Tables and Figures | 41 |
| Table 2: Efficacy Data | 42 |
| Table 3: Safety Data | 43 |
| Table 4: Pharmacokinetic/Pharmacodynamic Data | 46 |
| Table 5: Planned Listings | 46 |
| Table 6: Planned Figures | 50 |
| List of Figures | |
| Figure 1: Standardized Lavout | 52 |





## **List of Abbreviations**

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| ADA | Anti-Drug Antibody |
| AE | Adverse Event |
| AIC | Akaike Information Criterion |
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| BOCF | Baseline Observation Carried Forward |
| CI | Confidence Interval |
| СМН | Cochran-Mantel-Haenszel |
| COVID-19 | Coronavirus Disease 2019 |
| CSR | Clinical Study Report |
| DSIS | Daily Sleep Interference Scale |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| ED50, ED90 | The Dose to achieve 50%, 90% of the Maximum Effect. |
| EMA | European Medicines Agency |

AD-ST-33.06 Effective date: 12-Nov-2020





| Abbreviation | Definition |
|--------------|---------------------------------------------------------|
| Emax | The Model-Based Maximum Treatment Effect Versus Placebo |
| ePRO | Electronic Patient-Reported Outcome System |
| FDA | Food and Drug Administration |
| gCV% | Geometric Coefficient of Variation |
| GEE | Generalized Estimating Equation |
| gmean | Geometric Mean |
| gSD | Geometric Standard Deviation |
| HL | Hy's Law |
| HR | Heart Rate |
| ICH | International Council for Harmonization |
| IP | Investigational Product |
| IV | Intravenous |
| IWRS | Interactive Web Response System |
| LLOQ | Lower Limit of Quantification |
| LOCF | Last Observation Carried Forward |
| LS | Least Squares |
| MCP-mod | Multiple Comparison Procedure Modelling |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-Treat |





| Abbreviation | Definition |
|--------------|----------------------------------------|
| MMRM | Mixed Effects Models Repeated Measures |
| NC | Not Calculable |
| NCA | Noncompartmental Analysis |
| NPS | Neuropathic Pain Scale |
| NQ | Not Quantifiable |
| NRS | Numeric Rating Scale |
| PD | Pharmacodynamics |
| PDN | Painful Diabetic Neuropathy |
| PGIC | Patient Global Impression of Change |
| CCI | |
| PHT | Potential Hy's Law |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| QTcF | QT Fridericia's Correction |
| CCI | |
| RPOA | Rapidly Progressive Osteoarthritis |
| SAE | Serious Adverse Event |
| SAF | Safety |
| SAP | Statistical Analysis Plan |





| Abbreviation | Definition |
|--------------|------------------------------------------|
| SAS® | a Software System Used for Data Analysis |
| SDTM | Study Data Tabulation Model |
| SF-36 | 36-Item Short Form Health Survey |
| SiAP | Statistical Interim Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TBL | Total Bilirubin |
| TEAE | Treatment-Emergent Adverse Event |
| tNGF | Total Nerve Growth Factor |
| TNSn | Total Neuropathy Score-Nurse |
| ULN | Upper Limit of Normal |
| ULOQ | Upper Limit of Quantification |





#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for AstraZeneca protocol number D5680C00002 (A Randomised, Double-Blind, Placebo-Controlled, Dose-Response Study of the Efficacy and Safety of MEDI7352 in Subjects with Painful Diabetic Neuropathy), dated 13-Apr-2022 version 7.0. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials (ICH, 1998). All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association (ASA, 2018) and the Royal Statistical Society (RSS, 2014), for ethical statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts.

The statistical plan described hereafter has been developed by blinded study team members prior to the Interim Analysis but after the Administrative Analysis has been conducted. It will be approved before final unblind, performing inferential or descriptive analysis of hard-locked data from AstraZeneca's study D5680C00002.

### 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

#### 2.1.1. Primary Objective

The primary objective is to assess the efficacy of MEDI7352 versus placebo on chronic pain in subjects with painful diabetic neuropathy (PDN) currently taking standard of care medication for their PDN pain.

#### 2.1.2. Secondary Objectives

The secondary objectives are:

- To assess the safety and tolerability of MEDI7352 in subjects with PDN
- To assess the pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of MEDI7352 in subjects with PDN

AD-ST-33.06 Effective date: 12-Nov-2020



 To characterise the dose-response relationship of MEDI7352 on chronic pain in subjects with PDN

#### 2.1.3. Exploratory Objectives



## 2.2. Study Endpoints

## 2.2.1. Efficacy Endpoints

#### 2.2.1.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is the change in the weekly average of the average daily pain scores from the baseline week to Week 12 of MEDI7352 compared to placebo, as measured on an 11-point (0-10) numeric rating scale (NRS).

The target population is the entire patient population, i.e., the collection of all patients eligible to be included in the randomized clinical trial based on prespecified (and duly justified) inclusion/exclusion criteria.

The study was not designed using the Estimand framework. However, the following general aspects of an Estimand can be inferred: the Estimand can be generically defined as the true between-treatment difference in the target population endpoint means for the change from baseline for the Pain NRS at Week 12, while-on-treatment and regardless of prohibited or rescue medication use.

#### 2.2.1.2. Secondary Efficacy Endpoint(s)

The secondary efficacy endpoints of this study include the following:

- Change in the weekly average of the average daily pain score, as measured on an 11-point (0-10) NRS, from baseline to Weeks 2, 4, 6, 8, and 10 of treatment and the week before the follow-up visit.
- Percentage of subjects who have achieved ≥30% and ≥50% reductions in the weekly average of the average daily pain score from baseline during Weeks 4, 8, and 12 of treatment and the week before follow-up.

AD-ST-33.06 Effective date: 12-Nov-2020



- Change in Galer Neuropathic Pain Scale (NPS) from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in Daily Sleep Interference Scale (DSIS) from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Proportion of subjects who have 'improved', 'much improved,' or 'very much improved' relative to baseline on the Patient Global Impression of Change (PGIC) on Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in the 36-item Short-Form Health Survey (SF-36) from baseline to Day 84 of treatment.
- Usage of rescue medication (yes/no) from baseline to Week 12 of treatment.

#### 2.2.1.3. Exploratory Efficacy Endpoint(s)



#### 2.2.2. Safety Endpoints

The safety endpoints of this study include the following:

- Adverse events (AEs) and serious adverse events (SAEs)
- Physical and neurological examinations
- Neuropathy assessments Total Neuropathy Score-Nurse (TNSn) S
- Strength (dorsiflexion), and deep tendon reflex (knee and ankle) assessments
- Vital signs
- 12 lead digital electrocardiogram (ECGs)
- Clinical laboratory testing (hematology, chemistry, coagulation, and immunology)
- Motor and sensory nerve conduction studies
- Concomitant medications and therapies
- Injection site reactions and infusion reactions

## 2.2.3. Pharmacokinetic/Pharmacodynamic Variable(s)

The pharmacokinetic (PK) endpoints of the study include the MEDI7352 concentrations measurements in serum/plasma.

The pharmacodynamic (PD) endpoints of the study include total nerve growth factor (tNGF) measurements in serum/plasma.

AD-ST-33.06 Effective date: 12-Nov-2020





## 2.2.4. Other Endpoints

The following endpoints will be assessed:

- Change in the weekly average of the average daily pain scores from the baseline week to Week 12, as measured on an 11-point (0-10) NRS, versus dose.
- Immunogenicity (ADA) assessments.

#### 3. Overall Study Design and Plan

This is a randomised, double-blind, placebo-controlled study of MEDI7352 in subjects with moderate to severe chronic PDN persistent for 6 months or longer, not adequately controlled by standard of care treatments, caused by type 1 or type 2 diabetes mellitus. The study incorporates a screening period of up to 45 days and a 12-week double-blind treatment period during which MEDI7352 or placebo will be administered intravenously (IV) on 6 occasions, with each dose separated by 14 days. There will be a 6-week follow-up period.

#### 3.1. Overall Design

#### 3.2. Sample Size and Power

There will be 4 stages in the study: in the first stage, subjects will be randomly assigned to placebo or the lowest dose (CCI) until at least 10 subjects have been recruited. In the second stage, up to 30 subjects will be randomly assigned to a placebo or CCI of MEDI7352; prior to commencing the third stage, the safety and tolerability experience following administration of multiple doses of CCI in the Phase 1 study of MEDI7352 will be evaluated. In stage 3 of the study, approximately 67 subjects will be randomly assigned to placebo or CCI of MEDI7352. The third stage will include an interim analysis to enable decision making for stage 4 with respect to the sample size and dose allocation ratio. If no changes are made following the interim analysis, in stage 4 of the study, approximately 165 eligible subjects will be randomly assigned to treatment across 3 dose levels of MEDI7352 (CCI) or placebo, to ensure that approximately 236 subjects are evaluable for the efficacy analysis of stages 2 to 4 combined. The number of subjects in the fourth stage is currently planned to follow an equal treatment allocation to each of the 4 treatment groups. However, the exact number of subjects and the allocation to each dose in stage 4 will be determined after the interim analysis.

There is no formal sample size calculation for stage 1; 10 subjects in stage 1 are considered sufficient for the initial assessment of safety. The sample size for stages 2-4 combined was determined by a formal power calculation (see below) and the size of stage 3 was defined to enable decision making for the stage 4 sample size and dose allocation ratio.

This study is powered at greater than 80% to detect a statistically significant (1-sided alpha = 0.025) dose-response relationship when the true Week 12 placebo-corrected change from baseline difference at the  $\boxed{\text{CCI}}$  dose is 1.25 on the 11-point NRS scale (MEDI7352-placebo treatment) and the true dose-response follows a hyperbolic Emax relationship, with ED50 within the range 1-750 µg/kg. This calculation also assumes:

AD-ST-33.06 Effective date: 12-Nov-2020



- The true standard deviation (SD) is 2.4, which is based on other studies undertaken with pregabalin in PDN (Satoh et al. 2011, Lesser et al. 2004, Rosenstock et al. 2004, Tölle et al. 2008).
- The data from stages 2, 3, and 4 are combined so that the number of subjects for the dose-response analysis is 236 with the total number evaluable for placebo, column doses equal to 81, 37, 51, and 67, respectively. This is comprised of, assuming an overall 10% non-evaluability rate:
  - o 28 out of 30 randomised in stage 2; 14 per arm
  - o 60 out of 67 randomised in stage 3; 30 per arm, and
  - o 148 out of 165 randomised in stage 4; 37 per arm
- The dose-response hypothesis test is multiplicity adjusted as described by Pinheiro et al. 2006 in order to control the type 1-error.

The above calculations were performed using the software R and the R-package 'DoseFinding' [https://cran.r-project.org/web/packages/DoseFinding/DoseFinding.pdf] with the following parameters:

- Population SD (of change from baseline to week 12) = 2.4
- Placebo effect = 1 point reduction in NRS and CCl effect = 2.25 reduction from baseline, ie, delta= 1.25
- Linear contrasts were determined from 5 'candidate dose' response models which are all E<sub>max</sub> models with decreasing potency/increasing ED50: 7.5, 15, 30, 60, 750 μg/kg. The 5<sup>th</sup> case is essentially linear in dose. E<sub>max</sub> models were chosen following the recommendations in a recent meta-analysis of dose response studies by Thomas et al., 2014.
- Power was assessed across 16 alternative true dose response curves, 12 E<sub>max</sub> with ED50 ranging from 0.375 to 750 μg/kg, 3 logistic and 1 quadratic, all having a Week 12 placebo-corrected change from baseline difference at the column dose of 1.25.

The overall withdrawal rate is anticipated to be approximately 10%. However, since the primary analysis will use Last Observation Carried Forward (LOCF) for withdrawn subjects, and the SD estimate is taken from studies which also used the LOCF approach, the only additional subjects recruited will be to account for withdrawals in stages 2, 3, and 4 if withdrawal occurs at, or prior to, the Week 2 visit.

The number of subjects who will agree to participate in the genetic research is unknown. It is therefore not possible to establish whether sufficient data will be collected to allow a formal statistical evaluation or whether only descriptive statistics will be generated.

#### 3.3. Study Population

Male or female (postmenopausal or surgically sterile) subjects aged ≥18 to ≤80 years with

AD-ST-33.06 Effective date: 12-Nov-2020





chronic PDN persistent for 6 months or longer, not adequately controlled by standard of care treatments.

#### 3.4. Treatments Administered

Once randomized, subjects will be dosed with either MEDI7352 or placebo on Day 1, Day 14, Day 28, Day 42, Day 56, and Day 70. MEDI7352 or placebo will be administered IV over a 60-minute period. To maintain the blind, a placebo volume equivalent to the MEDI7352 volume will be administered for each dosing.

#### 3.5. Method of Assigning Subjects to Treatment Groups

The randomisation schedule will be computer generated using a permuted block algorithm appropriate to the treatment groups included in each stage and will randomly allocate investigational product (IP) to randomisation numbers. The randomisation numbers will be assigned sequentially through a central interactive web response system (IWRS) as subjects are entered into the study. The randomisation schedule will not be stratified, and study centre will not be a blocking factor in the randomisation schedule.

The randomisation schedule has been prepared by Premier Research before the start of the study. No one involved in the study performance will have access to the randomisation schedule before official unblinding of treatment assignment. No subject will be randomised into this study more than once.

#### 3.6. Blinding and Unblinding

All subjects, investigators, and study personnel involved in the conduct of the study, including data management, will be blinded to treatment assignment with the exception of a specified unblinded statistician and programmer from Premier Research who will have access to the randomization code, unblinded site monitors and clinical manager from Premier Research, and the unblinded pharmacist at each study site. The unblinded study personnel will not participate in study procedures or data analysis prior to unblinding of the study data to all study related personnel. Unblinded personnel who are not otherwise involved in the study will prepare data for review and interim analysis.

Study personnel will make every effort to safeguard the integrity of the study blind to minimize bias in the conduct of the study. Treatment unblinding is discouraged if knowledge of the treatment assignment will not materially change the planned management of a medical emergency. Unblinding will be permitted in a medical emergency that requires immediate knowledge of the subject's treatment assignment.

Unblinding should be discussed in advance with the medical monitor if possible. For emergency unblinding, study personnel will use the IWRS. Only authorized users will have access to the unblinding function in the IWRS, and the IWRS will reveal the treatment information for the selected subject only. If the investigator is not able to discuss treatment unblinding in advance, then he/she must notify the medical monitor as soon as possible about the unblinding incident without revealing the subject's treatment assignment. The IWRS will also send a blinded notification to the clinical team alerting them that a break blind occurred.





The investigator or designee must record the date and reason for treatment unblinding on the appropriate electronic case report form (eCRF) for that subject. In all cases that are not emergencies, the investigator must discuss the event with the medical monitor prior to unblinding the subject's treatment assignment.

If treatment assignment is unblinded for an individual subject, study personnel will be notified of that subject's treatment assignment without unblinding the treatment assignments for the remaining subjects in the study. Thus, the overall study blind will not be compromised. If a subject's treatment assignment is unblinded, he/she will be asked to withdraw from the study. The investigator will make this decision after consultation with the medical monitor.

Overall unblinding will take place at the end of the study only after database lock has been achieved.

#### 3.7. Schedule of Events

Please see the protocol Tables 2-1, 2-2 for a detailed schedule of events.

#### 4. Statistical Analysis and Reporting

All efficacy and safety statistical analysis will be based on data from stages 1, 2, 3 and 4 combined, unless specified otherwise.

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will primarily use SAS (release 9.4 or higher). The multiple comparison and modelling (MCP-Mod) analysis will be performed using R (release 4.2.1 or higher) and the DoseFinding package (version 1.0-3 or higher). If a use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, the number of missing values, arithmetic mean, SD, median, 1<sup>st</sup>, and 3<sup>rd</sup> quartiles (where applicable), minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment group, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population with non-missing data at each visit, unless otherwise specified.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be





reported to 1 degree of precision more than the observed data and measures of spread will be reported to 2 degrees of precision more than the observed data.

For derived data, minimum and maximum will be reported to 2 degrees of precision. Measures of location (mean and median) will be reported to 3 degree of precision, and measures of spread will be reported to 4 degrees of precision.

Percentages will be presented to 1 decimal place, unless otherwise specified.

Unless otherwise indicated, all statistical tests will be conducted at the 0.025 significance level using 1-tailed tests, and *P* values will be reported. For estimation purposes, 2-sided 95% confidence intervals (CI) will be presented.

Total NGF and PK concentration data will be summarized by dose as per the quantitative variables and presenting the number (n) of non-missing observations, and the n < lower limit of quantification (LLOQ). PD and PK parameters will be summarized by dose and will include the arithmetic mean, SD, geometric mean (gmean), gmean  $\pm$  geometric SD, geometric coefficient of variation (gCV%), median, minimum and maximum.

#### 4.2. Interim Analysis and Data Monitoring

Details of the interim analysis have been included in the Statistical Interim Analysis Plan (SiAP) version 1.0 dated 10-Feb-2023.

## 5. Analysis Populations

The following analysis populations are planned for this study:

- Screening Population (Screened): All subjects who provide informed consent and/or assent and provide demographic and/or baseline screening assessments, regardless of the subject's randomisation and treatment status in the study. The Screening Set will be analysed as randomised, according to planned treatment.
- Safety Population (SAF): The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication. The Safety Set will be analysed according to actual treatment.
- Modified Intent-To-Treat Population (mITT): The modified intent-to-treat population will be used for all efficacy analyses and will include all randomised subjects who receive at least 1 dose of double-blind study medication and have at least 1 daily NRS assessment while receiving double-blind treatment. The mITT Set will be analysed as randomised, according to planned treatment.
- Pharmacokinetic Population (PK): The PK Population will include all subjects for who a PK sample was obtained and analysed. The PK Set will be analysed according to actual treatment.

Assignment of subjects to populations will be confirmed at a blinded data review meeting to be

AD-ST-33.06 Effective date: 12-Nov-2020





held before the study database is locked.

If a subject is randomised incorrectly or is administered the incorrect IP, analyses of the mITT population will be based on the IWRS-assigned treatment whereas all other analyses will be based on the actual treatment.

## 6. General Issues for Statistical Analysis

#### 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Baseline

For all safety endpoints, the last observation recorded prior to the first dose of treatment will be used as the baseline observation for calculations of change from baseline.

For pain diary data the baseline period is defined as the seven-day period prior to randomization, i.e., Day -7 to Day -1, inclusive. A subject is considered to have an evaluable baseline pain score if there are at least 4 days of recorded diary pain scores in the 7-day period.

#### **6.1.2.** Adjustments for Covariates

In addition to treatment group, the baseline value of the variable undergoing analysis and the co-medication type (Anticonvulsant versus Antidepressant) will be included in the analysis of covariance (ANCOVA) model as additive covariates. Co-medication type will be determined by blinded clinical review of each subject's medication record at baseline.

Covariates in the mixed effects models repeated measures (MMRM) and generalized estimating equations (GEE) analyses include those specified for the ANCOVA analyses, together with time and its interaction with dose group.

The crossing of co-medication type and median baseline pain score will be used as strata in the Cochran-Mantel-Haenszel (CMH) model tests. Assuming two co-medication types, the strata will be:

- 1) Anticonvulsant (Baseline NRS < Median),
- 2) Anticonvulsant (Baseline NRS > Median),
- 3) Antidepressant (Baseline NRS < Median),
- 4) Antidepressant (Baseline NRS > Median).

Where the median baseline NRS is calculated over all subjects.

#### 6.1.3. Multiple Comparisons

A multiple comparison procedure modelling approach (MCP-Mod) on LOCF data will be used for primary efficacy endpoints.

AD-ST-33.06 Effective date: 12-Nov-2020





No adjustments will be made for multiple comparisons outside the MCP-Mod approach.

## 6.1.4. Handling of Dropouts or Missing Data

For the analyses of the primary efficacy endpoints based on the mITT Population, a variety of methods will be used to deal with missing data, including:

- Primary Method: LOCF.
- Observed cases analysis.
- Baseline observation carried forward (BOCF)

Subjects with missing weekly average NRS baseline data (i.e., zero or 1-3 days of diary pain scores) will not be included in the efficacy analysis because the primary analysis is change-from-baseline. If a subject has zero or  $\leq 3$  days of diary pain data in each of the possible post-baseline seven day periods ending within the protocol definition of week 12 (day  $84 \pm 3$ ), then an imputed 'week 12 LOCF' weekly average NRS pain score will be calculated from the latest 7 'non-missing' entries of the subject's diary closest to their nominal week 12 visit (i.e., the latest 7 day period containing at least 4 NRS values), provided that this would qualify as at least 'week 2' according to the windowing outlined in Section 6.1.5. Otherwise, the week 12 LOCF weekly average NRS pain score will be set to missing.

#### 6.1.5. Analysis Visit Windows

Statistical analyses will be based on scheduled visits and windows as per Protocol Table 2-1: Schedule of Events. If an assessment falls between 2 windows, then the closest visit will be used only if an assessment result is not provided within that window. All other visits will be listed only as unscheduled visits. For presentation purposes these will be mapped to the visit prior and labeled, e.g., Unscheduled Visit 3.1, if Visit 3 was the closest date prior.

For pain diary data the following analysis periods will be defined:

• Week X<sub>i</sub>: the 7-day period ending within the protocol window Day Y<sub>i</sub>±3 where at least 4 days out of 7 have recorded diary pain scores. Where several such windows exist the one ending closest to day Y<sub>i</sub> will be selected. If there are two such windows that are equidistant from day Y<sub>i</sub>, then the one with the largest number of diary entries will take precedence. If they have the same number of entries, then the later of the two end dates will be chosen. If no such window exists, then week X<sub>i</sub> will be considered missing for the purposes of weekly average scoring.

Where:

- $X_1=2, Y_1=14$
- $X_2=4, Y_2=28$
- $X_3=6, Y_3=42$

AD-ST-33.06 Effective date: 12-Nov-2020

Version 1.1 | Date 31-Aug-2023 | AD-PR-109.02 Effective date: 17-Aug-2020




- $X_4=8, Y_4=56$
- $X_5=10, Y_5=70$
- $X_6=12, Y_6=84$
- The week before follow-up is defined as the 7-day period prior to the last day of pain diary data for subjects completing the study (i.e., entering in the Week 18) where at least 4 days out of 7 have recorded diary pain scores.

#### 6.1.6. Pooling of Sites

Analysis by investigative site will not be conducted.

## 6.1.7. Efficacy Variables

#### 6.1.7.1. Pain Numerical Rating Scale

Subjects will assess their perceived average neuropathic pain over the previous 24 hours using an 11-point NRS, with 0 representing no pain and 10 representing the worst pain imaginable. Subjects will be instructed to assess their average daily pain at approximately the same time every morning, and to record their response in a subject diary (ePRO).

#### 6.1.7.2. Neuropathic Pain Scale

Subjects will assess their neuropathic pain using the Galer NPS. The NPS includes 2 descriptors of pain, including intensity and unpleasantness, and 8 descriptors that assess specific qualities of neuropathic pain: sharp, hot, dull, cold, sensitive, itchy, deep, and surface pain. Each of these 10 dimensions has a 0 to 10 NRS in which 0 is equal to no pain and 10 equals the most intense pain. There is an additional descriptor about duration and frequency of pain, which has a 1 to 3 NRS. In which 1 = I feel a background pain all the time and occasional flare-ups (breakthrough pain) some of the time, 2 = I feel a single type of pain all the time, and 3 = I feel a single type of pain only sometimes. Other times, I am pain free.

#### 6.1.7.3. Daily Sleep Interference Scale

Subjects will assess how their neuropathic pain interferes with their sleep using the DSIS. The DSIS is an 11-point Likert scale, with 0 indicating that pain did not interfere with sleep and 10 indicating that pain completely interfered with sleep. The DSIS is completed by subjects once a day (upon awakening) to accurately capture variability in sleep interference due to pain on a daily basis, thus minimizing recall bias.

#### 6.1.7.4. Patient Global Impression of Change

Subjects will rate their overall improvement in health status using the PGIC. The PGIC consists of a 7-point scale where 1 = "very much improved" and 7 = "very much worse." Subjects will be asked the following question: "How would you rate your overall improvement with treatment

AD-ST-33.06 Effective date: 12-Nov-2020





during the clinical study?" The response options include the following:

- Very Much Improved 1
- Much Improved 2
- Minimally Improved 3
- No Change 4
- Minimally Worse 5
- Much Worse 6
- Very Much Worse 7

## 6.1.7.5. Short-Form Health Survey

The subject's health status and quality of life will be assessed using the SF-36. The SF-36 assesses 8 health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. The items use Likert-type scales with either 5 or 6 points, or 2 or 3 points. Scores will be derived by the validated built-in scoring tool. Higher SF-36 scores indicate a better state of health.

#### 6.1.7.6. Rescue Medication Use

Subjects will record all rescue medications they take for neuropathic pain in a paper diary. This will be transcribed in to the eCRF collecting usage, date and time of rescue medication, medication administered, dose, frequency and route.

Subjects will be grouped by the following for rescue medication use:

- Compliant with protocol guidance on permitted therapies
- Non-compliant with protocol guidance on permitted therapies

A review of medications will be conducted at a blinded data review meeting to be held before the study database is locked.



AD-ST-33.06 Effective date: 12-Nov-2020



#### 6.1.8. Derived Variables

- Change from baseline = value at current time point value at baseline.
- Reference End Date = Date of completion/discontinuation.
- Study duration = Reference end date date of first dose of treatment + 1
- Duration of exposure (days) = min(date of last dose of treatment + 14 days or date of death) date of first dose of treatment + 1.
- Treatment-emergent AEs (TEAEs) are defined as:
  - o AEs with onset at the time of or following the start of treatment with IP, or
  - AEs starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with IP.
- Average Baseline Pain NRS = the arithmetic average of the 'non-missing' daily pain scores within the baseline period defined in Section 6.1.1. For example, if a subject has 5 days of non-missing pain scores their average will be calculated over 5 days, not the full 7-day baseline period.
- Average Week X Pain NRS = the arithmetic average of the 'non-missing' daily pain scores within each subject's specific week X period defined in Section 6.1.5.
- Average Week 12 Pain NRS (LOCF) = the arithmetic average of the 'non-missing' daily pain scores within each subject's specific week 12 period or according to the imputed LOCF/BOCF approach defined in Section 6.1.4.
- Change from Baseline to Week X Pain NRS = for each subject 'Average Week X Pain NRS' minus 'Average Baseline Pain NRS'.
- Change from Baseline to Week 12 Pain NRS (LOCF/BOCF) = for each subject 'Average Week 12 Pain NRS (LOCF)' minus 'Average Baseline Pain NRS'.
- Galer NPS Total Score (ranges from 0 to 100): sum of Pain Intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, and Surface Pain Intensity (All in an 11-point NRS).
- Change from Baseline to Week X Galer NPS Total Score = for each subject 'Galer NPS Total Score' minus 'Baseline Galer NPS Total Score'.
- Total number of days rescue medication was used = End Date of Medication Start Date





of medication + 1. Each day on which rescue medication was used at least once is counted.

- Cumulative consumption (mg) of paracetamol rescue medication use = Total dose of rescue medication (mg) consumed during the days in which paracetamol was used.
- Average daily dose (mg) of paracetamol rescue medication use = Cumulative consumption of paracetamol rescue medication (mg) /total number of days paracetamol rescue medication was used.

#### 6.1.9. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

All P values will be displayed in four decimals and rounded using standard scientific notation (e.g., 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as <0.0001.

AEs and medical histories will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) thesaurus available at time of programming.

If partial dates of AEs occur, the convention for replacing missing dates for the purpose of TEAE is as follows: if just day is missing then the day assigned is the first day of the month or the date of first dose (if in the same month), whichever is later; if just month is missing then the month assigned is the month of the first dose, unless that results in a date prior to the first dose in which case the month after the first dose is used; and if both month and day are missing then the month assigned is the month of the first dose and the day assigned is either the first day of the month or the first dose date, whichever is later.

If partial times occur, the convention is as follows: if the missing time occurs on the day of the first dose and both the hour and minute are missing then the time assigned is the time of the first dose, otherwise if both the hour and minute are missing and the date is not the date of first dose the time assigned is 12:00; if the date is the same as the date of the first dose and only hour is missing the hour assigned is 12 or the hour of first dose, whichever is later, and if the date is the same as the date of first dose and only the minute is missing the minute assigned is 30 or the minute of first dose, whichever is later. Otherwise the hour assigned is 12 if the hour is missing and the date is not the same as the date of first dose and the minute assigned is 30 is the the date is not the same as the date of first dose.

These conventions will be applied only to AE onset dates and times with the following precaution: if the missing date and time reflect the date and time of onset of an AE, the modified date and time will be constructed to match the first documented date/time post drug administration while preserving the order in which the AE was reported in the eCRF.

In general, for quantitative laboratory values reported as ' $\leq$ X' or ' $\leq$ X', the LLOQ will be used

AD-ST-33.06 Effective date: 12-Nov-2020





for analysis (i.e., the value of X will be used in the analysis for lab values reported as '<X' or ' $\le$ X'). Similarly, for quantitative laboratory values reported as '>X' or ' $\ge$ X', the upper limit of quantification (ULOQ) will be used for analysis (i.e., the value of X will be used in the analysis for lab values reported as '>X' or ' $\ge$ X').

For analysis purposes, repeat laboratory test results will not be used unless the original laboratory value is missing or indicated as invalid, in which case the first non-missing repeated laboratory value will be used for data analysis.

ADA titre reported as <30 (below the minimum required dilution) is a negative result for the presence of ADA.

For descriptive statistics of serum concentration summaries:

- At a time-point where less than or equal to 50% of the values are not quantifiable (NQ, below LLOQ), all NQ values will be set to the LLOQ, and all descriptive statistics will be calculated accordingly.
- If more than 50%, but not all, of the concentrations are NQ, the geometric mean, geometric mean ± geometric SD and gCV% will be reported as not calculable (NC). The maximum value is reported from the individual data, and the minimum and median are set as NO.
- If all concentrations are NQ at a time-point, the geometric mean, minimum, median and maximum are reported as NQ and the gCV% and geometric mean ± geometric SD as NC.

#### 7. Study Patients/Subjects and Demographics

#### 7.1. Disposition of Patients/Subjects and Withdrawals

The total number of subjects for each of the following analysis populations will be presented for the Screening Population by randomized treatment group and overall:

- Screening Population
- Safety Population
- mITT Population
- Included in the mITT population
  - Evaluable Week 12 efficacy
  - Evaluable LOCF efficacy
- Not efficacy evaluable
- PK Population

For the Screening Population, disposition will include tabulation of:

- the number of screened subjects
- the number of re-screened subjects
- the number of enrolled subjects

The output will be further presented by treatment group and overall summarising:

AD-ST-33.06 Effective date: 12-Nov-2020





- the number of randomized subjects
- the number of subjects who completed study treatment
- the number of completed subjects
- the number of subjects withdrawing (discontinued)
- the reasons for discontinuation from study treatment and withdrawal from the study.

For all categories of subjects by treatment group, percentages will be calculated using the number of subjects randomized as the denominator.

#### 7.2. Protocol Deviations

Major protocol deviations, as determined by a Sponsor blinded review of the data prior to database lock and unblinding of the study will be reported in listings.

The Sponsor or designee will be responsible for producing the final deviation file. This file will be finalized prior to database lock, and all information will be included in the SDTM.DV domain (deviations domain).

All protocol deviations will be presented in a data listing, with a flag to indicate if a deviation was considered major.

A summary table by treatment group and overall will be generated based on protocol deviation severity (minor/major) and the classification of protocol using the following categories:

- Inclusion
- o Exclusion
- Study drug
- Assessment safety
- Assessment– efficacy
- Lab/endpoint data
- Visit window
- Informed consent
- o Prohibited co-medication
- o Overdose/misuse
- o Other

#### 7.3. Demographics and Other Baseline Characteristics

Descriptive summaries of the demographic and other baseline characteristics will be presented for all analysis populations. All demographic and baseline characteristics will be presented both overall and by treatment group.

The following demographic and baseline data will be presented in tables:

AD-ST-33.06 Effective date: 12-Nov-2020





- Demographics: age, gender, ethnicity, race, height, weight, and body mass index (BMI)
- For female the number and percentage of women surgically sterile and postmenopausal will be described.
- Diagnosis of osteoarthritis: number of subjects with osteoarthritis diagnosis and area affected, clinical significance, radiological investigations, radiological significance, Kellgren-Lawrence score.

The number and percent of subjects reporting various medical histories, grouped by MedDRA system organ class (SOC) and preferred term (PT), will be tabulated by treatment group.

This analysis will be conducted for the Safety Population.

## 7.4. Exposure

The following parameters of study drug exposure and compliance will be summarized by treatment group for the Safety Population:

- Maximum number of doses administered
- Total duration of exposure
- Total (cumulative) dose infused

In addition, any incomplete infusions will be listed.

#### 8. Efficacy Analysis

All efficacy variables will be summarized descriptively including number of observations, number of missing values, mean, SD, minimum, median, and maximum for continuous variables, and frequency of observations in each category and percentage for categorical variables.

Primary and secondary endpoint efficacy data will be tabulated according to the observed cases, LOCF, and BOCF approaches.

#### 8.1. Primary Efficacy Analysis

The primary efficacy endpoint of this study is the change in the weekly average of the average daily pain scores from the baseline week to Week 12 measured on an 11-point (0-10) NRS.

MCP-Mod approach. The main statistical analysis of the primary efficacy endpoint will use the MCP-Mod approach on LOCF data, which is a well-established statistical methodology for establishing both the existence of a dose response and modelling the underlying dose-response relationship. The modelling step ('MOD' step) from the MCP-MOD approach will only be conducted if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

There are two steps to MCP-Mod:

AD-ST-33.06 Effective date: 12-Nov-2020





- 1. The 'MCP' step is a rigorous method to establish presence of a dose response while protecting the type I error and, if the dose-response relationship is statistically significant, then
- 2. The 'MOD' step estimates the dose response function and associated model parameters.

The MCP test will use linear contrasts corresponding to the five candidate models described in Section 3.2. The test will use pre-specified model parameters and optimal contrasts for each will be generated. The hypotheses are as follows:

Null hypothesis (H<sub>0</sub>): Optimal contrasts  $\mu \ge 0$  for all models

Alternative hypothesis (H<sub>A</sub>): Optimal contrasts  $\mu$  <0 for at least one model

where  $\mu$  is the true event rate.

The underlying model will be an ANCOVA with dependent variable 'change from baseline to Week 12 (LOCF)', and independent variables will include:

- dose group as a factor variable with the placebo group as the reference level
- baseline score, i.e. baseline weekly average pain (NRS), as a continuous variable
- co-medication type.

The random error is assumed to be normally and independently distributed with constant variance. The parameter estimates of the difference between each dose group and placebo, least square (LS) Means estimates of change from baseline to Week 12 for each dose, standard errors, 95% unadjusted, 'Lalonde-type' asymmetric CI (i.e., lower limit of 1-sided 90% CI and upper limit of 1-sided 80% CI), and *P* values will be presented.

If the MCP test is statistically significant, then the MOD step will select the most appropriate model from hyperbolic  $E_{max}$ , sigmoidal  $E_{max}$  or linear using the ' $E_{maxlin}$ ' approach as described by Kirby et al (2011). From this model (including the same covariates as the ANCOVA model), various estimates will be derived (together with CI) of parameters of interest such as ED50, effective dose to achieve 90% of maximum effect (ED90), dose to achieve selected target effects, and model estimates of the treatment effect at doses studied (see Appendix in Section 15).

**MMRM:** In addition, changes from baseline in continuous endpoints will be compared between treatment groups using mixed models repeated measures including terms for:

- co-medication type (as a factor)
- treatment (as a factor)
- time (as a factor)
- the interaction between treatment and time point
- and the baseline value of the variable undergoing analysis

The mixed model for repeated measure will use average of average daily pain score of observed data at week 2, 4, 6, 8, 10, and 12. An unstructured covariance matrix will be used to model the

AD-ST-33.06 Effective date: 12-Nov-2020





within-subject errors. The Kenwards-Roger method will be used to estimate degrees of freedom. If this analysis fails to converge, a simpler structure (e.g., first-order ante-dependent or heterogeneous compound symmetry structures) will be found using Akaike information criterion (AIC).

The results will be presented using LS Means estimates, corresponding 95% CI for each treatment group and timepoint, along with the LS Means of differences with Placebo, standard error, 95% CI and p-values.

The primary efficacy analysis will be based on the mITT population.

## 8.1.1. Sensitivity Analyses of the Primary Efficacy Endpoint

To complement the MCP-MOD outputs, estimates and CI of each pairwise comparison versus placebo from the ANCOVA model described in the MCP step will be produced.

#### 8.2. Secondary Efficacy Analysis

The MMRM model outlined in Section 8.1 will be applied for secondary endpoints using observed cases:

- Change in Galer NPS total score from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in DSIS from baseline to Days 28, 56, and 84 of treatment and the follow-up visit.
- Change in the eight SF-36 parameters from baseline to Day 84 of treatment.

A GEE approach for binary data will be used for the following dichotomous endpoints:

- Percentage of subjects who have achieved ≥30% reductions in the weekly average of the average daily pain score from baseline during Weeks 4, 8, and 12 of treatment and the week before follow-up.
- Percentage of subjects who have achieved ≥50% reductions in the weekly average of the average daily pain score from baseline during Weeks 4, 8, and 12 of treatment and the week before follow-up.

The GEE model specification will include a binomial distribution, a logit link function, and an unstructured covariance matrix. If this analysis fails to converge, a simpler structure (e.g. first-order autoregressive or compound symmetry structures) will be found using AIC. The model will include terms for:

- co-medication type (as a factor)
- treatment (as a factor)
- time (as a factor)
- the interaction between treatment and time





A CMH test stratified by the crossing of co-medication subgroup and median baseline pain score will also be carried out for the above dichotomous endpoints. The CMH risk difference at Week 12 will be estimated between the treatment group and placebo. The number and percentage of subjects meeting the reduction response will be displayed, along with the risk difference, 95% CI and *P* value.

The proportion of subjects who have 'improved', 'much improved,' or 'very much improved' relative to baseline on the PGIC on Days 28, 56, and 84 of treatment and the follow-up visit will be tested using a CMH statistics.

The efficacy analysis of secondary endpoints will be based on the observed cases and on the mITT population.

Usage of rescue medication (yes/no) will be summarized by dose group for each visit from baseline to Week 12 of treatment and over the whole treatment period. The following additional variables will be derived and summarised:

- Total number of days rescue medication was used.
  - Each day on which rescue medication was used at least once is counted.
- Cumulative consumption (mg) of paracetamol rescue medication use.
  - Calculated as the total dose of rescue medication (mg).
- Average daily dose (mg) of paracetamol rescue medication use.
  - Calculated as: cumulative consumption of rescue medication (mg)/total number of days rescue medication was used.

#### 8.3. Exploratory Efficacy Analysis



#### 9. Safety and Tolerability Analysis

All safety analyses will be performed on the Safety Population using descriptive statistics. Descriptive summaries by treatment group and overall will be produced. No inferential statistical tests will be performed.

AD-ST-33.06 Effective date: 12-Nov-2020





The analysis of safety assessments in this study will include summaries of the following categories of safety and tolerability data collected for each patient:

- Adverse events
  - o TEAEs
  - o SAEs
  - Significant AEs
    - TEAEs leading to discontinuation of IP
  - AEs of Special Interest
    - Positively-adjudicated possible or probable rapidly progressive osteoarthritis (RPOA), subchondral insufficiency fractures, primary osteonecrosis, or pathological fracture
    - Infections that meet SAE and/or severe AE criteria
    - Anaphylactic reactions or infusion-related reactions that lead to permanent discontinuation of administration of IP
  - o TEAEs associated with abnormal liver
  - o Any deaths
  - o Drug induced liver injury

Clinical laboratory investigations

- Vital signs
- Electrocardiograms (ECG)
- COVID-19 screening
- Physical and neurological examination
- Total neuropathy score-nurse
- Motor and sensory nerve conduction studies
- Strength and deep tendon reflexes
- Hypersensitivity /Anaphylactic reactions
- Injection site or infusion reactions
- Liver diagnostic investigations, risk factors, signs and symptoms.
- Infection diagnostic investigations, risk factors, signs and symptoms.
- Prior and concomitant medications and therapies





#### 9.1. Adverse Events

A summary table by treatment group will present the number and percent of subjects reporting:

- Any AEs
- Non-serious AEs occurring in more than 5% of subjects
- Any TEAEs
- Any SAEs
- Any TEAEs possibley related to study drug
- Any TEAEs leading to discontinuation of IP
- Any SAEs possibley related to study drug
- Life-threatenings SAEs
- SAEs resulting in death

Summaries of the incidence of TEAEs will be displayed by treatment group, by ADA status, by severity and by:

- SOC and PT
- SOC, PT, and maximum severity (mild, moderate, severe)
- SOC, PT, and maximum causality (not related, possibly related) to the study drug

In the summaries showing severity and relationship to study drug the event with the maximum severity or strongest relationship will be reported. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = related).

In the case of multiple occurrences of the same AE within the same subject, each subject will only be counted once for each level of summarization.

All AEs will be presented in a by-treatment and by-subject listing, detailing the verbatim term given by the Investigator, the PT, SOC, onset date and time, end date and time, severity, outcome, relationship to study drug, action taken with study drug, other action taken, seriousness, and criteria for seriousness.

#### 9.1.1. Adverse Events Leading to Discontinuation of IP

A summary of incidence rates (frequencies and percentages) of TEAEs leading to discontinuation of IP, by treatment group, SOC, and PT will be prepared. The table will also be produced separately by maximum severity and maximum causality.




A data listing of TEAEs leading to discontinuation of IP will also be provided, displaying details of the event(s) captured on the rCRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study and serious adverse events will be listed.

A summary of incidence rates (frequencies and percentages) of SAEs by treatment group, SOC, and PT will be prepared. The table will also be produced separately for life-threatening SAEs, for SAEs with outcome death and for SAEs by relationship to study medication.

#### 9.1.3. Drug-Induced Liver Injury

A summary of incidence rates of TEAEs associated with abnormal liver by treatment group, SOC, and PT will be prepared.

The type and the results of the liver diagnostic investigation performed will be tabulated by treatment group.

The number and percentage of subjects within each type of liver risk factors and style events will be tabulated by treatment group. Liver signs and symptoms will be presented in the same way.

#### 9.1.4. Infection Risk

A summary of incidence rates of infections that meet SAE or severe AE criteria by treatment group, SOC, and PT will be prepared.

The type and the results of infection diagnostic investigation performed will be tabulated by treatment group.

The number and percentage of subjects within each type of infection risk factors and style events will be tabulated by treatment group. Infection signs and symptoms will be presented in the same way.

#### 9.2. COVID-19 Vaccination and Screening

The number and percentage of fully vaccinated subjects at baseline will be summarized by treatment group.

The symptoms, tests, and results from coronavirus disease 2019 (COVID-19) screening will be tabulated for each visit by treatment group.

COVID-19 vaccination, signs, symptoms and impact will be presented in listings.

#### 9.3. Clinical Laboratory Evaluations

Absolute values and changes from baseline will be summarized using descriptive statistics by

AD-ST-33.06 Effective date: 12-Nov-2020

Version 1.1 | Date 31-Aug-2023 | AD-PR-109.02 Effective date: 17-Aug-2020 P





treatment group and visit for chemistry, hematology, coagulation, and urinalysis tests.

The number of subjects with clinical laboratory values (chemistry, hematology, coagulation, and urinalysis) categorized as below, within, or above normal ranges (or as either normal or abnormal for urinalysis variables that do not have quantitative ranges) and whether they are clinically significant or not will be tabulated for each clinical laboratory analyte by treatment group and visit. A shift table showing change from baseline in range categories for each clinical laboratory analyte will be produced by treatment group and by visit.

The number of subjects with values for Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)  $\geq 3 \times \text{upper limit of normal (ULN)}$ , and with values for total bilirubin (TBL)  $\geq 2 \times \text{ULN}$  will be summarized in AST, ALT vs. TBL shift tables to identify Potential Hy's Law (PHL) and Hy's Law (HL) cases by treatment group.

Diagnostic immunology, urine pregnancy, and urine drug tests will be presented in by-subject listings only.

All laboratory values will be displayed in the data listings and those that are outside the normal range will be flagged, along with corresponding normal ranges.

#### 9.4. Vital Signs

Descriptive summaries of actual values and changes from baseline by treatment group, visit and time point will be presented for:

- Supine heart rate
- Supine systolic blood pressure
- Supine diastolic blood pressure
- Respiratory rate
- Body temperature
- Standing heart rate
- Standing systolic blood pressure
- Standing diastolic blood pressure

Height, weight, and BMI will be presented at baseline only.

#### 9.5. Electrocardiograms

The number and percentage of subjects with normal, abnormal not clinically significant, and abnormal clinically significant ECG results will be summarized by treatment group and by visit.

If applicable (digital ECGs), descriptive summaries will be presented by treatment group, visit and time point (for Day 1 only) for ECG measures of PR, QRS, QT, RR intervals and for the calculated variables QTcF and HR for each treatment group and time point.

Heart rate (HR) and Fridericia's correction (QTcF) will be derived as follows:

AD-ST-33.06 Effective date: 12-Nov-2020






Heart Rate (HR) 
$$HR = 10^{3} \frac{60}{RR_{msec}}$$
Fridericia's Correction 
$$QTc_{f} = \frac{QT_{msec}}{\sqrt[3]{RR}}$$
(QTcF)

## 9.6. Physical and Neurological Examination

The physical and neurological examination findings will be presented in listings.

#### 9.7. Total Neuropathy Score-Nurse

Descriptive summaries of the TNSn will be presented by treatment groups and by visit. Additionally, the number and percentage of subjects within each category (0, 1, 2, 3, and 4) for each sub-score (sensory symptom, motor symptom, autonomic symptom, pin sensibility, vibration sensibility) will be summarized by treatment group and by visit.

#### 9.8. Motor and Sensory Nerve Conduction Studies

Amplitude, peak latency, conduction velocity, and duration of nerve action potentials will be summarized by treatment group and visit for each location and evaluation type. The number of subjects with normal and abnormal evaluation will be tabulated by treatment group and by visit.

#### 9.9. Strength and Deep Tendon Reflexes

The number and percentage of subjects within each category of the ankle dorsiflexion strength and the deep tendon reflexes will be tabulated by treatment group and by visit.

#### 9.10. Hypersensitivity/Anaphylactic Reactions, Injection Site or Infusion Reactions

The type and symptoms of hypersensitivity/ anaphylactic reactions will be tabulated by treatment group.

Injection site reactions will be tabulated describing the severity of pain, tenderness, erythema/redness, and induration/swelling by treatment group and by visit.

Anaphylactic reactions and infusion related reactions will be summarized in line with AEs, displayed by treatment group and by:

- SOC and PT
- SOC, PT, and maximum severity (mild, moderate, severe)

Hypersensitivity/anaphylactic and infusion related reactions will also be presented in a by-

AD-ST-33.06 Effective date: 12-Nov-2020






treatment and by-subject listings, detailing type of reaction, severity grade for symptom with highest severity and onset time for hypersensitivity/anaphylactic reactions, and assessment result for injection site or infusion related reactions.

#### 9.11. Prior and Concomitant Medication and Procedures

Prior medications will be presented separately from concomitant medications.

Medications will be coded using the latest version of the WHO Drug Dictionary.

Medications that started before first dose of study medication will be considered prior, whether they were stopped before first dose of study medication or not.

A concomitant medication is defined as any medication continuing or starting after first dose of study medication. This includes medications which start before first dose of study medication and continue while on-treatment, and medications that started after first dose of study medication.

The frequency and percentage of concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) class 2 and preferred name by treatment groups, unless otherwise specified.

In listings, all medications will be displayed.

If the start/stop dates of a medication are partially or completely missing, then the medication will be assumed to be concomitant if it cannot be definitely shown from the start/stop dates that it was not administered while on-treatment (from first exposure to treatment till last dose of study medication + 14 exposure days). Missing dates will not be replaced.

Thus, the following approach will be taken for exclusion from concomitant medications because of discontinuation before start of treatment:

- If the stop day is missing but the month is complete, then the medication will be excluded from concomitant medications only if the stop month is before the month of the first dose of study medication.
- If the stop day and month are missing but the year is complete, then the medication will be excluded from concomitant medications only if the stop year is before the year of the first dose of study medication.
- If the stop date is completely missing, then the medication will not be excluded.

For concomitant medication exclusion (because of the late start after the end of the treatment period):

• If the start day is missing but the month is complete, then the medication will be excluded from concomitant medications only if the start month is after the last month of the treatment period.





- If the start day and month are missing but the year is complete, then the medication will be excluded from concomitant medications only if the start year is after the year of the treatment period.
- If the start date is completely missing, then the medication will not be excluded.

A similar approach will be used for summarizing concomitant procedures.

#### 10. Changes from Planned Analysis



The PK endpoints involving derivation of PK parameters for each dose and for each subject will be conducted by a population PK analysis of the data as part of a pooled data analysis instead of by a noncompartmental analysis (NCA). This will be documented in the CSR as a change in planned analysis. The pooled data analysis will be described in a separate modelling analysis plan. As a result, description of TLFs related to PK parameters are removed from this SAP.

Additional analyses with pooled site as a covariate are not going to be conducted and as such, they are removed from this SAP.

It was planned to have a supplementary analysis to the primary using an adaptive MCP-MOD method. In this analysis, stages 2+3 and stage 4 were going to be analysed separately and the results combined using an inverse-normal *P* value combination function (with weights related to the original planned sample sizes). This supplementary analysis is removed from this SAP.

The Cochran-Mantel-Haenszel test for the non-binary categorical endpoints has been extended to include the secondary endpoint of pain response.

The definition of TEAE from the protocol has been changed in this SAP, eliminating the condition for the AE onset not being more than 30 days after the last administration of IP to be regarded as a TEAE. The change in the definition of TEAE has been made upon Sponsor request, to enable transparency, adequate safety reporting and oversight of safety profile/risks.

## 11. Other Planned Analysis

#### 11.1. **CC**



AD-ST-33.06 Effective date: 12-Nov-2020






| CCI |
|-----|
| CCI |
| COI |

#### 11.2. Immunogenicity

Blood samples will be collected for assessment of ADA levels. Anti-Drug Antibody response during the entire study period and at each study assessment will be summarised according to ADA category and titre value for the Safety population with evaluable ADA results. A listing of the ADA test results will be produced.

For immunogenicity analysis, the presence of detectable (i.e., positive) ADAs against MEDI7352 will be reported. ADA results from each sample are reported as either positive or negative. In addition, the ADA titer result will be reported for samples confirmed positive for the presence of ADAs. A participant is defined as being ADA-positive if a positive ADA result is available at any time, including baseline and all post-baseline measurements, otherwise ADA negative.

The following ADA categories will be determined:

- ADA positive if a collected sample is tested positive at any time during the study, including baseline and/or post-baseline. (The percentage of these participants in a population is known as ADA prevalence).
- Treatment-emergent ADA positive (TE-ADA+): A positive post-baseline result and either of the following statements holds:
  - Baseline is ADA negative and at least one post-baseline assessment is ADA positive. This is called treatment-induced ADA positive.
  - o Baseline is ADA positive, and the baseline titre is boosted by greater than the variability of the assay (i.e., ≥X-fold increase, commonly 4-fold) at ≥1 post-baseline timepoint. This is called treatment-boosted ADA positive.

(The percentage of these participants in a population is known as ADA incidence)

- Only baseline positive if a collected sample is tested positive at baseline.
- Non-Treatment-emergent ADA positive (non-TE-ADA+): Participants who are ADA positive but not fulfilling the conditions for TE-ADA+.
- Treatment-emergent Persistently ADA positive: ADA negative at baseline and having at least 2 post-baseline ADA positive measurements with ≥16 weeks (112 days) between first and last positive, or an ADA positive result at the last available post-baseline assessment.
- Treatment-emergent Transiently ADA positive: ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive





• ADA positive post-baseline and positive at baseline.

## 11.3. Pharmacokinetic Analysis

Pharmacokinetic concentration data will be summarized using descriptive statistics by dose and treatment visit overall and by ADA status (positive/negative) presenting the number (n) of non-missing observations, and the n < LLOQ. A figure of geometric mean (with and without gSD) serum MEDI7352 concentration over time by treatment group will be generated (overall and by ADA status (positive/negative)). Additionally, pharmacokinetic concentration data will be listed and presented graphically as spaghetti plots of individual participant profiles by treatment group and ADA status (positive/negative).

#### 12. References

- 1. ICH (1998) ICH Harmonised Tripartite Guideline. Statistical Principles for Clinical Trials E9; 1998. https://database.ich.org/sites/default/files/E9\_Guideline.pdf
- 2. ASA. (2018) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2018. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 4. Satoh J, Yagihashi S, Baba M, Suzuki M, Arakawa A, Yoshiyama T. Efficacy and safety evaluation of pregabalin treatment over 52 weeks in patients with diabetic neuropathic pain extended after a double-blind placebo-controlled trial. *J Diabetes Investig*. 2011;2(6):457-463. Doi: 10.1111/j.2040-1124.2011.00122.x.
- 5. Lesser H, Sharma U, LaMoreaux L, Poole RM. Pregabalin relieves symptoms of painful diabetic neuropathy: a randomized controlled trial. *Neurology*. 2004;63(11):2104-2110.
- 6. Rosenstock J, Tuchman M, LaMoreaux L, Sharma U. Pregabalin for the treatment of painful diabetic peripheral neuropathy: a double-blind, placebo-controlled trial. *Pain*. 2004;110(3):628-638.
- 7. Tölle T, Freynhagen R, Versavel M, Trostmann U, Young JP Jr. Pregabalin for relief of neuropathic pain associated with diabetic neuropathy: a randomized, double-blind study. *Eur J Pain*. 2008;12(2):203-213.
- 8. Pinheiro J, Bornkamp B, Bretz F. Design and analysis of dose-finding studies combining multiple comparisons and modelling procedures. *J Biopharm Stat.* 2006;16(5):639-656. Doi: 10.1080/10543400600860428.
- 9. Thomas N, Sweeney K, Somayaji V. Meta-analysis of clinical dose–response in a large drug development portfolio. *Stat Biopharm Res.* 2014;6(4):302-317. Doi: 10.1080/19466315.2014.924876.





10. Kirby S, Brain P, Jones B. Fitting E(max) models to clinical trial dose-response data. Pharma Stat. 2011;10(2):143-149. Doi: 10.1002/pst.432.





## 13. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (eCRF page or listing number).

The following are planned summary tables for protocol number D5680C00002. The table numbers and page numbers are place holders only and will be determined when the tables are produced.

#### 13.1. Demographic Data

Table 1: Demographic Data Summary Tables and Figures

| Table Number | Population | Table Title/Summary |
|---|---|---|
| Table 14.1.2 | Screening | Subject Disposition |
| Table 14.1.3 | Screen Failure | Summary of Reasons for Screening Failure |
| Table 14.1.4.1 | Screening | Demographics and Baseline Characteristics |
| Table 14.1.4.2 | Safety | Demographics and Baseline Characteristics |
| Table 14.1.4.3 | mITT | Demographics and Baseline Characteristics |
| Table 14.1.4.4 | PK | Demographics and Baseline Characteristics |
| Table 14.1.5.1 | Screening | Osteoarthritis Characteristics |
| Table 14.1.5.2 | Safety | Osteoarthritis Characteristics |
| Table 14.1.5.3 | mITT | Osteoarthritis Characteristics |
| Table 14.1.5.4 | PK | Osteoarthritis Characteristics |
| Table 14.1.6 | Safety | Medical History by System Organ Class and Preferred Term |
| Table 14.1.7 | Safety | Prior Medications by ATC Class and Preferred Name |
| Table 14.1.8 | Safety | Protocol Deviations |
| Table 14.1.9 | Safety | Overall Study Drug Exposure |

117 of 762

AD-ST-33.06 Effective date: 12-Nov-2020




# 13.2. Efficacy Data

**Table 2: Efficacy Data** 

| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.2.1.1.1 | mITT | Daily Pain NRS: Summary Statistics (Observed Cases) |
| Table 14.2.1.1.2 | mITT | Daily Pain NRS: Summary Statistics (LOCF) |
| Table 14.2.1.1.3 | mITT | Daily Pain NRS: Summary Statistics (BOCF) |
| Table 14.2.1.2.1 | mITT | Daily Pain NRS: Primary MCP-Mod Analysis (LOCF) |
| Table 14.2.1.2.2 | mITT | Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) |
| Table 14.2.1.3.1 | mITT | Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) |
| Table 14.2.1.3.2 | mITT | Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) |
| Table 14.2.2.1 | mITT | Galer NPS: Summary Statistics (Observed Cases) |
| Table 14.2.2.2 | mITT | Galer NPS: MMRM Analysis (Observed Cases) |
| Table 14.2.3.1 | mITT | DSIS: Summary Statistics (Observed Cases) |
| Table 14.2.3.2 | mITT | DSIS: MMRM Analysis (Observed Cases) |
| Table 14.2.4.1 | mITT | SF-36: Summary Statistics (Observed Cases) |
| Table 14.2.4.2 | mITT | SF-36: MMRM Analysis (Observed Cases) |
| Table 14.2.5.1 | mITT | Rescue Medication Use: Summary Statistics |
| Table 14.2.6.1 | mITT | Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel-Haenszel (Observed Cases) |
| Table 14.2.6.2 | mITT | Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) |
| Table 14.2.7.1 | mITT | Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel-Haenszel (Observed Cases) |
| Table 14.2.7.2 | mITT | Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) |
| Table 14.2.8.1 | mITT | Patient Global Impression of Change: Summary Statistics |
| Table 14.2.8.2 | mITT | Patient Global Impression of Change: Cochran-Mantel-Haenszel |
| CCI | | |

AD-ST-33.06 Effective date: 12-Nov-2020






# 13.3. Safety Data

**Table 3: Safety Data** 

| Table Number | Population | Table Title / Summary |
|---|---|---|
| 14.3.1 Displays of Adverse Events | | |
| Table 14.3.1.1 | Safety | Summary of Overall Adverse Events |
| Table 14.3.1.2 | Safety | Treatment Emergent Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.1.3 | Safety | Treatment Emergent Adverse Events by Severity, System Organ Class and Preferred Term |
| Table 14.3.1.4 | Safety | Treatment Emergent Adverse Events by Relationship to Study<br>Medication, System Organ Class and Preferred Term |
| Table 14.3.1.5 | Safety | Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term |
| Table 14.3.1.6 | Safety | Treatment Emergent Adverse Events Leading to Discontinuation of Study drug by System Organ Class and Preferred Term |
| Table 14.3.1.7 | Safety | Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term |
| Table 14.3.1.8 | Safety | Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term |
| Table 14.3.1.9 | Safety | Treatment Emergent Adverse Events by Preferred Term |
| 14.3.2 Summary | of Deaths, Other Se | erious and Significant Adverse Events |
| Table 14.3.2.1.1 | Safety | Serious Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.2.1.2 | Safety | Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.2.1.3 | Safety | Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term |
| Table 14.3.2.1.4 | Safety | Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term |
| 14.3.2.2 Displays of Significant Adverse Events and Adverse Events of Special Interest | | |
| Table 14.3.2.2.1 | Safety | Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term |
| Table 14.3.2.2.2 | Safety | Potential Joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term |
| Table 14.3.2.2.3 | Safety | Serious and/or severe Infections by System Organ Class and Preferred Term |

AD-ST-33.06 Effective date: 12-Nov-2020




| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.3.2.2.4 | Safety | Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions<br>Leading to Discontinuation of IP by System Organ Class and Preferred<br>Term |
| 14.3.3 Narrative | es of Deaths and Oth | ner Serious Adverse Events |
| Table 14.3.3.1 | Safety | Listing of Serious Adverse Events |
| Table 14.3.3.2 | Safety | Listing of Deaths |
| 14.3.4 Laborato | ry Data Summary | Γables |
| Table 14.3.4.1 | Safety | Descriptive Summary of Clinical Chemistry |
| Table 14.3.4.2 | Safety | Shift Table of Clinical Chemistry Results |
| Table 14.3.4.3 | Safety | Descriptive Summary of Hematology |
| Table 14.3.4.4 | Safety | Shift Table of Hematology Results |
| Table 14.3.4.5 | Safety | Descriptive Summary of Coagulation |
| Table 14.3.4.6 | Safety | Shift Table of Coagulation Results |
| Table 14.3.4.7 | Safety | Descriptive Summary of Urinalysis |
| Table 14.3.4.8 | Safety | Shift Table of Urinalysis Results |
| Table 14.3.4.9 | Safety | Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin |
| 14.3.6 Other Safety Data Summary Tables | | |
| Table 14.3.5.1 | Safety | Descriptive Summary of Vital Signs |
| Table 14.3.5.2 | Safety | Descriptive Summary of ECG Digital Data |
| Table 14.3.5.3 | Safety | Summary of Overall Evaluation of Safety ECG Data |
| Table 14.3.5.4 | Safety | Covid-19 Screening |
| Table 14.3.5.5 | Safety | Summary of Sub-Scores for Total Neuropathy Score-Nurse |
| Table 14.3.5.6 | Safety | Descriptive Summary of Total Neuropathy Score-Nurse |
| Table 14.3.5.7 | Safety | Summary of Motor and Sensory Nerve Conduction Studies |
| Table 14.3.5.8 | Safety | Summary of Strength and Deep Tendon Reflexes |
| Table 14.3.5.9 | Safety | Summary of Local Injection Site Reactions |
| Table 14.3.5.10 | Safety | Summary of Anaphylactic Reactions |
| Table 14.3.5.11 | Safety | Summary of Liver Diagnostic Investigations |
| Table 14.3.5.12 | Safety | Summary of Liver Risk Factors and Lifestyle Events |
| Table 14.3.5.13 | Safety | Summary of Liver Signs and Symptoms |

AD-ST-33.06 Effective date: 12-Nov-2020






| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.3.5.14 | Safety | Summary of Infection Diagnostic Investigations |
| Table 14.3.5.15 | Safety | Summary of Infection Risk Factors and Lifestyle Events |
| Table 14.3.5.16 | Safety | Summary of Infection Signs and Symptoms |
| Table 14.3.5.17 | Safety | Summary of Concomitant Medications by ATC Level 2 and Preferred Term |
| Table 14.3.5.18 | Safety | Summary of Concomitant Procedures |
| Table 14.3.5.19 | Safety | Anti-Drug Antibody Results and Titre Summary by Timepoint |
| Table 14.3.5.20 | Safety | Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories |



## 13.4. Pharmacokinetic/Pharmacodynamic Data

Table 4: Pharmacokinetic/Pharmacodynamic Data

| <b>Table Number</b> | Population | Table Title / Summary |
|---|---|---|
| 14.4 Pharmacokinetic and Pharmacodynamic Data Summary Tables | | |
| Table 14.4.1 PK Summary of Serum MEDI7352 Concentrations | | |
| Table 14.4.2 | Safety | Summary of Serum total NGF Concentrations |

#### 13.5. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number D5680C00002.

In general, one listing will be produced per eCRF domain. All listings will be sorted by treatment, site, and subject number. All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 5: Planned Listings** 

| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data Listi | 16.2 Subject Data Listings | |
| 16.2.1 Subject Disconti | nuations/Completio | ons |
| Listing 16.2.1.1 | Screening | Subject Disposition |
| Listing 16.2.1.2 | Screening | Assignment to Analysis Populations |
| Listing 16.2.1.3 | Safety | Reason for IP Discontinuation and Withdrawal from the Study |
| Listing 16.2.1.4 | Screen Failure | List of Reasons for Screening Failure |
| Listing 16.2.1.5 | Screening | Visits List and COVID-19 Impact |
| 16.2.2 Protocol Deviations | | |
| Listing 16.2.2.1 | Screening | Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria |
| Listing 16.2.2.2 | Safety | Protocol Deviations |
| 16.2.3 Randomization | 16.2.3 Randomization | |
| Listing 16.2.3 | Safety | Randomization and Treatment Group |

AD-ST-33.06 Effective date: 12-Nov-2020




| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data Listin | ngs | |
| 16.2.4 Demographic Data and Other Baseline Characteristics | | |
| Listing 16.2.4.1 | Screening | Demographic and Baseline Characteristics |
| Listing 16.2.4.2 | Safety | Medical History |
| Listing 16.2.4.3 | Screening | Osteoarthritis Characteristics |
| 16.2.5 Compliance and | or Drug Concentra | ation Data |
| Listing 16.2.5.1 | Safety | Study Drug Administration: Individual Doses |
| 16.2.6 Individual Effic | acy Response Data | |
| Listing 16.2.6.1 | mITT | Daily Pain NRS |
| Listing 16.2.6.2 | mITT | Galer NPS |
| Listing 16.2.6.3 | mITT | DSIS |
| Listing 16.2.6.4 | mITT | SF-36 |
| Listing 16.2.6.5 | mITT | Rescue Medication Usage |
| Listing 16.2.6.6 | mITT | Patient Global Impression of Change |
| CCI | | |
| 16.2.7 Adverse Event L | istings (by Patient/ | Subject) |
| Listing 16.2.7.1 | Safety | Adverse Events |
| Listing 16.2.7.2 | Safety | Treatment Emergent Adverse Events Leading to Study Drug<br>Discontinuation |
| Listing 16.2.7.3 | Safety | Treatment Emergent Adverse Events Associated with Abnormal Liver |
| Listing 16.2.7.4 | Safety | Joint Related Adverse Events of Special Interest |
| Listing 16.2.7.5 | Safety | Serious and/or Severe Infections |
| Listing 16.2.7.6 | Safety | Anaphylactic Reactions, Hypersensitivity or Infusion-Related<br>Reactions Leading to Discontinuation of Study Drug |
| 16.2.8 Laboratory Value | ues (by Patient/Subj | ject) |
| Listing 16.2.8.1 | Safety | Clinical Chemistry Laboratory Evaluations |
| Listing 16.2.8.2 | Safety | Hematology Laboratory Evaluations |
| Listing 16.2.8.3 | Safety | Coagulation Laboratory Evaluations |
| Listing 16.2.8.4 | Safety | Urinalysis Laboratory Evaluations |
| Listing 16.2.8.5 | Safety | Serology Laboratory Evaluations |
| Listing 16.2.8.6 | Safety | Pregnancy Test Results |

AD-ST-33.06 Effective date: 12-Nov-2020




| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data Listings | | |
| Listing 16.2.8.7 | Safety | Drug Test Results |
| Listing 16.2.8.8 | Safety | COVID-19 Screening |
| 16.2.9 Other Clinical O | bservations and M | leasurements (by Patient/Subject) |
| Listing 16.2.9.1 | Safety | Vital Signs Measurements |
| Listing 16.2.9.2.1 | Safety | 12-Lead Digital ECG Results |
| Listing 16.2.9.2.2 | Safety | 12-Lead Safety ECG Results |
| Listing 16.2.9.3 | Safety | Physical Examination Results |
| Listing 16.2.9.4 | Safety | Neurological Examination Results |
| Listing 16.2.9.5 | Safety | Total Neuropathy Score-Nurse |
| Listing 16.2.9.6 | Safety | Motor and Sensory Nerve Conduction Studies |
| Listing 16.2.9.7 | Safety | Strength and Deep Tendon Reflexes |
| Listing 16.2.9.8 | Safety | Injection Site Reactions |
| Listing 16.2.9.9 | Safety | Anaphylactic Reactions |
| Listing 16.2.9.10 | Safety | Liver Diagnostic Investigations |
| Listing 16.2.9.11 | Safety | Liver Risk Factors and Lifestyle Events |
| Listing 16.2.9.12 | Safety | Liver Signs and Symptoms |
| Listing 16.2.9.13 | Safety | Infection Diagnostic Investigations |
| Listing 16.2.9.14 | Safety | Infection Risk Factors and Lifestyle Events |
| Listing 16.2.9.15 | Safety | Infection Signs and Symptoms |
| Listing 16.2.9.16 | Safety | Prior and Concomitant Medications |
| Listing 16.2.9.17 | Safety | Prohibited Concomitant Medications |
| Listing 16.2.9.18 | Safety | Concomitant Procedures |
| Listing 16.2.9.19 | Safety | Anti-drug Antibody Test Results |
| 16.2.10 Pharmacokinet | 16.2.10 Pharmacokinetic/Pharmacodynamic Measurements | |
| Listing 16.2.10.1 | PK | Serum MEDI7352 Concentrations |
| Listing 16.2.10.2 | Safety | Serum total NGF Concentrations |





# 13.6. Planned Figure Descriptions

The following are planned summary figures for protocol number D5680C00002. The figure numbers and page numbers are place holders only and will be determined when the figures are produced.





**Table 6: Planned Figures** 

| Figure Number | Population | Figure Title/Summary |
|---|---|---|
| Figure 14.2.1.1 | mITT | Daily Pain NRS: MCP-Mod Dose Response Model |
| Figure 14.2.1.2 | mITT | Daily Pain NRS: Boxplots at Week 12 by Treatment<br>Group and Missing Data Handling |
| Figure 14.2.1.3 | mITT | Daily Pain NRS: Boxplots at Week 12 by Treatment<br>Group and Co-Medication Subgroup |
| Figure 14.2.1.4 | mITT | Daily Pain NRS: MMRM LS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases) |
| Figure 14.3.6.1.1 | Safety | Vita1Sign Profiles: Mean (±SD) Systolic Blood Pressure over time |
| Figure 14.3.6.1.2 | Safety | Vital Sign Profiles: Mean (±SD) Diastolic Blood<br>Pressure over time |
| Figure 14.3.6.1.3 | Safety | Vital Sign Profiles: Mean (±SD) Heart Rate over time |
| Figure 14.3.6.1.4 | Safety | Vital Sign Profiles: Mean (±SD) Respiratory Rate over time |
| Figure 14.3.6.1.5 | Safety | Vital Sign Profiles: Mean (±SD) Temperature over time |
| Figure 14.4.1.1 | PK | Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 over time |
| Figure 14.4.1.2 | PK | Pharmacokinetics: Individual Plot of Serum MEDI7352<br>Concentrations over time |
| Figure 14.4.2.1 | Safety | Pharmacodynamics: Line Plot of Geometric Mean (with and without gSD) Serum total NGF over time |
| Figure 14.4.2.2 | Safety | Pharmacodynamics: Individual Plot of Serum total NGF over time |





## 14. Tables, Listing and Figure Shells

# 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all Tables, Listings, and Figures in support of this study. Note that programming notes may be added if appropriate after each table, listing and figure shell. All shells will be provided as a separate document.





# Figure 1: Standardized Layout

| Astra Zeneca | Page xx of xx |
|---|---|
| Protocol: D5680C00002 | Version |
| <table, figure="" listing,=""> xx.x.x</table,> | |
| Title of Table, Listing or Figure | |
| Study Population and if applicable subgroup Description | |
| Body of Table, Listing or Figure | |
| Note: If directly Applicable | |
| Footnote 1 | |
| Footnote 2 | |
| Footnote n | |
| Footnote n+1 SAS program path and name Executed on ddmmmyyyy at hh:mm on data from ddmmmyy | ууу |



# 15. Appendix: Calculation of Dose to achieve target effects

Although only one dose-response model type (Emax) is pre-specified in the protocol for the primary analysis, on

Let us assume the R® *DoseFinding* package original parametrization for these two dose-response model functions below:

Journal of Statistical Software

9

| Name | $f(d, oldsymbol{	heta})$ | $f^0(d,oldsymbol{	heta^*})$ | (*) | (#) |
|---|---|---|---|---|
| linear | $E_0 + \delta d$ | d | | |
| linlog | $E_0 + \delta \log(d+c)$ | $\log(d+c)$ | | c |
| quadratic | $E_0 + \beta_1 d + \beta_2 d^2$ | $d + \delta d^2$ if $\beta_2 < 0$ | δ | |
| emax | $E_0 + E_{\rm max} d / (ED_{50} + d)$ | $d/(ED_{50} + d)$ | $ED_{50}$ | |
| logistic | $E_0 + E_{\text{max}} / \{1 + \exp[(ED_{50} - d)/\delta]\}$ | $1/\{1 + \exp[(ED_{50} - d)/\delta]\}$ | $(ED_{50}, \delta)^{\top}$ | |
| exponential | $E_0 + E_1(\exp(d/\delta) - 1)$ | $\exp(d/\delta) - 1$ | δ | |
| sigEmax | $E_0 + E_{\rm max} d^h / (ED_{50}^h + d^h)$ | $d^h/(ED_{50}^h + d^h)$ | $(ED_{50}, h)^{\top}$ | |
| betaMod | $E_0 + E_{\text{max}} B(\delta_1, \delta_2) (d/D)^{\delta_1} (1 - d/D)^{\delta_2}$ | $B(\delta_1, \delta_2)(d/D)^{\delta_1}(1 - d/D)^{\delta_2}$ | $(\delta_1, \delta_2)^{\top}$ | D |

Table 1: Dose-response models implemented in the MCPMod package. Column (\*) lists for

1. Equations for Target Dose  $D_{\Delta}$  to achieve a Delta ( $\Delta$ ) versus placebo

Emax:  $TD_{\Delta} = ED_{50}/((E_{max}/\Delta) - 1)$ , where  $ED_{50}$  and  $E_{max}$  are estimated from the fitted Emax model

Exponential:  $TD_{\Delta} = \delta * \log((\Delta/E_1) + 1)$ , where  $\delta$  and  $E_1$  are estimated from the fitted exponential model

(The function TD from the DoseFinding package will be used for the above)

2. Equations for Dose (ED<sub>P</sub>) to achieve a certain proportion P of the effect of the maximum dose studied versus placebo (See DoseFinding manual page 51 where ED is 'Effective Dose')





Emax:  $ED_P = (P * ED_{50} * max(doses))/(ED_{50} + (1-P) * max(doses)) = (P * ED_{50} * 150)/(ED_{50} + (1-P) * 150)$ 

Exponential:  $ED_P = \delta * log((P*exp(max(doses)/\delta) + 1-P)) = \delta * log((P*exp(150/\delta) + 1-P))$ 

(The function ED from the DoseFinding package will be used for the above)

3. Equation for Dose (asym ED<sub>P</sub>) to achieve a certain proportion P of the asymptotic maximum effect (E<sub>max</sub>) versus placebo

Emax: asymptotic  $ED_P = (P*ED_{50})/(1-P)$ 

Simulation-based CI will be created for each of the above quantities from the mean and covariance matrix of the model parameters, assuming multivariate normality. Therefore 10,000 samples from the multivariate distribution will be taken, and for each simulation the TD and ED estimates calculated. The 2.5% and 97.5% percentiles will then form the appropriate 95% two-sided CI.





| Sponsor: | AstraZeneca |
|---|---|
| Protocol Title | A Randomised, Double-Blind, Placebo-Controlled, Dose-<br>Response Study of the Efficacy and Safety of MEDI7352 in<br>Subjects with Painful Diabetic Neuropathy |
| Development Phase | 2 |
| Protocol Numbers: | D5680C00002 |
| Premier Research PCNs: | MEDU177093 |
| Document Version: | Final Version 1.0 |
| Document Date: | 12-Jul-2023 |

# **Document History**

| Version | Date | Author | Description |
|---------|-------------|--------|---------------|
| 0.1 | 24-Mar-2023 | PPD | Draft Version |
| 0.2 | 21-Apr-2023 | PPD | Draft Version |
| 0.3 | 24-May-2023 | PPD | Draft Version |
| 0.4 | 20-Jun-2023 | PPD | Draft Version |

Final 1.0 | 12-Jul-2023 | 





#### **Tables, Listings, and Figures Conventions**

All listings, tables, and graphs will have a header showing the sponsor company name, protocol and version of delivery and a footer showing the version of SAS, the file name and path, and the source of the data (listing number).

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

#### **General Reporting Conventions**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text will not be used in tables, figures, and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing.
- Adverse events with missing MedDRA coding will have their system organ class preferred term presented as "Not Coded" and the Preferred Term presented as verbatim in the tables. The "Not Coded" frequencies will be sorted to the end of the tables. This will only be applicable for any deliveries sent before database lock (e.g., for dry runs).
- Programming notes may be inserted into the shells, these notes will not appear in the final output.

#### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xx), where appropriate.
- All population summaries for categorical variables will include all categories that were planned and for which the participants may have had a response.
- All population summaries for continuous variables will include: n, mean, SD, median, quartiles, minimum, and maximum. Other summaries (e.g., number missing, geometric mean, 95% CIs, and coefficient of variation [CV] or % CV) may be used as appropriate. The precision of the maximum and minimum will match the maximum precision in the observed data and 2 decimals for derived data unless specifically mentioned in the corresponding shell. The mean and median will have 1 additional decimal place. The SD will have 2 additional decimal places. For derived data, minimum and maximum will be reported to 2 degrees of precision. Measures of location (mean and median) will be reported to 3 degree of precision, and measures of spread will be reported to 4 degrees of precision.

Final 1.0 | 12-Jul-2023 | 





• All percentages are rounded and reported to a single decimal point (xx.x%). Exceptions are 0 and 100 that will be displayed as 0 and 100% respectively.

#### **Planned Tables, Figures and Listings**

- The table and listing numbers are place holders only and will be determined when the outputs are produced.
- In all listings a blank line will be placed between each participant. Within a data listing, if an item appears line after line (e.g., repetition of participant number), then only the first occurrence will be displayed.
- In data listings, the information for 1 participant will be kept on 1 page, if possible, rather than splitting a Subjects's information across pages.

Final 1.0 | 12-Jul-2023 | 





# **Planned Table Descriptions and Shells**

| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.1.2 Screening Population | U |
| Table 14.1.3 - Summary of Reasons for Screening Failure - Screen Failure Population | U |
| Table 14.1.4.1 - Demographics and Baseline Characteristics - Screening Population | U |
| Table 14.1.4.2 - Demographics and Baseline Characteristics - Safety Population | R |
| Table 14.1.4.3 - Demographics and Baseline Characteristics - mITT Population | R |
| Table 14.1.4.4 - Demographics and Baseline Characteristics - PK Population | R |
| Table 14.1.5.1 - Osteoarthritis Characteristics - Screening Population | U |
| Table 14.1.5.2 - Osteoarthritis Characteristics - Safety Population | R |
| Table 14.1.5.3 - Osteoarthritis Characteristics - mITT Population | R |
| Table 14.1.5.4 - Osteoarthritis Characteristics - PK Population | R |
| Table 14.1.6 - Medical History by System Organ Class and Preferred Term - Safety Population | U |
| Table 14.1.7 - Prior Medications by ATC Level 2 and Preferred Name - Safety Population | U |
| Table 14.1.8 - Protocol Deviations - Safety Population | U |
| Table 14.1.9 - Overall Study Drug Exposure - Safety Population | U |
| Table 14.2.1.1.1 - Daily Pain NRS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.1.1.2 - Daily Pain NRS: Summary Statistics (LOCF) - mITT Population | R |
| Table 14.2.1.1.3 - Daily Pain NRS: Summary Statistics (BOCF) - mITT Population | R |
| Table 14.2.1.2.1 - Daily Pain NRS: Primary MCP-Mod Analysis (LOCF) - mITT Population | U |
| Table 14.2.1.2.2 - Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) - mITT Population | U |
| Table 14.2.1.3.1 - Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) - mITT Population | U |
| Table 14.2.1.3.2 - Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) - mITT Population | R |
| Table 14.2.2.1 - Galer NPS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.2.2 - Galer NPS: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.3.1 - DSIS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.3.2 - DSIS: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.4.1 - SF-36: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.4.2 - SF-36: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.5.1 - Rescue Medication Use: Summary Statistics - mITT Population | U |

Final 1.0 | 12-Jul-2023 | 





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.2.6.1 - Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel Haenszel (Observed Cases) - mITT Population | U |
| Table 14.2.6.2 - Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.7.1 - Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases) - mITT Population | R |
| Table 14.2.7.2 - Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) - mITT Population | R |
| Table 14.2.8.1 - Patient Global Impression of Change: Summary Statistics - mITT Population | U |
| Table 14.2.8.2 - Patient Global Impression of Change: Cochran-Mantel Haenszel - mITT Population | U |
| CCI | U |
| Table 14.3.1.1 - Summary of Overall Adverse Events - Safety Population | U |
| Table 14.3.1.2 - Treatment Emergent of Adverse Events by System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.3 - Treatment Emergent of Adverse Events by Severity, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.4 - Treatment Emergent Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.5 - Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.6 - Treatment Emergent Adverse Events Leading to Discontinuation of Study drug by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.1.7 - Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.1.8 - Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term - Safety Population | R |
| Table 14.3.1.9 - Treatment Emergent Adverse Events by Preferred Term - Safety Population | R |
| Table 14.3.2.1.1 - Serious Adverse Events by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.2 - Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.2 - Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.4 - Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.3.1 - Listing of Serious Adverse Events - Safety Population | U |
| Table 14.3.3.2 - Listing of Deaths - Safety Population | U |

Final 1.0 | 12-Jul-2023 | 





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.3.2.2.1 - Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.2 - Potential Joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.3 - Serious and/or severe Infections by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.4 - Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions<br>Leading to Discontinuation of IP by System Organ Class and Preferred Term - Safety<br>Population | R |
| Table 14.3.4.1 - Descriptive Summary of Clinical Chemistry - Safety Population | U |
| Table 14.3.4.2 - Shift Table of Clinical Chemistry Results - Safety Population | U |
| Table 14.3.4.3 - Descriptive Summary of Hematology - Safety Population | R |
| Table 14.3.4.4 - Shift Table of Hematology Results - Safety Population | R |
| Table 14.3.4.5 - Descriptive Summary of Coagulation - Safety Population | R |
| Table 14.3.4.6 - Shift Table of Coagulation Results - Safety Population | R |
| Table 14.3.4.7 - Descriptive Summary of Urinalysis - Safety Population | U |
| Table 14.3.4.8 - Shift Table of Urinalysis Results - Safety Population | R |
| Table 14.3.4.9 - Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin - Safety Population | U |
| Table 14.3.5.1 - Descriptive Summary of Vital Signs - Safety Population | U |
| Table 14.3.5.2 - Descriptive Summary of ECG Data - Safety Population | U |
| Table 14.3.5.3 - Summary of Overall Evaluation of safety ECG Data - Safety Population | U |
| Table 14.3.5.4 - Covid-19 Screening - Safety Population | U |
| Table 14.3.5.5 - Summary of Sub-Scores for Total Neuropathy Score-Nurse - Safety Population | U |
| Table 14.3.5.6 - Descriptive Summary of Total Neuropathy Score-Nurse - Safety Population | U |
| Table 14.3.5.7 - Summary of Motor and Sensory Nerve Conduction Studies - Safety Population | U |
| Table 14.3.5.8 - Summary of Strength and Deep Tendon Reflexes - Safety Population | U |
| Table 14.3.5.9 - Summary of Local Injection Site Reactions - Safety Population | U |
| Table 14.3.5.10 - Summary of Hypersensitivity/Anaphylactic Reactions - Safety Population | U |
| Table 14.3.5.11 - Summary of Liver Diagnostic Investigations - Safety Population | U |
| Table 14.3.5.12 - Summary of Liver Risk Factors and Lifestyle Events - Safety Population | U |
| Table 14.3.5.13 - Summary of Liver Signs and Symptoms - Safety Population | U |
| Table 14.3.5.14 - Summary of Infection Diagnostic Investigations - Safety Population | U |
| Table 14.3.5.15 - Summary of Infection Risk Factors and Lifestyle Events - Safety Population | U |

Final 1.0 | 12-Jul-2023 | 





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.3.5.16 - Summary of Infection Signs and Symptoms - Safety Population | U |
| Table 14.3.5.17 - Summary of Concomitant Medications by ATC Level 2 and Preferred Name - Safety Population | R |
| Table 14.3.5.18 - Summary of Concomitant Procedures - Safety Population | R |
| Table 14.3.5.19 - Anti-Drug Antibody Results and Titre Summary by Timepoint - Safety Population | U |
| Table 14.3.5.20 - Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories - Safety Population | U |
| Table 14.4.1 - Summary of Serum MEDI7352 Concentrations - PK Population | U |
| Table 14.4.2 - Summary of Serum total NGF Concentrations - PD Population | U |

Final 1.0 | 12-Jul-2023 | 





# **Table Change Log**

| Output<br>Number | Change Made<br>By (initials) | Description/Rationale |
|------------------|------------------------------|-----------------------|

Final 1.0 | 12-Jul-2023 | 





# 1. Demographic Data

Table 14.1.2 Subject Disposition Screening Population

| Screening Population | | | | | |
|---|---|---|---|---|---|
| | Placebo MEDI7352 | | | Total | |
| _ | | CCI | CCI | CCI | |
| Status | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Screening Population [1] | | | | | xx (100%) |
| Enrolled Subjects | | | | | xx (xx.x %) |
| Re-screened Subjects | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Randomized Subjects | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Safety Population [2] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| nITT Population [3] | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Evaluable Week 12 Efficacy | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Evaluable LOCF Efficacy [4] | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Efficacy Evaluable | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| PK Population [5] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Completed Study Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Study Treatment Reason for Discontinuation: | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lack of Efficacy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to Follow-up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Non-compliance with Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Physician Decision | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pregnancy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Progressive Disease | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Protocol Violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Study Terminated by Sponsor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Technical Problems | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Withdrawal by Subject | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

 Final 1.0 | 12-Jul-2023 |





| Completed Study Withdrawn from the Study | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
|---|---|---|---|---|---|
| Reason for Discontinuation: | , | , | , | , | , |
| Adverse Event | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Death | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lack of Efficacy | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to Follow-up | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| ••• | | | | | |

COVID-19 = Coronavirus disease 2019; LOCF = Last Observation Carried Forward; mITT = modified intent-to-treat; N = number of subjects per treatment group; PK = pharmacokinetic.

Note: Percentages are n/Number of subjects randomized\*100 as displayed in column header N, except for the screened, enrolled, re-screened and randomized, where n/Number of Screening subjects\*100.

- [1] The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments.
- [2] The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication.
- [3] The mITT Population includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.
- [4] Subjects in the mITT Population with LOCF applied for missing efficacy data at week 12,
- [5] The PK Population includes all subjects for who a pharmacokinetic sample was obtained and analyzed.

Reference Listings: 16.2.1.1, 16.2.1.2, 16.2.1.3,

## **Programming Notes:**

- Display only reasons for early discontinuation with non-missing value.
- A column for column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.1.3 Summary of Reasons for Screening Failure Screen Failure Population

| | Total |
|----------------------------------------------------------------|------------|
| | (N=xx) |
| Number of Subjects Who Don't Meet Inclusion/Exclusion Criteria | xx (xx.x%) |
| Reason 1 | xx (xx.x%) |
| Reason 2 | xx (xx.x%) |
| Reason 3 | xx(xx.x%) |
| Reason 4 | xx (xx.x%) |

N = number of subjects.

Note: subject can be counted in more than one criterion.

Reference Listing 16.2.1.4

Final 1.0 | 12-Jul-2023 | 





Table 14.1.4.1 Demographics and Baseline Characteristics Screening Population

| Variable | Placebo | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | (N=xx) | | | (N=xx) |
| Age (years) [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | XX.X | XX.X | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Age Category | | | | | |
| ≥18 - <65 years | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| ≥65 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Gender | | | | | |
| Male | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ethnicity | | | | | |
| Hispanic or Latino | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Race | | | | | |
| American Indian or Alaska Native | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Black or African American | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Not Specified | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Screening Height (cm) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Final 1.0 | 12-Jul-2023 | 





| Screening Weight (kg) | | | | | |
|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Screening BMI (kg/m²) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx |
| Female characteristics [2] | | | | | |
| Surgically sterile | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Postmenopausal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Fully vaccinated for COVID-19 | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

BMI = Body Mass Index; COVID-19 = Coronavirus disease 2019; n = number of subjects by treatment group with collected parameter; N = number of subjects per treatment group; SD = standard deviation.

## **Programming Notes:**

- If a variable is between 2 pages, start the variable in the second page.
- Keep all possible values for each category even if no subject.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

<sup>[1]</sup> Age was calculated as age at time of consent.

<sup>[2]</sup> Percentages are n/Number of Female subjects from Analysis Population\*100 Reference Listing: 16.2.4.1





# Table 14.1.4.2 Demographics and Baseline Characteristics Safety Population

## **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.1.4.3
Demographics and Baseline Characteristics
mITT Population

## **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.1.4.4
Demographics and Baseline Characteristics
PK Population

## **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 




Table 14.1.5.1 Osteoarthritis Characteristics Screening Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Variable | | CCI | CCI | CCI | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects diagnosed with Osteoarthritis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Joint(s)/Area(s) affected: | | | | | |
| Shoulder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Elbow | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hip | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Knee | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ankle | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Spine | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hands | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Feet | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Osteoarthritis clinically significant | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Radiologic investigations conducted [1] | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Plain radiography | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MRI | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Joint(s)/Area(s) investigated: | | | | | |
| Shoulder | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Elbow | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hip | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Knee | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ankle | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Spine | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1.0 | 12-Jul-2023 | 





| Hands | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|
| Feet | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Osteoarthritis radiologically significant | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Kellgren-Lawrence score reported | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 0 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Grade 2 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 3 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Grade 4 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| No/Not applicable | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Radiologic Scoring System Used? | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Grade 2 Grade 3 Grade 4 No/Not applicable Radiologic Scoring System Used? Yes | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

MRI = magnetic resonance imaging; N = number of subjects per treatment group.

## **Programming Notes:**

- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column dosing (column for column for col

<sup>[1]</sup> Subjects who reported more than one radiologic investigation within each category were only counted once. Reference Listing: 16.2.4.3





#### Table 14.1.5.2 Osteoarthritis Characteristics Safety Population

## **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column

Table 14.1.5.3 Osteoarthritis Characteristics mITT Population

## **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column for column dosing (column dosing (column for column for

Table 14.1.5.4 Osteoarthritis Characteristics PK Population

## **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column dosing (column for column for col

Final 1.0 | 12-Jul-2023 | 





Table 14.1.6

Medical History by System Organ Class and Preferred Term
Safety Population

| System Organ Class | Placebo | | MEDI7352 | | |
|---|---|---|---|---|---|
| Preferred Term | (N=xxx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| Any Medical History | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N = number of subjects per treatment group.

Note: All medical history terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 26.0. At each level of summarization (system organ class or preferred term), subjects having more than one medical history term were counted only once. System organ class and preferred terms are sorted in descending order of frequency of Total column, and alphabetically if same frequency.

Reference Listing: 16.2.4.2

#### **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Sort SOC and PT (within SOC) in descending order of frequency in the Total column. Sort alphabetically in case of ties.
- Uncoded Medical History Events
  - O When there are uncoded Medical History Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] will be sorted at the end of the table.
- A column for column

Final 1.0 | 12-Jul-2023 | 





Table 14.1.7
Prior Medications by ATC Class and Preferred Name
Safety Population

| ATC Class [1] | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Preferred Term | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with at Least One Prior<br>Medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Level 2 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name 1 | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name n | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Level 2 n | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name n | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |

ATC = Anatomical Therapeutic Class; N = number of subjects per treatment group.

Note: Prior medications are defined as medications that started before first dose of study, whether they were stopped before first dose of study medication or not. All prior medications are coded using WHO drug dictionary version vMar2023. At each level of summarization (ATC Level 2 or Preferred Name), subjects who reported more than one prior medication were only counted once. ATC Level 2 and Preferred Term are sorted in in descending order of frequency of total, and alphabetically if same frequency.

Reference Listing: 16.2.9.16

#### **Programming Notes:**

- If uncoded ATC Level or Preferred Name, please put them as [Not Coded]
- ATC and Preferred Name texts should be in proper case in table.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> ATC Class is defined as ATC Level 2.





Table 14.1.8 Protocol Deviations Safety Population

| | Placebo | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects With Any Important Protocol Deviation/Violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 2 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 5 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 6 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group.

Notes: Percentages are n/Number of subjects by treatment group\*100.

Subjects with one or more deviations within a type of protocol deviation were counted only once.

Reference Listing 16.2.2.1

## **Programming Notes:**

• A column for column for dosing (column for dosing

Final 1.0 | 12-Jul-2023 | 





## 2. Exposure and Compliance

Table 14.1.9
Overall Study Drug Exposure
Safety Population

| | Placebo | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| Category/ Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Maximum Number of Doses Administered [1] | | | | | |
| 1 Dose | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 Doses | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 Doses | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 Doses | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 5 Doses | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 6 Doses | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total Duration of Exposure (days) [2] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| Total (cumulative) dose infused (mL) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | xx, xx | xx, xx |

n = number of subjects by treatment group with collected parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Subjects are counted once for each level of dose administered.

<sup>[2]</sup> Duration of exposure (days) = min(date of last dose of treatment + 14 days or date of death) – date of first dose of treatment + 1. Reference Listing: 16.2.5.1





## **Programming Notes:**

- Add all categories even if count is 0.
- A column for column

Final 1.0 | 12-Jul-2023 | 





## 3. Primary Efficacy Analysis

Table 14.2.1.1.1

Daily Pain NRS: Summary Statistics (Observed Cases)

mITT Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx |
| Week 2 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | XX, XX | xx, xx |
| Week 2 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | XX, XX | XX, XX |

CFB = Change from Baseline; DPS = Daily Pain Score; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NRS = Numeric Rating Scale; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are weekly averages of the average daily pain scores on an 11-point (0-10) NRS and CFB for the same variable.

[1] Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

Reference Listing: 16.2.6.1

Final 1.0 | 12-Jul-2023 | 





## **Programming Notes:**

- Include all observed data (Not the LOCF) on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, 12 and 18.
- A column for column

Final 1.0 | 12-Jul-2023 | 





# Table 14.2.1.1.2 Daily Pain NRS: Summary Statistics (LOCF) mITT Population

#### **Programming Notes:**

- Same shell as Table 14.2.1.1.1.
- Include all observed and LOCF data on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Add abbreviation in footnote: LOCF = Last Observation Carried Forward.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Table 14.2.1.1.3

Daily Pain NRS: Summary Statistics (BOCF)

mITT Population

## **Programming Notes:**

- Same shell as Table 14.2.1.1.1.
- Include all observed and BOCF data on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Add abbreviation in footnote: BOCF = Baseline Observation Carried Forward.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





# Table 14.2.1.2.1 Daily Pain NRS: Primary MCP-Mod Analysis (LOCF) mITT Population

| 'MCP' step | | |
|-----------------------------|---------|------------------------------|
| Model | | |
| Contrast [1] | t value | 1-sided adjusted P-value [2] |
| Hyperbolic E <sub>max</sub> | · | |
| ED50 = 7.5 | XX.XX | 0.xxxx |
| ED50 = 15 | XX.XX | 0.xxxx |
| ED50 = 30 | XX.XX | 0.xxxx |
| ED50 = 60 | XX.XX | 0.xxxx |
| ED50 = 750 | XX.XX | 0.xxxx |
| Exponential | | |
| $\delta = 100$ | XX.XX | 0.xxxx |
| $\delta = 200$ | XX.XX | 0.xxxx |

CFB = Change from Baseline; LOCF = Last Observation Carried Forward; MCP = Multiple Comparisons; Procedure; NRS = Numeric rating scale.

<sup>[1]</sup> ED50 = Effective Dose giving half of the asymptotic maximum effect.

<sup>[2]</sup> Multiplicity Adjusted P-value





#### 'MOD' step [3] Selected Model xxxxxxxxx

| Parameter | Estimate | 95% CI of Estimate [6] |
|---|---|---|
| ED50 | XX.X | [ x.xx to x.xx ] |
| ED90 [4] | XX.X | [ x.xx to x.xx ] |
| Asymptotic ED90 [5] | XX.X | [ x.xx to x.xx ] |
| Dose to achieve target (-1.25) effect | XX.X | [ x.xx to x.xx ] |
| Treatment effect at dose = $5 \text{ mcg}$ | XX.X | [ x.xx to x.xx ] |
| Treatment effect at dose = 50 mcg | XX.X | [ x.xx to x.xx ] |
| Treatment effect at dose = 150 mcg | XX.X | [ x.xx to x.xx ] |
| Treatment effect at dose = 450 mcg | xx.x | [ x.xx to x.xx ] |

CI: Confidence Interval; LOCF = Last Observation Carried Forward; MCP = Multiple Comparisons; Procedure; MOD = Modelling; NRS = Numeric rating scale.

## **Programming Notes:**

• The 'MOD' step will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

Final 1.0 | 12-Jul-2023 | 

<sup>[3]</sup> Results from the 'MOD' step will only be available in case any of the MCP tests is statistically significant.

<sup>[4]</sup> ED90 = Effective Dose giving 90% of the effect of the maximum dose studied.

<sup>[5]</sup> Asymptotic ED90 = Effective Dose giving 90% of the asymptotic maximum effect.

<sup>[6] 2.5%</sup> and 97.5% quantiles taken from 100000 samples from the multivariate normal distribution for model fitted estimates and its covariance matrix. Reference Listing: 16.2.6.1





# Table 14.2.1.2.2 Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjusted Asymmetric CL | | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | • | xx.xxx | [ x.xx to x.xx ] | | |
| Co-Medication Type | | | 2 | | | | 0.xxxx |
| Baseline pain NRS | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| Active 5 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Active 150 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Active 450 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | | |

ANCOVA = analysis of covariance; CFB = Change from Baseline;

CL = Confidence limits; LOCF = Last Observation Carried Forward; NRS = Numeric rating scale.

[2] P-value is derived from the following model: ANCOVA by dose using NRS baseline value and co-medication as covariates, with CFB to Week 12 (LOCF) as dependent variable.

## Least Square Means

| Treatment | Number of Subjects | LS mean [3] | 95% CI of LS mean |
|----------------|--------------------|-------------|-------------------|
| Active 450 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Placebo | XX | X.XX | [ x.xx to x.xx ] |

CI = Confidence interval; LOCF = Last Observation Carried Forward; LS = least square; NRS = Numeric rating scale.

[3] The LS mean is a model estimate using fitted group parameter and the baseline weekly average pain NRS parameter evaluated at the grand mean over each group.

Reference Listing: 16.2.6.1

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.





## **Programming Notes:**

• Concomitant co-medication Type indicated for Painful Diabetic Neuropathy: either anticonvulsant class (pregabalin or gabapentin) or antidepressant class (duloxetine, venlafaxine, or amitriptyline).

• Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





#### Table 14.2.1.3.1 Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | d Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | | | |
| Co-medication type | | | 1 | | | | 0.xxxx |
| Week | | | 7 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 21 | | | | 0.xxxx |
| Baseline pain NRS | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| Active 5 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Active 150 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Active 450 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | xx.xx | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM = Mixed Model for Repeated Measures; NRS = Numeric rating scale.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, NRS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: week xxxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Active 450 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg | xx | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg | xx | X.XX | [ x.xx to x.xx ] |
| Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 450 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg - Placebo | xx | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LS = least square; NRS = Numeric rating scale.

## **Programming Notes:**

- Include LSmeans and difference in Lsmean with Placebo in repeated tables for the Treatment\*Week interaction.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline weekly average pain NRS parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.1





# Table 14.2.1.3.2 Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) mITT Population

#### **Programming Notes:**

- Same shell as Table 14.2.1.2.1, substituting "LOCF = Last Observation Carried Forward" by "BOCF = Baseline Observation Carried Forward".
- The MCP-MOD approach will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

Final 1.0 | 12-Jul-2023 | 





## 4. Secondary Efficacy Analysis

Table 14.2.2.1
Galer NPS: Summary Statistics (Observed Cases)
mITT Population

| Parameter: xxxxx | | | | | |
|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | Total |
| Visit/ | | CCI | CCI | CCI | _ |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | XX, XX | XX, XX |
| Week 4 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Week 4 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

•••

Final 1.0 | 12-Jul-2023 | 



feel a single type of pain only sometimes



xx(xx.x%)

xx (xx.x%) xx (xx.x%)

xx(xx.x%)

#### For Pain Duration Frequency

| Baseline [1] | | | | |
|---|---|---|---|---|
| I feel a background pain all of the time and occasional flare-ups | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| I feel a single type of pain all the time | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Week 4

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NPS = Neuropathic Pain Scale; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

xx(xx.x%)

xx (xx.x%)

xx (xx.x%)

Note: Data shown are Pain Intensity, Unpleasantness, and Descriptor scores on an 11-point (0-10) NRS, and Pain Duration/Frequency on a 3-point NRS (1-3), plus CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.6.2

#### **Programming Notes:**

- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Repeat for the Parameters: Pain intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, Surface Pain Intensity (All in an 11-point NRS), and Pain Duration/Frequency (in a 3-point NRS).
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





#### Table 14.2.2.2 Galer NPS: MMRM Analysis (Observed Cases) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | · | XX.XXX | | | |
| Co-Medication type | | | 1 | | | | 0.xxxx |
| Week | | | 4 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 12 | | | | 0.xxxx |
| Baseline NPS | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | | 0.xxxx |
| Active 5 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Active 150 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Active 450 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | xx.xx | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; NPS = Neuropathic Pain Scale.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, NPS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: week: xxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Active 450 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 450 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |

CI = Confidence interval; LS = least square; NPS = Neuropathic Pain Scale.

## **Programming Notes:**

- Include Lsmeans and difference in Lsmean with Placebo in repeated tables for the Treatment\*Week interaction.
- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Analysis is done for Galer NPS Total Score.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline NPS parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.2





Table 14.2.3.1
DSIS: Summary Statistics (Observed Cases)
mITT Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| | (= : ====) | (= : ===) | (= : ::::) | (= : ::::) | (= - = -) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | xx, xx |
| Week 4 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Week 4 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX |

CFB = Change from Baseline; DSIS = Daily Sleep Interference; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are weekly averages of the average daily sleep interference scores on an 11-point (0-10) NRS and CFB for the same variable.

[1] Baseline is defined as the average of the 'non-missing' DSIS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

Reference Listing: 16.2.6.3

Final 1.0 | 12-Jul-2023 | 





## **Programming Notes:**

- Include all observed data on weekly averages of the average daily Sleep Interference score for Baseline, Week 4, 8, 12, and 18.
- A column for column

Final 1.0 | 12-Jul-2023 | 





#### Table 14.2.3.2 DSIS: MMRM Analysis (Observed Cases) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | d Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | | | |
| Co-medication type | | | 1 | | | | 0.xxxx |
| Week | | | 4 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 12 | | | | 0.xxxx |
| Baseline DSIS | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | | 0.xxxx |
| Active 5 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Active 150 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Active 450 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | xx.xx | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; DSIS = Daily Sleep Interference.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, DSIS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: week xxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Active 450 mcg | xx | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg | XX | X.XX | [ x.xx to x.xx ] |
| Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 450 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |

CI = Confidence interval; LS = least square.

#### **Programming Notes:**

- Include LS means and difference in LS mean with Placebo in repeated tables for the Treatment\*Week interaction.
- Include all observed data on weekly average DSIS for Baseline, Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline weekly average DSIS parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.1





Table 14.2.4.1 SF-36: Summary Statistics (Observed Cases) mITT Population

Parameter: xxxxx

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx |
| Week 12 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Week 12 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

•••

Final 1.0 | 12-Jul-2023 | 





#### When parameter is "Change in general Health"

#### Baseline [1]

| Much better now than one year ago | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|
| Somewhat better now than one year ago | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| About the same as one year ago | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Somewhat worse now than one year ago | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Much worse now than one year ago | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

#### Week 12

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NRS = numeric rating scale; SD = standard deviation; SF-36 = 36-Item Short-Form Health Survey; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are derived SF-36 scores and Change in General Health on a 5-point NRS (1-5), plus CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.6.4

## **Programming Notes:**

- Include all observed data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Vitality (Energy/fatigue), Emotional well-being, Social functioning, Pain and General Health (from 0 to 100), Physical Health Summary, Mental Health Summary, and Change in general Health (in a 5-point NRS).
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





#### Table 14.2.4.2 SF-36: MMRM Analysis (Observed Cases) mITT Population

Model parameter estimates: xxxxxxxx

| | | | | | 2-sided 95% unadjuste | d Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | | | |
| Co-medication type | | | XX | | | | 0.xxxx |
| Week | | | 1 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 3 | | | | 0.xxxx |
| Baseline SF-36 | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| Active 5 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [ x.xx to x.xx ] | 0.xxxx |
| Active 150 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [ x.xx to x.xx ] | 0.xxxx |
| Active 450 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [ x.xx to x.xx ] | 0.xxxx |
| Model residual standard deviation | xx.xx | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; SF-36 = 36-Item Short-Form Health Survey.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, SF-36 baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: xxxxxxxx / week xxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Active 450 mcg | xx | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg | xx | X.XX | [x.xx to x.xx] |
| Active 5 mcg | xx | X.XX | [ x.xx to x.xx ] |
| Placebo | xx | X.XX | [ x.xx to x.xx ] |
| Active 450 mcg - Placebo | xx | X.XX | [ x.xx to x.xx ] |
| Active 150 mcg - Placebo | xx | X.XX | [ x.xx to x.xx ] |
| Active 5 mcg - Placebo | XX | X.XX | [ x.xx to x.xx ] |

CI = Confidence interval; LS = least square.

## **Programming Notes:**

- Include Lsmeans and difference in Lsmean with Placebo in repeated tables for the Treatment\*Week interaction.
- Include all observed data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Vitality (Energy/fatigue), Emotional well-being, Social functioning, Pain and General Health. Add parameter name after 'Model parameter estimates:' and after 'Least Square Means:'
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline SF-36 parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.4





Table 14.2.5.1 Rescue Medication Use: Summary Statistics mITT Population

| Variable | Placebo | | MEDI7352 | | |
|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | (N=xx) | | |
| Statistic of Category | (11-XX) | (11-11) | (N=xx) | (N=xx) | (11-XX) |
| Number of subjects taking any rescue medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of subjects taking any permitted rescue medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of days rescue medication was used [1] | | | | | |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | xx, xx |
| Cumulative consumption of | | | | | |
| Paracetamol Rescue Medication | | | | | |
| (mg) [2] | | | | | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Paracetamol Rescue Medication | | | | | |
| Average Daily Dose (mg) [3] | | | | | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Final 1.0 | 12-Jul-2023 | 





Number of subjects taking any prohibited rescue medication

xx (xx.x%)

xx (xx.x%)

xx(xx.x%)

xx(xx.x%)

xx (xx.x%)

N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

- [1] Each day on which permitted rescue medication was used at least once is counted.
- [2] Calculated as the total dose of paracetamol rescue medication (mg).
- [3] Calculated as: cumulative consumption of paracetamol rescue medication (mg) /total number of days rescue medication was used.

Reference Listing: 16.2.6.5

## **Programming Notes:**

- A column for column dosing (column for column for col
- Refer to

Final 1.0 | 12-Jul-2023 | 





#### Cochran-Mantel-Haenszel Test

| Number of | | 95% CI of Risk | 2-sided |
|---|---|---|---|
| Subjects (%) | Risk Difference [1] | Difference | P-value [2] |
| • | - | • | |
| xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| | xx (xx.x%) xx (xx.x%) xx (xx.x%) | Subjects (%) Risk Difference [1] xx (xx.x%) x.xx xx (xx.x%) x.xx xx (xx.x%) x.xx | Subjects (%) Risk Difference [1] Difference xx (xx.x%) x.xx [x.xx to x.xx] xx (xx.x%) x.xx [x.xx to x.xx] xx (xx.x%) x.xx [x.xx to x.xx] |

CI = confidence interval; NRS = numeric rating scale.

### **Programming notes:**

• Include all observed data for Week 4, 8, 12, 18.

<sup>[1]</sup> Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability across strata.

<sup>[2]</sup> P-value < 0.05 indicates a significant association between number of subjects with >=30% decrease from Baseline and treatment across strata. Reference Listing: 16.2.6.1





Table 14.2.6.2 Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) mITT Population

#### Model parameter estimates

| Parameter | Estimate | Z value | Degrees of freedom | Standard Error | 2-sided 95% CL | 2-sided<br>P-value [2] |
|---|---|---|---|---|---|---|
| Intercept | XX.XX | XX.XX | | XX.XXX | | • |
| Co-medication type | | | XX | | | 0.xxxx |
| Week | | | 4 | | | 0.xxxx |
| Treatment | | | 3 | | | 0.xxxx |
| Treatment*Week | | | 12 | | | 0.xxxx |
| Active 5 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | 0.xxxx |
| Active 150 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | 0.xxxx |
| Active 450 mcg vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | 0.xxxx |
| Dispersion | XX.XX | | | | | |

CL = Confidence limits; GEE: Generalized Estimation Equations; NRS = Numeric rating scale.

Reference Listing: 16.2.6.1

## **Programming notes:**

- Include all observed data for Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: GEE using Time, Treatment, Treatment\*Time and Co-medication type as covariates, with dependent binary variable indicating whether weekly average pain NRS has >=30% decrease from Baseline.





# Table 14.2.7.1 Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases) mITT Population

#### Cochran-Mantel-Haenszel Test

| Visit/ | Number of | | 95% CI of Risk | 2-sided |
|---|---|---|---|---|
| Category | Subjects (%) | Risk Difference [1] | Difference | P-value [2] |
| Week 4 | | | • | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [ x.xx to x.xx ] | 0.xxxx |
| Week 8 | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [ x.xx to x.xx ] | 0.xxxx |
| Week 12 | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| | , | | | |
| Week 18 | ( 0/) | | | 0 |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |

CI = confidence interval; NRS = numeric rating scale.

## **Programming notes:**

• Include all observed data for Week 4, 8, 12, and 18.

<sup>[1]</sup> Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability across strata.

<sup>[2]</sup> P-value < 0.05 indicates a significant association between number of subjects with >=50% decrease from Baseline and treatment across strata. Reference Listing: 16.2.6.1





#### Table 14.2.7.2 Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) mITT Population

## **Programming notes:**

- Same shell as Table 14.2.6.3. Change footnote in [2] as: "p-value is derived from the following model: GEE using Time, Treatment, Treatment\*Time and Co-medication type as covariates, with dependent binary variable indicating whether weekly average pain NRS has >=50% decrease from Baseline".
- Include all observed data for Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 




Table 14.2.8.1
Patient Global Impression of Change: Summary Statistics
mITT Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Week 4 | | | | | |
| Number of PGIC Responders | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Very Much Improved | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Much Improved | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Minimally Improved | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No change | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Minimally Worse | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Much Worse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Very Much Worse | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Week 8

. . .

N = number of subjects per treatment group; PGIC = Patient Global Impression of Change.

Note: Percentages for Number of subjects in the different improvement categories relative to baseline are n/Number of Subjects by treatment group at each visit \*100.

Reference Listing: 16.2.6.6

#### **Programming notes:**

- Include all observed data on PGIC scores for Week 4, 8, 12 and 18.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





# Table 14.2.8.2 Patient Global Impression of Change: Cochran-Mantel Haenszel mITT Population

Cochran-Mantel-Haenszel Test

| Visit/ | Number of | | 95% CI of Risk | 2-sided |
|---|---|---|---|---|
| Category | Patients (%) | Risk Difference [1] | Difference | P-value [2] |
| Week 4 | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Much Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Very Much improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Week 8 | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Much Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Very Much improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Week 12 | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Much Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Very Much improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |

Final 1.0 | 12-Jul-2023 | 





#### Week 18

| Improved relative to Baseline | xx (xx.x%) | X.XX | [ x.xx to x.xx ] | 0.xxxx |
|---|---|---|---|---|
| Much Improved relative to Baseline | xx (xx.x%) | x.xx | [ x.xx to x.xx ] | 0.xxxx |
| Very Much improved relative to Baseline | xx (xx.x%) | X.XX | [ x.xx to x.xx ] | 0.xxxx |

CI = confidence interval; NRS = numeric rating scale.

## **Programming Notes:**

• Include all observed data on PGIC scores for Week 4, 8, 12 and 18.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability across strata.

<sup>[2]</sup> P-value < 0.05 indicates a significant association between improvement relative to Baseline and treatment across strata. Reference Listing: 16.2.6.6





## 5. Exploratory Efficacy Analyses



Final 1.0 | 12-Jul-2023 | 







Final 1.0 | 12-Jul-2023 | 





## 6. Safety and Tolerability

## 6.1. Displays of Adverse Events

Table 14.3.1.1 Summary of Overall Adverse Events Safety Population

| | Placebo | | ME | DI7352 | | Total |
|---|---|---|---|---|---|---|
| Character | (NI) | CCI | CCI<br>(N) | CCI | All MEDI7352 | (NI) |
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with any AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE categorized as Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE categorized as Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE categorized as Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any SAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any SAE possibly related to IP [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE leading to Discontinuation of IP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE related to IP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE categorized as Mild related to IP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE categorized as Moderate related to IP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE categorized as Severe related to IP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any SAE leading to Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1.0 | 12-Jul-2023 | 





AE = adverse event; IP = Investigational product, N = number of subjects per treatment group; SAE = serious adverse event; TEAE = treatment emergent adverse event.

[1] Possibly related is defined as with reasonable possibility that the AE was caused by the IP, as assessed by investigator Note: Subjects who reported more than one adverse event within each category were only counted once. A TEAE is defined as an adverse event with an onset at the time of or following the start of treatment with IP.

Reference Listing: 16.2.7.1, 16.2.7.2, 16.2.7.3, 16.2.7.4

### **Programming Notes:**

• A column for doing (column f

Final 1.0 | 12-Jul-2023 | 





Table 14.3.1.2
Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| System Organ Class | Placebo | | M | IEDI7352 | | Total |
|---|---|---|---|---|---|---|
| | | CCI | CCI | CCI | All MEDI7352 | |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx(xx.x%)xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 3 Preferred Term 1 | xx (xx.x%) xx<br>xx (xx.x%) xx | XX (XX.X%) XX | xx (xx.x%) xx | $XX (XX.X^{0}\%) XX$ | XX (XX.X%) XX | XX (XX.X%) XX |
| Preferred Term 2 | ` / | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx $xx (xx.x%) xx$ | xx (xx.x%) xx $xx (xx.x%) xx$ | xx (xx.x%) xx<br>xx (xx.x%) xx |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT category; N = number of subjects per treatment group; IP = investigational product; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Note: Results are n (n/N \* 100) then the total number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

Aes were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

Aes are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing: 16.2.7.1

Final 1.0 | 12-Jul-2023 | 





- SOC and PT texts should be in proper case in table.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table.
- A column for column for column dosing (column for column for col

Final 1.0 | 12-Jul-2023 | 





Table 14.3.1.3

Treatment Emergent Adverse Events by Severity, System Organ Class and Preferred Term
Safety Population

| System Organ Class Preferred Term | Placebo MEDI7352 | | | | | |
|---|---|---|---|---|---|---|
| Severity | | CCI | CCI CCI All MEDI7352 | | | |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; ; n = number of subjects within each SOC/PT/Severity category; N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Note: Results are n (n/N \* 100).

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

Aes were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT at the maximum severity.

Aes are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing 16.2.7.1

Final 1.0 | 12-Jul-2023 | 





- SOC and PT texts should be in proper case in table.
- Present only severity categories with at least one subject.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.1.4

Treatment Emergent Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term Safety Population

| | | | outery I opulation | | | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Placebo MEDI7352 | | | | | |
| Relatedness | (N=xx) | (N=xx) | | | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Related [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Related [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Related [1] | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

. . .

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT/Relatedness category; N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

[1] Related is defined as reasonable possibility that the AE was caused by investigational product, as assessed by the investigator. Note: Results are n (n/N \*100).

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

Aes were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT for the most related AE.

Aes are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing 16.2.7.1

Final 1.0 | 12-Jul-2023 | 





- SOC and PT texts should be in proper case in table.
- Present only severity categories with at least one subject.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.1.5

Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term Safety Population

Treatment: xxxxxxx

| | ADA | | TE-ADA | Non-TE- | TE<br>Persistently | TE<br>Transiently | Post-Baseline and Baseline | Only Baseline |
|---|---|---|---|---|---|---|---|---|
| System Organ Class | Negative | ADA Positive | Positive | ADA Positive | ADA Positive | ADA Positive | Positive | Positive |
| Preferred Term | (N=xx) | (N=xx) | | (N=xx) | | | (N=xx) | (N=xx) |
| Freiened Tenn | (IN-XX) | (IN-XX) | (N=xx) | (IN-XX) | (N=xx) | (N=xx) | (IN-XX) | (IN-XX) |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) xx | , | ` / | xx (xx.x%) xx | ` / | ` / | ` / | ` / |
| Preferred Term 2 | ` / | xx (xx.x%) xx | | , , | | | | |
| Preferred Term 3 | ` / | xx (xx.x%) xx | ` / | ` / | ` / | ` / | ` / | ` / |
| System Organ Class 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | ` / | xx (xx.x%) xx | ` / | ` / | ` / | ` / | ` / | ` / |
| Preferred Term 2 | ` / | xx (xx.x%) xx | ` / | ` / | ` / | ` / | ` / | ` / |
| Preferred Term 3 | | xx (xx.x%) xx | | | | | | |
| System Organ Class 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) xx | | | xx (xx.x%) xx | | | | |
| Preferred Term 2 | xx (xx.x%) xx | xx (xx.x%) xx | ` / | | ` / | ` / | ` / | ` / |
| Preferred Term 3 | ` / | xx (xx.x%) xx | ` / | ` / | ` / | ` / | ` / | ` / |

AE = adverse event; ADA = Anti-Drug Antibodies; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; ; n = number of subjects within each SOC/PT category; N = number of subjects per ADA status category; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

ADA categories are defined in the Statistical Analysis Plan.

Note: Results are n (n/N \*100) then the total number of events.

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

Aes were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

Table is sorted by international order for SOC, and alphabetically for PT.

Reference Listing: 16.2.7.1





- SOC and PT texts should be in proper case in table.
- Repeat for Placebo, occurrence and Overall.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A table for column dosing (column dosing (column dosing

#### Table 14.3.1.6

Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One TEAE leading to IP discontinuation".
- Update Reference Listing to 16.2.7.2.
- A column for column dosing (Column dosing will only be added if Stage 4 is initiated.

#### Table 14.3.1.7

Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term Safety Population

### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One Non-Serious AE" and remove references to TEAEs.
- Update Reference Listing to 16.2.7.1.
- A column for column for dosing (column for dosing

Final 1.0 | 12-Jul-2023 | 





Table 14.3.1.8

Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term Safety Population

| | | | Safety I opulation | I . | | |
|---|---|---|---|---|---|---|
| | Placebo | Placebo MEDI7352 | | | | |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| ••• | | | | | | |

 $AE = adverse \ event; IP = investigational \ product; MedDRA = Medical \ Dictionary \ for \ Regulatory \ Activities; n = number \ of \ subjects \ within \ each \ PT \ category;$ 

N = number of subjects per treatment group; PT = Preferred Term; TEAE = treatment-emergent adverse event.

Note: Results are n (n/Number of subjects in the Safety population within each PT\*100) then the total number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

Aes were coded using MedDRA version 26.0. Subjects are counted once for each PT.

Aes are displayed by descending frequency of PT based on 'All MEDI7352' column, and alphabetically for PT of same frequency. Reference Listing: 16.2.7.1

## **Programming Notes:**

- PT texts should be in proper case in table.
- In case a term is not coded (e.g., in a dry run) it will be labelled as Not Coded [PT]", and sorted at the end of the table.
- A column for column dosing (column for column for col





## Table 14.3.1.9 Treatment Emergent Adverse Events by Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.8.
- Display all TEAEs, not only the most common.
- PT texts should be in proper case in table.
- In case a term is not coded (e.g., in a dry run) it will be labelled as Not Coded [PT]", and sorted at the end of the table.
- A column for column dosing column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





## 6.2. Summary of Deaths and Other Serious Adverse Events

Table 14.3.2.1.1
Serious Adverse Events by System Organ Class and Preferred Term
Safety Population

### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One SAE", add "SAE = Serious Adverse Event" to abbreviations, and remove references to TEAEs.
- Change footnote for "Reference Table 14.3.3.1".
- A column for column

Table 14.3.2.1.2
Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One Life-Threatening SAE", add "SAE = Serious Adverse Event" to abbreviations, and remove references to TEAEs.
- Add "Note: Life-threatening SAEs as judged by the investigator".
- Change footnote for "Reference Table 14.3.3.1".
- A column for column dosing (column for column for col

Final 1.0 | 12-Jul-2023 | 





## Table 14.3.2.1.3 Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One SAE with Outcome Death", add "SAE = Serious Adverse Event" to abbreviations, and remove references to TEAEs.
- Change footnote for "Reference Table 14.3.3.2".
- A column for column dosing (CC) will only be added if Stage 4 is initiated.

Table 14.3.2.1.4
Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.4. Change first row to be "Number of subjects with at Least One SAE", add "SAE = Serious Adverse Event" to abbreviations, and remove references to TEAEs.
- Change footnote for "Reference Table 14.3.3.1".
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





Table 14.3.3.1 Listing of Serious Adverse Events Safety Population

| Subject ID/<br>Treatment Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time<br>(Study Day) | Severity/<br>Relationship | Outcome/<br>Action Taken/<br>Therapy? | SAE Leading to Study DC? | | Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXXXXXXXX<br>XXXXXXXXXXX | DDMMMYYYY/<br>HH:MM (X)/<br>DDMMMYYYY/<br>HH:MM (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/<br>Yes | No | No | XX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>HH:MM (X)/<br>DDMONYYYY<br>/HH:MM (X) | XXXXXXXXX/<br>XXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/<br>No | Yes | XX | XX /<br>XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXX<br>XXXXXXXXXX | DDMONYYYY/<br>HH:MM (X)/<br>Ongoing | XXXXXXXXX/<br>XXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/N<br>o | No | XX | XX /<br>XXX |

DC = discontinuation; ID = identification; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Study Day = date of interest – date of first infusion. A TEAE is defined as an adverse event with an onset at the time of or following the start of treatment with IP.

SAEs were coded using MedDRA version 26.0

Final 1.0 | 12-Jul-2023 | 





- If time missing, display "- -:- -".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e., no AEs occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment ID/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g., in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.3.2 Listing of Deaths Safety Population

| Subject ID/<br>Treatment<br>Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time<br>(Study Day) | Severity/<br>Relationship | Outcome/<br>Action Taken/<br>Therapy? | AE<br>Leading<br>to IP DC? | TEAE? | Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>DDMMMYYYY/H<br>H:MM (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/<br>Yes | No | No | XX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>DDMMMYYYY/H<br>H:MM (X) | XXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX/No | Yes | XX | XX / XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>Ongoing | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXX/<br>No | No | XX | XX / XXX |

DC = discontinuation; ID = identification; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Study Day = date of interest – date of first infusion. A TEAE is defined as an adverse event with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0

Final 1.0 | 12-Jul-2023 | 





- If time missing, display "- -:- -".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e., no AEs occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g., in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Final 1.0 | 12-Jul-2023 | 





## 6.3. Displays of Significant Adverse Events and Adverse Events of Special Interest

Table 14.3.2.2.1
Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at least One TEAE Associated with Abnormal Liver". Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.3.
- A column for dosing (CC) will only be added if Stage 4 is initiated.

Table 14.3.2.2.2

Potential joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at least One Potential Joint Related AESI"
- Add abbreviation for AESI = Adverse Event of Special Interest. Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.4
- A column for column dosing (CC) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





#### Table 14.3.2.2.3 Serious and/or severe Infections by System Organ Class and Preferred Term Safety Population

### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One SAE or Severe AE Related to Infection". Add "SAE = Serious Adverse Event" to abbreviations. Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.5.
- A column for doing (CC) will only be added if Stage 4 is initiated.

#### Table 14.3.2.2.4

Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One Anaphylactic Reaction, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP". Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.6.
- A column for column dosing (cc) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





## 6.4. Laboratory Data

Table 14.3.4.1 Descriptive Summary of Clinical Chemistry Safety Population

Parameter: xxxxx (unit)

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| | VV | VV | VV | VV | V.V | VV |
| n<br>Maan (SD) | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Low CS | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Low CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High NCS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| | | | 1 | | | |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Final 1.0 | 12-Jul-2023 | 





Day 1 CFB

| n | XX | XX | XX | XX | XX | XX |
|---|---|---|---|---|---|---|
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

CFB = change from baseline; CS = clinically Significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = not clinically significant; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Note: Percentages are n/Number of subjects by treatment group at each visit\*100.

Reference Listing: 16.2.8.1

#### **Programming Notes:**

- Present only scheduled visits.
- Sort Parameters in the following Order: Albumin, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Bicarbonate, Calcium, Chloride, Creatinine, High-Sensitivity C-Reactive Protein (hs-CRP), Estimated Glomerular Filtration Rate (eGFR by Cockcroft Gault), Serum Glucose, Lactate Dehydrogenase (LDH), Potassium, Sodium, Total Bilirubin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





Table 14.3.4.2 Shift Table of Clinical Chemistry Results Safety Population

| Normal | Placebo<br>(N=xxx)<br>High | Missing | Total | e Grade [1] | ME<br>Normal | DI7352, CC<br>(N=xxx)<br>High | Missing | Total |
|---|---|---|---|---|---|---|---|---|
| | (N=xxx) | Missing | Total | Low | | (N=xxx) | | Total |
| | High | Missing | Total | Low | Normal | High | Missing | Total |
| v (vv v0/) | | | | | | | | |
| ·· (**** ··*0/) | | | | | | | | |
| v (vv v0/) | | | | | | | | |
| ** (**** **0/) | | | | | | | | |
| x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | | ` / | . , | | | ` / | x (xx.x%) | x (xx.x%) |
| x (xx.x%) | ` / | ` / | x (xx.x%) | 1 | 1 | ` / | 1 | x (xx.x%) |
| x (xx.x%) | | , , | x (xx.x%) | | , , | ` / | x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%) | x (xx.x%) x (xx.x%) | x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) | x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) | x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) | x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) | x (xx.x%) x (xx.x%) | x (xx.x%) x (xx.x%) |

Percentages are n/Number of subjects by treatment group at each visit for the parameter\*100.

Reference Listing 16.2.8.1

## **Programming Notes:**

- Repeat above in new pages for MEDI7352, CCI MEDI7352, MEDI7352, CCI and All MEDI7352.
- Repeat the above for dosing only if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.5.1.

Final 1.0 | 12-Jul-2023 | 

n = number of subjects within each category; N = number of subjects per treatment group.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





## Table 14.3.4.3 Descriptive Summary of Hematology Safety Population

### **Programming Notes:**

- Same shell as Table 14.3.5.1
- Present only scheduled visits.
- Sort Parameters in the following Order: Absolute basophil count, absolute eosinophil count, absolute lymphocytes count, Absolute Monocyte Count, Absolute Neutrophil Count, Basophils %, Eosinophils %, Hematocrit (HCT), Hemoglobin (HGB), hemoglobin A1C (HgbA1C), Lymphocytes %, mean corpuscular hemoglobin (MHC), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), Monocytes %, Neutrophils %, Platelets, Red blood cell count (RBC), Red Cell Distribution Width, white blood cell Count (WBC).
- Update Reference listing to 16.2.8.2.
- A column for column for column dosing (column dosing (column for column for

Table 14.3.4.4 Shift Table of Hematology Results Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.5.2
- Repeat the shell for occurred dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.5.3.
- Update Reference listing to 16.2.8.2

Final 1.0 | 12-Jul-2023 | 





## Table 14.3.4.5 Descriptive Summary of Coagulation Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.5.1
- Present only scheduled visits.
- Sort Parameters in the following Order: Activated Partial Thromboplastin Clotting Time (APTT), Fibrinogen, International normalized ratio (INR), Prothrombin Time (PT).
- Update Reference listing to 16.2.8.3.
- A column for column for column dosing (column dosing (column for column for

Table 14.3.4.6 Shift Table of Coagulation Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.5.2
- Repeat for column dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.5.4.
- Update Reference listing to 16.2.8.3.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.4.7 Descriptive Summary of Urinalysis Safety Population

Parameter: xxxxx (unit)

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Low NCS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Low CS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| Low CS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Final 1.0 | 12-Jul-2023 | 





٠.

#### Repeat for all visits for Parameters: Specific Gravity and pH

| Baseline [1] | | | | | | |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Negative | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Positive | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| If Positive, Specify [2] | | | | | | |
| 100 mg/dL | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| 250 mg/dL | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| 500 mg/dL | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| >= 1000 mg/dL | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Negative | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Positive | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High NCS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

...

#### Repeat for all visits for Parameters: Blood, Glucose, Ketones and Protein

CFB = change from baseline; CS = clinically significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = not clinically significant; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Percentages are n/Number of subjects by treatment group at each visit\*100.

Reference Listing: 16.2.8.4

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

<sup>[2]</sup> Percentages are n/Number of Subjects with a Positive Result\*100.





- Present only scheduled visits.
- Sort Parameters in the following Order: Blood Urine, Glucose, Ketones, pH, Protein, Specific Gravity.
- Categories for If Positive, Specify:
  - o Blood, Urine: Trace, Small, Moderate.
  - O Glucose: 100 mg/dL, 250 mg/dL, 500 mg/dL, >= 1000 mg/dL.
  - o Ketones: Trace, 15 mg/dL.
  - o Protein: Trace, 30 mg/dL, 100 mg/dL.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





#### Table 14.3.4.8 Shift Table of Urinalysis Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.5.2
- Repeat for column dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.5.3.
- Update Reference listing to 16.2.8.4

Final 1.0 | 12-Jul-2023 | 





Table 14.3.4.9

Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin Safety Population

| Accebo =xxx | | | | Total E | Bilirubin |
|---|---|---|---|---|---|
| Acebo =xxx | | | | <2 x ULN | >=2 x ULN |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Group | Nobs | | n (%) | n (%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Placebo | | | | |
| $ >=3 - <5 \text{ x ULN} & \text{x (xx.x\%)} & \text{x (xx.x\%)} \\ >=5 - <10 \text{ x ULN} & 0 & 0 \\ >=10 \text{ x ULN} & 0 & 0 \\ \hline \\ AST & \\ <3 \text{ x ULN} & & \text{x (xx.x\%)} & & \text{x (xx.x\%)} \\ >=3 - <5 \text{ x ULN} & & \text{x (xx.x\%)} & & \text{x (xx.x\%)} \\ >=5 - <10 \text{ x ULN} & 0 & 0 & 0 \\ >=10 \text{ x ULN} & 0 & 0 & 0 \\ \hline >=10 \text{ x ULN} & 0 & 0 & 0 \\ \hline $ | N=xxx | XXX | ALT | | |
| | | | <3 x ULN | x (xx.x%) | x (xx.x%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | | | >=3 - <5 x ULN | x(xx.x%) | x (xx.x%) |
| AST $<3 \text{ x ULN}$ $>=3 - <5 \text{ x ULN}$ $>=5 - <10 \text{ x ULN}$ $>=10 \text{ x ULN}$ | | | >=5 - <10 x ULN | 0 | |
| <3 x ULN $x (xx.x%)$ $x (xx.x.x%)$ $x (xx.x.x%)$ | | | >=10 x ULN | 0 | 0 |
| >=3 - <5 x ULN | | | AST | | |
| >=5 - <10 x ULN 0 0 0 0 0 | | | <3 x ULN | x(xx.x%) | x (xx.x%) |
| >=5 - <10 x ULN 0 0 0 0 | | | >=3 - <5 x ULN | x (xx.x%) | x (xx.x%) |
| | | | >=5 - <10 x ULN | | |
| | | | >=10 x ULN | 0 | 0 |

Repeat for: CC All MEDI7352

ALT = alanine aminotransferase; AST = aspartate aminotransferase; IP = investigational product; n = number of subjects per category; N = number of subjects per treatment group; Nobs = number of subjects per treatment group with at least one post-baseline assessment on treatment; ULN = upper limit of normal.

Note: On-treatment assessments include assessments on or after the date of first dose of IP. Baseline is defined as the last observation recorded prior to the first dose of treatment.

Percentages are based on Nobs.

Reference Listing: 16.2.8.1





• Per Protocol, the elevations of ALT or AST and Total Bilirubin do not have to occur at the same time or within a specified time frame. That is the reason why the table is presented by Subject instead of by visit. So, if for example, one subject has ALT >= 3 - <5 x ULN at Day 1, and TBL >= 2 x ULN at Week 18, n in that cell will increase by one.

• A column for column for column dosing (column for column for col

Final 1.0 | 12-Jul-2023 | 




# 6.5. Other Safety Data

Table 14.3.5.1
Descriptive Summary of Vital Signs
Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Day 1: 15 Minutes Post-<br>Dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Day 1: 15 Minutes Post- | | | | | | |
| Dose CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

<sup>• • • •</sup> 

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment. Reference Listing: 16.2.9.1





## **Programming Notes:**

- Repeat for Supine Heart Rate, Supine Systolic Blood Pressure, Supine Diastolic Blood Pressure, Respiratory Rate, Body Temperature, Standing Heart Rate, Standing Systolic Blood Pressure, Standing Diastolic Blood Pressure.
- After Week 2 (inclusive), Supine measure are taken in sitting position. We will consider them as supine (in resting position) for calculating Change from Baseline (always at supine position).
- Include the following timepoints: Baseline, Day 1: 5 Minutes Post-Dose, Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: Pre-Dose, Week 10: 5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that Body To, and standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- A column for dosing (c) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





# Table 14.3.5.2 Descriptive Summary of ECG Data Safety Population

Parameter: xxxxx

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 1: 1 hour Post-Dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX |
| Day 1: 1 hour Post-Dose | | | | | | |
| CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are averages of the 3 replicates taken for each parameter and timepoint, and CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.9.2





## **Programming Notes:**

- Repeat for PR, QRS, QT, RR, HR (Heart Rate) and QTcF taken from external data.
- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.
- A column for column dosing (column for column for col

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.3 Summary of Overall Evaluation of Safety ECG Data

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| | , , | , | , | , , , | , , | , |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal CS | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 1: 1 hour Post-Dose | : | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal CS | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal NCS | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

CS = clinically significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = Not clinically significant.

Note: Data are taken as the most conservative from the 3 replicates taken by timepoint.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.9.2

#### **Programming Notes:**

- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.
- A column for CC dosing (CC) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.4 Covid-19 Screening Safety Population

| | | Safety Populati | | | | |
|---|---|---|---|---|---|---|
| Visit/ | Placebo | | MEDI7352 | | | Total |
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Day 1 | | | | | | |
| Subjects Screened for COVID-19 Symptoms | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Symptoms Screened: | | | | | | |
| Fever | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Cough | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Dyspnoea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Sore Throat | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Loss of Taste | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Loss of Smell | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Body Temperature Check | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Subjects with COVID-19 Swab Performed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with COVID-19 Antibody Testing Performed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Confirmed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Suspected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1.0 | 12-Jul-2023 | 





| Subjects with COVID-19 A | Antigen Testing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|---|
| Performed | | | | | | | |
| COVID-19 Positive<br>COVID-19 Negative | to<br>C | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |

COVID-19 = coronavirus disease 2019; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Percentages are n/Number of subjects by treatment group at each visit\*100.

Reference Listing: 16.2.8.8

#### **Programming Notes:**

- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.5
Summary of Sub-Scores for Total Neuropathy Score-Nurse
Safety Population

| | | Safety Populati | | | | |
|---|---|---|---|---|---|---|
| Visit/ | Placebo | | MEDI7352 | | | Total |
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| | ···· (···· ··· 0/) | ···· (···· ··0/) | ···· (···· ··0/) | (0/) | ···· (···· ···0/) | · |
| Subjects performing TNSn | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Sensory Symptom Score | | | | | | |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 3 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 3 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Motor Symptom Score | | | | | | |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Autonomic Symptom Score | | | | | | |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pin Sensibility Score | | | | | | |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 3 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1.0 | 12-Jul-2023 | 





| Vibration Sensibility Score | Vibration | Sensibility | Score |
|-----------------------------|-----------|-------------|-------|
|-----------------------------|-----------|-------------|-------|

| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 3 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

•••

Note: Percentages for subjects performing TNSn are n/Number of subjects by treatment group at each visit\*100. Percentages for each Score are n/Number of subjects by treatment group at each visit without missing score\*100

Reference Listing: 16.2.9.5

#### **Programming Notes:**

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12 and Week 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

N = number of subjects per treatment group; TNSn = Total Neuropathy Score-Nurse.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





Table 14.3.5.6

Descriptive Summary of Total Neuropathy Score-Nurse
Safety Population

| Score: xxxxx | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX |
| Day 1 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |

TNSn = Total Neuropathy Score-Nurse; n = number of subjects by treatment group at each visit for the parameter; <math>N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment. Reference Listing: 16.2.9.5

## **Programming Notes:**

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12 and Week 18.
- Include the following scores: Sensory Symptom Score, Motor Symptom Score, Autonomic Symptom Score, Pin Sensibility Score, Vibration Sensibility Score, and TNSn Total.
- A column for column

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.7 Summary of Motor and Sensory Nerve Conduction Studies Safety Population

Parameter: xxxxx

| Parameter: xxxxx | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| Week 18 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| Week 18 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Final 1.0 | 12-Jul-2023 | 





xx(xx.x%)

| Evaluation Result Baseline [1] | | | | | | |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 18 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

xx(xx.x%)

xx (xx.x%)

xx (xx.x%)

xx (xx.x%)

Note: Percentages are number of subjects by treatment group at each visit for each category /Number of subjects by treatment group for each visit\*100 Reference Listing: 16.2.9.6

## **Programming Notes:**

Abnormal

- Repeat for the following Parameters: Lower Limb right side/Motor evaluation/Amplitude, Lower Limb right side/Sensory evaluation/Amplitude, Lower Limb left side/ Sensory evaluation/Amplitude, Upper Limb right side /Motor evaluation/Amplitude, Upper Limb right side /Sensory evaluation/Amplitude, Upper Limb left side/ Motor evaluation/Amplitude, Upper Limb left side /Sensory evaluation/Amplitude. (Repeat the same combination of Location Laterality/Evaluation for Peak Latency, Conduction Velocity, Duration of action Potential).
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

xx(xx.x%)

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





Table 14.3.5.8 Summary of Strength and Deep Tendon Reflexes Safety Population

| Visit/ | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| Subjects performing SDTR assessment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ankle Dorsiflexion Strength | | | | | | |
| 0 - Normal Power | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 - Mild Weakness | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 - Moderate Weakness | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 - Severe Weakness | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 4 - Paralysis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Deep Tendon Reflexes | | | | | | |
| 0 - Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 - Ankle reflex reduced | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 - Ankle reflex absent | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 - Ankle reflex absent and knee reflex | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| reduced | 4 | | 4 00 | | ( 0() | , |
| 4 - All reflexes (both ankle and knee) absent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

n = number of subjects by treatment group at each visit for each category; N = number of subjects per treatment group; SDTR = strength and deep tendon reflexes.

Note: Percentages for each Score are n/Number of subjects by treatment group at each visit\*100

Reference Listing: 16.2.9.7

#### **Programming Notes:**

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





Table 14.3.5.9
Summary of Local Injection Site Reactions
Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Day 1: 15 Minutes after | | | | | | |
| Start of Infusion | | | | | | |
| Subjects with injection<br>Site Assessed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pain | | | | | | |
| None | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tenderness | | | | | | |
| None | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Mild | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Erythema/ Redness | | | | | | |
| None | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1.0 | 12-Jul-2023 | 





#### Induration/ Swelling

...

| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|
| Mild | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

n = number of subjects by treatment group at each visit for each category; N = number of subjects per treatment group.

Note: Percentages for each Score are n/Number of subjects by treatment group at each visit\*100

Reference Listing: 16.2.9.8

# **Programming Notes:**

- Include the following timepoints: Day 1: 15 Minutes after Start of Infusion, Day 1: 30 Minutes after Start of Infusion, Day 1: 45 Minutes after Start of Infusion, Day 1: 60 Minutes after Start of Infusion, Day 1: 2 hours after Start of Infusion, Day 1: 4 hours after Start of Infusion, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.10
Summary of Hypersensitivity/Anaphylactic Reactions
Safety Population

| | | Si | afety Population | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with any | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypersensitivity/ | AA (AA.A/0) | AA (AA.A70) | AA (AA.A/0) | AA (AA.A70) | AA (AA.A/0) | AA (AA.A70) |
| Anaphylaxis | | | | | | |
| Highest Severity Grade | | | | | | |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 20.010 | ( | (, 0) | () | ( | () | 111 (1111117,0) |
| Type of Reaction | | | | | | |
| Urticaria | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pruritus | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Rash | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Flushing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Swollen Lips, Tongue, | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Uvula and/or Vulva | | | | | | |
| Dyspnoea | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Wheeze-Bronchospasm | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Stridor | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypoxia | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypotension | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Crampy Abdominal Pain | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Vomiting | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Diarrhoea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

...

N = number of subjects per treatment group.

Reference Listing: 16.2.9.9

Final 1.0 | 12-Jul-2023 | 





# **Programming Notes:**

- Display only Type of reaction with non-missing value.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.11 Summary of Liver Diagnostic Investigations Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Liver Diagnostics<br>Performed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Type of Diagnostic Investigation | | | | | | |
| Ultrasound | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| CT | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MRI/MRCP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Flushing | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ERCP | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X-Ray | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tox Screening for | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Acetaminophen/Paracetamol | | | | | | |
| Tox Screening for Ethanol | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tox Screening, Other | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Specialist Consulted | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serology for Hepatitis A | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serology for Hepatitis B | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serology for Hepatitis C | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serology for Hepatitis D | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serology for Hepatitis E | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) |
| Serology for Cytomegalovirus | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Serology for Epstein Barr Virus | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Autoimmune Serology | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

CT = Computerized tomography; ERCP = Endoscopic retrograde cholangiopancreatography; MRI = Magnetic resonance imaging; MRCP = Magnetic resonance cholangiopancreatography; N = number of subjects per treatment group.

Reference Listing: 16.2.9.10

Final 1.0 | 12-Jul-2023 | 





# **Programming Notes:**

- Display only Diagnostic Investigations with non-missing value.
- A column for column for dosing (column for dosing (column for dosing dosing (column for dosing dos

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.12 Summary of Liver Risk Factors and Lifestyle Events Safety Population

| Safety Population | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Liver Risk Factors | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Assessed | | | | | | |
| Liver Risk Factor | | | | | | |
| Alcohol Abuse | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Increased Alcohol Consumption | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| within 1 Month of Reported Event | , | | , , | , , , | , , | , , |
| IV Drug Abuse | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tattoo | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Acupuncture | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Sexually Transmitted Diseases | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Toxic/Chemical Agent Exposure | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Travel (Areas at Risk in the Last Year) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pregnancy | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Parenteral Nutrition | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Excessive Physical Exercise | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Changes Diet/Fasting Episodes/Weight | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Loss Diet | | | | | | |
| Previous Drug Reaction | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Blood Transfusion | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Patient Exposed to Anyone with | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) |
| Jaundice in the Last Month | | | | | | |
| History of Hypotension | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |

Final 1.0 | 12-Jul-2023 | 





| Low Blood Pressure at Time of Event of Liver Injury and/or Abnormal Liver | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|
| Laboratory Value History of Liver Disease Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

IV = intravenous; N = number of subjects per treatment group.

Reference Listing: 16.2.9.10

# **Programming Notes:**

- Display only Liver Risk Factor with non-missing value.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.13 Summary of Liver Signs and Symptoms Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Liver Signs/Symptoms | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Assessed | | | | | | |
| Liver Sign/Symptom | | | | | | |
| Anorexia | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Asthenia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pyrexia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pruritus | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Jaundice | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Arthralgia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abdominal Pain | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abdominal Tenderness | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Nausea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Vomiting | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Rash | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mucosal Inflammation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Purpura | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Hepatomegaly | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Splenomegaly | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) |
| Lymphadenopathy | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Ascites | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Confusional State | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Coma | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Upper Quadrant Tenderness | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) |
| Biliary Obstruction | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Eosinophilia | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Dark Urine | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group.

Reference Listing: 16.2.9.12

Final 1.0 | 12-Jul-2023 | 





# **Programming Notes:**

- Display only Liver Signs/Symptoms with non-missing value.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.14
Summary of Infection Diagnostic Investigations
Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Infection Diagnostic Investigations | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Method | | | | | | |
| Microscopy, Culture and Sensitivity | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serological Tests | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Nucleic Acid Based Tests | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| X-Ray | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group.

Reference Listing: 16.2.9.13

## **Programming Notes:**

- Display only Methods with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.15 Summary of Infection Risk Factors and Lifestyle Events Safety Population

| | D11 | Safety Population | | | | Т-4-1 |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Infection Risk Factor Occurred | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Infection risk factor | | | | | | |
| Extensive Burns within the Last Year | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Tattoo, Piercing or Acupuncture within the | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| last Year | | | | | | |
| Sexually Transmitted Diseases | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Travel to Areas at Risk of Tuberculosis or | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tropical Diseases | | | | | | |
| Infections Related to Travel | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Blood Transfusion (within the Last Year) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Exposure to Nosocomial Pathogens within the | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Last Year | | | | | | |
| Contact History with Infection Source | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Previous BCG Immunization | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Evidence of BCG Scar | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tuberculin Skin or Quantiferon Test Confirms | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Previous Exposure or Immunity to | | | | | | |
| Tuberculosis | | | | | | |

BCG = Bacillus Calmette-Guerin; N = number of subjects per treatment group.

Reference Listing: 16.2.9.14

# **Programming Notes:**

Display only infection risk factors with non-missing value.

A column for column dosing (cc) ) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.16 Summary of Infection Signs and Symptoms Safety Population

| | Placebo | Safety Population | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| | Placedo | | | | All MEDI7352 | Total |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | (= : :::=) | (= : ===) | (= : ====) | (= : ===) | (= : :::) | (= : ===) |
| Subjects with Infection Sign/Symptom | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Occurred | | | | | | |
| Infection Sign/Symptoms | | | | | | |
| Pyrexia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Headache | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Confusional State | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Convulsion | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Rhinitis | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Oropharyngeal Pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Cough | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Productive Cough | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Haemoptysis | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Wheezing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Dyspnoea | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pleuritic Pain | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Vomiting | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Diarrhoea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Genital Discharge | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Haematuria | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Dysuria | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Hepatosplenomegaly | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Jaundice | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lymphadenopathy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1.0 | 12-Jul-2023 | 





| Rash | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|
| Petechial | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Vesicular | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Macular | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Papular | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Urticaria | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Erythema | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Blanching | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Splinter Haemorrhages | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Night sweats | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Chills | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Myalgia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Weight Decrease | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group.

Reference Listing: 16.2.9.15

# **Programming Notes:**

- Display only infection Signs/Symptoms with non-missing value.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1.0 | 12-Jul-2023 | 





#### Table 14.3.5.17 Summary of Concomitant Medications by ATC Level 2 and Preferred Name Safety Population

## **Programming Notes:**

- Same shell as Table 14.1.7.
- Change footnote Note by: "Note: Concomitant medications are defined as medications continuing or starting on or after first dose of study medication. All concomitant medications are coded using WHO drug dictionary version vMar2023. At each level of summarization (ATC Level 2 or Preferred Name), subjects who reported more than one concomitant medication were only counted once. ATC Level 2 and Preferred Name are sorted in in descending order of frequency of total, and alphabetically if same frequency".
- If uncoded ATC Level or Preferred Name, please put them as [Not Coded]
- ATC and Preferred Name texts should be in proper case in table.
- A column for column for dosing (column for dosing

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.18
Summary of Concomitant Procedures
Safety Population

| System Organ Class | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Preferred Term | (N=xxx) | CCI<br>(N=xx) | (N=xx) | CCI<br>(N=xx) | (N=xxx) |
| Any Concomitant Procedure | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| ••• | ••• | | | ••• | |
| System Organ Class n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N = number of subjects per treatment group.

Note: All Procedure terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 26.0. At each level of summarization (system organ class or preferred term), subjects having more than one Procedure term were counted only once. System organ class and preferred terms are sorted in descending order of frequency of Total column, and alphabetically if same frequency.

Reference Listing: 16.2.9.18

#### **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Sort SOC and PT (within SOC) in descending order of frequency in the Total column. Sort alphabetically in case of ties.
- Uncoded Procedure events
  - When there are uncoded Procedure Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] will be sorted at the end of the table.
- A column for column for dosing (column for dosing

Final 1.0 | 12-Jul-2023 | 





Table 14.3.5.19
Anti-Drug Antibody Results and Titre Summary by Timepoint Safety Population

| | Placebo | | MEDI7352 | | |
|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | |
| n [2] | XX | XX | XX | XX | XX |
| ADA Positive: n (%) [3] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ADA Titre | ` / | ` ' | , , | , , | , |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| Week 2 | | | | | |
| n [2] | XX | XX | XX | XX | XX |
| ADA Positive: n (%) [3] | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| ADA Titre | , | , | | , , | , |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

ADA = Anti-Drug Antibodies; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Reference Listing: 16.2.9.19

# **Programming Notes:**

- Keep in mind that in this table 'Total' column does not include placebo.
- Repeat for all scheduled post-baseline visits.
- A column for CC dosing (CC) will only be added if Stage 4 is initiated.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

<sup>[2]</sup> Number of subjects with at least one ADA assessment at the specific visit.

<sup>[3]</sup> Number of subjects with a positive result at the specific visit. The denominator for all percentages is the number of subjects with an ADA result for each visit.





Table 14.3.5.20
Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories
Safety Population

| | Salet | y Population | | | |
|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | |
| ADA Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) |
| ADA positive at baseline and/or post-baseline (ADA | | | | | |
| prevalence)<br>n/Nobs (%) [1] [2]<br>Maximum ADA Titre | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| TE-ADA positive (ADA incidence) [5] n/Nobs (%) [1] [3] Maximum ADA Titre | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |
| Treatment Induced ADA Positive | | | | | |
| n/Nobs (%) [1] [3]<br>Maximum ADA Titre | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |

Final 1.0 | 12-Jul-2023 | 





| Treatment-Boosted ADA Positive n/Nobs (%) [1] [3] | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
|---|---|---|---|---|---|
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Non-TE-ADA Positive | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx (xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | , | | , | , | , |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx |
| Both baseline and post-baseline positive | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx(xx.x%) | xx/xxx (xx.x%) |
| Maximum ADA Titre | ( ( | () | ( ) | () | ( |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Only baseline positive | | | | | |
| n/Nobs (%) [1] [4] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx (xx.x%) |
| Maximum ADA Titre | , | , | , | , | , |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx |
| TE-persistently ADA positive [6] | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | ` , | , , | , , | , , | ` / |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| • | Ť | • | ŕ | • | * |

Final 1.0 | 12-Jul-2023 | 





| TE-transiently ADA positive [7] | | | | | |
|---|---|---|---|---|---|
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |

ADA = Anti-Drug Antibodies; N = number of subjects per treatment group; TE-ADA = Treatment Emergent ADA; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

- [1] n represents the number of subjects satisfying the conditions of the specified ADA category
- [2] Nobs represents the number of subjects with any ADA result at baseline and/or post-baseline.
- [3] Nobs represents the number of subjects with an ADA result at baseline and at least one post-baseline ADA assessment.
- [4] Nobs represents the number of subjects with an ADA result at baseline.
- [5] TE-ADA positive is defined as either ADA negative at baseline and post-baseline ADA positive (Treatment Induced ADA Positive), or as ADA positive at baseline with pre-existing titre boosted during the study period (Treatment Induced ADA Positive). ADA incidence is the proportion of TE-ADA+ subjects in a population.
- [6] ADA negative at baseline and having at least 2 post-baseline ADA positive measurements with ≥16 weeks (112 days) between first and last positive, or an ADA positive result at the last available post-baseline assessment.
- [7] ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.

Reference Listing: 16.2.9.19

#### **Programming Notes:**

- If a participant has more than 1 non-missing titre during the study, the maximum titre for each participant is summarized.
- Only present summary statistics if titre is available.
- If no positive results for a particular block of the table, then the summary statistics for the titres for that particular block would not appear.
- It is assumed that participants with a missing baseline ADA result are ADA negative at baseline.
- A column for column dosing (CC) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 



Min, Max



# 7. Pharmacokinetic/Pharmacodynamic Data

Table 14.4.1 Summary of Serum MEDI7352 Concentrations PK Population

| | Tit i opulation | 11 | |
|------------------------|-----------------|--------------|--------------|
| ADA Status: xxxxxxxxxx | | | |
| | | MEDI7352 | |
| Visit/ | CCI | CCI | CCI |
| Statistic | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean $\pm$ gSD | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx |
| gCV% | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Week 2 | xx (xx) | xx (xx) | xx (xx) |
| $n (n \le LLOQ)$ | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Mean (SD) | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx |
| $gMean \pm gSD$ | XX.X | XX.X | XX.X |
| gCV% | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Median | XX, XX | XX, XX | xx, xx |
| Min, Max | | | |
| Week 4 | xx (xx) | xx (xx) | xx (xx) |
| $n (n \le LLOQ)$ | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Mean (SD) | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx |
| $gMean \pm gSD$ | XX.X | XX.X | XX.X |
| gCV% | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Median | XX, XX | XX, XX | xx, xx |

Final 1.0 | 12-Jul-2023 | 

gCV% = Geometric Coefficient of Variation (%); gMean = Geometric Mean; gSD = Geometric SD; LLOQ = Lower Limit of Quantification; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment. Reference Listing: 16.2.10.1





#### **Programming Notes:**

- Include the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours/ Pre-Dose, Week 11/ Pre-Dose, Week 10 + 14 Days/Pre-Dose; Week 18.
- Repeat the table for 'ADA Positive', 'ADA Negative' and 'Overall'.
- Any values reported as NRR (not reportable) or NS (missing) will be excluded from the summary tables.
- At a time point where less than or equal to 50% of the concentration values are NQ (below LLOQ), all NQ values will be set to the LLOQ, and all descriptive statistics will be calculated accordingly.
- At a time point where more than 50% (but not all) of the values are NQ, the gmean, gmean ± gSD and gCV% will be set to NC. The maximum value will be reported from the individual data, and the minimum and median will be set to NQ.
- If all concentrations are NQ at a time point, no descriptive statistics will be calculated for that time point. The gmean, minimum, median and maximum will be reported as NQ and the gCV% and gmean ± gSD as NC.

Final 1.0 | 12-Jul-2023 | 





#### Table 14.4.2 Summary of Serum total NGF Concentrations Safety Population

ADA Status: xxxxxxxxxx

| | Placebo | | MEDI7352 | |
|------------------|--------------|--------------|--------------|--------------|
| Visit/ | | CCI | CCI | CCI |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| $gMean \pm gSD$ | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx |
| gCV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx, xx | XX, XX | XX, XX | xx, xx |
| Week 2 | | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| $gMean \pm gSD$ | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx |
| gCV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | xx, xx |
| Week 4 | | | | |
| $n (n \le LLOQ)$ | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| $gMean \pm gSD$ | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx | x.xx to x.xx |
| gCV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX |

• • •

gCV% = Geometric Coefficient of Variation (%); gMean = Geometric Mean; gSD = Geometric SD; LLOQ = Lower Limit of Quantification; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NGF = Nerve-Growth Factor.

Reference Listing: 16.2.10.3

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.




## **Programming Notes:**

- Repeat for ADA Status: "ADA Positive", "ADA Negative" and "Overall".
- Include the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





## **Planned Listing Descriptions and Shells**

| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| Listing 16.2.1.1 - Subject Disposition - Screening Population | U |
| Listing 16.2.1.2 - Assignment to Analysis Populations - Screening Population | U |
| Listing 16.2.1.3 - Reason for IP Discontinuation and Withdrawal from the Study - Safety Population | U |
| Listing 16.2.1.4 - List of Reasons for Screening Failure - Screen Failure Population | U |
| Listing 16.2.1.5 - Subject Visits and COVID-19 Impact - Screening Population | U |
| Listing 16.2.2.1 - Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria - Screening Population | U |
| Listing 16.2.2.2 - Protocol Deviations - Safety Population | U |
| Listing 16.2.3 - Randomization and Treatment Group - Safety Population | U |
| Listing 16.2.4.1 - Demographic and Baseline Characteristics - Screening Population | U |
| Listing 16.2.4.2 - Medical History - Safety Population | U |
| Listing 16.2.4.3 - Osteoarthritis Characteristics - Screening Population | U |
| Listing 16.2.5.1 - Study Drug Administration: Individual Doses - Safety Population | U |
| Listing 16.2.6.1 - Daily Pain NRS - mITT Population | U |
| Listing 16.2.6.2 - Galer NPS - mITT Population | U |
| Listing 16.2.6.3 - DSIS - mITT Population | U |
| Listing 16.2.6.4 - SF-36 - mITT Population | U |
| Listing 16.2.6.5 - Rescue Medication Usage - mITT Population | R |
| Listing 16.2.6.6 - Patient Global Impression of Change - mITT Population | U |

Final 1.0 | 12-Jul-2023 | 





| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| CCI | U |
| Listing 16.2.7.1 - Adverse Events - Safety Population | U |
| Listing 16.2.7.2 - Treatment Emergent Adverse Events Leading to Study Drug Discontinuation Safety Population | R |
| Listing 16.2.7.3 - Treatment Emergent Adverse Events Associated with Abnormal Liver - Safety Population | R |
| Listing 16.2.7.4 - Joint Related Adverse Events of Special Interest - Safety Population | R |
| Listing 16.2.7.5 - Serious and/or Severe Infections - Safety Population | R |
| Listing 16.2.7.6 - Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of Study Drug - Safety Population | R |
| Listing 16.2.8.1 - Clinical Chemistry Laboratory Evaluations - Safety Population | U |
| Listing 16.2.8.2 - Hematology Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.3 - Coagulation Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.4 - Urinalysis Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.5 - Serology Laboratory Evaluations - Safety Population | U |
| Listing 16.2.8.6 - Pregnancy Test Results - Safety Population | U |
| Listing 16.2.8.7 - Drug Test Results - Safety Population | U |
| Listing 16.2.8.8 - COVID-19 Screening and Vaccination - Safety Population | U |
| Listing 16.2.9.1 - Vital Signs Measurements - Safety Population | U |
| Listing 16.2.9.2 - ECG Results - Safety Population | U |
| Listing 16.2.9.3 - Physical Examination Results - Safety Population | U |
| Listing 16.2.9.4 - Neurological Examination Results - Safety Population | U |
| Listing 16.2.9.5 - Total Neuropathy Score-Nurse - Safety Population | U |

Final 1.0 | 12-Jul-2023 | 





| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| Listing 16.2.9.6 - Motor and Sensory Nerve Conduction Studies - Safety Population | U |
| Listing 16.2.9.7 - Strength and Deep Tendon Reflexes - Safety Population | U |
| Listing 16.2.9.8 - Injection Site Reactions - Safety Population | U |
| Listing 16.2.9.9 - Hypersensitivity/Anaphylactic Reactions - Safety Population | U |
| Listing 16.2.9.10 - Liver Diagnostic Investigations - Safety Population | U |
| Listing 16.2.9.11 - Liver Risk Factors and Lifestyle Events - Safety Population | U |
| Listing 16.2.9.12 - Liver Signs and Symptoms - Safety Population | |
| Listing 16.2.9.13 - Infection Diagnostic Investigations - Safety Population | U |
| Listing 16.2.9.14 - Infection Risk Factors and Lifestyle Events - Safety Population | U |
| Listing 16.2.9.15 - Infection Signs and Symptoms - Safety Population | U |
| Listing 16.2.9.16 - Prior and Concomitant Medications - Safety Population | U |
| Listing 16.2.9.17 - Prohibited Concomitant Medications - Safety Population | R |
| Listing 16.2.9.18 - Concomitant Procedures - Safety Population | R |
| Listing 16.2.9.19 - Anti-drug Antibody Test Results - Safety Population | U |
| Listing 16.2.10.1 - Serum MEDI7352 Concentrations - PK Population | U |
| Listing 16.2.10.2 - Serum total NGF Concentrations - PD Population | U |

Final 1.0 | 12-Jul-2023 | 





## **Listing Change Log:**

| Output<br>Number | Date of<br>Change | Change<br>Made By<br>(initials) | Description/Rationale |
|---|---|---|---|

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.1.1 Subject Disposition Screening Population

| | D 19/ | | D | | Protocol | Consont for | Consent for | Comment |
|---|---|---|---|---|---|---|---|---|
| Culticat | Re-screened?/ | Tuaatmaant | Re-consent/ | Data/Time of | Version at | Consent for CCI | COVID-19 Safety | Current |
| Subject | Previous | Treatment | Date/Time of Initial IC/ | Date/Time of | consent/ | sample? /Date of | Measures /Date of | Protocol |
| | Subject ID | Arm | Initial Protocol Version | Informed Consent | Re-consent | Consent | Consent | version |
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | Yes/ XXXX | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | No | XXXX | Yes /<br>DDMMMYYYY/hh:mm<br>/ XXXX | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | No | XXXXX |
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | No | No | XXXXX |

COVID-19 = coronavirus disease 2019; IC = Informed Consent;

# **Programming Notes:**

• Sort by Treatment Arm/ Subject ID.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.1.2 Assignment to Analysis Populations Screening Population

| '- | Treatment | | | | | | Reason to Exclude from | Reason to Exclude from |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Arm | Screened [1] | Randomized | SAF [2] | mITT [3] | PK [4] | Safety [5] | mITT [6] |
| XXXXXX | XXXX | Yes | No | No | No | No | | |
| XXXXXX | XXXX | Yes | Yes | Yes | Yes | Yes | | |
| XXXXXX | XXXX | Yes | Yes | No | No | No | XXX | |
| XXXXXX | XXXX | Yes | Yes | Yes | Yes | Yes | | |
| XXXXXX | XXXX | Yes | Yes | Yes | No | No | XXX/ XXX | XXX/ XXX |

mITT = Modified Intent-To-Treat Population Set; NRS = numeric rating scale; PK = pharmacokinetics; SAF = Safety Population Set.

## **Programming Notes:**

- If there is more than one major deviation, please concatenate with "/"
- Sort by Treatment Arm/ Subject ID.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments.

<sup>[2]</sup> The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication.

<sup>[3]</sup> The mITT Population includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.

<sup>[4]</sup> The PK Population includes all subjects for who a pharmacokinetic sample was obtained and analysed.

<sup>[5]</sup> Major deviation reason/s to exclude from Safety Population for randomized subject.

<sup>[6]</sup> Major deviation reason/s to exclude from mITT Population for randomized subject.





# Listing 16.2.1.3 Reason for IP Discontinuation and Withdrawal from the Study Safety Population

| Subject ID/<br>Treatment<br>Arm | Study<br>Completion<br>Status | IP Discontinuation/ Study Withdrawal | Completion/<br>Discontinuation<br>Date/Time (Study Day) | Date of Last Dose | Primary<br>Reason for<br>DC/<br>Withdrawal | Blind Broken? /<br>Date/Time /<br>Reason | Reason for breaking the Blind | Study<br>Duration |
|---|---|---|---|---|---|---|---|---|
| XXXXXX<br>/XXXX | Discontinued<br>Early | IP<br>Discontinuation | DDMMMYYYY/hh:mm (XX) | | XXXXXX<br>X | Yes /<br>DDMMMYYYY<br>/hh:mm | XXXXXX | XX |
| XXXXXX<br>/XXXX | Discontinued<br>Early | IP<br>Discontinuation | DDMMMYYYY/hh:mm (XX) | | XXXXXX<br>X | No | | XX |
| XXXXXX<br>/XXXX | Completed | | DDMMMYYYY/hh:mm<br>(XX) | DDMMMYYYY | | No | | XX |
| XXXXXX<br>/XXXX | Discontinued<br>Early | Study<br>Withdrawal | DDMMMYYYY/hh:mm | | Other:<br>XXXXXX<br>X | No | | XX |
| XXXXXX<br>/XXXX | Completed | | DDMMMYYYY/hh:mm<br>(XX) | DDMMMYYYY | | No | | XX |

DC = Discontinuation; IP = Investigational product.

Note: Study Day is calculated relative to the date of first dose. Study Duration = Reference end date – date of first dose of treatment + 1.

## **Programming Notes:**

- If reason for non-completion is Other, concatenate the specify text as follows: "Other: XXXXXXXXX".
- If reason for non-completion is adverse event, concatenate with AE line number as follows: "Adverse event number X".
- For Physician decision, screen-fail and withdrawal by subject, please provide explanation if presented on the logic "Physician decision: XXX".
- Sort by Treatment Arm/ Subject ID.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Any withdrawal from the study before last IP dose (Week 10) is considered an IP discontinuation.





# Listing 16.2.1.4 List of Reasons for Screening Failure Screen Failure Population

| Subject ID | Treatment Arm | Screen failure Date<br>Date/Time | Primary Reason for Screen Failure |
|---|---|---|---|
| XXXXXX | Screen Failure | DDMMMYYYY/hh:mm | XXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY/hh:mm | XXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY/hh:mm | |
| XXXXXX | Screen Failure | DDMMMYYYY/hh:mm | Other: XXXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY/hh:mm | |

### **Programming Notes:**

- If reason for non-completion is Other, concatenate the "Primary Reason for Screen Failure" text as follows: "Other: XXXXXXXXX".
- Sort by Subject ID.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.1.5 Visits List and COVID-19 Impact Screening Population

| Subject ID/<br>Treatment<br>Arm | Visit<br>Name | Visit Date<br>(Study<br>Day) | Is COVID-<br>19<br>Pandemic<br>Ongoing? | Impacted<br>by<br>COVID-19 | Was visit<br>performed? /<br>Visit Type | Visit<br>Performe<br>d Via | VS Data<br>provided? /<br>Assessments<br>Missed? | IP dosing<br>missed due to<br>COVID-19 /<br>Details | End of<br>Treatment<br>linked to<br>COVID-19 | Subject<br>discontinued<br>due to<br>COVID-19? /<br>Details |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | Yes | Yes | Yes/<br>Delayed | On site | Y/<br>Efficacy | Y/ XXXX | Other: XXXX | Y/ XXXX |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | Yes | No | Yes | | N/ Safety | | | |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | No | Yes | Yes | Video | N/<br>Efficacy,<br>Safety | Y/ Other:<br>XXXX | | |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | No | No | No / Missed | | | | | |

COVID-19 = coronavirus disease 2019; IP = Investigational Product; VS = Vital Signs.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Visit Type: Missed, Abbreviated, Delayed.
- Visit Performed Via: Video, Phone, On Site Other: xxxxxx.
- Details on IP dosing missed: Treatment on hold due to Sponsor Decision, Subject infected with COVID-19, Subject decision, Other: xxxxxx.
- End of treatment, reason if due to COVID: Subject infected with COVID-19, Subject decision, Travel restrictions, Site closed, Study delayed/cancelled, Other: xxxxxx.
- Details on Subjects discontinuing due to COVID-19: Subject infected with COVID-19, Subject decision, End of Treatment due to Sponsor, Other: xxxxxx.
- Sort by Treatment Arm/ Subject ID.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.2.1 Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria Screening Population

| Subject ID | Treatment Arm | Enrolled | Randomized | Inclusion or Exclusion | Criteria<br>Number | Criteria Label |
|---|---|---|---|---|---|---|
| <u> </u> | TTOMINION THIN | Emoneu | Tundonnized | Entrasion | Tuniou | Cintina Bacci |
| XXXXXX | Screen Failure | Yes | No | Inclusion | XX | XXXXXXXXXXXXXXXXX |
| | | Yes | No | Exclusion | XX | XXXXXXXXXXXXXXXXX |

## **Programming Notes:**

• Sort by Subject ID.

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.2.2 Protocol Deviations Safety Population

| Subject ID Tr | eatment Arm | Analysis Population | Event Date (Study Day) | Event Type | Description | Category | Covid-<br>19<br>Related? |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Screened\RND\SAF\ I mITT | DDMMMYYYY (XX) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxx<br>xxxxxxxxxxxxxx | Non-<br>important<br>Important | Y |
| XXXXXX | XXXX | 1 | DDMMMYYYY (XX) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxx<br>xxxxx | |
| XXXXXX | XXXX | 1 | DDMMMYYYY (XX) | xxxxxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX | |

COVID-19 = Coronavirus disease 2019; mITT = Modified Intent-To-Treat Population; RND = Randomized Subjects; SAF = Safety Population. Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- The structure of this listing may change depending on the information in the protocol deviations file. In the analysis population column, include only the analysis population where subject is included in.
- Sort by Treatment Arm/ Subject ID. If date is present in file, add a column for date of event and sort by date. If no date is present, sort by category with non-important first and then important.
- Event Type: Inclusion Criteria, Exclusion Criteria, Study Drug, Assessment Safety, Assessment Efficacy, Lab/endpoint data, Visit Window, Informed Consent, Prohibited Co-Medication, Overdose/Misuse, Other.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.3 Randomization and Treatment group Safety Population

| Subject ID | Treatment Arm | Randomization Stage | Randomization Treatment | Randomization Date / Time<br>(Study Day) | Randomization<br>Number |
|---|---|---|---|---|---|
| XXXXXX | XXXX | Stage 1 | Active <b>CC</b> | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 3 | Active CCI | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 2 | Placebo | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 2 | Active OCI | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 3 | Placebo | DDMMMYYYY/hh:mm (-X) | XXXX |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

• Sort by Treatment Arm/ Subject ID.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.4.1 Demographic and Baseline Characteristics Screening Population

| Subject<br>ID | Treatment<br>Arm | Birth Date | Age<br>(years) | Sex | Surgically sterile?/ Postmenopausal? [1] | Ethnicity | Race | Weight<br>(kg) | Height (cm) | BMI<br>(kg/m²) | Fully<br>vaccinated<br>for COVID-<br>19? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | DDMMMYYY | XX | XX | | XXXXX | XXXX | XX.X | XX.X | XX.X | Y |
| XXX | XXX | MMMYYY | XX | XX | No/Yes | XXXXX | XXXX | XX.X | XX.X | XX.X | N |

COVID-19 = Coronavirus disease 2019.

Note: Height and weight are the values at Screening.

[1] Age was calculated as age at time of consent.

[2] For Female Subject Only.

## **Programming Notes:**

o Sort by Treatment Arm/ Subject ID

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.4.2 Medical History Safety Population

| | | System Organ Class/ | | _ |
|---|---|---|---|---|
| | | Preferred Term/ | Start Date (Study Day)/ | |
| Subject ID | Treatment Arm | Verbatim Term | End Date (Study Day)/ | |
| XXXXXX | XXXX | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | |
| | | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXX | MMMYYYY (X)/<br>Ongoing | |
| | | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXX | DDMMMYYYY (X)/<br>Ongoing | |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | |

MedDRA = Medical Dictionary for Regulatory Activities. Note: Study Day is calculated relative to the date of first dose. Medical History were coded using MedDRA version 26.0. Only subjects with medical history recorded are listed.

### **Programming Notes:**

- SOC & PT text should be in proper case in listing.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date of medical event.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.4.3 Osteoarthritis Characteristics Screening Population

| Subject ID | Treatment<br>Arm | Subject with OA? / Joint/<br>Area affected | Is OA<br>considered<br>CS? | Radiological<br>Investigations<br>Conducted? / Details | Joint Area<br>Investigated | Is OA<br>considered<br>RS? | K-L Score<br>Reported | Radiologic Scoring<br>System / Details/<br>Result |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Y / Shoulder | Y | Y/ Other: XXXXXX | Shoulder | Y | Grade 3 | XXXXXX/<br>XXXXXX/<br>XX |
| XXXXXX | XXXX | Y / Ankle | N | Y / MRI | Ankle | N | N | N |

CS = Clinically Significant; K-L = Kellgren-Lawrence; OA = Osteoarthritis; RS = Radiologically Significant.

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.5.1 Study Drug Administration: Individual Doses Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit<br>Name | Start<br>Date/<br>Time<br>(Study<br>Day) | End<br>Date/<br>Time<br>(Study<br>Day) | Was Infusion Performed?/ Infusion Volume (mL)[1]/ Reason not Performed | Actually<br>Administered<br>Volume (mL)<br>[2] | If Difference between [1] and [2] Volume, Reason | Any<br>Injection<br>Site<br>Reactions? | Any<br>Infusion<br>Related<br>Reactions | Infusion<br>Rate<br>(mL/<br>hour) | Rate Change<br>Justification | Reason<br>for<br>Infusion<br>Rate<br>Change |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX/<br>XXXX | XXX | DDMM<br>MYYYY<br>/hh:mm<br>(X) | DDMM<br>MYYYY<br>/hh:mm<br>(X) | Y/<br>XX | XX | | | | xx.x | | |
| XXXX/<br>XXXX | XXX | DDMM<br>MYYYY<br>/hh:mm<br>(X) | DDMM<br>MYYYY<br>/hh:mm<br>(X) | Y/<br>XX | XX | XXXXX | Y | Y | xx.x | XXXXX | XXXXX<br>XX |
| XXXX/<br>XXXX | XXX | | | N/<br>XXXXXX | | | | | | | |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / End Date.
- Rate Change Justification: Increased, Decreased, Interrupted.

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.6.1 Daily Pain NRS mITT Population

| Subject ID | Treatment Arm | Study Visit [1] | Subject Diary (ePRO) Date / Study Day | Baseline Flag [2] | DPS |
|---|---|---|---|---|---|
| XXXXXX | XXXX | Baseline | DDMMMYYYY/ (-7) | Y | X |
| | | Baseline | DDMMMYYYY/ (-6) | Y | XX |
| | | ••• | | | |
| | | Baseline | DDMMMYYYY/ (-2) | Y | XX |
| | | Baseline | DDMMMYYYY/ (-1) | Y | XX |
| | | Week 2 | DDMMMYYYY/ (13) | | XX |
| | | Week 2 | DDMMMYYYY/ (14) | | XX |
| | | ••• | | ••• | |
| | | Week X | DDMMMYYYY/(X) | | XX |
| | | ••• | | | |
| XXXXXX | XXXX | Baseline | DDMMMYYYY/ (-7) | Y | XX |
| DDG D II F | n' G DDO I | ••• | | ••• | ••• |

DPS = Daily Pain Score; ePRO = Electronic Patient-Reported Outcome; NRS = Numeric Rating Scale.

Note: Data shown in column 'DPS' are average daily pain scores on an 11-point (0-10) NRS. Study Day is calculated relative to the date of first dose.

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> Study Visit is defined as the 7-day period ending within the protocol window Day  $\pm$  3, where at least 4 days out of 7 have recorded diary pain scores.

<sup>[2]</sup> Baseline is defined as the 7-day period prior to randomization i.e., Day -7 to Day -1, inclusive. A subject is considered to have an evaluable baseline pain score if there are at least 5 days of recorded diary pain scores in the 7-day period.





#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Subject Diary Date.
- Display all measurement per Subject, starting on the Study Day = -7.
- Display Study Visit for days involved in weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Flag Baseline records only when there is at least 5 days of recorded diary pain scores in the 7-day Baseline period

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.6.2 Galer NPS mITT Population

| | | | | Collection Date / Study | | |
|---|---|---|---|---|---|---|
| Subject ID | Treatment Arm | Parameter | Study Visit | Day | Baseline Flag [1] | NPS |
| XXXXXX | XXXX | Pain intensity | Baseline | DDMMMYYYY/(X) | Y | XX |
| | | | Week 4 | $DDMMMYYYY/\left( X\right)$ | | XX |
| | | | Week 8 | $DDMMMYYYY/\left( X\right)$ | | XX |
| | | | | ••• | | XX |
| | | | Week X | $DDMMMYYYY/\left( X\right)$ | | XX |
| | | | | ••• | | XX |
| | | XXXX | Baseline | $DDMMMYYYY/\left( X\right)$ | Y | XX |
| | | ••• | ••• | | ••• | ••• |
| XXXXXX | XXXX | Pain intensity | Baseline | $DDMMMYYYY/\left( X\right)$ | Y | XX |
| | | | ••• | | ••• | |
| | | XXXX | Week X | $DDMMMYYYY/\left( X\right)$ | | XX |
| | | ••• | ••• | | ••• | |

NPS = Neuropathic Pain Scale; NRS = Numeric Rating Scale.

Note: Data shown in column 'NPS' are Pain Intensity, Unpleasantness, and Descriptor scores on an 11-point (0-10) NRS, and Pain Duration/Frequency on a 3-point NRS (1-3).

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Final 1.0 | 12-Jul-2023 | 





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter /Collection Date.
- Keep Parameter sorting from the last bullet point in this programming notes.
- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Repeat for the Parameters: Pain intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, Surface Pain Intensity (All in an 11-point NRS), and Pain Duration/Frequency (in a 3-point NRS).

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.6.3 DSIS mITT Population

#### **Programming Notes:**

- Same shell as Listing 16.2.6.1.
- Update footnote as:
  - DSIS = Daily Sleep Interference Scale; ePRO = Electronic Patient-Reported Outcome; NRS = Numeric Rating Scale.
  - Note: Data shown in column 'DSIS' are average daily Sleep Interference scores on an 11-point (0-10) NRS. Study Day is calculated relative to the date of the day of first dose.
  - [1] Study Visit is defined as the seven-day period ending within the protocol window Day  $\pm$  3.
  - [2] Baseline is defined as the seven-day period prior to randomization i.e., Day -7 to Day -1,.
- Sort by Treatment Arm/ Subject ID / Subject Diary Date.
- Display all measurement per Subject, starting on the Study Day = -7.
- Display Study Visit for days involved in weekly averages of the average Sleep interference scores for Baseline, Week 4, 8, 12, and 18.
- Flag Baseline records only when there is at least 5 days of recorded diary Sleep interference scores in the 7-day Baseline period.

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.6.4 SF-36 mITT Population

| Subject ID | Treatment<br>Arm | Parameter | Item<br>Number | Item name | Study Visit | Collection Date / Study<br>Day | Baseline<br>Flag [1] | SF-36 |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Physical functioning | 3 | Vigorous<br>Activities | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | | | | Week 12 | DDMMMYYYY/(X) | | XX |
| | | | 4 | Moderate<br>Activities | Baseline | DDMMMYYYY/(X) | Y | XX |
| | | ••• | | ••• | | | | |
| | | | - | Total | Baseline | DDMMMYYYY/(X) | Y | |
| | | | | | Week 12 | DDMMMYYYY/(X) | | XX |
| XXXXXX | XXXX | Role<br>limitations<br>due to<br>physical | | Cut Amount<br>of Time<br>Spent on<br>Work/Act | Baseline | | | |
| | | health | 13 | WOIK/ACT | | DDMMMYYYY/(X) | Y | XX |
| | | | | | Week 12 | DDMMMYYYY/(X) | | XX |
| | | | | | ••• | ••• | | |
| | | ••• | ••• | | ••• | | ••• | ••• |

SF-36 = 36-Item Short-Form Health Survey; NRS = Numeric Rating Scale.

Note: Data shown in column 'SF-36' are derived SF-36 scores and Change in General Health on a 5-point NRS (1-5).

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Final 1.0 | 12-Jul-2023 | 





#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter / Item /Collection Date.
- Keep Parameter sorting from the last bullet point in this programming notes.
- Include all data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical functioning (items 3, 4, 5, 6, 7, 8, 9, 10, 11, 12), Role limitations due to physical health (items: 13, 14, 15, 16), Role limitations due to emotional problems (items: 17, 18, 19), Vitality (Energy/fatigue) (items: 23, 27, 29, 31), Emotional well-being (items: 24, 25, 26, 28, 30), Social functioning (20, 32), Pain (items: 21, 22) and General Health (items: 1, 33, 34, 35, 36), all with values ranging from 0 to 100. Change in general Health (in a 5-point NRS, item: 2).

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.6.5 Rescue Medication Usage mITT Population

| Subject<br>ID | Treatment Arm | ATC Class (Level 2)/<br>Preferred Name/<br>Verbatim Term | Primary<br>Indication | Start Date (Study Day)/<br>End Date (Study Day) | Dose<br>(unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXX | Painful<br>Diabetic<br>Neuropathy | MMMYYYY (-XX)/<br>DDMMMYYYY (-X) | XXXX<br>unit | XXXXXXXX | XXXXX |
| | XXXX | XXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | MMMYYYY (-X)/<br>Ongoing | XXXX<br>unit | XXXXXXXX | XXXXX |
| | XXXX | XXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | DDMMMYYYY (X)/<br>DDMMMYYYY<br>(XX) | XXXX<br>unit | XXXXXXXX | XXXXX |

ATC = anatomical therapeutic chemical.

Note: Study Day is calculated relative to the date of first dose.

Medications were coded using WHO drug dictionary version vMar2023.

### **Programming Notes:**

- ATC & Preferred Name text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name .
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.6.6 Patient Global Impression of Change mITT Population

| Subject ID | Treatment Arm | Study Visit | Collection Date / Study Day | PGIC |
|---|---|---|---|---|
| XXXXXX | XXXX | Week 4 | DDMMMYYYY/(X) | XXXXXXXX |
| | | Week 8 | DDMMMYYYY/(X) | XXXXXXXX |
| | | Week 12 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 18 | DDMMMYYYY/(X) | XXXXXXX |
| XXXXXX | XXXX | Week 4 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 8 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 12 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 18 | DDMMMYYYY/(X) | XXXXXXX |

PGIC =Patient Global Impression of Change.

Note: Data shown in column 'PGIC' are Subjects ratings about overall improvement in health status.

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include all observed data on PGIC scores for Week 4, 8, 12, and 18.

Final 1.0 | 12-Jul-2023 | 







Final 1.0 | 12-Jul-2023 | 





CCI



Final 1.0 | 12-Jul-2023 | 





Listing 16.2.7.1 Adverse Events Safety Population

| Subject ID/<br>Treatment<br>Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time<br>(Study Day) | Severity/<br>Relationship | Outcome/<br>Action Taken/<br>Therapy? | AE Leading to Study DC | TEAE | Serious/<br>Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMMMYYYY/HH<br>MM (X)/<br>X DDMMMYYYY/HH<br>MM (X) | XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>Yes | No | Yes | No |
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMMMYYYY/HH<br>MM (X)/<br>X DDMONYYYY/HH:<br>MM (X) | XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>No | Yes | No | Yes / XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXX | DDMONYYYY/HH:<br>MM (X)/<br>X Ongoing | XXXXXX/<br>XXXXXX | XXXXXXXXX/<br>XXXXXXX/<br>No | No | No | Yes / XXX |

AE = adverse event; DC = discontinuation; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Study Day is calculated relative to the date of first dose. A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0





#### **Programming Notes:**

- If time missing, display "- -:- -".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e, no AEs occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).

In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Listing 16.2.7.2

Treatment Emergent Adverse Events Leading to Study Drug Discontinuation
Safety Population

#### **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update listing deleting seventh and eight columns

Listing 16.2.7.3

Treatment Emergent Adverse Events Associated with Abnormal Liver Safety Population

#### **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update listing deleting eighth column.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.7.4 Joint Related Adverse Events of Special Interest Safety Population

### **Programming Notes:**

• Same shell as Listing 16.2.7.1.

Listing 16.2.7.5 Serious and/or Severe Infections Safety Population

### **Programming Notes:**

• Same shell as Listing 16.2.7.1.

Listing 16.2.7.6

Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of Study Drug Safety Population

## **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update listing by deleting seventh column.

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.8.1 Clinical Chemistry Laboratory Evaluations Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Parameter | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Original<br>Result<br>(Unit) | Standard<br>Results<br>(unit) | Reference<br>Range<br>[1] | Baseline<br>Flag | CFB | Results<br>Assessment<br>/ Reason<br>CS | Lab ID<br>Number | Fasting<br>Status | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | Chemistry panel | XXXXXX | | | | | | | ND: xxx | | | |
| XXXXX/<br>XXXX | Albumin | XXXXXX<br>XXXXXX | DDMMMYYYY/<br>HH:MM (X)<br>DDMMMYYYY/ | XX<br>(XX)<br>XX | XX<br>(XX)<br>XX | XX - YY<br>XX - YY | Y | XX.X | H-CS/ | XXXXXXX<br>XXXXXXX | Y<br>Y | XXXX |
| | | XXXXXX | HH:MM (X)<br>DDMMMYYYY/<br>HH:MM (X) | (XX)<br>XX<br>(XX) | (XX)<br>XX<br>(XX) | XX - YY | | XX.X | XXX | XXXXXXX | Y | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX (XX) | XX (XX) | XX - YY | | XX.X | H-NCS | XXXXXXX | N | |

CFB = change from baseline; CS = clinically significant; H = High; L = Low; NCS = not clinically significant; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

[1] Reference range is used to identify potentially clinically significant laboratory values.

#### **Programming Notes:**

- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Chemistry panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Albumin, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Bicarbonate, Calcium, Chloride, Creatinine, High-Sensitivity C-Reactive Protein (hs-CRP), Estimated Glomerular Filtration Rate (eGFR by Cockcroft Gault), Serum Glucose, Lactate Dehydrogenase (LDH), Potassium, Sodium, Total Bilirubin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid.

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.8.2 Hematology Laboratory Evaluations Safety Population

#### **Programming Notes:**

- Same shell as Listing 16.2.8.1.
- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Hematology panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Absolute basophil count, absolute eosinophil count, absolute lymphocytes count, Absolute Monocyte Count, Absolute Neutrophil Count, Basophils %, Eosinophils %, Hematocrit (HCT), Hemoglobin (HGB), hemoglobin A1C (HgbA1C), Lymphocytes %, mean corpuscular hemoglobin (MHC), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), Monocytes %, Neutrophils %, Platelets, Red blood cell count (RBC), Red Cell Distribution Width, white blood cell Count (WBC).

Listing 16.2.8.3 Coagulation Laboratory Evaluations Safety Population

## **Programming Notes:**

- Same shell as Listing 16.2.8.1.
- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Coagulation panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Activated Partial Thromboplastin Clotting Time (APTT), Fibrinogen, International normalized ratio (INR), Prothrombin Time (PT).

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.8.4 Urinalysis Laboratory Evaluations Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Parameter | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Original<br>Result<br>(Unit) | Standard<br>Results<br>(unit) | Reference<br>Range<br>[1] | Baseline<br>Flag | CFB | Results<br>Assessment<br>/ Reason<br>CS | Lab ID<br>Number | Fasting<br>Status | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Urinalysis<br>panel | XXXXXX | | | | | | | ND: xxx | | | |
| XXXXX | pH/<br>Specific<br>Gravity | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX<br>(XX) | XX<br>(XX) | XX - YY | Y | | | XXXXXXX | Y | |
| | Glavity | XXXXXX | DDMMMYYYY/ | XX | XX | XX - YY | | XX.X | H-CS/ | XXXXXXX | Y | XXXX |
| | | XXXXXX | HH:MM (X) DDMMMYYYY/ | (XX)<br>XX | (XX)<br>XX | XX - YY | | XX.X | XXX | XXXXXXX | Y | |
| | | XXXXXX | HH:MM (X)<br>DDMMMYYYY/<br>HH:MM (X) | (XX)<br>XX<br>(XX) | (XX)<br>XX<br>(XX) | XX - YY | | XX.X | H-NCS | XXXXXXX | N | |
| | Blood<br>Urine/<br>Glucose/<br>Ketones/<br>Protein | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Trace | | | Y | | H-NCS | XXXXXXX | Y | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | 100<br>(mg/dL) | 100<br>(mg/dL) | | | | H-CS /<br>XXX | XXXXXXX | Y | XXXX |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Negative | | | | | | XXXXXXX | N | |

Final 1.0 | 12-Jul-2023 | 





CFB = change from baseline; CS = clinically significant; H = High; L = Low; NCS = not clinically significant; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

[1] Reference range is used to identify potentially clinically significant laboratory values.

#### **Programming Notes:**

- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Urinalysis panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Blood Urine, Glucose, Ketones, pH, Protein, Specific Gravity.

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.8.5 Serology Laboratory Evaluations Safety Population

| Subject<br>ID | Treatment<br>Arm | Was<br>Serology<br>Test<br>Collected? | Date/Time of<br>Collection<br>(Study Day) | Test (Unit) [1] | Result | Lab ID<br>Number | Fasting<br>Status | Reason not collected | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXX | Yes | DDMMMYYY<br>Y/HH:MM (X) | Hepatitis B Ag | Negative | XXXX | Y | | XXXXXXXX |
| | | | | Hepatitis C Ab | Positive | XXXX | Y | | |
| | | | | HIV-1/ -2 Ag | Not Done | XXXX | Y | XXXXXXX | |
| | | | | Quantiferon<br>Gold Plus NIL | X.XX (IU/mL) | XXXX | Y | | |

Ab = antibody; Ag = antigen; HIV = human immunodeficiency virus; TB = tuberculosis.

Note: Study Day is calculated relative to the date of first dose.

[1] if Applicable

#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date of collection / Test.
- Keep parameter sorting from the last bullet point below
- Sort Parameters in the following Order: Hepatitis B Antigen, Hepatitis C Virus Antigen, Hepatitis C Virus Antibody, HIV-1/-2 Antigen, Quantiferon Gold Plus NIL, Quantiferon Gold Plus TB, Quantiferon Gold Plus Mitogen minus NIL, Quantiferon Gold Plus TB1 minus NIL, Quantiferon Gold Plus TB2 minus NIL

Final 1.0 | 12-Jul-2023 | 




#### Listing 16.2.8.6 Pregnancy Test Results Safety Population

| | Treatment | | Was a Urine pregnancy test | Date/Time Performed (Study Day) | | |
|---|---|---|---|---|---|---|
| Subject ID | Arm | Visit | performed? | | If not, Reason | Result |
| xxxxx | xxxx | XXXXX | Xxxx | $Ddmmmyyyy/\ hh:mm\ (XX)$ | xxxx | xxxx |
| | | XXXXX | Xxxx | Ddmmmyyyy/ hh:mm (XX) | Other: xxxx | XXXX |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment.

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.8.7 Drug Test Results Safety Population

| Subject ID | Treatment<br>Arm | Was Drug Test<br>Performed? | Date/ Time Assessment<br>(Study Day) | Result | Findings | Reason Test<br>not Performed |
|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Yes | DDMMMYYYY/ HH:MM<br>(XX) | Negative | Negative | |
| XXXXXX | XXXX | Yes | DDMMMYYYY/ HH:MM<br>(XX) | Positive | Cocaine /<br>Opiates | |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Concatenate all findings by "/"
- Sort by Treatment Arm/ Subject ID / Date of assessment.

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.8.8 COVID-19 Screening Safety Population

| Subject ID/ | | COVID-19 Sx<br>Screening?/Date | | Body To Check?/ Date/ | Pody Tº | COVID-19<br>swab?/ Date/ | Cresch | COVID-19 Ab testing?/ Date/ | Ab | COVID-19 Ag testing?/ | Ag |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Arm | Visit | / Time (Study<br>Day) | Sx | Time (Study<br>Day) | Body T <sup>o</sup><br>(Unit) | Time (Study<br>Day) | Swab<br>result | Time (Study<br>Day) | testing results | Date/ Time (Study Day) | testing results |
| xxxxx/<br>xxxx | xxxx | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XXX/<br>XXX | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XX (XX) | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Yes/<br>Ddmmmyyyy<br>/ hh:mm (XX) | Xxxx |
| | xxxx | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XXX | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XX (XX) | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Yes/<br>Ddmmmyyyy<br>/ hh:mm (XX) | Xxxx |

Ab = Antibody; Ag = Antigen; COVID-19 = Coronavirus disease 2019; Sx = Symptoms; To = Temperature.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Concatenate all Symptoms by "/"
- Sort by Treatment Arm/ Subject ID / Date of assessment





#### Listing 16.2.9.1 Vital Signs Measurements Safety Population

| Subject<br>ID | Treatment<br>Arm | Parameter | Study<br>Visit | Position [1] /<br>T <sup>o</sup> Method | Date/Time of<br>Collection<br>(Study Day) | Original Result<br>(Unit) | Baseline Flag | CFB |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Body<br>Temperature | XXXXXX | XXXX | DDMMMYYYY/<br>HH:MM (X) | XX (XX) | Y | |
| | | | XXXXXX | XXXX | DDMMMYYYY/<br>HH:MM (X) | XX (XX) | | XX |
| | | | | | | ••• | | |
| | | Resting<br>Heat Rate | Screening | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | | |
| | | | Day 1:<br>Pre-Dose | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | Y | XX |
| | | | XXXXXX | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | | XX |
| | | | XXXXXX<br>XXXXXX | Sitting<br>Sitting | DDMMMYYYY/ | ND<br>XX | | XX |
| | | | ΑΛΛΑΛ | Sitting | HH:MM (X) | $\Lambda\Lambda$ | | $\Lambda\Lambda$ |

CFB = change from baseline; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

[1] Resting position measurements encompass Sitting and Supine position measurements.

Final 1.0 | 12-Jul-2023 | 





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter (Order in the second bullet point)/ Date time of collection.
- Repeat for Resting Heart Rate, Resting Systolic Blood Pressure, Resting Diastolic Blood Pressure, Respiratory Rate, Body Temperature, Standing Heart Rate, Standing Systolic Blood Pressure, Standing Diastolic Blood Pressure.
- After Week 2 (inclusive), Supine measure are taken in sitting position. We will consider them as supine (in resting position) for calculating Change from Baseline (always at supine position).
- Include the following timepoints: Screening, Baseline (Day 1: Pre-Dose), Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: Pre-Dose, Week 10: 5 minutes after Infusion Completion, Week 11, Week 12, Week 18.
- Note that Body To, and standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.9.2 ECG Results Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit | ECG Date / Time<br>(Study Day) | Tracing | ECG Result/<br>Comment | PR<br>Interval<br>(msaec) | QRS<br>duration<br>(msec) | QT<br>Interval<br>(msec) | Heart<br>Rate<br>(bpm) | QTcF<br>Interval<br>(msec) | Reason<br>Not<br>Done |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Day 1: Pre-Dose | DDMMMYYYY /<br>HH:MM (XX) | 1 | Abnormal CS/<br>xxxx | XX | XX | xx | XX | XX | |
| | | , | 2 | Abnormal CS/ | XX | XX | XX | XX | XX | |
| | | | 3 | Abnormal NCS/<br>xxxx | XX | XX | XX | XX | XX | |
| XXXXX | XXXX | DDMMMYYYY/<br>HH:MM (XX) | 1 | Normal | XX | XX | XX | XX | XX | |
| | | , , | 2 3 | Normal<br>Normal | XX<br>XX | XX<br>XX | XX<br>XX | xx<br>xx | XX<br>XX | |

CS = clinically significant; ECG = electrocardiogram; NCS = Not clinically significant

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date time of collection / Tracing
- Include the following timepoints: Day 1: Pre-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.3 Physical Examination Results Safety Population

| Subject ID | Treatment<br>Arm | Visit | Examination<br>Type | Exam Date/ Time<br>(Study Day) | Body System | Result / Change<br>from previous<br>assessment [1] | If Abnormal,<br>findings /<br>Specify<br>Changes [2] | Reason Not<br>Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Screening | Complete | DDMMMYYYY<br>/ HH:MM (XX) | Head, Neck and<br>Thyroid<br>Ears, Eyes, Nose<br>and Throat | Normal Abnormal CS | XXXXXXX | |
| | | Day 1 | Targeted | DDMMMYYYY<br>/ HH:MM (XX) | Ears, Eyes, Nose<br>and Throat | XXXXXXXXX | XXXXXXX | |

CS = Clinically Significant, NCS = Not Clinically Significant

Note: Study Day is calculated relative to the date of first dose.

[2] For targeted examination type: Specify Changes.

### **Programming Notes:**

- Keep sorting from eCRF: Head, Neck and Thyroid/ Ears, Eyes, Nose and Throat/ Chest (including breasts)/ Lungs / Heart / Lymph Nodes / Abdomen / Hepatic / Gastrointestinal / Anorectal / Genitourinary/ Skin / Musculoskeletal/Extremities / Neurological / Other.
- Complete Physical examination only at Screening, Week 12, 18 (it can also be unscheduled).
- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Body system

Final 1.0 | 12-Jul-2023 | 

<sup>[1]</sup> For targeted examination type: Change from previous assessment.





# Listing 16.2.9.4 Neurological Examination Results Safety Population

| | Treatment | | Exam Date/ Time | | | If Abnormal, | Reason Not |
|---|---|---|---|---|---|---|---|
| Subject ID | Arm | Visit | (Study Day) | Body System | Result | findings | Done |
| XXXXX | XXXX | Screening | DDMMMYYYY /<br>HH:MM (XX) | Mental Status | Normal | | |
| | | | , | Cranial Nerves | Abnormal CS | XXXXXXX | |
| | | Day 1 | DDMMMYYYY /<br>HH:MM (XX) | Cranial Nerves | XXXXXXXXX | xxxxxxxx | |

CS = Clinically Significant, NCS = Not Clinically Significant

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Keep sorting from eCRF: Mental status/ Cranial Nerves/ Motor Function/ Reflexes / Sensation and Propioception / Coordination / Other.
- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Body system

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.9.5
Total Neuropathy Score-Nurse
Safety Population

| | | | | | recording to the second | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | | Sensory | Motor | | Pin | Vibration | | |
| ID/ | | Date/ Time of | Symptom | Symptom | Autonomic | Sensibility | Sensibility | | |
| Treatment | | collection | Score | Score | Symptom | Score | Score | TNSn Total | |
| Arm | Visit | (Study Day) | (0-4) | (0-4) | Score (0–4) | (0-4) | (0-4) | (0-20) | Reason Not Done |
| XXXXX/<br>XXXX | Screening Day 1 Week 2 | DDMMMYYYY / HH:MM (XX) DDMMMYYYY / HH:MM (XX) DDMMMYYYY | XX<br>XX | XX<br>XX | XX<br>XX | XX<br>XX | XX<br>XX | XX<br>XX | |
| | WCCK Z | / HH:MM (XX) | ND | ND | ND | ND | ND | ND | XXXXXXXXXXXX |

ND = Not Done; TNSn = Total Neuropathy Score-Nurse.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.6 Motor and Sensory Nerve Conduction Studies Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit | Date / Time of<br>Collection<br>(Study Day) | Location /<br>Evaluation | Was<br>Evaluation<br>Preformed<br>?/Nerve | Amplitude<br>(Motor =<br>mV; sensory<br>= microV) /<br>Range | Peak<br>Latency<br>(msec) /<br>Range | Conduction<br>velocity<br>(msec) /<br>Range | Duration<br>of action<br>potential<br>(msec) /<br>Range | Evaluation<br>Result | If<br>Abnormal,<br>Specify | Significant Changes from Baseline? / if Yes, Specify |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX/<br>XXXX | Screening | DDMMMYY<br>YY / HH:MM<br>(XX) | Lower Limb - right side/ | Y/<br>XXXXXX<br>Y/<br>XXXXXX<br>N | xx [x.xx to x.xx] xx [x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx] | Abnormal<br>Normal | XXXXX | NA<br>NA |
| | Week 18 | DDMMMYY<br>YY/ HH:MM<br>(XX) | XXXXXX/<br>XXXXXX/<br>XXXXXX/<br>XXXXXX/<br>XXXXXX/ | Y/<br>XXXXXX<br>Y/<br>XXXXXX<br>Y/<br>XXXXXX | xx [ x.xx to x.xx ] xx [ x.xx to x.xx ] xx [ x.xx to x.xx ] | xx [x.xx to x.xx] xx [x.xx to x.xx] xx [x.xx to x.xx] xx [x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx] xx [x.xx to x.xx] xx [x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx] xx [x.xx to x.xx] xx [x.xx to x.xx] | Abnormal Normal Abnormal | XXXXX<br>XXXXX | N<br>N<br>Y/<br>XXXXXXX |

NA = Not Applicable

Note: Study Day is calculated relative to the date of first dose.





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Location Evaluation
- Keep sorting from eCRF: Lower Limb right side/Motor evaluation, Lower Limb right side/Sensory evaluation, Lower Limb left side/ Sensory evaluation, Upper Limb right side/ Sensory evaluation, Upper Limb left side/ Motor evaluation, Upper Limb left side/ Sensory evaluation, Upper Limb left side/ Sensory evaluation.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.7 Strength and Deep Tendon Reflexes Safety Population

| Subject ID | Treatment<br>Arm | Visit | Date/ Time of collection (Study Day) | Ankle Dorsiflexion<br>Strength | Deep Tendon Reflexes | Reason Not Done |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | Screening | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | |
| | | Day 1 | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | |
| | | Week 2 | DDMMMYYYY /<br>HH:MM (XX) | ND | ND | XXXXXXXXXXXX |

ND = Not Done.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.8 Injection Site Reactions Safety Population

| Subject<br>ID | Treatment<br>Arm | Visit | Date/ Time of Assessment (Study Day) | Pain | Tenderness | Erythema/redness | Induration/<br>swelling | Reason Not Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Day 1: 15<br>Minutes<br>after Start of<br>Infusion | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | XXXX | XXXX | Reason Not Done |
| | | Day 1: 30<br>Minutes<br>after Start of<br>Infusion | DDMMMYYYY /<br>HH:MM (XX) | XX | XX | XX | XX | |
| | | Week 18 | DDMMMYYYY /<br>HH:MM (XX) | ND | ND | ND | ND | xxxxxxxxxxxx |

ND = Not Done.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment
- Include the following timepoints: Day 1: 15 Minutes after Start of Infusion, Day 1: 30 Minutes after Start of Infusion, Day 1: 45 Minutes after Start of Infusion, Day 1: 60 Minutes after Start of Infusion, Day 1: 2 hours after Start of Infusion, Day 1: 4 hours after Start of Infusion, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.9 Hypersensitivity/Anaphylactic Reactions Safety Population

| Subject<br>ID | Treatment<br>Arm | AE ID<br>Number | Onset Date/Time (Study Day)/<br>Resolution Date/Time (Study<br>Day) | Type of Reaction | Severity grade for<br>the Symptom<br>with Highest<br>Severity | Onset Time<br>for Highest<br>Severity | Leading to IP Discontinuation? |
|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXX | XXXX | /HH:MM | Yes |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXX | | | No |
| | | ••• | | | | | |
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXX | XXXX | /НН:ММ | No |

AE = Adverse Event.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Onset Date/Time / Resolution Date/Time / Reaction Type.
- Keep sorting from eCRF: Urticaria, Pruritus, Rash, Flushing, Swollen lips, tongue, uvula and/or vulva, Dyspnoea, Wheeze-bronchospasm, Stridor, Hypoxia, Hypotension, Crampy abdominal pain, Vomiting, Diarrhoea, Other.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.10 Liver Diagnostic Investigations Safety Population

| | | Potential Hy's | | | Liver Diagnostic | |
|---|---|---|---|---|---|---|
| Subject ID | Treatment<br>Arm | Law Case<br>Number | Liver Diagnostic Investigation Date (Study Day) | Liver Diagnostic<br>Investigation | Investigation<br>Results | Comments |
| XXXXX | XXXX | X | DDMMMYYYY (X) | XXXX | XXXX | XXXXX |
| | | X | DDMMMYYYY(X) | XXXXX | XXXXX | |
| XXXXX | XXXX | X | DDMMMYYYY (X) | XXXXX | XXXXX | |

CT = Computerized tomography; ERCP = Endoscopic retrograde cholangiopancreatography; MRI = Magnetic resonance imaging; MRCP = Magnetic resonance cholangiopancreatography.

Note: Study Day is calculated relative to the date of first dose.

#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Diagnostic Date / Liver Diagnostic Investigation.
- Keep sorting from eCRF: Ultrasound, CT, MRI/MRCP, ERCP, Liver Biopsy, X-Ray, Tox Screening for Acetaminophen/Paracetamol, Tox Screening for Ethanol, Tox Screening, Other, Specialist (e.g. Hepatologist) Consulted, Serology for Hepatitis A, Serology for Hepatitis B, Serology for Hepatitis C, Serology for Hepatitis D, Serology for Hepatitis E, for Cytomegalovirus (CMV), Serology for Epstein Barr Virus (EBV), Autoimmune Serology, Other.

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.9.11
Liver Risk Factors and Lifestyle Events
Safety Population

| | | Potential | A Dete | Liver Risk Factor Start Date | Liver Risk | | |
|---|---|---|---|---|---|---|---|
| | Treatment | Hy's Law<br>Case | Assessment Date (Study Day) | (Study Day)/<br>Liver Risk Factor Stop Date | Factor / Reference | Liver Risk | |
| Subject ID | Arm | Number | | (Study Day) | Period | Factor Details | Comments |
| XXXXX | XXXX | 37 | DDMMMYYYY | DDMMMYYYY (X)/ | XXXX/ | | |
| | | X | (X) | DDMMMYYYY (X) | XXX | XXXX | XXXXX |
| | | v | DDMMMYYYY | DDMMMYYYY (X)/ | XXXXX/ | | |
| | | X | (X) | DDMMMYYYY (X) | XXX | XXXXX | |
| | | ••• | | | | | |
| XXXXX | XXXX | X | DDMMMYYYY | DDMMMYYYY (X)/ | XXXXX/ | | |
| | | 71 | (X) | Ongoing | XXX | XXXXX | |

Note: Study Day is calculated relative to the date of first dose.

#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Assessment Date / Liver Risk Factor Start Date / Stop Date / Liver Risk Factor.
- Keep sorting from eCRF: Alcohol Abuse, Increased Alcohol Consumption within 1 Month of Reported Event, IV Drug Abuse, Tattoo, Acupuncture, Sexually Transmitted Diseases, Toxic/Chemical Agent Exposure, Travel (Areas at Risk in the Last Year), Pregnancy, Parenteral Nutrition, Excessive Physical Exercise, Changes Diet/Fasting Episodes/Weight Loss Diet, Previous Drug Reaction (Associated with an Elevation of Liver Tests), Blood Transfusion, Subject Exposed to Anyone with Jaundice in the Last Month, History of Hypotension, Low Blood Pressure at Time of Event of Liver Injury and/or Abnormal Liver Laboratory Value, History of Liver Disease, Other.
- Concatenate comments with "/".

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.9.12 Liver Signs and Symptoms Safety Population

| | | Potential Hy's | Start Date (Study Day)/ | Liver Sign/ | |
|---|---|---|---|---|---|
| Subject ID | Treatment Arm | Law Case Number | Stop Date (Study Day) | Symptom | Intermittent |
| XXXXX | XXXX | X | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXX | N |
| | | X | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXX | N |
| | | ••• | | | |
| XXXXX | XXXX | X | DDMMMYYYY (X)/<br>Ongoing | XXXXX | Y |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Liver Sign/Symptom.
- Keep sorting from eCRF: Anorexia, Asthenia, Pyrexia, Pruritus, Jaundice, Arthralgia, Abdominal Pain, Abdominal Tenderness, Nausea, Vomiting, Rash, Mucosal Inflammation, Purpura, Hepatomegaly, Splenomegaly, Lymphadenopathy, Ascites, Confusional State, Coma, Upper Quadrant Tenderness, Biliary Obstruction, Eosinophilia, Dark Urine, Other.
- If Rash, Lymphadenopathy or Other, Concatenate Symptom with Comment as: "Rash: xxxxxx". "Lymphadenopathy: xxxxxx", "Other: xxxxxxxx"

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.13 Infection Diagnostic Investigations Safety Population

| | | AE ID | Start Date/ Time (Study Day)/ | | Examination | |
|---|---|---|---|---|---|---|
| Subject ID | Treatment Arm | Number | Stop Date/ Time (Study Day) | Method | performed | Test Result |
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXX | Y | XXXXX |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X)) | XXXXX | Y | XXXXX |
| XXXXX | XXXX | <br>X | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXX | N | XXXXX |

AE = adverse event.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Method.
- Keep sorting from eCRF: Microscopy, Culture and Sensitivity, Serological Tests, Nucleic Acid Based Tests, X-Ray, Other.

Final 1.0 | 12-Jul-2023 | 





Listing 16.2.9.14
Infection Risk Factors and Lifestyle Events
Safety Population

| Subject ID | Treatment<br>Arm | AE ID<br>Number | Start Date/ Time (Study Day)/<br>Stop Date/ Time (Study Day) | Infection Risk<br>Factor | Infection Risk<br>Occurrence | Comments |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXX | Y | XXXXX |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X)) | XXXXX | Y | XXXXX |
| XXXXX | XXXX | <br>X | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXX | N | Ongoing |

AE = adverse event; BCG = Bacillus Calmette–Guérin.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Infection Risk Factor.
- Keep sorting from eCRF: Extensive Burns within the Last Year (Thermal Burn), Tattoo, Piercing or Acupuncture within the Last Year, Sexually Transmitted Diseases, Travel to Areas at Risk of Tuberculosis or Tropical Diseases, Infections Related to Travel (e.g. Tuberculosis and Tropical Diseases), Blood Transfusion (within the Last Year), Exposure to Nosocomial Pathogens within the Last Year, Contact History with Infection Source, Previous BCG Immunization, Evidence of BCG Scar, Tuberculin Skin or Quantiferon Test Confirms Previous Exposure or Immunity to Tuberculosis.
- Fill Comment column if Infection risk factor test = Unknown Previous BCG Immunization, not done, known Sexually Transmitted Disease reference Period, or Infection risk factor specifications.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.15 Infection Signs and Symptoms Safety Population

| | | | System Organ Class/ | | | Infection | |
|---|---|---|---|---|---|---|---|
| | Treatment | AE ID | Preferred Term/ | Start Date/ Time (Study Day)/ | Clinical | Sign/Symptom | |
| Subject ID | Arm | Number | Verbatim Term | Stop Date/ Time (Study Day) | Event | Occurrence | Comments |
| XXXXX | XXXX | X | XXXXXXXXXX/ | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM | | | |
| | | Α | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (X) | XXXXX | Y | XXXXX |
| | | X | XXXXXXXXXX/ | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM | | | |
| | | 11 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (X)) | XXXXX | Y | XXXXX |
| | | ••• | | | | | |
| XXXXX | XXXX | X | XXXXXXXXXX/ | DDMMMYYYY/HH:MM (X)/<br>Ongoing | | | |
| | | Α | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | XXXXX | N | Ongoing |

AE = adverse event.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Clinical Event.
- Keep sorting from eCRF: Pyrexia, Headache, Confusional State, Convulsion, Rhinitis, Oropharyngeal Pain, Cough, Productive Cough, Haemoptysis, Wheezing, Dyspnoea, Pleuritic Pain, Vomiting, Diarrhoea, Genital Discharge, Haematuria, Dysuria, Hepatosplenomegaly, Jaundice, Lymphadenopathy, Rash, Night sweats, Chills, Myalgia, Weight Decrease.
- Fill Comment column if Maximum To (Unit) available for Pyrexia, or if site for Rash or Lymphadenopathy is known.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.16 Prior and Concomitant Medications Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Prior/<br>Concomitant<br>[1] | ATC Class (Level 2)/ Preferred Name/ Verbatim Term | Given<br>for/as | Primary<br>Indication | Start Date (Study<br>Day)/<br>End Date (Study<br>Day) | Dose (unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|---|
| XXXXXX<br>/ XXXX | Prior | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXX | Medical<br>History | XXXXXXX | MMMYYYY<br>(-XX)/<br>DDMMMYYYY<br>(-X) | XXXX unit | XXXXXX<br>XXX | XXXXX |
| | Both | XXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Prophylaxis | XXXXXXX | MMMYYYY<br>(-X)/<br>Ongoing | XXXX unit | XXXXXX<br>XXX | XXXXX |
| | Concomitant | XXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Adverse event | XXXXXXX | DDMMMYYYY<br>(X)/<br>DDMMMYYYY<br>(XX) | XXXX unit | XXXXXX<br>XXX | XXXXX |

ATC = anatomical therapeutic chemical; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

Note: Study Day is calculated relative to the date of first dose.

Medications were coded using WHO-DDE version vMar2018.

[1] Prior medications are defined as medications that started before first dose of study, whether they were stopped before first dose of study medication or not. Concomitant medications are defined as medications starting on or after first dose of study medication Both indicates medication that was started before the day of first dose and continued after.

Final 1.0 | 12-Jul-2023 | 





### **Programming Notes:**

- ATC & Preferred Name text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name.
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by Treatment ID/ Subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications)

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.17 Prohibited Concomitant Medications Safety Population

### **Programming Notes:**

- Same Shell as Listing 16.2.9.16.
- Display prohibited prior and concomitant medications provided by the Medical Coder:
- Prohibited concomitant medications:
  - NSAIDs analgesic therapies (with acetylsalicylic acid with doses >= 325 mg/day).
  - COX-2 analgesic therapies.
  - o Immunotherapeutics.
  - o Live viral or attenuated bacterial vaccines.
  - Oral, IV, intramuscular, or any other parenteral (other than oral) steroids (inhaled or topical steroids are permitted).
  - o Biologic therapeutic agents.
- Prohibited prior and/or concomitant medications:
  - o Anti-NGF therapies.
  - o Anti-TNF therapies.
- ATC & PN text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name .
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications)

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.9.18 Concomitant Procedures Safety Population

| Subject | Treatment | System Organ Class/<br>Preferred Term/ | Start Date (Study Day)/ | | Reason (derived verbatim | · |
|---|---|---|---|---|---|---|
| ID | Arm | Verbatim Term | End Date (Study Day) | Reason for Procedure | term) | Specify |
| XXXXX | XXXX | XXXXXXXXXXX/<br>XXXXXXXXXXXXXX<br>XXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX | |
| XXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX | |
| XXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>Ongoing | OTHER | OTHER | XXXXXXXXXX |

MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study Day is calculated relative to the date of first dose. All Procedure terms were coded using the MedDRA version 26.0. Concomitant Procedures are defined as medications continuing or starting on or after first dose of study medication.

# **Programming Notes:**

- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Final 1.0 | 12-Jul-2023 | 





# Listing 16.2.9.19 Anti-drug Antibody Test Results Safety Population

| Subject<br>ID | Treatment<br>Arm | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Screening<br>Status Result | ADA Titer | Confirmatory<br>Status result | Lab ID<br>Number | Comments |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Positive | XX | Positive | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Positive | XX | Positive | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Negative | XX | Negative | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Missing | | NRR | XXXXXXX | XXXX |

ADA = Anti-Drug Antibodies; NA = Not Applicable; NRR = Not Reportable Result; QNS = Quantity Not Sufficient.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- ADA titre reported as <30 (below the minimum required dilution) is a negative result for the presence of ADA.
- Include Following timepoints: Screening, Weeks 2, 4, 8, 10, 12, 18.

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.10.1 Serum MEDI7352 Concentrations PK Population

| Subject<br>ID | Treatment<br>Arm | Parameter | Study<br>Visit | Date/Time of Collection (Study Day) | Result<br>(ng/mL) | Lab ID Number | Comments |
|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | MEDI7352<br>Concentration | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | NRR | XXXXXXX | XXXX |

NA = Not Applicable; NRR = Not Reportable Result.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours: after Week 10/ Pre-Dose, Week 11: after Week 10/ Pre-Dose, Week 10 + 14 Days: after Week 10/ Pre-Dose, Week 18.

Final 1.0 | 12-Jul-2023 | 





#### Listing 16.2.10.2 Serum total NGF Concentrations Safety Population

| Subject<br>ID | Treatment<br>Arm | Parameter | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Result<br>(pg/mL) | Lab ID Number | Comments |
|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | tNGF | XXXXXX | DDMMMYYYY/ | XX | XXXXXXX | |
| | | Concentration | | HH:MM(X) | | | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | NS | XXXXXXX | XXXX |

BLLOQ = Below the Lowest Limit of Quantitation; NA = Not Applicable; ND = Not Detected; NS = No Value due to Insufficient Volume or No Sample Received; SAT = Greater than the Top of the Standard Curve; tNGF = total Nerve-Growth Factor.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.

Final 1.0 | 12-Jul-2023 | 





# **Planned Figure Descriptions and Shells**

| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Figure 14.2.1.1 - Daily Pain NRS: MCP-Mod Dose Response Model - mITT Population | U |
| Figure 14.2.1.2 - Daily Pain NRS: Boxplots at Week 12 by Treatment Group and Missing Data Handling - mITT Population | U |
| Figure 14.2.1.3 - Daily Pain NRS: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup - mITT Population | R |
| Figure 14.2.1.4 - Daily Pain NRS: MMRM LS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases mITT Population | s) - U |
| Figure 14.3.6.1.1 - Vital Sign Profiles: Mean (±SD) Systolic Blood Pressure over time - Safety Population | U |
| Figure 14.3.6.1.2 - Vital Sign Profiles: Mean (±SD) Diastolic Blood Pressure over time - Safety Population | R |
| Figure 14.3.6.1.3 - Vital Sign Profiles: Mean (±SD) Heart Rate over time - Safety Population | R |
| Figure 14.3.6.1.4 - Vital Sign Profiles: Mean (±SD) Respiratory Rate over time - Safety Population | R |
| Figure 14.3.6.1.5 - Vital Sign Profiles: Mean (±SD) Temperature over time - Safety Population | R |
| Figure 14.4.1.1 - Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 over time - PK Population | on R |
| Figure 14.4.1.2 - Pharmacokinetics: Individual Plot of Serum MEDI7352 Concentrations over time - PK Population | U |
| Figure 14.4.2.1 - Pharmacodynamics: Line Plot of Geometric Mean (with and without gSD) total NGF over time - Safety Population | R |
| Figure 14.4.2.2 - Pharmacodynamics: Individual Plot of Serum total NGF over time - Safety Population | R |

Final 1.0 | 12-Jul-2023 | 





# **Figures Change Log**

| Output<br>Number | Date of<br>Change | Change<br>Made By<br>(initials) | Description/Rationale |
|---|---|---|---|

Final 1.0 | 12-Jul-2023 | 





Figure 14.2.1.1
Daily Pain NRS: MCP-Mod Dose Response Model mITT Population

#### Weekly Average to Week 12 Daily Pain NRS CFB, Emax dose-response model



CI = Confidence Interval; CFB = Change from Baseline; DPS = Daily Pain Score; NRS = Numeric Rating Scale.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e.,

Day -7 to Day -1, inclusive. Envelope depicts 95% CI of mean dose-response. Added dots are actual doses ± 95% CI.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.

Reference Listing: 16.2.6.1

Final 1.0 | 12-Jul-2023 | 





### **Programming Notes:**

- Insert the following text as legend: "Weekly Average to Week 12 Daily Pain NRS CFB, xxxx dose-response model", with 'xxxx' as the selected dose-response model (e.g., Hyperbolic  $E_{max}$ ).
- Dose (μg/kg) in x axis and Daily Pain NRS CFB in y axis.
- Add model parameter values as an inset plot. For e.g., Sigmoid  $E_{max}$ ;  $E_0 = xxx$ ,  $E_{max} = xxx$ , ED50 = xxx,  $\lambda = xxx$ .
- The MCP-MOD approach will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

Final 1.0 | 12-Jul-2023 | 





Figure 14.2.1.2

Daily Pain NRS: Boxplots at Week 12 by Treatment Group and Missing Data Handling mITT Population

# Weekly Average CFB to Week 12 Daily Pain NRS 0 Daily Pain NRS CFB Data OBS LOCF BOCF -6 0 5 150 450 Dose (µg/kg)

BOCF = Baseline Observation Carried Forward; CFB = Change from Baseline; DPS = Daily Pain Score; LOCF = Last Observation Carried Forward; NRS = Numeric Rating Scale; OBS = Observed Cases.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

Final 1.0 | 12-Jul-2023 | 





### **Programming Notes:**

- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS".
- Dose (μg/kg) and Observed/LOCF/BOCF in x axis and Daily Pain NRS CFB in y axis.
- A level for occurrence dosing (occurrence) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





# Figure 14.2.1.3 Daily Pain NRS: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup mITT Population

CFB = Change from Baseline; DPS = Daily Pain Score; NRS = Numeric Rating Scale.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.2
- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS".
- Dose (µg/kg) in x axis, Anticonvulsant/ Antidepressant/ Both/ None in right side Co-medication labels, and Daily Pain NRS CFB in y axis.
- A level for column dosing (between column ) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Figure 14.2.1.4

Daily Pain NRS: MMRM LS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases) mITT Population

#### Weekly Average CFB to Week 12 Daily Pain NRS ± 95% CI



CFB = Change from Baseline; CI = Confidence Interval; DPS = Daily Pain Score; LS = Least Square; MMRM = Mixed Model for Repeated Measures; NRS = Numeric Rating Scale.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

Final 1.0 | 12-Jul-2023 | 





### **Programming Notes:**

- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS  $\pm$  95% CI".
- Week in x axis and Daily Pain NRS CFB in y axis.
- Include a profile for each dose treatment group.
- Include the following timepoints: Week 2, 4, 6, 8, 10, and 12.
- Extract data for this figure from the MMRM of CFB Daily Pain NRS with Observed Cases.
- A profile for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 




#### Figure 14.3.6.1.1 Vital Sign Profiles: Mean (±SD) Systolic Blood Pressure over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; SBP = Systolic Blood Pressure; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average SBP ± Standard Deviation".
- Study Visit in x axis and Systolic Blood Pressure (mmHg) in y axis.
- Include a profile for Resting SBP and another for Standing SBP.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: 7 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 7 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





#### Figure 14.3.6.1.2 Vital Sign Profiles: Mean (±SD) Diastolic Blood Pressure over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; DBP = Diastolic Blood Pressure; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average DBP ± Standard Deviation".
- Study Visit in x axis and Diastolic Blood Pressure (mmHg) in y axis.
- Include a profile for Resting DBP and another for Standing DBP.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: 7 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 7 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing will only be added if Stage 4 is initiated)

Final 1.0 | 12-Jul-2023 | 





#### Figure 14.3.6.1.3 Vital Sign Profiles: Mean (±SD) Heart Rate over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; HR = Heart Rate; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average HR  $\pm$  Standard Deviation".
- Study Visit in x axis and Heart Rate (Beats/min) in y axis.
- Include a profile for Resting HR and another for Standing HR.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: Pre-Dose, Week 10: 5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





#### Figure 14.3.6.1.4 Vital Sign Profiles: Mean (±SD) Respiratory Rate over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 4H PD = 4 hours Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

# **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average Respiratory Rate ± Standard Deviation".
- Study Visit in x axis and Respiratory Rate (Breaths/min) in y axis.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 5 minutes after Infusion Completion, Week 10 + 24 hours, Week 11, Week 12, Week 18. (Do not include Screening records).
- Make one plot with 4 profiles (one for each treatment group).
- A profile for column dosing (CC) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





#### Figure 14.3.6.1.5 Vital Sign Profiles: Mean (±SD) Temperature over time Safety Population

1H PD = 1 Hour Post-Dose; 2H PD = 2 Hours Post-Dose; 4H PD = 4 hours Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; T° = Temperature; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average Body T° ± Standard Deviation".
- Study Visit in x axis and Body Temperature (°C) in y axis.
- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: Pre-Dose, Week 10: 5 minutes after Infusion Completion, Week 10: 4 hours, Week 11, Week 12, Week 18. (Do not include Screening records).
- Make one plot with 4 profiles (one for each treatment group).
- A plot for column dosing column dosing column will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Figure 14.4.1.1

Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 Concentrations over time PK Population



ADA = Antidrug Antibodies; gMean = Geometric Mean.

PK Population = includes all subjects for who a pharmacokinetic sample was obtained and analyzed.

ADA positive represents number of participants with at least one positive ADA result.

ADA negative represents number of participants with only negative ADA results (no positive).

Reference Listing: 16.2.10.1

Final 1.0 | 12-Jul-2023 | 





#### **Programming Notes:**

- Insert the following text as upper legend: "Geometric Mean serum MEDI7352 ± Geometric Standard Deviation" for the linear plot, and "Geometric Mean serum MEDI7352" for the semi-log plot. Below legend, add legend for ADA status: "Overall", "ADA Positive", "ADA Negative".
- Insert legend with different point symbols and colors for each treatment group (CC) for the Overall plot, and a legend with different point symbols and colors for each ADA status (ADA+, ADA-) for each treatment group plot by ADA status.
- Study Visit in x axis and Serum MEDI7352 concentration (ng/mL) in y axis (in linear and log<sub>10</sub> scale, for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10: Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 10 + 14 days, Week 18.
- Make one overall plot by treatment group, and a plot for each treatment group by ADA status for a total of 4 plots.
- A line for column dosing (CC) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Figure 14.4.1.2
Pharmacokinetics: Individual Plot of Serum MEDI7352 Concentrations over time PK Population



ADA = Antidrug Antibodies.

PK Population = includes all subjects for who a pharmacokinetic sample was obtained and analyzed.

ADA positive represents number of participants with at least one positive ADA result.

ADA negative represents number of participants with only negative ADA results (no positive).

Reference Listing: 16.2.10.1

Final 1.0 | 12-Jul-2023 | 





# **Programming Notes:**

- Insert the following text as upper legend: "MEDI7352 Concentration by Subject, Treatment group, and ADA status". Below legend, add legend for Treatment Group:
- Insert legend with different colors for each ADA status (Positive/ Negative).
- Time (days) in x axis and Serum MEDI7352 concentration (ng/mL) in y axis (in linear and log<sub>10</sub> scale, for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 10 + 14 days, Week 18.
- Make one plot for each Treatment group (CO), for a total of 3 plots.
- Plots for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





# Figure 14.4.2.1 Pharmacodynamics Line Plot of Geometric Mean (with and without gSD) Serum total NGF over time Safety Population

ADA = Antidrug Antibodies; gMean = Geometric Mean; NGF = Nerve-Growth Factor. Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication. ADA positive represents number of participants with at least one positive ADA result. ADA negative represents number of participants with only negative ADA results (no positive). Reference Listing: 16.2.10.3

#### **Programming Notes:**

- Same shell as Figure 14.4.1.1
- Insert the following text as upper legend: "Geometric Mean total NGF ± Geometric Standard Deviation" for the linear plot, and "Geometric Mean total NGF" for the semi-log plot. Below legend, add legend for ADA status: "Overall", "ADA Positive", "ADA Negative".
- Insert legend with different point symbols and colors for each treatment group (Placebo, CC) for the Overall plot, and a legend with different point symbols and colors for each ADA status (ADA+, ADA-) for each treatment group plot by ADA status.
- Study Visit in x axis and Serum tNGF (pg/mL) in y axis (in linear and log10 scale for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10: Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12, Week 18.
- Make one overall plot by treatment group, and a plot for each treatment group by ADA status for a total of 5 plots .
- A plot for column dosing (column) will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 





Figure 14.4.2.2
Pharmacodynamics: Individual Plot of Serum total NGF over time
Safety Population

ADA = Antidrug Antibodies; NGF = Nerve-Growth Factor.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

ADA positive represents number of participants with at least one positive ADA result.

ADA negative represents number of participants with only negative ADA results (no positive).

Reference Listing: 16.2.10.3

#### **Programming Notes:**

- Same shell as Figure 14.4.1.2
- Insert the following text as legend: "Total NGF by Subject, Treatment group, and ADA status". Below legend, add legend for Treatment Group: [66]
- Insert legend with different colors for each ADA status (Positive/ Negative).
- Time (days) in x axis and Serum tNGF concentration (pg/mL) in y axis (in linear and log10 scale for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.
- Make one plot for each Treatment group (CC) Placebo), for a total of 4 plots.
- Plots for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.0 | 12-Jul-2023 | 



Table, Listing and Figure Shells Sponsor AstraZeneca Protocol Number D5680C00002 PCN Number MEDU177093



| Sponsor: | AstraZeneca |
|---|---|
| Protocol Title | A Randomised, Double-Blind, Placebo-Controlled, Dose-Response Study of the Efficacy and Safety of MEDI7352 in Subjects with Painful Diabetic Neuropathy |
| Development Phase | 2 |
| Protocol Numbers: | D5680C00002 |
| Premier Research PCNs: | MEDU177093 |
| Document Version: | Final Version 1.1 |
| Document Date: | 31-Aug-2023 |

# **Document History**

| Version | Date | Author | Description |
|---------|-------------|--------|---------------|
| 0.1 | 24-Mar-2023 | PPD | Draft Version |
| 0.2 | 21-Apr-2023 | PPD | Draft Version |
| 0.3 | 24-May-2023 | PPD | Draft Version |
| 1 | 12-Jul-2023 | PPD | Final Version |

Draft 1.1 | 31-Aug-2023 | 





#### Tables, Listings, and Figures Conventions

All listings, tables, and graphs will have a header showing the sponsor company name, protocol and version of delivery and a footer showing the version of SAS, the file name and path, and the source of the data (listing number).

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

#### **General Reporting Conventions**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text will not be used in tables, figures, and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing.
- Adverse events with missing MedDRA coding will have their system organ class preferred term presented as "Not Coded" and the Preferred Term presented as verbatim in the tables. The "Not Coded" frequencies will be sorted to the end of the tables. This will only be applicable for any deliveries sent before database lock (e.g., for dry runs).
- Programming notes may be inserted into the shells, these notes will not appear in the final output.

#### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xx), where appropriate.
- All population summaries for categorical variables will include all categories that were planned and for which the participants may have had a response.
- All population summaries for continuous variables will include: n, mean, SD, median, quartiles, minimum, and maximum. Other summaries (e.g., number missing, geometric mean, 95% CIs, and coefficient of variation [CV] or % CV) may be used as appropriate. The precision of the maximum and minimum will match the maximum precision in the observed data and 2 decimals for derived data unless specifically mentioned in the corresponding shell. The mean and median will have 1 additional decimal place. The SD will have 2 additional decimal places. For derived data, minimum and maximum will be reported to 2 degrees of precision. Measures of location (mean and median) will be reported to 3 degree of precision, and measures of spread will be reported to 4 degrees of precision.

Draft 1.1 | 31-Aug-2023 | 





• All percentages are rounded and reported to a single decimal point (xx.x%). Exceptions are 0 and 100 that will be displayed as 0 and 100% respectively.

#### Planned Tables, Figures and Listings

- The table and listing numbers are place holders only and will be determined when the outputs are produced.
- In all listings a blank line will be placed between each participant. Within a data listing, if an item appears line after line (e.g., repetition of participant number), then only the first occurrence will be displayed.
- In data listings, the information for 1 participant will be kept on 1 page, if possible, rather than splitting a Subjects's information across pages.

Draft 1.1 | 31-Aug-2023 | 





# **Planned Table Descriptions and Shells**

| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.1.2 Screening Population | U |
| Table 14.1.3 - Summary of Reasons for Screening Failure - Screen Failure Population | U |
| Table 14.1.4.1 - Demographics and Baseline Characteristics - Screening Population | U |
| Table 14.1.4.2 - Demographics and Baseline Characteristics - Safety Population | R |
| Table 14.1.4.3 - Demographics and Baseline Characteristics - mITT Population | R |
| Table 14.1.4.4 - Demographics and Baseline Characteristics - PK Population | R |
| Table 14.1.5.1 - Osteoarthritis Characteristics - Screening Population | U |
| Table 14.1.5.2 - Osteoarthritis Characteristics - Safety Population | R |
| Table 14.1.5.3 - Osteoarthritis Characteristics - mITT Population | R |
| Table 14.1.5.4 - Osteoarthritis Characteristics - PK Population | R |
| Table 14.1.6 - Medical History by System Organ Class and Preferred Term - Safety Population | U |
| Table 14.1.7 - Prior Medications by ATC Level 2 and Preferred Name - Safety Population | U |
| Table 14.1.8 - Protocol Deviations - Safety Population | U |
| Table 14.1.9 - Overall Study Drug Exposure - Safety Population | U |
| Table 14.2.1.1.1 - Daily Pain NRS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.1.1.2 - Daily Pain NRS: Summary Statistics (LOCF) mITT Population | R |
| Table 14.2.1.1.3 - Daily Pain NRS: Summary Statistics (BOCF) - mITT Population | R |
| Table 14.2.1.2.1 - Daily Pain NRS: Primary MCP-Mod Analysis (LOCF) - mITT Population | U |
| Table 14.2.1.2.2 - Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) - mITT Population | U |
| Table 14.2.1.3.1 - Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) - mITT Population | U |
| Table 14.2.1.3.2 - Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) - mITT Population | R |
| Table 14.2.2.1 - Galer NPS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.2.2 - Galer NPS: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.3.1 - DSIS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.3.2 - DSIS: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.4.1 - SF-36: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.4.2 - SF-36: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.5.1 - Rescue Medication Use: Summary Statistics - mITT Population | U |

Draft 1.1 | 31-Aug-2023 | 





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.2.6.1 - Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel Haenszel (Observed Cases) - mITT Population | U |
| Table 14.2.6.2 - Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.7.1 - Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases) - mITT Population | R |
| Table 14.2.7.2 - Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) - mITT Population | R |
| Table 14.2.8.1 - Patient Global Impression of Change: Summary Statistics - mITT Population | U |
| Table 14.2.8.2 - Patient Global Impression of Change: Cochran-Mantel Haenszel - mITT Population | U |
| CCI | U |
| Table 14.3.1.1 - Summary of Overall Adverse Events - Safety Population | U |
| Table 14.3.1.2 - Treatment Emergent of Adverse Events by System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.3 - Treatment Emergent of Adverse Events by Severity, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.4-Treatment Emergent Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.5 - Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.6 - Treatment Emergent Adverse Events Leading to Discontinuation of Study drug by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.1.7 - Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.1.8 - Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term - Safety Population | R |
| Table 14.3.1.9 - Treatment Emergent Adverse Events by Preferred Term - Safety Population | R |
| Table 14.3.2.1.1 - Serious Adverse Events by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.2 - Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.3 - Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.4 - Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.3.1 - Listing of Serious Adverse Events - Safety Population | U |
| Table 14.3.3.2 - Listing of Deaths - Safety Population | U |





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.3.2.2.1 - Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.2 - Potential Joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.3 - Serious and/or severe Infections by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.4 - Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.4.1 - Descriptive Summary of Clinical Chemistry - Safety Population | U |
| Table 14.3.4.2 - Shift Table of Clinical Chemistry Results - Safety Population | U |
| Table 14.3.4.3 - Descriptive Summary of Hematology - Safety Population | R |
| Table 14.3.4.4 - Shift Table of Hematology Results - Safety Population | R |
| Table 14.3.4.5 - Descriptive Summary of Coagulation - Safety Population | R |
| Table 14.3.4.6 - Shift Table of Coagulation Results - Safety Population | R |
| Table 14.3.4.7 - Descriptive Summary of Urinalysis - Safety Population | U |
| Table 14.3.4.8 - Shift Table of Urinalysis Results - Safety Population | R |
| Table 14.3.4.9 - Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin - Safety Population | U |
| Table 14.3.5.1 - Descriptive Summary of Vital Signs - Safety Population | U |
| Table 14.3.5.2 - Descriptive Summary of Digital ECG Data - Safety Population | U |
| Table 14.3.5.3 - Summary of Overall Evaluation of safety ECG Data - Safety Population | U |
| Table 14.3.5.4 - Covid-19 Screening - Safety Population | U |
| Table 14.3.5.5 - Summary of Sub-Scores for Total Neuropathy Score-Nurse - Sa fety Population | U |
| Table 14.3.5.6 - Descriptive Summary of Total Neuropathy Score-Nurse - Safety Population | U |
| Table 14.3.5.7 - Summary of Motor and Sensory Nerve Conduction Studies - Safety Population | U |
| Table 14.3.5.8 - Summary of Strength and Deep Tendon Reflexes - Safety Population | U |
| Table 14.3.5.9 - Summary of Local Injection Site Reactions - Safety Population | U |
| Table 14.3.5.10 - Summary of Hypersensitivity/Anaphylactic Reactions - Safety Population | U |
| Table 14.3.5.11 - Summary of Liver Diagnostic Investigations - Safety Population | U |
| Table 14.3.5.12 - Summary of Liver Risk Factors and Lifestyle Events - Safety Population | U |
| Table 14.3.5.13 - Summary of Liver Signs and Symptoms - Safety Population | U |
| Table 14.3.5.14 - Summary of Infection Diagnostic Investigations - Safety Population | U |
| Table 14.3.5.15 - Summary of Infection Risk Factors and Lifestyle Events - Safety Population | U |





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.3.5.16 - Summary of Infection Signs and Symptoms - Safety Population | U |
| Table 14.3.5.17 - Summary of Concomitant Medications by ATC Level 2 and Preferred Name - Safety Population | R |
| Table 14.3.5.18 - Summary of Concomitant Procedures - Safety Population | R |
| Table 14.3.5.19 - Anti-Drug Antibody Results and Titre Summary by Timepoint - Safety Population | U |
| Table 14.3.5.20 - Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories - Safety Population | U |
| Table 14.4.1 - Summary of Serum MEDI7352 Concentrations - PK Population | U |
| Table 14.4.2 - Summary of Serum total NGF Concentrations - PD Population | U |

Draft 1.1 | 31-Aug-2023 | 





# **Table Change Log**

| Output | Date of | Change Made | Description/Rationale |
|--------|---------|---------------|-----------------------|
| Number | Change | By (initials) | |

Draft 1.1 | 31-Aug-2023 | 



# 1. Demographic Data

Table 14.1.2
Subject Disposition
Screening Population

| | | Screening Population | | | |
|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | Total |
| Status | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) |
| Screening Population [1] | | | | | xx (100%) |
| Screen Failures | | | | | xx (xx.x %) |
| Enrolled Subjects | | | | | xx (xx.x %) |
| Re-screened Subjects | | | | | xx (xx.x %) |
| Re-sereened Subjects | | | | | AA (AA.A 70) |
| Randomized Subjects | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Randomized and Not Treated Subjects | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Reason for Discontinuation | , | , , | , , | , | ` ' |
| Adverse Event | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Safety Population [2] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| nITT Population [3] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Evaluable Week 12 Efficacy | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Evaluable LOCF Efficacy [4] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Not Efficacy Evaluable | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| PK Population [5] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Completed Study Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Study Treatment | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Reason for Discontinuation: | | | | | |
| Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Death | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lack of Efficacy | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lost to Follow-up | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Non-compliance with Study Drug | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Physician Decision | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pregnancy | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Progressive Disease | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Violation | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Draft 1.1 | 31-Aug-2023 | 





| Study Terminated by Sponsor | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|
| Technical Problems | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal by Subject | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| COVID-19 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Sponsor Decision | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Completed Study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawn from the Study | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reason for Discontinuation: | | | | | |
| Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Death | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lack of Efficacy | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lost to Follow-up | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

COVID-19 = Coronavirus disease 2019; LOCF = Last Observation Carried Forward; mITT = modified intent-to-treat; N = number of subjects per treatment group; PK = pharmacokinetic.

Note: Percentages are n/Number of subjects randomized\*100 as displayed in column header N, except for the screened, enrolled and re-screened where n/Number of Screening subjects\*100, and for the randomized, where n/Number of Enrolled subjects\*100.

Re-screened subjects are a subset of the Screening population.

- [1] The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments.
- [2] The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication.
- [3] The mITT Population includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.
- [4] Subjects in the mITT Population with LOCF applied for missing efficacy data at week 12,
- [5] The PK Population includes all subjects for who a pharmacokinetic sample was obtained and analyzed.

Reference Listings: 16.2.1.1, 16.2.1.2, 16.2.1.3,

### **Programming Notes:**

- Display only reasons for early discontinuation with non-missing value.
- A column for column for dosing (column for dosing





### Table 14.1.3 Summary of Reasons for Screening Failure Screen Failure Population

| • | Total<br>(N=xx) |
|---|---|
| Number of Subjects Who Don't Meet Inclusion/Exclusion Criteria | xx (xx.x%) |
| IC 01: Xxxxxxxxxxx | xx (xx.x%) |
| IC 02: Xxxxxxxxxxx | xx (xx.x%) |
| EC 01: Xxxxxxxxxxx | xx (xx.x%) |
| EC 02: Xxxxxxxxxxx | xx (xx.x%) |
| ••• | |
| Number of Subjects Who are Screen Failure for other Reason than Eligibility Criteria | xx (xx.x%) |

EC = exclusion criteria; IC = inclusion criteria; N = number of subjects.

Note: subject can be counted in more than one criterion.

Reference Listing 16.2.1.4





Table 14.1.4.1 Demographics and Baseline Characteristics Screening Population

| Variable | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Age (years) [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Age Category | | | | | |
| ≥18 - <65 years | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| ≥65 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Gender | | | | | |
| Male | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Female | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ethnicity | | | | | |
| Hispanic or Latino | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Race | | | | | |
| American Indian or Alaska Native | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Asian | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Black or African American | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| White | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Not Specified | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Screening Height (cm) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |

Draft 1.1 | 31-Aug-2023 | 





| Screening Weight (kg) | | | | | |
|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx |
| Screening BMI (kg/m²) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Female characteristics [2] | | | | | |
| Surgically sterile | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Postmenopausal | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Fully vaccinated for COVID-19 | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

BMI = Body Mass Index; COVID-19 = Coronavirus disease 2019; n = number of subjects by treatment group with collected parameter; N = number of subjects per treatment group; SD = standard deviation.

Note: The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments.

Reference Listing: 16.2.4.1

# **Programming Notes:**

- If a variable is between 2 pages, start the variable in the second page.
- Keep all possible values for each category even if no subject.
- A column for on dosing (oc) will only be added if Stage 4 is initiated.

<sup>[1]</sup> Age was calculated as age at time of consent.

<sup>[2]</sup> Percentages are n/Number of Female subjects from Analysis Population\*100





# Table 14.1.4.2 Demographics and Baseline Characteristics Safety Population

# **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.1.4.3
Demographics and Baseline Characteristics
mITT Population

### **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Table 14.1.4.4
Demographics and Baseline Characteristics
PK Population

# **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Draft 1.1 | 31-Aug-2023 | 





Table 14.1.5.1 Osteoarthritis Characteristics Screening Population

| | Placebo | | MEDI7352 | | |
|---|---|---|---|---|---|
| Variable | | CCI | CCI | CCI | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects diagnosed with Osteoarthritis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Joint(s)/Area(s) affected: | | | | | |
| Shoulder | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Elbow | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Hip | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Knee | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Ankle | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Spine | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hands | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Feet | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Other | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Osteoarthritis clinically significant | | | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Radiologic investigations conducted [1] | | | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Plain radiography | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| MRI | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Joint(s)/Area(s) investigated: | | | | | |
| Shoulder | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Elbow | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hip | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Knee | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Ankle | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Spine | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Draft 1.1 | 31-Aug-2023 | 





| Hands<br>Feet<br>Other | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
|---|---|---|---|---|---|
| Osteoarthritis radiologically significant | ( | (, 0) | () | ( | (, 0) |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | XX (XX.X%)<br>XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| NO | XX (XX.X /0) | AA (AA.A /0) | AA (AA.A /0) | AA (AA.A /0) | AA (AA.A /0) |
| Kellgren-Lawrence score reported | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 0 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 1 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Grade 2 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| No/Not applicable | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Radiologic Scoring System Used? | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

MRI = magnetic resonance imaging; N = number of subjects per treatment group.

# **Programming Notes:**

- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

<sup>[1]</sup> Subjects who reported more than one radiologic investigation within each category were only counted once. Reference Listing: 16.2.4.3





#### Table 14.1.5.2 Osteoarthritis Characteristics Safety Population

### **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column for column dosing (column dosing (column for column for

Table 14.1.5.3 Osteoarthritis Characteristics mITT Population

# **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.1.5.4 Osteoarthritis Characteristics PK Population

# **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.1.6 Medical History by System Organ Class and Preferred Term Safety Population

| System Organ Class | Placebo | | Total | | |
|---|---|---|---|---|---|
| Preferred Term | (N=xxx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xxx) |
| Any Medical History | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N = number of subjects per treatment group.

Note: All medical history terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 26.0. At each level of summarization (system organ class or preferred term), subjects having more than one medical history term were counted only once. System organ class and preferred terms are sorted in descending order of frequency of Total column, and alphabetically if same frequency.

Reference Listing: 16.2.4.2

# **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Sort SOC and PT (within SOC) in descending order of frequency in the Total column. Sort alphabetically in case of ties.
- Uncoded Medical History Events
  - o When there are uncoded Medical History Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] will be sorted at the end of the table.
- A column for column for dosing (column for dosing

Draft 1.1 | 31-Aug-2023 | 





#### Table 14.1.7 Prior Medications by ATC Class and Preferred Name Safety Population

| ATC Class [1] | Placebo | | MEDI7352 | Total | |
|---|---|---|---|---|---|
| Preferred Term | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with at Least One Prior<br>Medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Level 2 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Preferred Name n | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Level 2 n | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name 1 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Preferred Name n | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |

ATC = Anatomical Therapeutic Class; N = number of subjects per treatment group.

Note: Prior medications are defined as medications that started before first dose of study, whether they were stopped before first dose of study medication or not. All prior medications are coded using WHO drug dictionary version vMar2023. At each level of summarization (ATC Level 2 or Preferred Name), subjects who reported more than one prior medication were only counted once. ATC Level 2 and Preferred Term are sorted in descending order of frequency of total, and alphabetically if same frequency.

Reference Listing: 16.2.9.16

# **Programming Notes:**

- If uncoded ATC Level or Preferred Name, please put them as [Not Coded]
- ATC and Preferred Name texts should be in proper case in table.
- A column for column for dosing (column for dosing

<sup>[1]</sup> ATC Class is defined as ATC Level 2.





Table 14.1.8 Protocol Deviations Safety Population

| | Placebo | MEDI7352 | | | Total (N=xx) |
|---|---|---|---|---|---|
| | (N=xx) | CCI<br>(N=xx) | | | |
| Subjects With Any Important Protocol<br>Deviation/Violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 5 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 6 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| | | | , | , | , |

N = number of subjects per treatment group.

Notes: Percentages are n/Number of subjects by treatment group\*100.

Subjects with one or more deviations within a type of protocol deviation were counted only once.

Reference Listing 16.2.2.1

# **Programming Notes:**

• A column for column for column dosing (column for column for col



# 2. Exposure and Compliance

Table 14.1.9
Overall Study Drug Exposure
Safety Population

| | Placebo | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| Category/ Statistic | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) |
| Maximum Number of Doses Administered [1] | | | | | |
| 1 Dose | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 2 Doses | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 Doses | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 4 Doses | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 5 Doses | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 6 Doses | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total Duration of Exposure (days) [2] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | xx, xx |
| Total (cumulative) IP volume infused (mL) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

n = number of subjects by treatment group with collected parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

<sup>[1]</sup> Subjects are counted once for each level of dose administered.

<sup>[2]</sup> Duration of exposure (days) = min(date of last dose of treatment + 14 days or date of death) – date of first dose of treatment + 1. Reference Listing: 16.2.5.1





# **Programming Notes:**

- Add all categories even if count is 0.
- A column for column for column dosing (column for column for col

Draft 1.1 | 31-Aug-2023 | 



# 3. Primary Efficacy Analysis

Table 14.2.1.1.1
Daily Pain NRS: Summary Statistics (Observed Cases)
mITT Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx |
| Week 2 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 2 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

CFB = Change from Baseline; DPS = Daily Pain Score; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NRS = Numeric Rating Scale; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are weekly averages of the average daily pain scores on an 11-point (0-10) NRS and CFB for the same variable. Total N for the mITT population = 106 at Week 2 as Subject PPD has < 4 days of diary pain data on that visit, completing the following visits till Week 12.

[1] Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

Reference Listing: 16.2.6.1

Draft 1.1 | 31-Aug-2023 | 





# **Programming Notes:**

• Include all observed data (Not the LOCF) on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, 12 and 18.

• A column for column dosing (cc) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





# Table 14.2.1.1.2 Daily Pain NRS: Summary Statistics (LOCF) mITT Population

# **Programming Notes:**

- Same shell as Table 14.2.1.1.1.
- Include all observed and LOCF data on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Add abbreviation in footnote: LOCF = Last Observation Carried Forward.
- Add the following note in footnote: "LOCF applied to Week 12 only".
- A column for column for dosing (column dosing (column dosing (column for column for co

Table 14.2.1.1.3
Daily Pain NRS: Summary Statistics (BOCF)
mITT Population

# **Programming Notes:**

- Same shell as Table 14.2.1.1.1.
- Include all observed and BOCF data on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Add abbreviation in footnote: BOCF = Baseline Observation Carried Forward.
- Add the following note in footnote: "BOCF applied to Week 12 only".
- A column for column dosing (column

Draft 1.1 | 31-Aug-2023 | 




Table 14.2.1.2.1
Daily Pain NRS: Primary MCP-Mod Analysis (LOCF)
mITT Population

| 'MCP' s | tep |
|---------|-----|
|---------|-----|

| t value | 1-sided adjusted P-value [2] |
|---------|-------------------------------------------|
| XX.XX | 0.xxxx |
| XX.XX | 0.xxxx |
| XX.XX | 0.xxxx |
| XX.XX | 0.xxxx |
| XX.XX | 0.xxxx |
| XX.XX | 0.xxxx |
| XX.XX | 0.xxxx |
| xx.xx | 0.xxxx |
| | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX |

CFB = Change from Baseline; LOCF = Last Observation Carried Forward; MCP = Multiple Comparisons; Procedure; NRS = Numeric rating scale.

<sup>[1]</sup> ED50 = Effective Dose giving half of the asymptotic maximum effect.

<sup>[2]</sup> Multiplicity Adjusted P-value.





#### 'MOD' step [3] Selected Model xxxxxxxxxx

| Parameter | Estimate | 95% CI of Estimate [6] |
|---------------------------------------|----------|------------------------|
| ED50 | XX.X | [x.xx to x.xx] |
| ED90 [4] | XX.X | [x.xx to x.xx] |
| Asymptotic ED90 [5] | XX.X | [x.xx to x.xx] |
| Dose to achieve target (-1.25) effect | XX.X | [x.xx to x.xx] |
| Treatment effect at dose = CC | XX.X | [x.xx to x.xx] |

CI: Confidence Interval; LOCF = Last Observation Carried Forward; MCP = Multiple Comparisons; Procedure; MOD = Modelling; NRS = Numeric rating scale.

- [3] Results from the 'MOD' step will only be available in case any of the MCP tests is statistically significant.
- [4] ED90 = Effective Dose giving 90% of the effect of the maximum dose studied.
- [5] Asymptotic ED90 = Effective Dose giving 90% of the asymptotic maximum effect.
- [6] 2.5% and 97.5% quantiles taken from 100000 samples from the multivariate normal distribution for model fitted estimates and its covariance matrix. Reference Listing: 16.2.6.1

### **Programming Notes:**

• The 'MOD' step will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.





Table 14.2.1.2.2
Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | [x.xx to x.xx] | | |
| Co-Medication Type | | | 3 | | | | 0.xxxx |
| Baseline pain NRS | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | | |

ANCOVA = analysis of covariance; CFB = Change from Baseline;

CL = Confidence limits; LOCF = Last Observation Carried Forward; NRS = Numeric rating scale.

Draft 1.1 | 31-Aug-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: ANCOVA by dose using NRS baseline value and co-medication as covariates, with CFB to Week 12 (LOCF) as dependent variable.





# Least Square Means

| Treatment | Number of Subjects | LS mean [3] | 95% CI of LS mean |
|--------------|--------------------|-------------|-------------------|
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| Placebo | XX | X.XX | [ x.xx to x.xx ] |

CI = Confidence interval; LOCF = Last Observation Carried Forward; LS = least square; NRS = Numeric rating scale.

weekly average pain NRS parameter evaluated at the grand mean over each group.

Reference Listing: 16.2.6.1

# **Programming Notes:**

- Concomitant co-medication Type indicated for Painful Diabetic Neuropathy: either anticonvulsant class (pregabalin or gabapentin) or antidepressant class (duloxetine, venla faxine, or amitripty line).
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline





Table 14.2.1.3.1 Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | | | |
| Co-medication type | | | 3 | | | | 0.xxxx |
| Week | | | 6 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 18 | | | | 0.xxxx |
| Baseline pain NRS | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 local vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM = Mixed Model for Repeated Measures; NRS = Numeric rating scale.

Note: model was fitted using an unstructured covariance structure. Estimates for difference vs Placebo at Week 12.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, NRS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: Week xxxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| Placebo | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |

CI = Confidence interval; LS = least square; NRS = Numeric rating scale.

Reference Listing: 16.2.6.1

## **Programming Notes:**

- Include LSmeans and difference in LSmean with Placebo in repeated tables for the Treatment\*Week interaction.
- Rows for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline weekly average pain NRS parameter evaluated at the grand mean over each group.





# Table 14.2.1.3.2 Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) mITT Population

# **Programming Notes:**

- Same shell as Table 14.2.1.2.1, substituting "LOCF = Last Observation Carried Forward" by "BOCF = Baseline Observation Carried Forward".
- The MCP-MOD approach will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

Draft 1.1 | 31-Aug-2023 | 





# 4. Secondary Efficacy Analysis

Table 14.2.2.1
Galer NPS: Summary Statistics (Observed Cases)
mITT Population

| Parameter: xxxxx | · | | | | |
|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | Total |
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| Week 4 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 4 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

• • •

Draft 1.1 | 31-Aug-2023 | 



feel a single type of pain only sometimes



xx(xx.x%)

xx (xx.x%)

#### For Pain Duration Frequency

| Baseline [1] | | | | | |
|---|---|---|---|---|---|
| I feel a background pain all of the time and occasional flare-ups | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| I feel a single type of pain all the time | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

#### Week 4

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NPS = Neuropathic Pain Scale; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

xx(xx.x%)

xx(xx.x%)

xx(xx.x%)

Note: Data shown are Pain Intensity, Unpleasantness, and Descriptor scores on an 11-point (0-10) NRS, and Pain Duration/Frequency on a 3-point NRS (1-3), plus CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.6.2

## **Programming Notes:**

- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Repeat for the Parameters: Pain intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, Surface Pain Intensity (All in an 11-point NRS), Galer NPS Total Score (ranging from 0 to 100), and Pain Duration/Frequency (in a 3-point NRS).
- A column for occurrence dosing (occurrence dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





## Table 14.2.2.2 Galer NPS: MMRM Analysis (Observed Cases) mITT Population

### Model parameter estimates

| | | | | 2-sided 95% unadjusted Asymmetric CI | 2-sided |
|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom Standard Erro | or CL [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | XX.XXX | | |
| Co-Medication type | | | 3 | | 0.xxxx |
| Week | | | 3 | | 0.xxxx |
| Treatment | | | 3 | | 0.xxxx |
| Treatment*Week | | | 9 | | 0.xxxx |
| Baseline NPS | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 cc vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] $[x.xx to x.xx]$ | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] $[x.xx to x.xx]$ | 0.xxxx |
| MEDI7352 vs Placebo | xx.xx | XX.XX | $1 \qquad \qquad xx.xxx$ | [x.xx to x.xx] $[x.xx to x.xx]$ | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; NPS = Neuropathic Pain Scale.

Note: model was fitted using an unstructured covariance structure.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, NPS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: Week: xxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| MEDI7352 CC | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CC | XX | X.XX | [ x.xx to x.xx ] |
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 - Placebo | XX | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LS = least square; NPS = Neuropathic Pain Scale.

# **Programming Notes:**

- Include LSmeans and difference in LSmean with Placebo in repeated tables for the Treatment\*Week interaction.
- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Analysis is done for Galer NPS Total Score.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline NPS parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.2





Table 14.2.3.1
DSIS: Summary Statistics (Observed Cases)
mITT Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 4 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX |
| Week 4 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |

• • •

Reference Listing: 16.2.6.3

CFB = Change from Baseline; DSIS = Daily Sleep Interference; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are weekly averages of the average daily sleep interference scores on an 11-point (0-10) NRS and CFB for the same variable.

<sup>[1]</sup> Baseline is defined as the average of the 'non-missing' DSIS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.





# **Programming Notes:**

• Include all observed data on weekly averages of the average daily Sleep Interference score for Baseline, Week 4, 8, 12, and 18.

• A column for column dosing (column dosing dosing (column dosing do

Draft 1.1 | 31-Aug-2023 | 





## Table 14.2.3.2 DSIS: MMRM Analysis (Observed Cases) mITT Population

### Model parameter estimates

| | | | | 2-sided 95% unadjusted Asymmetric CI | 2-sided |
|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom Standard Erro | or CL [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | XX.XXX | | |
| Co-medication type | | | 3 | | 0.xxxx |
| Week | | | 3 | | 0.xxxx |
| Treatment | | | 3 | | 0.xxxx |
| Treatment*Week | | | 9 | | 0.xxxx |
| Baseline DSIS | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] $[x.xx to x.xx$ | ] 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] $[x.xx to x.xx$ | ] 0.xxxx |
| MEDI7352 CCI vs Placebo | xx.xx | XX.XX | 1 xx.xxx | [x.xx to x.xx] $[x.xx to x.xx$ | ] 0.xxxx |
| Model residual standard deviation | XX.XX | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; DSIS = Daily Sleep Interference.

Note: model was fitted using an unstructured covariance structure.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, DSIS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: Week xxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | XX | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LS = least square.

# **Programming Notes:**

- Include LS means and difference in LS mean with Placebo in repeated tables for the Treatment\*Week interaction.
- Include all observed data on weekly average DSIS for Baseline, Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline weekly average DSIS parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.3





Table 14.2.4.1 SF-36: Summary Statistics (Observed Cases) mITT Population

Parameter: xxxxx

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | • |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| Week 12 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Week 12 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

• • •

Draft 1.1 | 31-Aug-2023 | 





## When parameter is "Change in general Health"

| Baseline [1] | | | | | |
|---|---|---|---|---|---|
| Much better now than one year ago | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Somewhat better now than one year ago | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| About the same as one year ago | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Somewhat worse now than one year a go | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Much worse now than one year ago | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

#### Week 12

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NRS = numeric rating scale; SD = standard deviation; SF-36 = 36-Item Short-Form Health Survey; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are derived SF-36 scores and Change in General Health on a 5-point NRS (1-5), plus CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.6.4

#### **Programming Notes:**

- Include all observed data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Vitality (Energy/fatigue), Emotional well-being, Social functioning, Pain and General Health (from 0 to 100), Physical Health Summary, Mental Health Summary, and Change in general Health (in a 5-point NRS).
- A column for column dosing (cc) will only be added if Stage 4 is initiated.





## Table 14.2.4.2 SF-36: MMRM Analysis (Observed Cases) mITT Population

Model parameter estimates: xxxxxxxx

| | | | | 2-sided 95% unadjuste | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom Standard Error | r CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | XX.XXX | | | |
| Co-medication type | | | 3 | | | 0.xxxx |
| Week | | | 1 | | | 0.xxxx |
| Treatment | | | 3 | | | 0.xxxx |
| Treatment*Week | | | 3 | | | 0.xxxx |
| Baseline SF-36 | XX.XX | XX.XX | 1 xx.xxx | [ x.xx to x.xx ] | | 0.xxxx |
| MEDI7352 cc vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [ x.xx to x.xx ] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; SF-36 = 36-Item Short-Form Health Survey.

Note: model was fitted using an unstructured covariance structure.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Treatment, SF-36 baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: xxxxxxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| MEDI7352 CC | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LS = least square.

#### **Programming Notes:**

- Include LSmeans and difference in LSmean with Placebo..
- Include all observed data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical Health Summary, and Mental Health Summary Add parameter name after 'Model parameter estimates:' and after 'Least Square Means:'
- Rows for column dosing (column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline SF-36 parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.4





Table 14.2.5.1 Rescue Medication Use: Summary Statistics mITT Population

| Variable | Placebo | | MEDI7352 | Total | |
|---|---|---|---|---|---|
| | • | CCI | CCI | CCI | • |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Number of subjects taking any rescue medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of subjects taking any permitted rescue medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of days rescue<br>medication was used [1] | | | | | |
| n<br>Mean (SD) | xx<br>xx.x (xx.xx) | xx<br>xx.x (xx.xx) | xx<br>xx.x (xx.xx) | xx<br>xx.x (xx.xx) | xx<br>xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Cumulative consumption of | | | | | |
| Paracetamol Rescue Medication | | | | | |
| (mg) [2] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Paracetamol Rescue Medication<br>Average Daily Dose (mg) [3] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Draft 1.1 | 31-Aug-2023 | 





Number of subjects taking any prohibited rescue medication

xx(xx.x%)

xx (xx.x%)

xx (xx.x%)

xx (xx.x%)

xx(xx.x%)

N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

- [1] Each day on which permitted rescue medication was used at least once is counted.
- [2] Calculated as the total dose of paracetamol rescue medication (mg).
- [3] Calculated as: cumulative consumption of paracetamol rescue medication (mg) /total number of days rescue medication was used.

Reference Listing: 16.2.6.5

# **Programming Notes:**

- A column for column dosing (column dosing (column dosing (column dosing (column dosing (column dosing (column dosing dosing (column dosing dosing dosing (column dosing
- Refer to

Draft 1.1 | 31-Aug-2023 | 





# Table 14.2.6.1 Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel Haenszel (Observed Cases) mITT Population

#### Cochran-Mantel-Haenszel Test

| Treatment/ Category | Number of<br>Subjects (%) | Risk Difference [1] | 95% CI of Risk<br>Difference | 2-sided<br>P-value [2] |
|---|---|---|---|---|
| Placebo (n = xx) >=30% decrease from Baseline | xx (xx.x%) | | | |
| MEDI7352 (n = xx)<br>>=30% decrease from Baseline | xx (xx.x%) | x.xx | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 (n = xx)<br>>=30% decrease from Baseline | xx (xx.x%) | x.xx | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 (n = xx)<br>>=30% decrease from Baseline | xx (xx.x%) | x.xx | [x.xx to x.xx] | 0.xxxx |

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

## **Programming notes:**

• Include all observed data for Week 12.

<sup>[1]</sup> Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

<sup>[2]</sup> P-value < 0.05 indicates a significant association between number of subjects with >=30% decrease from Baseline and treatment across strata. Note: a separate CMH test is performed for each dose versus placebo at Week 12. Reference Listing: 16.2.6.1





#### Table 14.2.6.2 Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) mITT Population

#### Model parameter estimates

| Parameter | Estimate | Z value | Degrees of freedom | Standard Error | 2-sided 95% CL | 2-sided<br>P-value [2] |
|---|---|---|---|---|---|---|
| Intercept | XX.XX | XX.XX | | XX.XXX | | |
| Co-medication type | | | 3 | | | 0.xxxx |
| Week | | | 3 | | | 0.xxxx |
| Treatment | | | 3 | | | 0.xxxx |
| Treatment*Week | | | 9 | | | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | 0.xxxx |
| Dispersion | XX.XX | | | | | |

CL = Confidence limits; GEE: Generalized Estimation Equations; NRS = Numeric rating scale.

Note: model was fitted using a first-order autoregressive covariance structure. Estimates for MEDI7352 dose vs placebo and for 2-sided 95% CL displayed in odds ratio scale.

Reference Listing: 16.2.6.1

# **Programming notes:**

- Include all observed data for Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: GEE using Time, Treatment, Treatment\*Time and Co-medication type as covariates, with dependent binary variable indicating whether weekly average pain NRS has >=30% decrease from Baseline.





Table 14.2.7.1
Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases)

#### mITT Population

#### Cochran-Mantel-Haenszel Test

| Treatment/ | Number of | D: 1 D:00 [1] | 95% CI of Risk | 2-sided |
|---|---|---|---|---|
| Category | Subjects (%) | Risk Difference [1] | Difference | P-value [2] |
| Placebo $(n = xx)$ | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | | | |
| MEDIA252 ( ) | | | | |
| MEDI7352 | ( 0() | | | |
| >=50% decrease from Baseline | XX (XX.X%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| $MEDI7352 \bigcirc (n = xx)$ | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| | , , | | | |
| MEDI7352 | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

# **Programming notes:**

• Include all observed data for Week 12.

<sup>[1]</sup> Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

<sup>[2]</sup> P-value < 0.05 indicates a significant association between number of subjects with >=50% decrease from Baseline and treatment across strata. Note: a separate CMH test is performed for each dose versus placebo at Week 12. Reference Listing: 16.2.6.1





#### Table 14.2.7.2 Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) mITT Population

# **Programming notes:**

- Same shell as Table 14.2.6.2. Change footnote in [2] as: "p-value is derived from the following model: GEE using Time, Treatment, Treatment\*Time and Co-medication type as covariates, with dependent binary variable indicating whether weekly average pain NRS has >=50% decrease from Baseline. Note: model was fitted using an unstructured covariance structure, with 'MEDI7352 color and 'MEDI7352 treatment groups, together with co-medication categories (both types at the same time and none) dropped from the analysis to make the generalized Hessian matrix positive definite. Estimates for MEDI7352 dose vs placebo and for 2-sided 95% CL displayed in odds ratio scale."
- Include all observed data for Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.2.8.1
Patient Global Impression of Change: Summary Statistics mITT Population

| | Placebo | Placebo MEDI7352 | | | |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Week 4 | | | | | |
| Number of PGIC Responders | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Very Much Improved | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Much Improved | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Minimally Improved | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No change | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Minimally Worse | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Much Worse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Very Much Worse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

Week 8

...

N = number of subjects per treatment group; PGIC = Patient Global Impression of Change.

Note: Percentages for Number of subjects in the different improvement categories relative to baseline are n/Number of Subjects by treatment group at each visit \*100.

Reference Listing: 16.2.6.6

# **Programming notes:**

- Include all observed data on PGIC scores for Week 4, 8, 12 and 18.
- A column for column for dosing (column for dosing

Draft 1.1 | 31-Aug-2023 | 





# Table 14.2.8.2 Patient Global Impression of Change: Cochran-Mantel Haenszel mITT Population

Cochran-Mantel-Haenszel Test: MEDI7352 xxx μg/kg vs Placebo

| Visit/ | Number of | | 95% CI of Risk | 2-sided |
|---|---|---|---|---|
| Category | Patients (%) | Risk Difference [1] | Difference | P-value [2] |
| Placebo, Week $4 (n = xx)$ | | | | |
| Improved relative to Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 4 $(n = xx)$ | | | | |
| Improved relative to Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 8 (n = xx) | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 12 $(n = xx)$ | | | | |
| Improved relative to Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |

Draft 1.1 | 31-Aug-2023 | 





Placebo, Week 18 (n = xx)

Improved relative to Baseline xx (xx.x%)

MEDI7352 xxx  $\mu$ g/kg, Week 4 (n = xx)

Improved relative to Baseline xx(xx.x%) x.xx [x.xx to x.xx] 0.xxxx

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

[1] Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

[2] P-value < 0.05 indicates a significant association between improvement relative to Baseline and treatment across strata.

Note: median Baseline Pain NRS was calculated from subjects having valid NRS data on at least one of the above four post-baseline visits. Note: a separate CMH test is performed for each dose versus placebo.

Reference Listing: 16.2.6.6

# **Programming Notes:**

• Include all observed data on PGIC scores for Week 4, 8, 12 and 18.

Draft 1.1 | 31-Aug-2023 | 





# 5. Exploratory Efficacy Analyses



Draft 1.1 | 31-Aug-2023 | 





CCI

Draft 1.1 | 31-Aug-2023 | 





# 6. Safety and Tolerability

# 6.1. Displays of Adverse Events

Table 14.3.1.1 Summary of Overall Adverse Events Safety Population

| - | Placebo | MEDI7352 | | | | Total |
|---|---|---|---|---|---|---|
| Category | (N=xx) | CCI<br>(N=xx) | (N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with any AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE TEAE categorized as Mild TEAE categorized as Moderate TEAE categorized as Severe | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Subjects with any SAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any SAE possibly related to IP [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE leading to Discontinuation of IP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE related to IP<br>TEAE categorized as Mild related to IP<br>TEAE categorized as Moderate related<br>to IP<br>TEAE categorized as Severe related to<br>IP | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Subjects with any SAE leading to Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Draft 1.1 | 31-Aug-2023 | 





AE = adverse event; IP = Investigational product, N = number of subjects per treatment group; SAE = serious adverse event; TEAE = treatment emergent adverse event.

[1] Possibly related is defined as with reasonable possibility that the AE was caused by the IP, as assessed by investigator.

Note: Subjects who reported more than one adverse event within each category were only counted once. A TEAE is defined as an adverse event with an onset at the time of or following the start of treatment with IP. For TEAEs categorized by severity, subjects were counted at the maximum severity. Reference Listing: 16.2.7.1, 16.2.7.2, 16.2.7.3, 16.2.7.4

# **Programming Notes:**

• A column for column for dosing (column for dosing

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.1.2
Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| System Organ Class Preferred Term | Placebo | | Total | | | |
|---|---|---|---|---|---|---|
| | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | All MEDI7352<br>(N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1 Preferred Term 1 | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx |
| Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx |
| System Organ Class 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 Preferred Term 2 | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx |
| Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 3 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT category; N = number of subjects per treatment group; IP = investigational product; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Note: Results are n (n/N \* 100) m is number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing: 16.2.7.1





# **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table.
- A column for column for column dosing (column for column for col

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.1.3
Treatment Emergent Adverse Events by Severity, System Organ Class and Preferred Term Safety Population

| System Organ Class | DI 1 | | Total | | | |
|---|---|---|---|---|---|---|
| Preferred Term | Placebo | | MEDI7352 | | | |
| Severity | | CCI | CCI | CCI | All MEDI7352 | (N=xx) |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | |
| Subjects with at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT/Severity category; N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Note: Results are n (n/N \* 100).

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT at the maximum severity.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing 16.2.7.1





# **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Present only severity categories with at least one subject.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 




Table 14.3.1.4

Treatment Emergent Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term Safety Population

| Placebo | | Total | | | |
|---|---|---|---|---|---|
| (N=vv) | (N=vv) | (N=vv) | (N=vv) | All MEDI7352 | (N=xx) |
| (11-11) | (11-XX) | (11-XX) | (IV-XX) | (IN-XX) | (11-11) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xx) CCI xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xx) CCI (N=xx) CCI (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xx) CCI (N=xx) CCI (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xx) CCI (N=xx) CCI (N=xx) All MEDI7352 (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) |

• • •

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT/Relatedness category; N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

[1] Related is defined as reasonable possibility that the AE was caused by investigational product, as a ssessed by the investigator. If investigator's assessment is missing the event is judged as related.

Note: Results are n (n/N \*100).

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT for the most related AE.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing 16.2.7.1





- SOC and PT texts should be in proper case in table.
- Present only severity categories with at least one subject.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A column for column for dosing (column for dosing

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.1.5
Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term Safety Population

Treatment: xxxxxxx

| | ADA | | | Non-TE- | TE<br>Persistently | TE<br>Transiently | Post-Baseline and Baseline | Only Baseline |
|---|---|---|---|---|---|---|---|---|
| System Organ Class Preferred Term | Negative (N=xx) n (n/N * 100) m | ADA Positive (N=xx) n (n/N * 100) m | TE-ADA + (N=xx) n (n/N * 100) m | NOII-1E-<br>ADA +<br>(N=xx)<br>n (n/N * 100) m | ADA + (N=xx) n (n/N * 100) m | ADA + (N=xx) n (n/N * 100) m | Positive (N=xx) n (n/N * 100) m | Positive (N=xx) n (n/N * 100) m |
| | II (II/14 100) III | 11 (11/11 100) 111 | II (II/IV 100) III | II (II/IV 100) III | II (II/I 100) III | II (II/14 100) III | II (II/11 100) III | 11 (11/11 100) 111 |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1<br>Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx |
| System Organ Class 2<br>Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx |
| System Organ Class 3 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx |

AE = adverse event; ADA = Anti-Drug Antibodies; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT category; N = number of subjects per ADA status category; PT = Preferred Term; SOC = System Organ Class; TE-ADA + = Treatment emergent ADA positive; TEAE = treatment-emergent adverse event.

ADA categories are defined in the Statistical Analysis Plan.

Note: Results are n (n/N \*100) m is number of events.

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

Table is sorted by international order for SOC, and alphabetically for PT.

Reference Listing: 16.2.7.1





- SOC and PT texts should be in proper case in table.
- Repeat for Placebo, CCI and Overall.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A table for column dosing (column dosing will only be added if Stage 4 is initiated.

#### Table 14.3.1.6

Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One TEAE leading to IP discontinuation".
- Update Reference Listing to 16.2.7.2.
- A column for CC dosing (CC) will only be added if Stage 4 is initiated.

#### Table 14.3.1.7

Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One Non-Serious TEAEAE".
- Update footnote adding: "The 5% threshold for an AE to be displayed is taken from the Total column."
- Update Reference Listing to 16.2.7.1.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.1.8

Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term Safety Population

| | | | Safety Topulatio | 11 | | |
|---|---|---|---|---|---|---|
| | Placebo | | M | EDI7352 | | Total |
| Preferred Term | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | All MEDI7352<br>(N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each PT category;

N = number of subjects per treatment group; PT = Preferred Term; TEAE = treatment-emergent adverse event.

Note: Results are n (n/Number of subjects in the Safety population within each PT\*100) m is number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each PT.

AEs are displayed by descending frequency of PT based on 'All MEDI7352' column, and alphabetically for PT of same frequency.

The 5% threshold for a TEAE to be displayed is taken from the Total column.

Reference Listing: 16.2.7.1

#### **Programming Notes:**

- PT texts should be in proper case in table.
- In case a term is not coded (e.g., in a dry run) it will be labelled as "Not Coded [PT]" and sorted at the end of the table.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi





# Table 14.3.1.9 Treatment Emergent Adverse Events by Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.8.
- Display all TEAEs, not only the most common.
- PT texts should be in proper case in table.
- In case a term is not coded (e.g., in a dry run) it will be labelled as Not Coded [PT]", and sorted at the end of the table.
- A column for column for dosing (column for dosing to the second dosing

Draft 1.1 | 31-Aug-2023 | 





## 6.2. Summary of Deaths and Other Serious Adverse Events

Table 14.3.2.1.1
Serious Adverse Events by System Organ Class and Preferred Term
Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One Treatment Emergent SAE", add "SAE = Serious Adverse Event" to abbreviations.
- Change footnote for "Reference Table 14.3.3.1".
- A column for column for column dosing (column dosing (column for column for

Table 14.3.2.1.2
Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One Life-Threatening SAE", add "SAE = Serious Adverse Event" to abbreviations.
- Add "Note: Life-threatening SAEs as judged by the investigator".
- Change footnote for "Reference Table 14.3.3.1".
- A column for column for column dosing (column dosing (column for column for

Draft 1.1 | 31-Aug-2023 | 





# Table 14.3.2.1.3 Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One SAE with Outcome Death", add "SAE = Serious Adverse Event" to abbreviations.
- Change footnote for "Reference Table 14.3.3.2".
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Table 14.3.2.1.4
Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term Safety Population

### **Programming Notes:**

- Same shell as Table 14.3.1.4. Change first row to be "Number of subjects with at Least One Treatment Emergent SAE", add "SAE = Serious Adverse Event" to abbreviations.
- Change footnote for "Reference Table 14.3.3.1".
- A column for column for dosing (column dosing (column dosing (column for column for co

Draft 1.1 | 31-Aug-2023 | 





#### Table 14.3.3.1 Listing of Serious Adverse Events Safety Population

| Subject ID/<br>Treatment Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | AE Start Date/Time<br>(Study Day)/<br>End Date/Time(Study S<br>Day) | Severity/<br>Relationship [1] | Outcome/<br>Action Taken with IP/<br>Therapy taken for this AE? | SAE<br>Leading<br>to Study<br>DC? | | Serious?/<br>Serious<br>?Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MX<br>M (X)/<br>DDMMMYYYY/HH:M<br>M (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/<br>Yes | No | No | XX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MX<br>M (X)/<br>DDMONYYYY/HH:<br>MM (X) | XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/<br>No | Yes | XX | XX /<br>XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/HH:M X<br>M (X)/<br>Ongoing | XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX/No | No | XX | XX /<br>XXX |

DC = discontinuation; ID = identification; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Study Day = date of interest – date of first infusion. A TEAE is defined as an adverse event with an onset at the time of or following the start of treatment with IP.

SAEs were coded using MedDRA version 26.0

<sup>[1]</sup> Reasonable possibility AE caused by IP as assessed by the investigator.





- If time missing, display "--:--".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e, no AEs occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment ID/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g.. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.3.2 Listing of Deaths Safety Population

| Subject ID/<br>Treatment<br>Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time<br>(Study Day) | Severity/<br>Relationship | Outcome/<br>Action Taken/<br>Therapy? | AE<br>Leading<br>to IP DC? | TEAE? | Serious? /<br>Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>DDMMMYYYY/H<br>H:MM (X) | XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX/<br>Yes | No | No | XX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>DDMMMYYYY/H:MM (X) | XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX/No | Yes | XX | XX / XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>Ongoing | H XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXX/<br>No | No | XX | XX / XXX |

DC = discontinuation; ID = identification; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Study Day = date of interest - date of first infusion. A TEAE is defined as an adverse event with an onset at the time of or following the start of treat ment with IP.

AEs were coded using MedDRA version 26.0

Draft 1.1 | 31-Aug-2023 | 





- If time missing, display "--:--".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e, no Aes occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g., in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Draft 1.1 | 31-Aug-2023 | 





#### 6.3. Displays of Significant Adverse Events and Adverse Events of Special Interest

Table 14.3.2.2.1
Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term Safety Population

### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at least One TEAE Associated with Abnormal Liver".
- Update Reference Listing to 16.2.7.3.
- A column for column for column dosing (column dosing (column for column for

Table 14.3.2.2.2
Potential joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at least One Potential Joint Related AESI"
- Add abbreviation for AESI = Adverse Event of Special Interest. Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.4
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





#### Table 14.3.2.2.3 Serious and/or severe Infections by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One SAE or Severe AE Related to Infection". Add "SAE = Serious Adverse Event" to abbreviations. Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.5.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.2.2.4

Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP by System Organ Class and Preferred Term Safety Population

| | | | Safety Population | П | | |
|---|---|---|---|---|---|---|
| System Organ Class | Placebo | | M | EDI7352 | | Total |
| Preferred Term | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | All MEDI7352<br>(N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m |
| Subjects with at Least<br>One Anaphylactic<br>Reaction,<br>Hypersensitivity or<br>Infusion-Related<br>Reactions Leading to<br>Discontinuation of IP | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx |
| Subjects with at Least One Anaphylactic Reaction, Hypersensitivity or Infusion-Related Reactions Not Leading to Discontinuation of IP[1] | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT category; N = number of subjects per treatment group; IP = investigational product; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Draft 1.1 | 31-Aug-2023 | 





[1] Anaphylactic reactions, hypersensitivity or infusion-related reactions not leading to discontinuation of IP were included in table as they were categorized as AE of special interest under Protocol Amendment 4 (V5.0). Definition for AE of special interest changed from Amendment 6 (V6.0) onwards, including anaphylactic reactions, hypersensitivity or infusion-related reactions leading to permanent discontinuation of IP..

Note: Results are n (n/N \* 100) m is number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing: 16.2.7.6

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One Anaphylactic Reaction, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP". Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.6.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Draft 1.1 | 31-Aug-2023 | 





## 6.4. Laboratory Data

Table 14.3.4.1
Descriptive Summary of Clinical Chemistry
Safety Population

Parameter: xxxxx (unit)

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Low CS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| High NCS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Low NCS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) |
| Low CS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| High NCS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |

Draft 1.1 | 31-Aug-2023 | 





Day 1 CFB

| n | XX | XX | XX | XX | XX | XX |
|---|---|---|---|---|---|---|
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |

CFB = change from baseline; CS = clinically Significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = not clinically significant; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Reference Listing: 16.2.8.1

### **Programming Notes:**

- Present only scheduled visits.
- Sort Parameters in the following Order: Albumin, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Bicarbonate, Calcium, Chloride, Creatinine, High-Sensitivity C-Reactive Protein (hs-CRP), Estimated Glomerular Filtration Rate (eGFR by Cockcroft-Gault), Serum Glucose, Lactate Dehydrogenase (LDH), Potassium, Sodium, Total Bilirubin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid.
- A column for on dosing (oc) will only be added if Stage 4 is initiated.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

Note: Percentages are n/Number of subjects with not missing data by treatment group at each visit\*100.





Table 14.3.4.2 Shift Table of Clinical Chemistry Results Safety Population

| Parameter (Unit)/ | | | | | Baseline | Grade [1] | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | | | Placebo | | | | ME | DI7352, 5 μg | /kg | |
| Post-Baseline | | | (N=xxx) | | | | | (N=xxx) | | |
| Grade | Low | Normal | High | Missing | Total | Low | Normal | High | Missing | Total |
| XXXXXX (Unit) | | | | | | | | | | |
| Week x | | | | | | | | | | |
| Low | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Missing | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Total | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Week x | | | | | | | | | | |
| Low | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High | x (xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Missing | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Total | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |

n = number of subjects within each category; N = number of subjects per treatment group.

Percentages are n/Number of subjects by treatment group at each visit for the parameter\*100.

Reference Listing 16.2.8.1

## **Programming Notes:**

- Repeat above in new pages for MEDI7352, CC MEDI7352, CC and All MEDI7352.
- Repeat the above for oclassical dosing only if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.1.

Draft 1.1 | 31-Aug-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





## Table 14.3.4.3 Descriptive Summary of Hematology Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.4.1
- Present only scheduled visits.
- Sort Parameters in the following Order: Absolute basophil count, absolute eosinophil count, absolute lymphocytes count, Absolute Monocyte Count, Absolute Neutrophil Count, Basophils %, Eosinophils %, Hematocrit (HCT), Hemoglobin (HGB), hemoglobin A1C (HgbA1C), Lymphocytes %, mean corpuscular hemoglobin (MHC), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), Monocytes %, Neutrophils %, Platelets, Red blood cell count (RBC), Red Cell Distribution Width, white blood cell Count (WBC).
- Update Reference listing to 16.2.8.2.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.3.4.4 Shift Table of Hematology Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.4.2
- Repeat the shell for column dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.3.
- Update Reference listing to 16.2.8.2

Draft 1.1 | 31-Aug-2023 | 





## Table 14.3.4.5 Descriptive Summary of Coagulation Safety Population

### **Programming Notes:**

- Same shell as Table 14.3.4.1
- Present only scheduled visits.
- Sort Parameters in the following Order: Activated Partial Thromboplastin Clotting Time (APTT), Fibrinogen, International normalized ratio (INR), Prothrombin Time (PT).
- Update Reference listing to 16.2.8.3.
- A column for column for column dosing (column dosing (column for column for

Table 14.3.4.6 Shift Table of Coagulation Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.4.2
- Repeat for column dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.5.
- Update Reference listing to 16.2.8.3.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.4.7 Descriptive Summary of Urinalysis Safety Population

Parameter: xxxxx (unit)

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Low CS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| ow NCS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| ow CS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High NCS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |

Draft 1.1 | 31-Aug-2023 | 





٠.

## Repeat for all visits for Parameters: Specific Gravity and pH

| Baseline [1] | | | | | | |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Negative | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Positive | x (xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| High NCS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| If Positive, Specify [2] | | | | | | |
| 100 mg/dL | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| 250 mg/dL | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| 500 mg/dL | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| >= 1000 mg/dL | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Negative | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| Positive | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| High NCS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |

• • •

#### Repeat for all visits for Parameters: Blood, Glucose, Ketones and Protein

CFB = change from baseline; CS = clinically significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = not clinically significant; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Percentages are n/Number of subjects with not missing data by treatment group at each visit\*100.

Reference Listing: 16.2.8.4

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

<sup>[2]</sup> Percentages are n/Number of Subjects with a Positive Result\*100.





- Present only scheduled visits.
- Sort Parameters in the following Order: Blood Urine, Glucose, Ketones, pH, Protein, Specific Gravity.
- Categories for If Positive, Specify:
  - o Blood, Urine: Trace, Small, Moderate.
  - O Glucose: 100 mg/dL, 250 mg/dL, 500 mg/dL,  $\geq 1000 \text{ mg/dL}$ .
  - o Ketones: Trace, 15 mg/dL, 40 mg/dL.
  - o Protein: Trace, 30 mg/dL, 100 mg/dL, 300 mg/dL.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





#### Table 14.3.4.8 Shift Table of Urinalysis Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.4.2
- Repeat for dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.7.
- Update Reference listing to 16.2.8.4

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.4.9

Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin Safety Population

| | | | Total F | Bilirubin |
|---------|------|-----------------|-----------|-----------|
| | | | <2 x ULN | >=2 x ULN |
| Group | Nobs | | n (%) | n (%) |
| Placebo | | | | |
| N=xxx | XXX | ALT | | |
| | | <3 x ULN | x (xx.x%) | x (xx.x%) |
| | | >=3 - <5 x ULN | x (xx.x%) | x (xx.x%) |
| | | >=5 -<10 x ULN | 0 | 0 |
| | | >=10 x ULN | 0 | 0 |
| | XXX | AST | | |
| | | <3 x ULN | x (xx.x%) | x (xx.x%) |
| | | >=3 -<5 x ULN | x (xx.x%) | x (xx.x%) |
| | | >=5 -<10 x ULN | 0 | 0 |
| | | >=10 x ULN | 0 | 0 |

Repeat for: Column All MEDI7352

ALT = a lanine aminotransferase; AST = a spartate a minotransferase; IP = investigational product; n = number of subjects per category; N = number of subjects per treatment group; Nobs = number of subjects per treatment group with at least one post-baseline a ssessment on treatment; ULN = upper limit of normal.

Note: On-treatment assessments include assessments on or after the date of first dose of IP. Baseline is defined as the last observation recorded prior to the first dose of treatment.

Percentages are based on Nobs.

Reference Listing: 16.2.8.1





• Per Protocol, the elevations of ALT or AST and Total Bilirubin do not have to occur at the same time or within a specified time frame. That is the reason why the table is presented by Subject instead of by visit. So, if for example, one subject has ALT >= 3 - <5 x ULN at Day 1, and TBL >= 2 x ULN at Week 18, n in that cell will increase by one.

• A column for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





## 6.5. Other Safety Data

Draft 1.1 | 31-Aug-2023 | 





#### Table 14.3.5.1 Descriptive Summary of Vital Signs Safety Population

Parameter: xxxxx

| Parameter: xxxxx | Dlacaba | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit | Placebo | | | | All MEDI7352 | 10181 |
| Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 1: 15 Minutes Pos | st- | | | | | |
| Dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| Day 1: 15 Minutes Pos | st- | | | | | |
| Dose CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

<sup>• • •</sup> 

Reference Listing: 16.2.9.1

CFB = Change from Baseline; eCRF = Electronic Case Report Form; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

Note: 'Day 1: 5 minutes after Infusion Completion' time point was only applied to subjects enrolled in Stage 1, with data collected under eCRF versions 4.0 (11DEC2018) or older.





- Repeat for Supine Heart Rate, Supine Systolic Blood Pressure, Supine Diastolic Blood Pressure, Respiratory Rate, Body Temperature, Standing Heart Rate, Standing Systolic Blood Pressure, Standing Diastolic Blood Pressure.
- After Week 2 (inclusive), Supine measure are taken in sitting position. We will consider them as supine (in resting position) for calculating Change from Baseline (always at supine position).
- Include the following timepoints: Baseline, Day 1: 5 Minutes Post-Dose, Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 7 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that Body To, and standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- A column for column for dosing (column for dosing

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.2 Descriptive Summary of Digital ECG Data Safety Population

Parameter: xxxxx

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Day 1: 1 hour Post-Dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX |
| Day 1: 1 hour Post-Dose | | | | | | |
| CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD =

Reference Listing: 16.2.9.2.1

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are averages of the 3 replicates taken for each parameter and timepoint, and CFB for the same variables.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





- Repeat for PR, QRS, QT, RR, HR (Heart Rate) and QTcF taken from external data.
- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.3 Summary of Overall Evaluation of Safety ECG Data Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal CS | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal NCS | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 1: 1 hour Post-Dose | ; | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal CS | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x% |
| Abnormal NCS | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

. . .

CS = clinically significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = Not clinically significant.

Note: Data are taken as the most conservative from the 3 replicates taken by timepoint.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.9.2.2

## **Programming Notes:**

- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.





Table 14.3.5.4 Covid-19 Screening Safety Population

| | | Safety Populat | | | | |
|---|---|---|---|---|---|---|
| Visit/ | Placebo | | MEDI7352 | | | Total |
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Day 1 | | | | | | |
| Subjects Screened for COVID-19 Symptoms | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| COVID-19 Symptoms Screened: | | | | | | |
| Fever | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Cough | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Dyspnoea | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Sore Throat | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Loss of Taste | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Loss of Smell | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Body Temperature Check | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | xx.x | XX.X | xx.x | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Subjects with COVID-19 Swab Performed | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Positive | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Subjects with COVID-19 Antibody Testing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Performed | ΛΛ (ΛΛ.Λ/0) | AA (AA.A /0) | ΛΛ (ΛΛ.Λ/0) | AA (AA.A /0) | AA (AA.A/0) | AA (AA.A /0) |
| COVID-19 Confirmed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Confirmed<br>COVID-19 Suspected | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| COVID-19 Suspected COVID-19 Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 INEgative | ΛΛ (ΛΛ.Λ/0) | AA (AA.A /0) | ΛΛ (ΛΛ.Λ/0) | AA (AA.A /0) | ΛΛ (ΛΛ.Λ/0) | AA (AA.A/0) |

Draft 1.1 | 31-Aug-2023 | 





| Subjects with COVID-19 Antigen Testing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|---|
| Performed | | | | | | |
| COVID-19 Positive | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| COVID-19 Negative | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

COVID-19 = coronavirus disease 2019; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Percentages are n/Number of subjects by treatment group at each visit\*100.

Reference Listing: 16.2.8.8

## **Programming Notes:**

- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10.
- A column for column dosing (column

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.5
Summary of Sub-Scores for Total Neuropathy Score-Nurse
Safety Population

| | | Safety Populat | | | | |
|---|---|---|---|---|---|---|
| Visit/ | Placebo | | MEDI7352 | | | Total |
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| Subjects performing TNSn | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Sensory Symptom Score | | | | | | |
| 0 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 3 | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 4 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Motor Symptom Score | | | | | | |
| 0 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 1 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 3 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 3 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 4 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Autonomic Symptom Score | | | | | | |
| 0 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 3 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pin Sensibility Score | | | | | | |
| 0 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 3 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

Draft 1.1 | 31-Aug-2023 | 




#### Vibration Sensibility Score

| 0 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|------------|-----------|------------|-----------|-----------|------------|
| 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 4 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group; TNSn = Total Neuropathy Score-Nurse.

Note: Percentages for subjects performing TNSn are n/Number of subjects by treatment group at each visit\*100. Percentages for each Score are n/Number of subjects by treatment group at each visit without missing score\*100

Reference Listing: 16.2.9.5

### **Programming Notes:**

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12 and Week 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





XX, XX

Table 14.3.5.6
Descriptive Summary of Total Neuropathy Score-Nurse
Safety Population

| | | 3 | safety ropulation | | | |
|---|---|---|---|---|---|---|
| Score: xxxxx | | | | | | |
| | Placebo | | MEDI7352 | | | Total |
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| Day 1 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

TNSn = Total Neuropathy Score-Nurse; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

XX, XX

XX, XX

XX, XX

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment. Reference Listing: 16.2.9.5

XX, XX

#### **Programming Notes:**

Min, Max

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12 and Week 18.
- Include the following scores: Sensory Symptom Score, Motor Symptom Score, Autonomic Symptom Score, Pin Sensibility Score, Vibration Sensibility Score, and TNSn Total.
- A column for column

XX, XX

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.7 Summary of Motor and Sensory Nerve Conduction Studies Safety Population

Parameter: xxxxx

| Tatameter. XXXXX | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X (XX.XX) |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | , and the second second | ŕ | ŕ | * | , and the second | , in the second second |
| IVIIII, IVIAX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Week 18 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Week 18 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| 1.111, 1.1011 | 1111, 1111 | 1111, 1111 | 11119 1111 | 1111, 1111 | 7177, 7171 | 7171, 7171 |

Draft 1.1 | 31-Aug-2023 | 





xx(xx.x%)

| Evaluation Result<br>Baseline [1] | | | | | | |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 18 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

...

Abnormal

xx(xx.x%)

xx(xx.x%)

xx(xx.x%)

xx(xx.x%)

Note: Percentages are number of subjects by treatment group at each visit for each category / Number of subjects with not missing data by treatment group for each visit\*100

Reference Listing: 16.2.9.6

## **Programming Notes:**

- Repeat for the following Parameters: Lower Limb right side/Motor evaluation/Amplitude, Lower Limb right side/Sensory evaluation/Amplitude, Lower Limb left side/ Motor evaluation/Amplitude, Upper Limb right side / Motor evaluation/Amplitude, Upper Limb right side / Sensory evaluation/Amplitude, Upper Limb left side/ Motor evaluation/Amplitude, Upper Limb left side / Sensory evaluation/Amplitude, Upper Limb left side / Sensory evaluation/Amplitude. (Repeat the same combination of Location Laterality/Evaluation for Peak Latency, Conduction Velocity, Duration of action Potential).
- A column for column dosing (column

xx (xx.x%)

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





Table 14.3.5.8 Summary of Strength and Deep Tendon Reflexes Safety Population

| Visit/ | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| Subjects performing SDTR assessment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ankle Dorsiflexion Strength | | | | | | |
| 0 - Normal Power | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 - Mild Weakness | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x% |
| 2 - Moderate Weakness | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x% |
| 3 - Severe Weakness | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| 4 - Paralysis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Deep Tendon Reflexes | | | | | | |
| 0 - Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 - Ankle reflex reduced | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x% |
| 2 - Ankle reflex absent | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x% |
| 3 - Ankle reflex absent and knee reflex reduced | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 4 - All reflexes (both ankle and knee) absent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

n = number of subjects by treatment group at each visit for each category; N = number of subjects per treatment group; SDTR = strength and deep tendon

Note: Percentages for each Score are n/Number of subjects by treatment group at each visit\*100

Reference Listing: 16.2.9.7

#### **Programming Notes:**

reflexes.

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.
- A column for column for dosing (column for dosing

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





Table 14.3.5.9 Summary of Local Injection Site Reactions Safety Population

| - | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/<br>Statistic or Category | (N=xx) | OCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Day 1: 15 Minutes after<br>Start of Infusion<br>Subjects with injection<br>Site Assessed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pain | | | | | | |
| | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Mild | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Severe | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tenderness | | | | | | |
| None | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Mild | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Moderate | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Erythema/ Redness | | | | | | |
| None | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Mild | | | | | • | |
| Moderate | | | | | | |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| None Mild Moderate Severe Tenderness None Mild Moderate Severe Erythema/ Redness None Mild Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Draft 1.1 | 31-Aug-2023 | 





#### Induration/ Swelling

...

| None | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|---|
| Mild | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Severe | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

n = number of subjects by treatment group at each visit for each category; N = number of subjects per treatment group.

Note: Percentages for each Score are n/Number of subjects by treatment group at each visit\*100

Reference Listing: 16.2.9.8

## **Programming Notes:**

- Include the following timepoints: Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.10 Summary of Hypersensitivity/Anaphylactic Reactions Safety Population

| Safety Population | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with any<br>Hypersensitivity/<br>Anaphylaxis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Highest Severity Grade | ( 0() | ( 0() | ( 0() | ( 0() | ( 0 () | ( 0() |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Type of Reaction | | | | | | |
| Urticaria | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pruritus | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Rash | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Flushing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Swollen Lips, Tongue,<br>Uvula and/or Vulva | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Dyspnoea | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Wheeze-Bronchospasm | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Stridor | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypoxia | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Hypotension | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Crampy Abdominal Pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Vomiting | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Diarrhoea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

. . .

N = number of subjects per treatment group.

Reference Listing: 16.2.9.9





## **Programming Notes:**

- Display only Type of reaction with non-missing value.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.11 Summary of Liver Diagnostic Investigations Safety Population

| Safety Population | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | • | MEDI7352 | | | Total |
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | $\overline{(N=xx)}$ | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Liver Diagnostics<br>Performed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Type of Diagnostic Investigation | | | | | | |
| Ültra sound | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| CT | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| MRI/MRCP | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Flushing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| ERCP | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| X-Ray | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Tox Screening for | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Acetaminophen/Paracetamol | | | | | | |
| Tox Screening for Ethanol | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tox Screening, Other | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Specialist Consulted | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis A | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis B | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis C | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis D | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis E | xx xx.x% | xx xx.x%) | xx xx.x%) | xx xx.x% | xx xx.x%) | xx xx.x%) |
| Serology for Cytomegalovirus | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Epstein Barr Virus | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Autoimmune Serology | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

CT = Computerized tomography; ERCP = Endoscopic retrograde cholangiopancreatography; MRI = Magnetic resonance imaging; MRCP = Magnetic resonance cholangiopancreatography; N = number of subjects per treatment group.

Reference Listing: 16.2.9.10

Draft 1.1 | 31-Aug-2023 | 





## **Programming Notes:**

- Display only Diagnostic Investigations with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.12 Summary of Liver Risk Factors and Lifestyle Events Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Liver Risk Factors<br>Assessed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Liver Risk Factor | | | | | | |
| Alcohol Abuse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Increased Alcohol Consumption | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| within 1 Month of Reported Event | | | | | | |
| IV Drug Abuse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tattoo | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Acupuncture | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Sexually Transmitted Diseases | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Toxic/Chemical Agent Exposure | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Travel (Areas at Risk in the Last Year) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pregnancy | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Parenteral Nutrition | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Excessive Physical Exercise | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Changes Diet/Fasting Episodes/Weight | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Loss Diet | | | | | | |
| Previous Drug Reaction | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Blood Transfusion | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Patient Exposed to Anyone with | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) |
| Jaundice in the Last Month | | | | | | |
| History of Hypotension | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Draft 1.1 | 31-Aug-2023 | 





| Low Blood Pressure at Time of Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|
| of Liver Injury and/or Abnormal Liver | | | | | | |
| Laboratory Value | | | | | | |
| History of Liver Disease | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

IV = intravenous; N = number of subjects per treatment group.

Reference Listing: 16.2.9.10

# **Programming Notes:**

- Display only Liver Risk Factor with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.13 Summary of Liver Signs and Symptoms Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Liver Signs/Symptoms<br>Assessed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Liver Sign/Symptom | | | | | | |
| Anorexia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Asthenia | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pyrexia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Pruritus | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Jaundice | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Arthra lgia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abdominal Pain | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Abdominal Tenderness | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Nausea | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Vomiting | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Rash | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Mucosal Inflammation | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Purpura | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Hepatomegaly | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Splenomegaly | xx xx.x% | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x% | xx xx.x% |
| Lymphadenopathy | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Ascites | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Confusional State | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Coma | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Upper Quadrant Tenderness | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x% | xx xx.x%) |
| Biliary Obstruction | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Eosinophilia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Dark Urine | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Other | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group.

Reference Listing: 16.2.9.12

Draft 1.1 | 31-Aug-2023 | 





# **Programming Notes:**

- Display only Liver Signs/Symptoms with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.14 Summary of Infection Diagnostic Investigations Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Infection Diagnostic Investigations | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Method | ( 0() | ( 0() | ( 0() | ( 0() | | ( 0() |
| Microscopy, Culture and Sensitivity | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serological Tests | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Nucleic Acid Based Tests | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| X-Ray | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

N = number of subjects per treatment group. Reference Listing: 16.2.9.13

# **Programming Notes:**

- Display only Methods with non-missing value.
- A column for column dosing (col ) will only be added if Stage 4 is initiated.

Draft 1.1 31-Aug-2023 





Table 14.3.5.15
Summary of Infection Risk Factors and Lifestyle Events
Safety Population

| | Placebo | Safety Fopulati | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| | Placedo | | | | A 11 N (ED) (72 52 | 10111 |
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Infection Risk Factor Occurred | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Infection risk factor | | | | | | |
| Extensive Burns within the Last Year | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tattoo, Piercing or Acupuncture within the | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| last Year | , | , , | . , | , | , , | , |
| Sexually Transmitted Diseases | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Travel to Areas at Risk of Tuberculosis or | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tropical Diseases | , | , | · · · · · · | | , , | , , , , , |
| Infections Related to Travel | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Blood Transfusion (within the Last Year) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Exposure to Nosocomial Pathogens within the | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Last Year | , | , | , | , | , | , |
| Contact History with Infection Source | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Previous BCG Immunization | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Evidence of BCG Scar | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tuberculin Skin or Quantiferon Test Confirms | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Previous Exposure or Immunity to | , | , , | , | , , | , , | , , |
| Tuberculosis | | | | | | |

BCG = Bacillus Calmette-Guerin; N = number of subjects per treatment group. Reference Listing: 16.2.9.14

# **Programming Notes:**

- Display only infection risk factors with non-missing value.
- A column for column for dosing (column for dosing

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.16 Summary of Infection Signs and Symptoms Safety Population

| | | Safety Populati | on | | | |
|---|---|---|---|---|---|---|
| | Placebo | - | MEDI7352 | | | Total |
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | $\overline{(N=xx)}$ | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Infection Sign/Symptom | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Occurred | | | | | | |
| Infection Sign/Symptoms | | | | | | |
| Pyrexia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Headache | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Confusional State | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Convulsion | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Rhinitis | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Oropharyngeal Pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Cough | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Productive Cough | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Haemoptysis | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Wheezing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Dyspnoea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pleuritic Pain | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Vomiting | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Diarrhoea | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Genital Discharge | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Haematuria | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Dysuria | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Hepatosplenomegaly | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Jaundice | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lymphadenopathy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Draft 1.1 | 31-Aug-2023 | 





| Rash | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|
| Petechial | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Vesicular | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Macular | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Papular | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Urticaria | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Erythema | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Blanching | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Splinter Haemorrhages | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Night sweats | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Chills | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Myalgia | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Weight Decrease | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |

N = number of subjects per treatment group.

Reference Listing: 16.2.9.15

# **Programming Notes:**

- Display only infection Signs/Symptoms with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





#### Table 14.3.5.17 Summary of Concomitant Medications by ATC Level 2 and Preferred Name Safety Population

### **Programming Notes:**

- Same shell as Table 14.1.7.
- Change footnote Note by: "Note: Concomitant medications are defined as medications continuing or starting on or after first dose of study medication. All concomitant medications are coded using WHO drug dictionary version vMar2023. At each level of summarization (ATC Level 2 or Preferred Name), subjects who reported more than one concomitant medication were only counted once. ATC Level 2 and Preferred Name are sorted in in descending order of frequency of total, and alphabetically if same frequency".
- If uncoded ATC Level or Preferred Name, please put them as [Not Coded]
- ATC and Preferred Name texts should be in proper case in table.
- A column for column for dosing (column for dosing

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.18
Summary of Concomitant Procedures
Safety Population

| System Organ Class | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Preferred Term | (N=xxx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| Any Concomitant Procedure | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class.

Note: All Procedure terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 26.0. At each level of summarization (system organ class or preferred term), subjects having more than one Procedure term were counted only once. System organ class and preferred terms are sorted in descending order of frequency of Total column, and alphabetically if same frequency.

When there are uncoded Procedure Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] are sorted at the end of the table.

Reference Listing: 16.2.9.18

#### **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Sort SOC and PT (within SOC) in descending order of frequency in the Total column. Sort alphabetically in case of ties.
- Uncoded Procedure events
  - When there are uncoded Procedure Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] will be sorted at the end of the table.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Table 14.3.5.19
Anti-Drug Antibody Results and Titre Summary by Timepoint Safety Population

| | Placebo | | MEDI | [7352 | |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) |
| Dagalina [1] | | | | | |
| Baseline [1] | | | | | |
| n [2] | XX | XX | XX | XX | XX |
| ADA Positive: n (%) [3] | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Week 2 | | | | | |
| n [2] | XX | XX | XX | XX | XX |
| ADA Positive: n (%) [3] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| ADA Titre | | | , | , | , |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

ADA = Anti-Drug Antibodies; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Reference Listing: 16.2.9.19

### **Programming Notes:**

- Keep in mind that in this table 'Total' column does not include placebo.
- Repeat for all scheduled post-baseline visits.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

<sup>[2]</sup> Number of subjects with at least one ADA assessment at the specific visit.

<sup>[3]</sup> Number of subjects with a positive result at the specific visit. The denominator for all percentages is the number of subjects with an ADA result for each visit.





Table 14.3.5.20
Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories
Safety Population

| | Placebo | y Population | MED | I7352 | |
|---|---|---|---|---|---|
| ADA Category | (N=xx) | CCI<br>(N=xx) | (N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) |
| ADA positive at baseline and/or post-baseline (ADA | | | | | |
| prevalence) | | | | | |
| n/Nobs (%) [1] [2] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| TE-ADA positive (ADA incidence) [5] | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | , | , | , | , | , |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX |
| Treatment Induced ADA Positive | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | , | • | | , | · · · · |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

Draft 1.1 | 31-Aug-2023 | 





| Treatment-Boosted ADA Positive<br>n/Nobs (%) [1] [3]<br>Maximum ADA Titre | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
|---|---|---|---|---|---|
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Non-TE-ADA Positive [6] | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Both baseline and post-baseline positive | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Only baseline positive | | | | | |
| n/Nobs (%) [1] [4] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| TE-persistently ADA positive [7] | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

Draft 1.1 | 31-Aug-2023 | 





TE-transiently ADA positive [8]
n/Nobs (%) [1] [3]
Maximum ADA Titre
Median
Q1, Q3
Min, Max

| $xx/xxx$ ( $xx.x^0$ | %) xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx(xx.x%) | xx/xxx (xx.x%) |
|---|---|---|---|---|
| xx.x | XX.X | XX.X | xx.x | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |

ADA = Anti-Drug Antibodies; N=number of subjects per treatment group; TE-ADA = Treatment Emergent ADA; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

- [1] n represents the number of subjects satisfying the conditions of the specified ADA category
- [2] Nobs represents the number of subjects with any ADA result at baseline and/or post-baseline.
- [3] Nobs represents the number of subjects with an ADA result at baseline and at least one post-baseline ADA assessment.
- [4] Nobs represents the number of subjects with an ADA result at baseline.
- [5] TE-ADA positive is defined as either ADA negative at baseline and post-baseline ADA positive (Treatment Induced ADA Positive), or as ADA positive at baseline with pre-existing titre boosted by 4-fold or greater during the study period (Treatment Induced ADA Positive). ADA incidence is the proportion of TE-ADA+ subjects in a population.
- [6] ADA post-baseline positive but not fulfilling the conditions for TE-ADA+
- [7] ADA negative at baseline and having at least 2 post-baseline ADA positive measurements with ≥16 weeks (112 days) between first and last positive, or an ADA positive result at the last available post-baseline assessment.
- [8] ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.

Reference Listing: 16.2.9.19

## **Programming Notes:**

- If a participant has more than 1 non-missing titre during the study, the maximum titre for each participant is summarized.
- Only present summary statistics if titre is available.
- If no positive results for a particular block of the table, then the summary statistics for the titres for that particular block would not appear.
- It is assumed that participants with a missing baseline ADA result are ADA negative at baseline.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.





# 7. Pharmacokinetic/Pharmacodynamic Data

Table 14.4.1 Summary of Serum MEDI7352 Concentrations PK Population

ADA Status: xxxxxxxxxx

| | | MEDI7352 | |
|---|---|---|---|
| Visit/ | CCI | CCI | CCI |
| Statistic | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean $[gMean \pm gSD]$ | x.xx [x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] |
| gCV% | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | xx, xx |
| Week 2 | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean [gMean $\pm$ gSD] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] |
| gCV% | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Week 4 | | | |
| n (n < LLOQ) | xx(xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean $[gMean \pm gSD]$ | x.xx [x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] |
| gCV% | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx |

gCV% = Geometric Coefficient of Variation (%); gMean = Geometric Mean; gSD = Geometric SD; LLOQ = Lower Limit of Quantification; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NC = not calculable; NQ = not quantifiable. [1] Baseline is defined as the last observation recorded prior to the first dose of treatment. Reference Listing: 16.2.10.1

Draft 1.1 | 31-Aug-2023 | 





## **Programming Notes:**

- Include the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours/ Pre-Dose, Week 11/ Pre-Dose, Week 10 + 14 Days/Pre-Dose; Week 18.
- Repeat the table for 'ADA Positive', 'ADA Negative' and 'Overall'.
- Any values reported as NRR (not reportable) or NS (missing) will be excluded from the summary tables.
- At a time point where less than or equal to 50% of the concentration values are NQ (below LLOQ), all NQ values will be set to the LLOQ, and all descriptive statistics will be calculated accordingly.
- At a time point where more than 50% (but not all) of the values are NQ, the gmean, gmean ± gSD and gCV% will be set to NC. The maximum value will be reported from the individual data, and the minimum and median will be set to NQ.
- If all concentrations are NQ at a time point, no descriptive statistics will be calculated for that time point. The gmean, minimum, median and maximum will be reported as NQ and the gCV% and gmean ± gSD as NC.

Draft 1.1 | 31-Aug-2023 | 





#### Table 14.4.2 Summary of Serum total NGF Concentrations Safety Population

ADA Status: xxxxxxxxxx

| | Placebo | | MEDI7352 | |
|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean [gMean $\pm$ gSD] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | · · · · · · |
| gCV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx |
| Week 2 | | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean [gMean ± gSD] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] | |
| gCV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx |
| Week 4 | | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean [gMean $\pm$ gSD] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | |
| gCV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |

gCV% = Geometric Coefficient of Variation (%); gMean = Geometric Mean; gSD = Geometric SD; LLOQ = Lower Limit of Quantification; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; ; NC = not calculable; NGF = Nerve-Growth Factor; NQ = not quantifiable.

Reference Listing: 16.2.10.3

Draft 1.1 | 31-Aug-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





## **Programming Notes:**

- Repeat for ADA Status: "ADA Positive", "ADA Negative" and "Overall".
- Include the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Draft 1.1 | 31-Aug-2023 | 





# **Planned Listing Descriptions and Shells**

| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| Listing 16.2.1.1 - Subject Disposition - Screening Population | U |
| Listing 16.2.1.2 - Assignment to Analysis Populations - Screening Population | U |
| Listing 16.2.1.3 - Reason for IP Discontinuation and Withdrawal from the Study - Safety Population | U |
| Listing 16.2.1.4 - List of Reasons for Screening Failure - Screen Failure Population | U |
| Listing 16.2.1.5 - Subject Visits and COVID-19 Impact - Screening Population | U |
| Listing 16.2.2.1 - Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria - Screening Population | U |
| Listing 16.2.2.2-Protocol Deviations - Sa fety Population | found.Error! U |
| Listing 16.2.3 - Randomization and Treatment Group - Safety Population | |
| Listing 16.2.4.1 - Demographic and Baseline Characteristics - Screening Population | U |
| Listing 16.2.4.2 - Medical History - Safety Population | U |
| Listing 16.2.4.3 - Osteoarthritis Characteristics - Screening Population | U |
| Listing 16.2.5.1 - Study Drug Administration: Individual Doses - Safety Population | U |
| Listing 16.2.6.1 - Daily Pain NRS - mITT Population | U |
| Listing 16.2.6.2 - Galer NPS - mITT Population | U |
| Listing 16.2.6.3 - DSIS - mITT Population | U |
| Listing 16.2.6.4 - SF-36 - mITT Population | U |
| Listing 16.2.6.5 - Rescue Medication Usage - mITT Population | R |
| Listing 16.2.6.6 - Patient Global Impression of Change - mITT Population | U |

Draft 1.1 | 31-Aug-2023 | 





| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| CCI | U |
| Listing 16.2.7.1 - Adverse Events - Safety Population | U |
| Listing 16.2.7.2 - Treatment Emergent Adverse Events Leading to Study Drug Discontinuation <b></b> - Sa fety Population | R |
| Listing 16.2.7.3 - Treatment Emergent Adverse Events Associated with Abnormal Liver - Safety Population | R |
| Listing 16.2.7.4 - Joint Related Adverse Events of Special Interest - Safety Population | R |
| Listing 16.2.7.5 - Serious and/or Severe Infections - Safety Population | R |
| Listing 16.2.7.6 - Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of Study Drug - Safety Population | R |
| Listing 16.2.8.1 - Clinical Chemistry Laboratory Evaluations - Safety Population | U |
| Listing 16.2.8.2 - Hematology Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.3 - Coagulation Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.4 - Urinalysis Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.5 - Serology Laboratory Evaluations - Safety Population | U |
| Listing 16.2.8.6 - Pregnancy Test Results - Safety Population | U |
| Listing 16.2.8.7 - Drug Test Results - Safety Population | U |
| Listing 16.2.8.8 - COVID-19 Screening and Vaccination - Safety Population | U |
| Listing 16.2.9.1 - Vital Signs Measurements - Safety Population | U |
| Listing 16.2.9.2.1 - <sup>12-Lead Digital ECG Results</sup> - Sa fety Population | U |
| Listing 16.2.9.2.2 - 12-Lead Safety ECG Results - Safety Population | U |
| Listing 16.2.9.3 - Physical Examination Results - Safety Population | U |
| Listing 16.2.9.4 - Neurological Examination Results - Safety Population | U |
| Listing 16.2.9.5 - Total Neuropathy Score-Nurse - Safety Population | U |

Draft 1.1 | 31-Aug-2023 | 





| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| Listing 16.2.9.6 - Motor and Sensory Nerve Conduction Studies - Safety Population | U |
| Listing 16.2.9.7 - Strength and Deep Tendon Reflexes - Safety Population | U |
| Listing 16.2.9.8 - Injection Site Reactions - Safety Population | U |
| Listing 16.2.9.9 - Hypersensitivity/Anaphylactic Reactions - Safety Population | U |
| Listing 16.2.9.10 - Liver Diagnostic Investigations - Safety Population | U |
| Listing 16.2.9.11 - Liver Risk Factors and Lifestyle Events - Safety Population | U |
| Listing 16.2.9.12 - Liver Signs and Symptoms - Safety Population | U |
| Listing 16.2.9.13 - Infection Diagnostic Investigations - Safety Population | U |
| Listing 16.2.9.14 - Infection Risk Factors and Lifestyle Events - Safety Population | U |
| Listing 16.2.9.15 - Infection Signs and Symptoms - Safety Population | U |
| Listing 16.2.9.16 - Prior and Concomitant Medications - Safety Population | U |
| Listing 16.2.9.17 - Prohibited Concomitant Medications - Safety Population | R |
| Listing 16.2.9.18 - Concomitant Procedures - Safety Population | R |
| Listing 16.2.9.19 - Anti-drug Antibody Test Results - Safety Population | U |
| Listing 16.2.10.1 - Serum MEDI7352 Concentrations - PK Population | U |
| Listing 16.2.10.2 - Serum total NGF Concentrations - PD Population | U |

Draft 1.1 | 31-Aug-2023 | 





# **Listing Change Log:**

| Output<br>Number | Date of<br>Change | Change<br>Made By<br>(initials) | Description/Rationale |
|---|---|---|---|

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.1.1 Subject Disposition Screening Population

| Subject<br>ID | Re-screened?/<br>Previous<br>Subject ID | Treatment<br>Arm | Re-consent/ Date/Time of Initial IC/ Initial Protocol Version | Date/Time of<br>Informed Consent | Protocol<br>Version at<br>consent/<br>Re-consent | Consent for Colsample? /Date of Consent | Consent for<br>COVID-19 Sa fety<br>Mea sures / Date of<br>Consent | Current<br>Protocol<br>version |
|---|---|---|---|---|---|---|---|---|
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | Yes/ XXXX | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | No | XXXX | Yes /<br>DDMMMYYYY/hh:mm<br>/ XXXX | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | No | XXXXX |
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | No | No | XXXXX |

COVID-19 = corona virus disease 2019; IC = Informed Consent;

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.1.2 Assignment to Analysis Populations Screening Population

| SubjectID | Treatment<br>Arm | Screened [1] | Randomized | SAF [2] | mITT[3] | PK [4] | Reason to Exclude from Safety [5] | Reason to Exclude from mITT [6] |
|---|---|---|---|---|---|---|---|---|
| | | <u> </u> | | | | | , [-] | |
| XXXXXX | XXXX | Yes | No | No | No | No | | |
| XXXXXX | XXXX | Yes | Yes | Yes | Yes | Yes | | |
| XXXXXX | XXXX | Yes | Yes | No | No | No | XXX | |
| XXXXXX | XXXX | Yes | Yes | Yes | Yes | Yes | | |
| XXXXXX | XXXX | Yes | Yes | Yes | No | No | XXX/ XXX | XXX/ XXX |

mITT = Modified Intent-To-Treat Population Set; NRS = numeric rating scale; PK = pharmacokinetics; SAF = Safety Population Set.

## **Programming Notes:**

- If there is more than one major deviation, please concatenate with "/"
- Sort by Treatment Arm/ Subject ID.

<sup>[1]</sup> The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments.

<sup>[2]</sup> The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication.

<sup>[3]</sup> The mITT Population includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.

<sup>[4]</sup> The PK Population includes all subjects for who a pharmacokinetic sample was obtained and analysed.

<sup>[5]</sup> Major deviation reason/s to exclude from Safety Population for randomized subject.

<sup>[6]</sup> Major deviation reason/s to exclude from mITT Population for randomized subject.





# Listing 16.2.1.3 Reason for IP Discontinuation and Withdrawal from the Study Safety Population

| Subject ID/<br>Treatment<br>Arm | IP<br>Discontinuation<br>[1]/ Study<br>Withdrawal | Completion/<br>Discontinuation<br>Date (Study Day) | Date of Last Dose | Number of doses | Primary<br>Reason for<br>DC/<br>Withdrawal | Blind Broken? /<br>Date/Time /<br>Reason | Reason for<br>breaking<br>the Blind | Study<br>Duratio<br>n |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXX | IP<br>Discontinuation | DDMMMYYYY(XX) | DDMMMYYYY | XX | XXXXXX<br>X | Yes /<br>DDMMMYYYY/<br>hh:mm | XXXXXX | XX |
| XXXXXX/<br>XXXX | IP<br>Discontinuation | DDMMMYYYY (XX) | DDMMMYYYY | XX | XXXXXX<br>X | No | | XX |
| XXXXXX/<br>XXXX | Study<br>Withdrawal | DDMMMYYYY (XX) | DDMMMYYYY | XX | Other:<br>XXXXXX<br>X | No | | XX |

DC = Discontinuation; IP = Investigational product.

Note: Study Day is calculated relative to the date of first dose. Study Duration = Reference end date – date of first dose of treatment + 1.

## **Programming Notes:**

- If reason for non-completion is Other, concatenate the specify text as follows: "Other: XXXXXXXXX".
- If reason for non-completion is adverse event, concatenate with AE line number as follows: "Adverse event number X".
- For Physician decision, screen-fail and withdrawal by subject, please provide explanation if presented on the logic "Physician decision: XXX".
- Do not include subjects who completed the study.
- Sort by Treatment Arm/ Subject ID.

<sup>[1]</sup> Any withdrawal from the study before last IP dose (Week 10) is considered an IP discontinuation.




### Listing 16.2.1.4 List of Reasons for Screening Failure Screen Failure Population

| Subject ID | Treatment Arm | Screen failure Date | Primary Reason for Screen Failure |
|---|---|---|---|
| XXXXXX | Screen Failure | DDMMMYYYY | XXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY | XXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY | |
| XXXXXX | Screen Failure | DDMMMYYYY | Other: XXXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY | |

# **Programming Notes:**

- If reason for non-completion is Other, concatenate the "Primary Reason for Screen Failure" text as follows: "Other: XXXXXXXXX".
- Sort by Subject ID.

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.1.5 Visits List and COVID-19 Impact Screening Population

| Subject ID/<br>Treatment<br>Arm | Visit<br>Name | Visit Date<br>(Study<br>Day) | Is COVID-<br>19<br>Pandemic<br>Ongoing? | Impacted<br>by<br>COVID-19 | Was visit<br>performed?/<br>Visit Type | Visit<br>Performe<br>d Via | VS Data<br>provided? /<br>Assessments<br>Missed? | IP dosing<br>missed due to<br>COVID-19 /<br>Details | End of<br>Treatment<br>linked to<br>COVID-19 | Subject<br>discontinued<br>due to<br>COVID-19?/<br>Details |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | Yes | Yes | Yes/<br>Delayed | On site | Y/<br>Efficacy | Y/ XXXX | Other: XXXX | Y/ XXXX |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | Yes | No | Yes | | N/ Safety | | | |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | No | Yes | Yes | Video | N/<br>Efficacy,<br>Safety | Y/ Other:<br>XXXX | | |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | No | No | No / Missed | | | | | |

COVID-19 = corona virus disea se 2019; IP = Investigational Product; VS = Vital Signs.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Visit Type: Missed, Abbreviated, Delayed.
- Visit Performed Via: Video, Phone, On Site Other: xxxxxx.
- Details on IP dosing missed: Treatment on hold due to Sponsor Decision, Subject infected with COVID-19, Subject decision, Other: xxxxxx.
- End of treatment, reason if due to COVID: Subject infected with COVID-19, Subject decision, Travel restrictions, Site closed, Study delayed/cancelled, Other: xxxxxx.
- Details on Subjects discontinuing due to COVID-19: Subject infected with COVID-19, Subject decision, End of Treatment due to Sponsor, Other: xxxxxx.
- Sort by Treatment Arm/ Subject ID/ Visit Date.

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.2.1
Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria
Screening Population

| SubjectID | Treatment Arm | Enrolled | Randomized | Inclusion or<br>Exclusion | Criteria<br>Number | Criteria Label |
|---|---|---|---|---|---|---|
| XXXXXX | Screen Failure | Yes | No | Inclusion | XX | XXXXXXXXXXXXXXXXX |
| | | Yes | No | Exclusion | XX | XXXXXXXXXXXXXXXXX |

# **Programming Notes:**

• Sort by Subject ID.

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.2.2 Protocol Deviations Safety Population

| | | | | | | Covid-<br>19 |
|---|---|---|---|---|---|---|
| SubjectIDTr | eatment An | m Analysis Population Event Date (Study Day) | Event Type | Description | Category | Related? |
| XXXXXX | XXXX | Screened\RND\SAF\DDMMMYYYY (XX) mITT | XXXXXXXXX | XXXXXXX | Non-<br>important | Y |
| | | | XXXXXXXXXXXX | XXXXXXXXXXXXXX | - | |
| XXXXXX | XXXX | DDMMMYYYY (XX) | XXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX | |
| | | | XXXXXXXXXXXXXXX | XXXXXXXXXX | XXXXX | |
| XXXXXX | XXXX | DDMMMYYYY (XX) | XXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX | |

COVID-19 = Corona virus disease 2019; mITT = Modified Intent-To-Treat Population; RND = Randomized Subjects; SAF = Safety Population. Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- The structure of this listing may change depending on the information in the protocol deviations file. In the analysis population column, include only the analysis population where subject is included in.
- o Sort by Treatment Arm/ Subject ID. If date is present in file, add a column for date of event and sort by date. If no date is present, sort by category with non-important first and then important.
- Event Type: Inclusion Criteria, Exclusion Criteria, Study Drug, Assessment Safety, Assessment Efficacy, Lab/endpoint data, Visit Window, Informed Consent, Prohibited Co-Medication, Overdose/Misuse, Other.





# Listing 16.2.3 Randomization and Treatment group Safety Population

| Subject ID | Treatment Arm | Randomization Stage | Randomization Treatment | Randomization Date / Time<br>(Study Day) | Randomization<br>Number |
|---|---|---|---|---|---|
| XXXXXX | XXXX | Stage 1 | Active CC | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 3 | Active <b>CC</b> | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 2 | Placebo | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 2 | Active <b>CC</b> | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 3 | Placebo | DDMMMYYYY/hh:mm (-X) | XXXX |

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

• Sort by Treatment Arm/ Subject ID.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.4.1 Demographic and Baseline Characteristics Screening Population

| Subject<br>ID | Treatment<br>Arm | Birth Date | Age<br>(years) | Sex | Surgically sterile?/ Postmenopausal? [2] | Ethnicity | Race | Weight (kg) | Height | BMI (kg/m²) | Fully<br>vaccinated<br>for COVID-<br>19? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | DDMMMYYY | XX | XX | Tostinenopausur. [2] | XXXXX | XXXX | XX.X | XX.X | XX.X | Y |
| XXX | XXX | MMMYYY | XX | XX | No/ Yes | XXXXX | XXXX | XX.X | XX.X | XX.X | N |

COVID-19 = Corona virus disease 2019.

Note: Height and weight are the values at Screening.

[1] Age was calculated as age at time of consent.

[2] For Female Subject Only.

# **Programming Notes:**

Sort by Treatment Arm/ Subject ID

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.4.2 Medical History Safety Population

| Subject ID | Treatment Arm | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day)/ |
|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |
| | | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXX | MMMYYYY (X)/<br>Ongoing |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>Ongoing |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |

MedDRA = Medical Dictionary for Regulatory Activities. Note: Study Day is calculated relative to the date of first dose. Medical History were coded using MedDRA version 26.0. Only subjects with medical history recorded are listed.

# **Programming Notes:**

- SOC & PT text should be in proper case in listing.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date of medical event.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.4.3 Osteoarthritis Characteristics Screening Population

| Subject ID | Treatment<br>Arm | Subject with OA? / Joint/<br>Area affected | Is OA<br>considered<br>CS? | Radiological<br>Investigations<br>Conducted? / Details | Joint Area<br>Investigated | Is OA<br>considered<br>RS? | K-L Score<br>Reported | Radiologic Scoring<br>System / Details/<br>Result |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Y / Shoulder | Y | Y/ Other: XXXXXX | Shoulder | Y | Grade 3 | XXXXXX/<br>XXXXXX/<br>XX |
| XXXXXX | XXXX | Y / Ankle | N | Y / MRI | Ankle | N | N | N |

CS = Clinically Significant; K-L = Kellgren-Lawrence; OA = Osteoarthritis; RS = Radiologically Significant.

# **Programming Notes:**

• Sort by Treatment Arm/ Subject ID

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.5.1 Study Drug Administration: Individual Doses Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit<br>Name | Start<br>Date/<br>Time<br>(Study<br>Day) | End<br>Date/<br>Time<br>(Study<br>Day) | Was Infusion Performed?/ Infusion Volume (mL)[1]/ Reason not Performed | Actually<br>Administered<br>Volume (mL)<br>[2] | If Difference between [1] and [2] Volume, Reason | Any<br>Injection<br>Site<br>Reactions? | Any<br>Infusion<br>Related<br>Reactions | Infusion<br>Rate<br>(mL/<br>hour) | Rate Change<br>Justification | Reason<br>for<br>Infusion<br>Rate<br>Change |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX/<br>XXXX | XXX | DDMM<br>MYYYY<br>/hh:mm<br>(X) | DDMM<br>MYYYY<br>/hh:mm<br>(X) | Y/<br>XX | XX | | | | xx.x | | |
| XXXX/<br>XXXX | XXX | DDMM<br>MYYYY<br>/hh:mm<br>(X) | DDMM<br>MYYYY<br>/hh:mm<br>(X) | Y/<br>XX | XX | XXXXX | Y | Y | xx.x | XXXXX | XXXXX<br>XX |
| XXXX/<br>XXXX | XXX | | | N/<br>XXXXXX | | | | | | | |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / End Date.
- Rate Change Justification: Increased, Decreased, Interrupted.





Listing 16.2.6.1 Daily Pain NRS mITT Population

| Subject ID | Treatment Arm | Study Visit [1] | Subject Diary (ePRO) Date / Study Day | Baseline Flag [2] | DPS |
|---|---|---|---|---|---|
| XXXXXX | XXXX | Baseline | DDMMMYYYY/ (-7) | Y | X |
| | | Baseline | DDMMMYYYY/ (-6) | Y | XX |
| | | ••• | ••• | ••• | ••• |
| | | Baseline | DDMMMYYYY/ (-2) | Y | XX |
| | | Baseline | DDMMMYYYY/ (-1) | Y | XX |
| | | ••• | | | |
| | | Week 2 | DDMMMYYYY/ (13) | | XX |
| | | Week 2 | DDMMMYYYY/ (14) | | XX |
| | | ••• | | | |
| | | Week X | DDMMMYYYY/ (X) | | XX |
| | | ••• | ••• | | |
| XXXXXX | XXXX | Baseline | DDMMMYYYY/ (-7) | Y | XX |
| DDG D 1 D | | | | ••• | ••• |

DPS = Daily Pain Score; ePRO = Electronic Patient-Reported Outcome; NRS = Numeric Rating Scale.

Note: Data shown in column 'DPS' are average daily pain scores on an 11-point (0-10) NRS. Study Day is calculated relative to the date of first dose. [1] Study Visit is defined as the 7-day period ending within the protocol window Day  $\pm 3$ , where at least 4 days out of 7 have recorded diary pain scores.

Draft 1.1 | 31-Aug-2023 | 

<sup>[2]</sup> Baseline is defined as the 7-day period prior to randomization i.e., Day -7 to Day -1, inclusive. A subject is considered to have an evaluable baseline pain score if there are at least 4 days of recorded diary pain scores in the 7-day period.





## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Subject Diary Date.
- Display all measurement per Subject, starting on the Study Day = -7.
- Display Study Visit for days involved in weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Flag Baseline records only when there is at least 5 days of recorded diary pain scores in the 7-day Baseline period

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.6.2 Galer NPS mITT Population

| Subject ID | Treatment Arm | Parameter | Study Visit | Collection Date / Study<br>Day | Baseline Flag [1] | NPS |
|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Pain intensity | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | j | Week 4 | DDMMMYYYY/ (X) | | XX |
| | | | Week 8 | DDMMMYYYY/ (X) | | XX |
| | | | | | | XX |
| | | | Week X | DDMMMYYYY/(X) | | XX |
| | | | | ••• | | XX |
| | | XXXX | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | ••• | | | | |
| XXXXXX | XXXX | Pain intensity | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | | ••• | | | |
| | | XXXX | Week X | DDMMMYYYY/ (X) | | XX |
| | | ••• | ••• | ••• | | |

NPS = Neuropathic Pain Scale; NRS = Numeric Rating Scale.

Note: Data shown in column 'NPS' are Pain Intensity, Unpleasantness, and Descriptor scores on an 11-point (0-10) NRS, and Pain Duration/Frequency on a 3-point NRS (1-3).

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Draft 1.1 | 31-Aug-2023 | 





## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter / Collection Date.
- Keep Parameter sorting from the last bullet point in this programming notes.
- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Repeat for the Parameters: Pain intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, Surface Pain Intensity (All in an 11-point NRS), and Pain Duration/Frequency (in a 3-point NRS).

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.6.3
DSIS
mITT Population

### **Programming Notes:**

- Same shell as Listing 16.2.6.1.
- Update footnote as:
  - DSIS = Daily Sleep Interference Scale; ePRO = Electronic Patient-Reported Outcome; NRS = Numeric Rating Scale. Note: Data shown in column 'DSIS' are daily Sleep Interference scores on an 11-point (0-10) NRS. Study Day is calculated relative to the date of the day of first dose.
  - [1] Study Visit is defined as the seven-day period ending within the protocol window Day  $\pm 3$ .
  - [2] Baseline is defined as the seven-day period prior to randomization i.e., Day -7 to Day -1,.
- Sort by Treatment Arm/ Subject ID / Subject Diary Date.
- Display all measurement per Subject, starting on the Study Day = -7.
- Display Study Visit for days involved in weekly averages of the average Sleep interference scores for Baseline, Week 4, 8, 12, and 18.

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.6.4 SF-36 mITT Population

| Subject ID | Treatment<br>Arm | Parameter | Item<br>Number | Item name | Study Visit | Collection Date / Study<br>Day | Baseline<br>Flag[1] | SF-36 |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Physical functioning | 3 | Vigorous<br>Activities | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | | | | Week 12 | DDMMMYYYY/ (X) | | XX |
| | | | 4 | Moderate<br>Activities | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | ••• | ••• | ••• | ••• | | | |
| | | | - | Total | Baseline | DDMMMYYYY/ (X) | Y | |
| | | | | | Week 12 | DDMMMYYYY/ (X) | | XX |
| XXXXXX | XXXX | Role<br>limitations<br>due to<br>physical | | Cut Amount<br>of Time<br>Spent on<br>Work/Act | Baseline | | | |
| | | health | 13 | WOIK/ACt | | DDMMMYYYY/(X) | Y | XX |
| | | | | | Week 12 | DDMMMYYYY/ (X) | | XX |
| | | | ••• | | ••• | ••• | | ••• |
| | | ••• | | | ••• | | ••• | |

SF-36 = 36-Item Short-Form Health Survey; NRS = Numeric Rating Scale.

Note: Data shown in column 'SF-36' are derived SF-36 scores and Change in General Health on a 5-point NRS (1-5).

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Draft 1.1 | 31-Aug-2023 | 





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter / Item /Collection Date.
- Keep Parameter sorting from the last bullet point in this programming notes.
- Include all data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical functioning (items 3, 4, 5, 6, 7, 8, 9, 10, 11, 12), Role limitations due to physical health (items: 13, 14, 15, 16), Role limitations due to emotional problems (items: 17, 18, 19), Vitality (Energy/fatigue) (items: 23, 27, 29, 31), Emotional well-being (items: 24, 25, 26, 28, 30), Social functioning (20, 32), Pain (items: 21, 22) and General Health (items: 1, 33, 34, 35, 36), all with values ranging from 0 to 100. Change in general Health (in a 5-point NRS, item: 2).

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.6.5 Rescue Medication Usage mITT Population

| Subject<br>ID | Treatment Arm | ATC Class (Level 2)/<br>Preferred Name/<br>Verbatim Term | Primary<br>Indication | Start Date (Study Day)/<br>End Date (Study Day) | Dose<br>(unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | MMMYYYY (-XX)/<br>DDMMMYYYY (-X) | XXXX<br>unit | XXXXXXXX | XXXXX |
| | XXXX | XXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | MMMYYYY (-X)/<br>Ongoing | XXXX<br>unit | XXXXXXXX | XXXXX |
| | XXXX | XXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | DDMMMYYYY (X)/<br>DDMMMYYYY<br>(XX) | XXXX<br>unit | XXXXXXXX | XXXXX |

ATC = anatomical therapeutic chemical.

Note: Study Day is calculated relative to the date of first dose.

Medications were coded using WHO drug dictionary version vMar2023.

### **Programming Notes:**

- ATC & Preferred Name text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name.
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX") but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications





# Listing 16.2.6.6 Patient Global Impression of Change mITT Population

| Subject ID | Treatment Arm | Study Visit | Collection Date / Study Day | PGIC |
|---|---|---|---|---|
| XXXXXX | XXXX | Week 4 | DDMMMYYYY/(X) | XXXXXXXX |
| | | Week 8 | DDMMMYYYY/(X) | XXXXXXXX |
| | | Week 12 | DDMMMYYYY/ (X) | XXXXXXX |
| | | Week 18 | DDMMMYYYY/(X) | XXXXXXX |
| XXXXXX | XXXX | Week 4 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 8 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 12 | DDMMMYYYY/ (X) | XXXXXXX |
| | | Week 18 | DDMMMYYYY/(X) | XXXXXXX |

PGIC =Patient Global Impression of Change.

Note: Data shown in column 'PGIC' are Subjects ratings about overall improvement in health status.

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include all observed data on PGIC scores for Week 4, 8, 12, and 18.

Draft 1.1 | 31-Aug-2023 | 







Draft 1.1 | 31-Aug-2023 | 





CCI



Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.7.1 Adverse Events Safety Population

| Subject ID/<br>Treatment<br>Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | AE Start Date/Time<br>(Study Day)/<br>End Date/Time<br>(Study Day) | Severity/<br>Relationship<br>[1] | Outcome/ Action Taken with IP/ Therapy taken for this AE | AE Leading<br>to Study DC | ?<br>TEAE | Serious? /<br>Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMMMYYYY/HH<br>MM (X)/<br>X DDMMMYYYY/HH<br>MM (X) | XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>Yes | No | Yes | No |
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMMMYYYY/HH<br>MM (X)/<br>X DDMONYYYY/HH:<br>MM (X) | XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>No | Yes | No | Yes / XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMONYYYY/HH:<br>MM (X)/<br>X Ongoing | XXXXXX/<br>XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>No | No | No | Yes / XXX |

AE = adverse event; DC = discontinuation; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Study Day is calculated relative to the date of first dose. A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0

<sup>[1]</sup> Reasonable possibility AE caused by IP as assessed by the investigator.





## **Programming Notes:**

- If time missing, display "--:--".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e, no AEs occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically by SOC /PT if same date for two events).

In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Listing 16.2.7.2
Treatment Emergent Adverse Events Leading to Study Drug Discontinuation
Safety Population

### **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update listing deleting seventh and eight columns

Listing 16.2.7.3
Treatment Emergent Adverse Events Associated with Abnormal Liver
Safety Population

## **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update listing deleting 8<sup>th</sup> column.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.7.4 Joint Related Adverse Events of Special Interest Safety Population

### **Programming Notes:**

• Same shell as Listing 16.2.7.1.

Listing 16.2.7.5 Serious and/or Severe Infections Safety Population

### **Programming Notes:**

• Same shell as Listing 16.2.7.1.

Listing 16.2.7.6

Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of Study Drug Safety Population

### **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update footnote: Anaphylactic reactions, hypersensitivity or infusion-related reactions not leading to discontinuation of IP were included in listing as they were categorized as AE of special interest under Protocol Amendment 4 (V5.0). Definition for AE of special interest changed from Amendment 6 (V6.0) onwards, including an applylactic reactions, hypersensitivity or infusion-related reactions leading to permanent discontinuation of IP.

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.8.1 Clinical Chemistry Laboratory Evaluations Safety Population

| Subject ID/<br>Treatment Arm | Parameter | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Original<br>Result<br>(Unit) | Standard<br>Results<br>(unit) | Reference<br>Range<br>[1] | Baseline<br>Flag | CFB | Results<br>Assessment<br>/ Reason<br>CS | Lab ID<br>Number | Fasting<br>Status | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | Chemistry panel | XXXXXX | | | | | | | ND: xxx | | | |
| XXXXX/<br>XXXX | Albumin | XXXXXX<br>XXXXXX<br>XXXXXX<br>XXXXXX | DDMMMYYYY/ HH:MM (X) DDMMMYYYY/ HH:MM (X) DDMMMYYYY/ HH:MM (X) DDMMMYYYY/ HH:MM (X) | XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX) | XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX) | XX - YY XX - YY XX - YY XX - YY | Y | XX.X<br>XX.X<br>XX.X | H-CS /<br>XXX<br>H-NCS | XXXXXXX<br>XXXXXXX<br>XXXXXXX<br>XXXXXXX | Y<br>Y<br>Y<br>N | XXXX |

CFB = change from baseline; CS = clinically significant; H = High; L = Low; NCS = not clinically significant; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

[1] Reference range is used to identify potentially clinically significant laboratory values.

# **Programming Notes:**

- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Chemistry panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Albumin, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Bicarbonate, Calcium, Chloride, Creatinine, High-Sensitivity C-Reactive Protein (hs-CRP), Estimated Glomerular Filtration Rate (eGFR by Cockcroft-Gault), Serum Glucose, Lactate Dehydrogenase (LDH), Potassium, Sodium, Total Bilirubin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid.

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.8.2 Hematology Laboratory Evaluations Safety Population

### **Programming Notes:**

- Same shell as Listing 16.2.8.1.
- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Hematology panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Absolute basophil count, absolute eosinophil count, absolute lymphocytes count, Absolute Monocyte Count, Absolute Neutrophil Count, Basophils %, Eosinophils %, Hematocrit (HCT), Hemoglobin (HGB), hemoglobin A1C (HgbA1C), Lymphocytes %, mean corpuscular hemoglobin (MHC), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), Monocytes %, Neutrophils %, Platelets, Red blood cell count (RBC), Red Cell Distribution Width, white blood cell Count (WBC).

Listing 16.2.8.3 Coagulation Laboratory Evaluations Safety Population

### **Programming Notes:**

- Same shell as Listing 16.2.8.1.
- Keep parameter sorting from the last bullet point below.
- · For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Coagulation panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Activated Partial Thromboplastin Clotting Time (APTT), Fibrinogen, International normalized ratio (INR), Prothrombin Time (PT).

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.8.4 Urinalysis Laboratory Evaluations Safety Population

| Subject ID/<br>Treatment Arm | Parameter | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Original<br>Result<br>(Unit) | Standard<br>Results<br>(unit) | Reference<br>Range<br>[1] | Baseline<br>Flag | CFB | Results<br>Assessment<br>/ Reason<br>CS | Lab ID<br>Number | Fasting<br>Status | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Urinalysis<br>panel | XXXXXX | | | | | | | ND: xxx | | | |
| XXXXX | pH/<br>Specific<br>Gravity | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX<br>(XX) | XX<br>(XX) | XX - YY | Y | | | XXXXXXX | Y | |
| | Glavity | XXXXXX | DDMMMYYYY/ | XX | XX | XX - YY | | XX.X | H-CS/ | XXXXXXX | Y | XXXX |
| | | XXXXXX | HH:MM (X)<br>DDMMMYYYY/ | (XX)<br>XX | (XX)<br>XX | XX - YY | | XX.X | XXX | XXXXXXX | Y | |
| | | XXXXXX | HH:MM (X)<br>DDMMMYYYY/<br>HH:MM (X) | (XX)<br>XX<br>(XX) | (XX)<br>XX<br>(XX) | XX - YY | | XX.X | H-NCS | XXXXXXX | N | |
| | Blood<br>Urine/<br>Glucose/<br>Ketones/<br>Protein | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Trace | | | Y | | H-NCS | XXXXXXX | Y | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | 100<br>(mg/dL) | 100<br>(mg/dL) | | | | H-CS /<br>XXX | XXXXXXX | Y | XXXX |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Negative | | | | | | XXXXXXX | N | |

Draft 1.1 | 31-Aug-2023 | 





CFB = change from baseline; CS = clinically significant; H = High; L = Low; NCS = not clinically significant; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

[1] Reference range is used to identify potentially clinically significant laboratory values.

### **Programming Notes:**

- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Urinalysis panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Blood Urine, Glucose, Ketones, pH, Protein, Specific Gravity.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.8.5 Serology Laboratory Evaluations Safety Population

| Subject<br>ID | Treatment<br>Arm | Was<br>Serology<br>Test<br>Collected? | Date/Time of<br>Collection<br>(Study Day) | Test (Unit) [1] | Result | Lab ID<br>Number | Fasting<br>Status | Reason not collected | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXX | Yes | DDMMMYYY<br>Y/HH:MM (X) | Hepatitis B Ag | Negative | XXXX | Y | | XXXXXXXX |
| | | | | Hepatitis C Ab | Positive | XXXX | Y | | |
| | | | | HIV-1/ -2 Ag | Not Done | XXXX | Y | XXXXXXX | |
| | | | | Quantiferon<br>Gold Plus NIL | X.XX (IU/mL) | XXXX | Y | | |

Ab = antibody; Ag = antigen; HIV = human immunodeficiency virus; TB = tuberculosis.

Note: Study Day is calculated relative to the date of first dose.

[1] if Applicable

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date of collection / Test.
- Keep parameter sorting from the last bullet point below
- Sort Parameters in the following Order: Hepatitis B Antigen, Hepatitis C Virus Antigen, Hepatitis C Virus Antibody, HIV-1/-2 Antigen, Quantiferon Gold Plus NIL, Quantiferon Gold Plus TB, Quantiferon Gold Plus Mitogen minus NIL, Quantiferon Gold Plus TB1 minus NIL, Quantiferon Gold Plus TB2 minus NIL

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.8.6 Pregnancy Test Results Safety Population

| Subject ID | Treatment<br>Arm | Visit | Was a Urine pregnancy test performed? | Date/Time Performed (Study Day) | If not, Reason | Result |
|---|---|---|---|---|---|---|
| XXXXX | xxxx | xxxxx | Xxxx | Ddmmmyyyy/ hh:mm (XX) | xxxx | XXXX |
| | | xxxxx | Xxxx | Ddmmmyyyy/ hh:mm (XX) | Other: xxxx | xxxx |

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment.

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.8.7 Drug Test Results Safety Population

| Subject ID | Treatment<br>Arm | Was Drug Test<br>Performed? | Date/ Time Assessment<br>(Study Day) | Result | Findings | Reason Test<br>not Performed |
|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Yes | DDMMMYYYY/ HH:MM<br>(XX) | Negative | Negative | |
| XXXXXX | XXXX | Yes | DDMMMYYYY/ HH:MM<br>(XX) | Positive | Cocaine /<br>Opiates | |

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Concatenate all findings by "/"
- Sort by Treatment Arm/ Subject ID / Date of assessment.

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.8.8 COVID-19 Screening Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit | COVID-19 Sx<br>Screening?/Date<br>/ Time (Study<br>Day) | Sx | Body T°<br>Check?/Date/<br>Time (Study<br>Day) | Body T°<br>(Unit) | COVID-19<br>swab?/ Date/<br>Time (Study<br>Day) | Swab<br>result | COVID-19 Ab<br>testing?/ Date/<br>Time (Study<br>Day) | Ab<br>testing<br>results | COVID-19<br>Ag testing?/<br>Date/ Time<br>(Study Day) | Ag<br>testing<br>results |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx/<br>xxxx | xxxx | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XXX/<br>XXX | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XX (XX) | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Yes/ Ddmmmyyyy/ hh:mm (XX) | Xxxx | Yes/ Ddmmmyyyy / hh:mm(XX) | Xxxx |
| | xxxx | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XXX | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | XX (XX) | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Yes/<br>Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Yes/<br>Ddmmmyyyy<br>/ hh:mm(XX) | Xxxx |

Ab = Antibody; Ag = Antigen; COVID-19 = Corona virus disease 2019; Sx = Symptoms; T° = Temperature.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Concatenate all Symptoms by "/"
- Sort by Treatment Arm/ Subject ID / Date of assessment

Draft 1.1 | 31-Aug-2023 | 





### Listing 16.2.9.1 Vital Signs Measurements Safety Population

| Subject<br>ID | Treatment<br>Arm | Parameter | Study<br>Visit | Position [1] /<br>T° Method | Date/Time of<br>Collection<br>(Study Day) | Original Result<br>(Unit) | Baseline Flag | CFB |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Body<br>Temperature | XXXXXX | XXXX | DDMMMYYYY/<br>HH:MM (X) | XX (XX) | Y | |
| | | • | XXXXXX | XXXX | DDMMMYYYY/<br>HH:MM (X) | XX (XX) | | XX |
| | | | | | | ••• | | |
| | | Resting<br>Heat Rate | Screening | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | | |
| | | | Day 1:<br>Pre-Dose | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | Y | XX |
| | | | XXXXXX | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | | XX |
| | | | XXXXXX<br>XXXXXX | Sitting<br>Sitting | DDMMMYYYY/<br>HH:MM (X) | ND<br>XX | | XX |

CFB = change from baseline; eCRF = Electronic Case Report Form; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

'Day 1:5 minutes after Infusion Completion' time point was only applied to subjects enrolled in Stage 1, with data collected under eCRF versions 4.0 (11DEC2018) or older.

[1] Resting position measurements encompass Sitting and Supine position measurements.

Draft 1.1 | 31-Aug-2023 | 





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter (Order in the second bullet point)/ Date time of collection.
- Repeat for Resting Heart Rate, Resting Systolic Blood Pressure, Resting Dia stolic Blood Pressure, Respiratory Rate, Body Temperature, Standing Heart Rate, Standing Systolic Blood Pressure, Standing Dia stolic Blood Pressure.
- After Week 2 (inclusive), Supine measure are taken in sitting position. We will consider them as supine (in resting position) for calculating Change from Baseline (always at supine position).
- Include the following timepoints: Screening, Baseline (Day 1: Pre-Dose), Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: Pre-Dose, Week 10: 5 minutes after Infusion Completion, Week 11, Week 12, Week 18.
- Note that Body To, and standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.9.2.1 12-Lead Digital ECG Results Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Visit | ECG Date / Time<br>(Study Day) | Tracin<br>g | PR Interval (msec) | QRS<br>duration<br>(msec) | QT<br>Interval<br>(msec) | RR<br>interval<br>(bpm) | Heart Rate<br>(beats/min) | QTcF<br>Interval<br>(msec) | Findings | Reason<br>Not<br>Done |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Day 1:<br>Pre-Dose | DDMMMYYYY<br>/ HH:MM (XX) | 1 | XX | XX | xx | xx | XX | XX | xx:<br>xxxxx | |
| | | • | 2 | XX | XX | XX | XX | XX | XX | | |
| | | | 3 | XX | XX | XX | XX | XX | XX | xx:<br>xxxxx | |
| XXXXX | XXXX | DDMMMYYYY/<br>HH:MM (XX) | 1 | xx | XX | XX | xx | XX | XX | xx:<br>xxxxx | |
| | | | 2 | XX | XX | XX | XX | XX | XX | | |
| | | | 3 | XX | XX | XX | XX | XX | XX | | |

CS = clinically significant; ECG = electrocardiogram; NCS = Not clinically significant

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date time of collection / Tracing.
- For Findings, concatenate test name with test result for category "FINDINGS".
- Include the following timepoints: Day 1: Pre-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.

Draft 1.1 | 31-Aug-2023 | 





### 00Listing 16.2.9.2.2 12-Lead Safety ECG Results Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit | ECG Date / Time<br>(Study Day) | Tracing | ECG Result/<br>Comment | PR Interval (msec) | QRS duration (msec) | QTcF<br>Interval<br>(msec) | Reason<br>Not Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | Day 1: Pre-<br>Dose | DDMMMYYYY /<br>HH:MM (XX) | 1 | AbnormalCS/ xxxx | XX | xx | XX | |
| | | ` ' | 2 | Abnormal CS/xxxx | XX | XX | XX | |
| | | | 3 | Abnormal NCS/<br>xxxx | XX | XX | XX | |
| XXXXX | XXXX | DDMMMYYYY/<br>HH:MM (XX) | 1 | Normal | XX | XX | xx | |
| | | , | 2 | Normal | XX | XX | XX | |
| | | | 3 | Normal | XX | XX | XX | |

CS = clinically significant; ECG = electrocardiogram; NCS = Not clinically significant

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date time of collection / Tracing.
- Include the following timepoints: Screening, Day 1: Pre-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.3 Physical Examination Results Safety Population

| Subject ID | Treatment<br>Arm | Visit | Examination<br>Type | Exam Date/ Time<br>(Study Day) | Body System | Result / Change<br>from previous<br>assessment [1] | If Abnormal,<br>findings /<br>Specify<br>Changes [2] | Reason Not<br>Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Screening | Complete | DDMMMYYYY<br>/ HH:MM (XX) | Head, Neck and<br>Thyroid<br>Ears, Eyes, Nose<br>and Throat | Normal<br>Abnormal CS | XXXXXXX | |
| | | Day 1 | Targeted | DDMMMYYYY<br>/ HH:MM (XX) | Ears, Eyes, Nose<br>and Throat | xxxxxxxxx | XXXXXXXX | |

CS = Clinically Significant, NCS = Not Clinically Significant

Note: Study Day is calculated relative to the date of first dose.

[1] For targeted examination type: Change from previous assessment.

[2] For targeted examination type: Specify Changes.

# **Programming Notes:**

- Keep sorting from eCRF: Head, Neck and Thyroid/Ears, Eyes, Nose and Throat/ Chest (including breasts)/ Lungs/Heart/LymphNodes/Abdomen/Hepatic/Gastrointestinal/Anorectal/Genitourinary/Skin/Musculoskeletal/Extremities/Neurological/Other.
- Complete Physical examination only at Screening, Week 12, 18 (it can also be unscheduled).
- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Body system

Draft 1.1 | 31-Aug-2023 | 




# Listing 16.2.9.4 Neurological Examination Results Safety Population

| | Treatment | | Exam Date/ Time | | | If Abnormal, | Reason Not |
|---|---|---|---|---|---|---|---|
| Subject ID | Arm | Visit | (Study Day) | Body System | Result | findings | Done |
| XXXXX | XXXX | Screening | DDMMMYYYY /<br>HH:MM (XX) | Mental Status | Normal | | |
| | | | , | Cranial Nerves | AbnormalCS | XXXXXXX | |
| | | Day 1 | DDMMMYYYY /<br>HH:MM (XX) | Cranial Nerves | XXXXXXXXX | XXXXXXXX | |

CS = Clinically Significant, NCS = Not Clinically Significant

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Keep sorting from eCRF: Mental status/ Cranial Nerves/ Motor Function/ Reflexes / Sensation and Propioception / Coordination / Other.
- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Body system

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.9.5
Total Neuropathy Score-Nurse
Safety Population

| | | | | ~ ~ . | 100 T op 6.716.110 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | | Sensory | Motor | | Pin | Vibration | | |
| ID/ | | Date/ Time of | Symptom | Symptom | Autonomic | Sensibility | Sensibility | | |
| Treatment | | collection | Score | Score | Symptom | Score | Score | TNSn Total | |
| Arm | Visit | (Study Day) | (0-4) | (0-4) | Score (0–4) | (0-4) | (0-4) | (0-20) | Reason Not Done |
| XXXXX/<br>XXXX | Screening Day 1 | DDMMMYYYY<br>/HH:MM (XX)<br>DDMMMYYYY | XX | XX | XX | XX | XX | XX | |
| | | / HH:MM (XX) | XX | XX | XX | XX | XX | XX | |
| | Week 2 | DDMMMYYYY<br>/ HH:MM (XX) | ND | ND | ND | ND | ND | ND | XXXXXXXXXXXX |

ND = Not Done; TNSn = Total Neuropathy Score-Nurse.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.6 Motor and Sensory Nerve Conduction Studies Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit | Date/Time of<br>Collection<br>(Study Day) | Location /<br>Evaluation | Was<br>Evaluation<br>Preformed<br>? / Nerve | Amplitude<br>(Motor =<br>mV; sensory<br>= microV)/<br>Range | Peak<br>Latency<br>(msec)/<br>Range | Conduction<br>velocity<br>(msec) /<br>Range | Duration<br>of action<br>potential<br>(msec) /<br>Range | Evaluation<br>Result | If<br>Abnomal,<br>Specify/<br>Reason<br>Not Done | Significant<br>Changes<br>from<br>Baseline? /<br>if Yes,<br>Specify |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX/<br>XXXX | Screening | DDMMMYY<br>YY / HH:MM<br>(XX) | Lower Limb - Right Side/ | Y/<br>XXXXXX<br>Y/<br>XXXXXX<br>N | xx [x.xx to x.xx] xx [x.xx to x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx to | xx [x.xx to x.xx] xx [x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx] | Abnormal<br>Normal | XXXXX | NA<br>NA |
| | Week 18 | DDMMMYY<br>YY/ HH:MM<br>(XX) | XXXXXX/<br>XXXXXX/<br>XXXXXX/<br>XXXXXX/<br>XXXXXX/ | Y/<br>XXXXXX<br>Y/<br>XXXXXX<br>Y/<br>XXXXXX | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | Abnormal Normal Abnormal | XXXXX | N<br>N<br>Y/<br>XXXXXXX |

NA = Not Applicable

Note: Study Day is calculated relative to the date of first dose.





## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Location Evaluation
- Keep sorting from eCRF: Lower Limb right side/Motor evaluation, Lower Limb right side/Sensory evaluation, Lower Limb left side/ Motor evaluation, Upper Limb right side/Sensory evaluation, Upper Limb left side/ Motor evaluation, Upper Limb left side/ Sensory evaluation, Upper Limb left side/ Sensory evaluation.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.7 Strength and Deep Tendon Reflexes Safety Population

| Subject ID | Treatment<br>Arm | Visit | Date/ Time of<br>collection<br>(Study Day) | Ankle Dorsiflexion<br>Strength | Deep Tendon Reflexes | Reason Not Done |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | Screening | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | |
| | | Day 1 | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | |
| | | Week 2 | DDMMMYYYY /<br>HH:MM (XX) | ND | ND | XXXXXXXXXXXX |

ND = Not Done.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.8 Injection Site Reactions Safety Population

| Subject<br>ID | Treatment<br>Arm | Visit | Date/Time of Assessment<br>(Study Day) | Pain | Tenderness | Erythema/redness | Induration/<br>swelling | Reason Not Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Day 1: 15<br>Minutes<br>after Start of<br>Infusion | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | XXXX | XXXX | |
| | | Day 1: 30<br>Minutes<br>after Start of<br>Infusion | DDMMMYYYY /<br>HH:MM (XX) | XX | XX | XX | XX | |
| | | <br>Week 18 | DDMMMYYYY /<br>HH:MM (XX) | ND | ND | ND | ND | XXXXXXXXXXXX |

ND = Not Done.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment
- Include the following timepoints: Day 1: 15 Minutes after Start of Infusion, Day 1: 30 Minutes after Start of Infusion, Day 1: 45 Minutes after Start of Infusion, Day 1: 60 Minutes after Start of Infusion, Day 1: 4 hours after Start of Infusion, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.9.9 Hypersensitivity/Anaphylactic Reactions Safety Population

| Subject<br>ID | Treatment<br>Arm | AE ID<br>Number | Onset Date/Time (Study Day)/<br>Resolution Date/Time (Study<br>Day) | Type of<br>Reaction | Severity grade for<br>the Symptom<br>with Highest<br>Severity | Onset Time<br>for Highest<br>Severity | Leading to IP<br>Discontinuation? |
|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXX | XXXX | /HH:MM | Yes |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXX | | | No |
| | | ••• | | | | | |
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXX | XXXX | /НН:ММ | No |

AE = Adverse Event.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Onset Date/Time / Resolution Date/Time / Reaction Type.
- Keep sorting from eCRF: Urticaria, Pruritus, Rash, Flushing, Swollen lips, tongue, uvula and/or vulva, Dyspnoea, Wheeze-bronchospasm, Stridor, Hypoxia, Hypotension, Crampy abdominal pain, Vomiting, Diarrhoea, Other.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.10 Liver Diagnostic Investigations Safety Population

| Subject ID | Treatment<br>Arm | Potential Hy's<br>Law Case<br>Number | Liver Diagnostic Investigation<br>Date (Study Day) | Liver Diagnostic<br>Investigation | Liver Dia gnostic<br>Investigation<br>Results | Comments |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY (X) | XXXX | XXXX | XXXXX |
| | | X | DDMMMYYYY (X) | XXXXX | XXXXX | |
| XXXXX | XXXX | X | DDMMMYYYY (X) | XXXXX | XXXXX | |

CT = Computerized tomography; ERCP = Endoscopic retrograde cholangiopancreatography; MRI = Magnetic resonance imaging; MRCP = Magnetic resonance cholangiopancreatography.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Diagnostic Date / Liver Diagnostic Investigation.
- Keep sorting from eCRF: Ultra sound, CT, MRI/MRCP, ERCP, Liver Biopsy, X-Ray, Tox Screening for Acetaminophen/Paracetamol, Tox Screening for Ethanol, Tox Screening, Other, Specialist (e.g. Hepatologist) Consulted, Serology for Hepatitis A, Serology for Hepatitis B, Serology for Hepatitis C, Serology for Hepatitis D, Serology for Hepatitis E, for Cytomegalovirus (CMV), Serology for Epstein Barr Virus (EBV), Autoimmune Serology, Other.

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.9.11
Liver Risk Factors and Lifestyle Events
Safety Population

| | | Potential | | Liver Risk Factor Start Date | Liver Risk | | |
|---|---|---|---|---|---|---|---|
| | | Hy's Law | Assessment Date | (Study Day)/ | Factor/ | | |
| | Treatment | Case | (Study Day) | Liver Risk Factor Stop Date | Reference | Liver Risk | |
| Subject ID | Arm | Number | | (Study Day) | Period | Factor Details | Comments |
| XXXXX | XXXX | X | DDMMMYYYY<br>(X) | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXX/<br>XXX | XXXX | XXXXX |
| | | X | DDMMMYYYY<br>(X) | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXX/<br>XXX | XXXXX | |
| | | ••• | | | | | |
| XXXXX | XXXX | X | DDMMMYYYY<br>(X) | DDMMMYYYY (X)/<br>Ongoing | XXXXX/<br>XXX | XXXXX | |

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Assessment Date / Liver Risk Factor Start Date / Stop Date / Liver Risk Factor.
- Keep sorting from eCRF: Alcohol Abuse, Increased Alcohol Consumption within 1 Month of Reported Event, IV Drug Abuse, Tattoo, Acupuncture, Sexually Transmitted Diseases, Toxic/Chemical Agent Exposure, Travel (Areas at Risk in the Last Year), Pregnancy, Parenteral Nutrition, Excessive Physical Exercise, Changes Diet/Fasting Episodes/Weight Loss Diet, Previous Drug Reaction (Associated with an Elevation of Liver Tests), Blood Transfusion, Subject Exposed to Anyone with Jaundice in the Last Month, History of Hypotension, Low Blood Pressure at Time of Event of Liver Injury and/or Abnormal Liver Laboratory Value, History of Liver Disease, Other.
- Concatenate comments with "/".

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.9.12 Liver Signs and Symptoms Safety Population

| | | Potential Hy's | Start Date (Study Day)/ | Liver Sign/ | |
|---|---|---|---|---|---|
| Subject ID | Treatment Arm | Law Case Number | Stop Date (Study Day) | Symptom | Intermittent |
| XXXXX | XXXX | X | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXX | N |
| | | X | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXX | N |
| | | ••• | | | |
| XXXXX | XXXX | X | DDMMMYYYY (X)/<br>Ongoing | XXXXX | Y |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Liver Sign/Symptom.
- Keep sorting from eCRF: Anorexia, Asthenia, Pyrexia, Pruritus, Jaundice, Arthralgia, Abdominal Pain, Abdominal Tenderness, Nausea, Vomiting, Rash, Mucosal Inflammation, Purpura, Hepatomegaly, Splenomegaly, Lymphadenopathy, Ascites, Confusional State, Coma, Upper Quadrant Tenderness, Biliary Obstruction, Eosinophilia, Dark Urine, Other.
- If Rash, Lymphadenopathy or Other, Concatenate Symptom with Comment as: "Rash: xxxxxx". "Lymphadenopathy: xxxxxx", "Other: xxxxxxxx"

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.9.13
Infection Diagnostic Investigations
Safety Population

| Subject ID | Treatment Arm | AE ID<br>Number | Start Date/ Time (Study Day)/<br>Stop Date/ Time (Study Day) | Method | Examination performed | Test Result |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXX | Y | XXXXX |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X)) | XXXXX | Y | XXXXX |
| XXXXX | XXXX | <br>X | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXX | N | XXXXX |

AE = adverse event.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Method.
- Keep sorting from eCRF: Microscopy, Culture and Sensitivity, Serological Tests, Nucleic Acid Based Tests, X-Ray, Other.

Draft 1.1 | 31-Aug-2023 | 





Listing 16.2.9.14
Infection Risk Factors and Lifestyle Events
Safety Population

| Subject ID | Treatment<br>Arm | AE ID<br>Number | Start Date/ Time (Study Day)/<br>Stop Date/ Time (Study Day) | Infection Risk<br>Factor | Infection Risk<br>Occurrence | Comments |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXX | Y | XXXXX |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X)) | XXXXX | Y | XXXXX |
| XXXXX | XXXX | <br>X | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXX | N | Ongoing |

AE = adverse event; BCG = Bacillus Calmette-Guérin.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Infection Risk Factor.
- Keep sorting from eCRF: Extensive Burns within the Last Year (Thermal Burn), Tattoo, Piercing or Acupuncture within the Last Year, Sexually Transmitted Diseases, Travel to Areas at Risk of Tuberculosis or Tropical Diseases, Infections Related to Travel (e.g. Tuberculosis and Tropical Diseases), Blood Transfusion (within the Last Year), Exposure to Nosocomial Pathogens within the Last Year, Contact History with Infection Source, Previous BCG Immunization, Evidence of BCG Scar, Tuberculin Skin or Quantiferon Test Confirms Previous Exposure or Immunity to Tuberculosis.
- Fill Comment column if Infection risk factor test = Unknown Previous BCG Immunization, not done, known Sexually Transmitted Disease reference Period, or Infection risk factor specifications.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.15 Infection Signs and Symptoms Safety Population

| | | | System Organ Class/ | · · · | | Infection | |
|---|---|---|---|---|---|---|---|
| | Treatment | AE ID | Preferred Term/ | Start Date/ Time (Study Day)/ | Clinical | Sign/Symptom | |
| Subject ID | Arm | Number | Verbatim Term | Stop Date/ Time (Study Day) | Event | Occurrence | Comments |
| XXXXX | XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM<br>(X) | | Y | |
| | | | XXXXXXXXXX | | XXXXX | | XXXXX |
| | | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM<br>(X)) | XXXXX | Y | XXXXX |
| | | ••• | | | | | |
| XXXXX | XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXX | N | Ongoing |

AE = adverse event.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Clinical Event.
- Keep sorting from eCRF: Pyrexia, Headache, Confusional State, Convulsion, Rhinitis, Oropharyngeal Pain, Cough, Productive Cough, Haemoptysis, Wheezing, Dyspnoea, Pleuritic Pain, Vomiting, Diarrhoea, Genital Discharge, Haematuria, Dysuria, Hepatosplenomegaly, Jaundice, Lymphadenopathy, Rash, Night sweats, Chills, Myalgia, Weight Decrease.
- Fill Comment column if Maximum To (Unit) available for Pyrexia, or if site for Rash or Lymphadenopathy is known.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.16 Prior and Concomitant Medications Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Prior/<br>Concomitant<br>[1] | ATC Class (Level 2)/<br>Preferred Name/<br>Verbatim Term | Given<br>for/as | Primary<br>Indication | Start Date (Study<br>Day)/<br>End Date (Study<br>Day) | Dose (unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|---|
| XXXXXX<br>/ XXXX | Prior | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXX | Medical<br>History | XXXXXXX | MMMYYYY<br>(-XX)/<br>DDMMMYYYY<br>(-X) | XXXX unit | XXXXXX<br>XXX | XXXXX |
| | Both | XXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXX | Prophylaxis | XXXXXXX | MMMYYYY<br>(-X)/<br>Ongoing | XXXX unit | XXXXXX<br>XXX | XXXXX |
| | Concomitant | XXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Adverse<br>event | XXXXXXX | DDMMMYYYY<br>(X)/<br>DDMMMYYYY<br>(XX) | XXXX unit | XXXXXX<br>XXX | XXXXX |

 $ATC = anatomical\ the rapeutic\ chemical;\ WHO-DDE = World\ Health\ Organization-Drug\ Dictionary\ Enhanced.$ 

Note: Study Day is calculated relative to the date of first dose.

Medications were coded using WHO-DDE version vMar2023.

[1] Prior medications are defined as medications that started before first dose of study, whether they were stopped before first dose of study medication or not. Concomitant medications are defined as medications starting on or after first dose of study medication Both indicates medication that was started before the day of first dose and continued after.

Draft 1.1 | 31-Aug-2023 | 





### **Programming Notes:**

- ATC & Preferred Name text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name.
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX") but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by Treatment ID/ Subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications)

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.17 Prohibited Concomitant Medications Safety Population

### **Programming Notes:**

- Same Shell as Listing 16.2.9.16.
- Display prohibited prior and concomitant medications provided by the Medical Coder:
- Prohibited concomitant medications:
  - $\circ$  NSAIDs analgesic therapies (with acetylsalicylic acid with doses  $\geq 325$  mg/day).
  - COX-2 analgesic therapies.
  - o Immunotherapeutics.
  - o Live viral or attenuated bacterial vaccines.
  - o Oral, IV, intramuscular, or any other parenteral (other than oral) steroids (inhaled or topical steroids are permitted).
  - o Biologic therapeutic agents.
- Prohibited prior and/or concomitant medications:
  - o Anti-NGF therapies.
  - o Anti-TNF therapies.
- ATC & PN text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name.
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications)

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.9.18 Concomitant Procedures Safety Population

| | | | J : | | | |
|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Arm | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day) | Reason for Procedur | Reason (derived verbating term) | n If Reason is Other,<br>Specify |
| XXXXX | XXXX | XXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXXXXXX/<br>XXXXXXXX | XXXXXXXXX | |
| XXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX | |
| XXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>Ongoing | OTHER | OTHER | XXXXXXXXXX |

MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study Day is calculated relative to the date of first dose. All Procedure terms were coded using the MedDRA version 26.0. Concomitant Procedures are defined as medications continuing or starting on or after first dose of study medication.

## **Programming Notes:**

- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Draft 1.1 | 31-Aug-2023 | 





# Listing 16.2.9.19 Anti-drug Antibody Test Results Safety Population

| Subject<br>ID | Treatment<br>Arm | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Screening<br>Status Result | Confirmatory<br>Status result | ADA Titer | Lab ID<br>Number | Comments |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Positive | Positive | XX | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Positive | Positive | XX | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Negative | Negative | XX | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Missing | Not<br>Reportable<br>Result | NRR | XXXXXXX | XXXX |

ADA = Anti-Drug Antibodies; NA = Not Applicable; NRR = Not Reportable Result; QNS = Quantity Not Sufficient. Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- ADA titre reported as <30 (below the minimum required dilution) is a negative result for the presence of ADA.
- Include Following timepoints: Screening, Weeks 2, 4, 8, 10, 12, 18.

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.10.1 Serum MEDI7352 Concentrations PK Population

| Subject<br>ID | Treatment<br>Arm | Study<br>Visit | PK Blood<br>Sample<br>Collected? /<br>Reason Not<br>Collected | Date/Time of<br>Collection<br>(Study Day) | MEDI7352<br>Concentration<br>(ng/mL) | Lab ID Number | Comments |
|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | NRR | XXXXXXX | XXXX |
| | | XXXXXX | No /<br>XXXXXX | | | | |

NA = Not Applicable; NRR = Not Reportable Result.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours: after Week 10/Pre-Dose, Week 11: after Week 10/Pre-Dose, Week 10 + 14 Days: after Week 10/Pre-Dose, Week 18.

Draft 1.1 | 31-Aug-2023 | 





#### Listing 16.2.10.2 Serum total NGF Concentrations Safety Population

| | | | | <i>j</i> <u>F</u> | | | |
|---|---|---|---|---|---|---|---|
| | | | PD Blood Sample | | | | |
| | | | Collected? / | Date/Time of | Total NGF | | |
| Subject | Treatment | Study | Reason Not | Collection | Concentration | | |
| ID | Arm | Visit | Collected | (Study Day) | (pg/mL) | Lab ID Number | Comments |
| XXXXX | XXXX | XXXXXX | Yes | DDMMMYYYY/ | XX | XXXXXXX | |
| | | | | HH:MM(X) | | | |
| | | XXXXXX | Yes | DDMMMYYYY/ | XX | XXXXXXX | |
| | | | | HH:MM(X) | | | |
| | | XXXXXX | Yes | DDMMMYYYY/ | NS | XXXXXXX | XXXX |
| | | | | HH:MM(X) | | | |
| | | XXXXXX | No / | ( ) | | | |
| | | | XXXXXX | | | | |

BLLOQ = Below the Lowest Limit of Quantitation; NA = Not Applicable; ND = Not Detected; NS = No Value due to Insufficient Volume or No Sample Received; PD: Pharmacodynamic; SAT = Greater than the Top of the Standard Curve; tNGF = total Nerve-Growth Factor. Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.

Draft 1.1 | 31-Aug-2023 | 





## **Planned Figure Descriptions and Shells**

| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Figure 14.2.1.1 - Daily Pain NRS: MCP-Mod Dose Response Model - mITT Population | U |
| Figure 14.2.1.2 - Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Missing Data Handling - mITT Population | U |
| Figure 14.2.1.3 - Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup - mITT Population | R |
| Figure 14.2.1.4 - Daily Pain NRS: MMRMLS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases) - mITT Population | U |
| Figure 14.3.6.1.1 - Vital Sign Profiles: Mean (±SD) Systolic Blood Pressure over time - Safety Population | U |
| Figure 14.3.6.1.2 - Vital Sign Profiles: Mean (±SD) Diastolic Blood Pressure over time - Safety Population | |
| Figure 14.3.6.1.3 - Vital Sign Profiles: Mean (±SD) Heart Rate over time - Safety Population | |
| Figure 14.3.6.1.4 - Vital Sign Profiles: Mean (±SD) Respiratory Rate over time - Safety Population | |
| Figure 14.3.6.1.5 - Vital Sign Profiles: Mean (±SD) Temperature over time - Safety Population | R |
| Figure 14.4.1.1 - Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 over time - PK Population | R |
| Figure 14.4.1.2 - Pharmacokinetics: Individual Plot of Serum MEDI7352 Concentrations over time - PK Population | |
| Figure 14.4.2.1 - Pharmacodynamics: Line Plot of Geometric Mean (with and without gSD) total NGF over time - Safety Population | R |
| Figure 14.4.2.2 - Pharmacodynamics: Individual Plot of Serum total NGF over time - Safety Population | R |

Draft 1.1 | 31-Aug-2023 | 





## **Figures Change Log**

| Output<br>Number | Date of<br>Change | Change<br>Made By<br>(initials) | Description/Rationale |
|---|---|---|---|

Draft 1.1 | 31-Aug-2023 | 





Figure 14.2.1.1
Daily Pain NRS: MCP-Mod Dose Response Model mITT Population

#### Weekly Average to Week 12 Daily Pain NRS CFB, Emax dose-response model



CI = Confidence Interval; CFB = Change from Baseline; DPS = Daily Pain Score; NRS = Numeric Rating Scale.
Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e.,
Day -7 to Day -1, inclusive. Envelope depicts 95% CI of mean dose-response. Added dots are actual doses ± 95% CI.
mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.
Reference Listing: 16.2.6.1

Draft 1.1 | 31-Aug-2023 | 





## **Programming Notes:**

- Insert the following text as legend: "Weekly Average to Week 12 Daily Pa in NRS CFB, xxxx dose-response model", with 'xxxx' as the selected dose-response model (e.g., Hyperbolic E<sub>max</sub>).
- Dose (μg/kg) in x axis and Daily Pain NRS CFB in y axis.
- Add model parameter values as an inset plot. For e.g., Sigmoid  $E_{max}$ ;  $E_0 = xxx$ ,  $E_{max} = xxx$ , ED50 = xxx,  $\lambda = xxx$ .
- The MCP-MOD approach will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

Draft 1.1 | 31-Aug-2023 | 





Figure 14.2.1.2
Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Missing Data Handling mITT Population

# Weekly Average CFB to Week 12 Daily Pain NRS 0 Daily Pain NRS CFB Data OBS LOCF BOCF -6 5 150 450 Dose (µg/kg)

BOCF = Baseline Observation Carried Forward; CFB = Change from Baseline; DPS = Daily Pain Score; LOCF = Last Observation Carried Forward; NRS = Numeric Rating Scale; OBS = Observed Cases.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1





## **Programming Notes:**

- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS".
- Dose (μg/kg) and Observed/LOCF/BOCF in x axis and Daily Pain NRS CFB in y axis.
- A level for column dosing (column dosing (column) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





# Figure 14.2.1.3 Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup mITT Population

CFB = Change from Baseline; DPS = Daily Pain Score; NRS = Numeric Rating Scale. Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

### **Programming Notes:**

- Same shell as Figure 14.2.1.2
- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS".
- Dose (μg/kg) in x axis, Anticonvulsant/ Antidepressant/ Both/ None in right side Co-medication labels, and Daily Pain NRS CFB in y axis.
- A level for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Figure 14.2.1.4

Daily Pain NRS: MMRM LS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases) mITT Population

#### Weekly Average CFB to Week 12 Daily Pain NRS ± 95% CI



CFB = Change from Baseline; CI = Confidence Interval; DPS = Daily Pain Score; LS = Least Square; MMRM = Mixed Model for Repeated Measures; NRS = Numeric Rating Scale.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

Draft 1.1 | 31-Aug-2023 | 





### **Programming Notes:**

- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS  $\pm$  95% CI".
- Week in x axis and Daily Pain NRS CFB in y axis.
- Include a profile for each dose treatment group.
- Include the following timepoints: Week 2, 4, 6, 8, 10, and 12.
- Extract data for this figure from the MMRM of CFB Daily Pain NRS with Observed Cases.
- A profile for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





#### Figure 14.3.6.1.1 Vital Sign Profiles: Mean (±SD) Systolic Blood Pressure over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes a fter Infusion Completion; BASE = Baseline; D1 = Day 1; SBP = Systolic Blood Pressure; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average SBP  $\pm$  Standard Deviation".
- Study Visit in x axis and Systolic Blood Pressure (mmHg) in y axis.
- Include a profile for Resting SBP and another for Standing SBP.
- Include the following timepoints: Baseline, Day 1:15 Minutes Post-Dose, Day 1:30 Minutes Post-Dose, Day 1:45 Minutes Post-Dose, Day 1:1 hour Post-Dose, Day 1:2 hours Post-Dose, Day 1:4 hours Post-Dose, Week 2: Pre-Dose, Week 2:5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4:5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6:5 minutes a fter Infusion Completion, Week 8: Pre-Dose, Week 8:5 minutes a fter Infusion Completion, Week 10: Pre-Dose, Week 10:5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





#### Figure 14.3.6.1.2 Vital Sign Profiles: Mean (±SD) Diastolic Blood Pressure over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes a fter Infusion Completion; BASE = Baseline; D1 = Day 1; DBP = Diastolic Blood Pressure; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11: W12 = Week 12: W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average DBP ± Standard Deviation".
- Study Visit in x axis and Diastolic Blood Pressure (mmHg) in y axis.
- Include a profile for Resting DBP and another for Standing DBP.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1:30 Minutes Post-Dose, Day 1:45 Minutes Post-Dose, Day 1:1 hour Post-Dose, Day 1:2 hours Post-Dose, Day 1:4 hours Post-Dose, Week 2: Pre-Dose, Week 2:5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4:5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6:5 minutes a fter Infusion Completion, Week 8: Pre-Dose, Week 8:5 minutes a fter Infusion Completion, Week 10: Pre-Dose, Week 10:5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing (column)) will only be added if Stage 4 is initiated)

Draft 1.1 | 31-Aug-2023 | 





# Figure 14.3.6.1.3 Vital Sign Profiles: Mean (±SD) Heart Rate over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes a fter Infusion Completion; BASE = Baseline; D1 = Day 1; HR = Heart Rate; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average HR  $\pm$  Standard Deviation".
- Study Visit in x axis and Heart Rate (Beats/min) in y axis.
- Include a profile for Resting HR and another for Standing HR.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1:30 Minutes Post-Dose, Day 1:45 Minutes Post-Dose, Day 1:1 hour Post-Dose, Day 1:2 hours Post-Dose, Day 1:4 hours Post-Dose, Week 2: Pre-Dose, Week 2:5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4:5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6:5 minutes a fter Infusion Completion, Week 8: Pre-Dose, Week 8:5 minutes a fter Infusion Completion, Week 10: Pre-Dose, Week 10:5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





#### Figure 14.3.6.1.4 Vital Sign Profiles: Mean (±SD) Respiratory Rate over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 4H PD = 4 hours Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average Respiratory Rate ± Standard Deviation".
- Study Visit in x axis and Respiratory Rate (Breaths/min) in y axis.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 5 minutes after Infusion Completion, Week 10 + 24 hours, Week 11, Week 12, Week 18. (Do not include Screening records).
- Make one plot with 4 profiles (one for each treatment group).
- A profile for column dosing (CC) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





Figure 14.3.6.1.5
Vital Sign Profiles: Mean (±SD) Temperature over time
Safety Population

1H PD = 1 Hour Post-Dose; 2H PD = 2 Hours Post-Dose; 4H PD = 4 hours Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; T° = Temperature; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average Body To ± Standard Deviation".
- Study Visit in x axis and Body Temperature (°C) in y axis.
- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 5 minutes after Infusion Completion, Week 10: 4 hours, Week 11, Week 12, Week 18. (Do not include Screening records).
- Make one plot with 4 profiles (one for each treatment group).
- A plot for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 



Figure 14.4.1.1
Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 Concentrations over Time PK Population



ADA = Antidrug Antibodies; gSD = Geometric Standard Deviation; LLOQ = Lower Limit of Quantification.

Draft 1.1 | 31-Aug-2023 | 





PK Population = includes all subjects for who a pharmacokinetic sample was obtained and analyzed. ADA positive represents participants with at least one positive ADA result. ADA negative represents participants with only negative ADA results (no positive). Reference Listing: 16.2.10.1

## **Programming Notes:**

- Insert the following text as upper legend: "Geometric Mean serum MEDI7352± Geometric Standard Deviation (Linear Scale)" followed by "Geometric Mean serum MEDI7352" for the linear plot, and "Geometric Mean serum MEDI7352 ± Geometric Standard Deviation (Semi-Logarithmic Scale)" followed by "Geometric Mean serum MEDI7352" for the semi-log plot. Below legend, add legend for ADA status: "Overall", "ADA Positive", "ADA Negative".
- Insert legend with different point symbols and colors for each treatment group (CC) for the Overall plot, and a legend with different point symbols and colors for each ADA status (ADA+, ADA-) for each treatment group plot by ADA status.
- Time (Days) in x axis and Serum MEDI7352 concentration (ng/mL) in y axis (in linear and log<sub>10</sub> scale, for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10: Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 10 + 14 days, Week 18.
- Make one overall plot by treatment group, and a plot for each treatment group by ADA status for a total of 4 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (1.00 ng/mL)".
- A line for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 




Figure 14.4.1.2
Pharmacokinetics: Individual Plot of Serum MEDI7352 Concentrations over time PK Population



ADA = Antidrug Antibodies; LLOQ = Lower Limit of Quantification.

PK Population = includes all subjects for who a pharmacokinetic sample was obtained and analyzed.

ADA positive represents number of participants with at least one positive ADA result.

ADA negative represents number of participants with only negative ADA results (no positive).

Reference Listing: 16.2.10.1

Draft 1.1 | 31-Aug-2023 | 





#### **Programming Notes:**

- Insert the following text as upper legend: "MEDI7352 Concentration by Subject, Treatment group, and ADA status" followed by "(Linear Scale)" or "(Semi-Logarithmic Scale)" depending on the plot (linear or semi-log). Below legend, add legend for Treatment Group: CCI
- Insert legend with different colors for each ADA status (Positive/ Negative).
- Time (days) in x axis and Serum MEDI7352 concentration (ng/mL) in y axis (in linear and log<sub>10</sub> scale, for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 10 + 14 days, Week 18.
- Make one plot for each Treatment group (CC), for a total of 3 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (1.00 ng/mL)".
- Plots for column dosing (column dosing will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





# Figure 14.4.2.1 Pharmacodynamics Line Plot of Geometric Mean (with and without gSD) Serum total NGF over time Safety Population

ADA = Antidrug Antibodies; gSD = Geometric Standard Deviation; LLOQ = Lower Limit of Quantification, NGF = Nerve-Growth Factor.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

ADA positive represents participants with at least one positive ADA result.

ADA negative represents participants with only negative ADA results (no positive).

Reference Listing: 16.2.10.3

#### **Programming Notes:**

- Same shell as Figure 14.4.1.1
- Insert the following text as upper legend: "Geometric Mean Serum Concentration of tNGF ± Geometric Standard Deviation (Linear Scale)" followed by "Geometric Mean Serum Concentration of tNGF" for the linear plot, and "Geometric Mean Serum Concentration of tNGF (Semi-Logarithmic Scale)" followed by "Geometric Mean Serum Concentration of tNGF" for the semi-log plot. Below legend, add legend for ADA status: "Overall", "ADA Positive", "ADA Negative".
- Insert legend with different point symbols and colors for each treatment group (Placebo, CC) for the Overall plot, and a legend with different point symbols and colors for each ADA status (ADA+, ADA-) for each treatment group plot by ADA status.
- Time (Days) in x axis and Serum tNGF Concentration (pg/mL) in y axis (in linear and log<sub>10</sub> scale for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10: Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12, Week 18.
- Make one overall plot by treatment group, and a plot for each treatment group by ADA status for a total of 5 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (10.00 pg/mL)".
- A plot for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.





Figure 14.4.2.2
Pharmacodynamics: Individual Plot of Serum total NGF over time
Safety Population

ADA = Antidrug Antibodies; LLOQ = Lower Limit of Quantification; NGF = Nerve-Growth Factor. Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication. ADA positive represents number of participants with at least one positive ADA result. ADA negative represents number of participants with only negative ADA results (no positive). Reference Listing: 16.2.10.3

#### **Programming Notes:**

- Same shell as Figure 14.4.1.2
- Insert the following text as legend: "Total NGF by Subject, Treatment group, and ADA status" followed by "(Linear Scale)" or "(Semi-Logarithmic Scale)" depending on the plot (linear or semi-log). Below legend, add legend for Treatment Group: GCI.
- Insert legend with different colors for each ADA status (Positive/ Negative).
- Time (days) in x axis and Serum tNGF concentration (pg/mL) in y axis (in linear and log<sub>10</sub> scale for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.
- Make one plot for each Treatment group (CC) Placebo), for a total of 4 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (10.00 pg/mL)".
- Plots for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Draft 1.1 | 31-Aug-2023 | 





| Sponsor: | AstraZeneca |
|---|---|
| Protocol Title | A Randomised, Double-Blind, Placebo-Controlled, Dose-<br>Response Study of the Efficacy and Safety of MEDI7352 in<br>Subjects with Painful Diabetic Neuropathy |
| Development Phase | 2 |
| Protocol Numbers: | D5680C00002 |
| Premier Research PCNs: | MEDU177093 |
| Document Version: | Final Version 1.2 |
| Document Date: | 04-Oct-2023 |

# **Document History**

| Version | Date | Author | Description |
|---------|-------------|--------|---------------|
| 0.1 | 24-Mar-2023 | PPD | Draft Version |
| 0.2 | 21-Apr-2023 | PPD | Draft Version |
| 0.3 | 24-May-2023 | PPD | Draft Version |
| 1 | 12-Jul-2023 | PPD | Final Version |
| 1.1 | 31-Aug_2023 | PPD | Final Version |

Final 1 2 | 04-Oct-2023 | 





#### Tables, Listings, and Figures Conventions

All listings, tables, and graphs will have a header showing the sponsor company name, protocol and version of delivery and a footer showing the version of SAS, the file name and path, and the source of the data (listing number).

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

#### **General Reporting Conventions**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text will not be used in tables, figures, and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing.
- Adverse events with missing MedDRA coding will have their system organ class preferred term presented as "Not Coded" and the Preferred Term presented as verbatim in the tables. The "Not Coded" frequencies will be sorted to the end of the tables. This will only be applicable for any deliveries sent before database lock (e.g., for dry runs).
- Programming notes may be inserted into the shells, these notes will not appear in the final output.

#### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xx), where appropriate.
- All population summaries for categorical variables will include all categories that were planned and for which the participants may have had a response.
- All population summaries for continuous variables will include: n, mean, SD, median, quartiles, minimum, and maximum. Other summaries (e.g., number missing, geometric mean, 95% CIs, and coefficient of variation [CV] or % CV) may be used as appropriate. The precision of the maximum and minimum will match the maximum precision in the observed data and 2 decimals for derived data unless specifically mentioned in the corresponding shell. The mean and median will have 1 additional decimal place. The SD will have 2 additional decimal places. For derived data, minimum and maximum will be reported to 2 degrees of precision. Measures of location (mean and median) will be reported to 3 degree of precision, and measures of spread will be reported to 4 degrees of precision.
- All percentages are rounded and reported to a single decimal point (xx.x%). Exceptions are 0 and 100 that will be displayed as 0 and 100% respectively.

Final 1.2 | 04-Oct-2023 | 





### Planned Tables, Figures and Listings

- The table and listing numbers are place holders only and will be determined when the outputs are produced.
- In all listings a blank line will be placed between each participant. Within a data listing, if an item appears line after line (e.g., repetition of participant number), then only the first occurrence will be displayed.
- In data listings, the information for 1 participant will be kept on 1 page, if possible, rather than splitting a Subjects's information across pages.

Final 1 2 | 04-Oct-2023 | 





# **Planned Table Descriptions and Shells**

| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.1.2 Screening Population | U |
| Table 14.1.3 - Summary of Reasons for Screening Failure - Screen Failure Population | U |
| Table 14.1.4.1 - Demographics and Baseline Characteristics - Screening Population | U |
| Table 14.1.4.2 - Demographics and Baseline Characteristics - Safety Population | R |
| Table 14.1.4.3 - Demographics and Baseline Characteristics - mITT Population | R |
| Table 14.1.4.4 - Demographics and Baseline Characteristics - PK Population | R |
| Table 14.1.5.1 - Osteoarthritis Characteristics - Screening Population | U |
| Table 14.1.5.2 - Osteoarthritis Characteristics - Safety Population | R |
| Table 14.1.5.3 - Osteoarthritis Characteristics - mITT Population | R |
| Table 14.1.5.4 - Osteoarthritis Characteristics - PK Population | R |
| Table 14.1.6 - Medical History by System Organ Class and Preferred Term - Safety Population | U |
| Table 14.1.7 - Prior Medications by ATC Level 2 and Preferred Name - Safety Population | U |
| Table 14.1.8 - Protocol Deviations - Safety Population | U |
| Table 14.1.9 - Overall Study Drug Exposure - Safety Population | U |
| Table 14.2.1.1.1 - Daily Pain NRS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.1.1.2 - Daily Pain NRS: Summary Statistics (LOCF) <b></b> - mITT Population | R |
| Table 14.2.1.1.3 - Daily Pain NRS: Summary Statistics (BOCF) - mITT Population | R |
| Table 14.2.1.2.1 - Daily Pain NRS: Primary MCP-Mod Analysis (LOCF) - mITT Population | U |
| Table 14.2.1.2.2 - Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) - mITT Population | U |
| Table 14.2.1.3.1 - Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) - mITT Population | U |
| Table 14.2.1.3.2 - Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) - mITT Population | R |
| Table 14.2.2.1 - Galer NPS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.2.2 - Galer NPS: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.3.1 - DSIS: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.3.2 - DSIS: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.4.1 - SF-36: Summary Statistics (Observed Cases) - mITT Population | U |
| Table 14.2.4.2 - SF-36: MMRM Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.5.1 - Rescue Medication Use: Summary Statistics - mITT Population | U |

Final 1.2 | 04-Oct-2023 |





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.2.6.1.1 - Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel Haenszel (Observed Cases) - mITT Population | U |
| Table 14.2.6.1.2 - Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel Haenszel (Observed Cases): All Visits - mITT Population | CCI |
| Table 14.2.6.2 - Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) - mITT Population | U |
| Table 14.2.7.1.1 - Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases) - mITT Population | R |
| Table 14.2.7.1.2 - Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases): All Visits - mITT Population | CCI |
| Table 14.2.7.2 - Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) - mITT Population | R |
| Table 14.2.8.1 - Patient Global Impression of Change: Summary Statistics - mITT Population | U |
| Table 14.2.8.2 - Patient Global Impression of Change: Cochran-Mantel Haenszel - mITT Population | U |
| CCI | U |
| Table 14.3.1.1 - Summary of Overall Adverse Events - Safety Population | U |
| Table 14.3.1.2 - Treatment Emergent of Adverse Events by System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.3 - Treatment Emergent of Adverse Events by Severity, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.4-Treatment Emergent Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.5 - Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term - Safety Population | U |
| Table 14.3.1.6 - Treatment Emergent Adverse Events Leading to Discontinuation of Study drug by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.1.7 - Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.1.8 - Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term - Safety Population | R |
| Table 14.3.1.9 - Treatment Emergent Adverse Events by Preferred Term - Safety Population | R |
| Table 14.3.2.1.1 - Serious Adverse Events by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.2 - Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.1.3 - Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term - Safety Population | R |





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.3.2.1.4 - Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.3.1 - Listing of Serious Adverse Events - Safety Population | U |
| Table 14.3.3.2 - Listing of Deaths - Safety Population | U |
| Table 14.3.2.2.1 - Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.2 - Potential Joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.3 - Serious and/or severe Infections by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.2.2.4 - Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP by System Organ Class and Preferred Term - Safety Population | R |
| Table 14.3.4.1 - Descriptive Summary of Clinical Chemistry - Safety Population | U |
| Table 14.3.4.2 - Shift Table of Clinical Chemistry Results - Safety Population | U |
| Table 14.3.4.3 - Descriptive Summary of Hematology - Safety Population | R |
| Table 14.3.4.4 - Shift Table of Hematology Results - Safety Population | R |
| Table 14.3.4.5 - Descriptive Summary of Coagulation - Safety Population | R |
| Table 14.3.4.6 - Shift Table of Coagulation Results - Safety Population | R |
| Table 14.3.4.7 - Descriptive Summary of Urinalysis - Safety Population | U |
| Table 14.3.4.8 - Shift Table of Urinalysis Results - Safety Population | R |
| Table 14.3.4.9 - Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin - Safety Population | U |
| Table 14.3.5.1 - Descriptive Summary of Vital Signs - Safety Population | U |
| Table 14.3.5.2 - Descriptive Summary of Digital ECG Data - Safety Population | U |
| Table 14.3.5.3 - Summary of Overall Evaluation of safety ECG Data - Safety Population | U |
| Table 14.3.5.4 - Covid-19 Screening - Safety Population | U |
| Table 14.3.5.5 - Summary of Sub-Scores for Total Neuropathy Score-Nurse - Sa fety Population | U |
| Table 14.3.5.6 - Descriptive Summary of Total Neuropathy Score - Nurse - Safety Population | U |
| Table 14.3.5.7.1 - Summary of Motor and Sensory Nerve Conduction Studies - Safety Population | U |
| Table 14.3.5.7.2 - Shift Table of Motor and Sensory Nerve Conduction Results - Safety Population | CCI |
| Table 14.3.5.8 - Summary of Strength and Deep Tendon Reflexes - Safety Population | U |
| Table 14.3.5.9 - Summary of Local Injection Site Reactions - Safety Population | U |





| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Table 14.3.5.10 - Summary of Hypersensitivity/Anaphylactic Reactions - Safety Population | U |
| Table 14.3.5.11 - Summary of Liver Diagnostic Investigations - Safety Population | U |
| Table 14.3.5.12 - Summary of Liver Risk Factors and Lifestyle Events - Safety Population | U |
| Table 14.3.5.13 - Summary of Liver Signs and Symptoms - Safety Population | U |
| Table 14.3.5.14 - Summary of Infection Diagnostic Investigations - Safety Population | U |
| Table 14.3.5.15 - Summary of Infection Risk Factors and Lifestyle Events - Safety Population | U |
| Table 14.3.5.16 - Summary of Infection Signs and Symptoms - Safety Population | U |
| Table 14.3.5.17 - Summary of Concomitant Medications by ATC Level 2 and Preferred Name - Safety Population | R |
| Table 14.3.5.18 - Summary of Concomitant Procedures - Safety Population | R |
| Table 14.3.5.19 - Anti-Drug Antibody Results and Titre Summary by Timepoint - Safety Population | U |
| Table 14.3.5.20 - Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories - Safety Population | U |
| Table 14.4.1 - Summary of Serum MEDI7352 Concentrations - PK Population | U |
| Table 14.4.2 - Summary of Serum total NGF Concentrations - PD Population | U |

Final 1 2 | 04-Oct-2023 | 





# **Table Change Log**

| Output | Date of | Change Made | Description/Rationale |
|--------|---------|---------------|-----------------------|
| Number | Change | By (initials) | |

Final 1 2 | 04-Oct-2023 | 





# 1. Demographic Data

Table 14.1.2 Subject Disposition Screening Population

| | | Screening Population | | | |
|---|---|---|---|---|---|
| | Placebo MEDI7352 | | | | Total |
| Status | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Screening Population [1] | | | | | xx (100%) |
| Screen Failures | | | | | xx (xx.x %) |
| Enrolled Subjects | | | | | xx (xx.x %) |
| Re-screened Subjects | | | | | xx (xx.x %) |
| Randomized Subjects | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Randomized and Not Treated Subjects Reason for Discontinuation | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Adverse Event | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Safety Population [2] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| mITT Population [3] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Evaluable Week 12 Efficacy | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Evaluable LOCF Efficacy [4] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Not Efficacy Evaluable | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| PK Population [5] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Completed Study Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Study Treatment Reason for Discontinuation: | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Death | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lack of Efficacy | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lost to Follow-up | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Non-compliance with Study Drug | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Physician Decision | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pregnancy | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Progressive Disease | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Violation | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |

Final 1.2 | 04-Oct-2023 





| Study Terminated by Sponsor | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|
| Technical Problems | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal by Subject | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| COVID-19 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Sponsor Decision | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Completed Study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawn from the Study | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reason for Discontinuation: | | | | | |
| Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Death | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lack of Efficacy | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lost to Follow-up | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

COVID-19 = Coronavirus disease 2019; LOCF = Last Observation Carried Forward; mITT = modified intent-to-treat; N = number of subjects per treatment group; PK = pharmacokinetic.

Note: Percentages are n/Number of subjects randomized\*100 as displayed in column header N, except for the screened, enrolled and re-screened where n/Number of Screening subjects\*100, and for the randomized, where n/Number of Enrolled subjects\*100.

Re-screened subjects are a subset of the Screening population.

- [1] The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments.
- [2] The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication.
- [3] The mITT Population includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.
- [4] Subjects in the mITT Population with LOCF applied for missing efficacy data at week 12,
- [5] The PK Population includes all subjects for who a pharmacokinetic sample was obtained and analyzed.

Reference Listings: 16.2.1.1, 16.2.1.2, 16.2.1.3,

#### **Programming Notes:**

- Display only reasons for early discontinuation with non-missing value.
- A column for column for dosing (column for dosing





#### Table 14.1.3 Summary of Reasons for Screening Failure Screen Failure Population

| | Total<br>(N=xx) |
|---|---|
| Number of Subjects Who Don't Meet Inclusion/Exclusion Criteria | xx (xx.x%) |
| IC 01: Xxxxxxxxxxx | xx (xx.x%) |
| IC 02: Xxxxxxxxxxx | xx (xx.x%) |
| EC 01: Xxxxxxxxxxx | xx (xx.x%) |
| EC 02: Xxxxxxxxxxx | xx (xx.x%) |
| ••• | |
| Number of Subjects Who are Screen Failure for other Reason than Eligibility Criteria | xx (xx.x%) |

EC = exclusion criteria; IC = inclusion criteria; N = number of subjects.

Note: subject can be counted in more than one criterion.

Reference Listing 16.2.1.4

Final 1 2 | 04-Oct-2023 | 





Table 14.1.4.1 Demographics and Baseline Characteristics Screening Population

| Variable | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Age (years) [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Age Category | | | | | |
| ≥18 - <65 years | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| ≥65 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Gender | | | | | |
| Male | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ethnicity | | | | | |
| Hispanic or Latino | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Race | | | | | |
| American Indian or Alaska Native | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Asian | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Black or African American | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| White | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Not Specified | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Screening Height (cm) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |

Final 1 2 | 04-Oct-2023 | 





| Screening Weight (kg) | | | | | |
|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx |
| Screening BMI (kg/m²) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Female characteristics [2] | | | | | |
| Surgically sterile | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Postmenopausal | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Fully vaccinated for COVID-19 | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

BMI = Body Mass Index; COVID-19 = Coronavirus disease 2019; n = number of subjects by treatment group with collected parameter; N = number of subjects per treatment group; SD = standard deviation.

Note: The Screening Population includes all subjects who are enrolled and provide informed consent and demographic and/or baseline screening a ssessments.

Reference Listing: 16.2.4.1

#### **Programming Notes:**

- If a variable is between 2 pages, start the variable in the second page.
- Keep all possible values for each category even if no subject.
- A column for column for dosing (column for dosing to the second dosing

<sup>[1]</sup> Age was calculated as age at time of consent.

<sup>[2]</sup> Percentages are n/Number of Female subjects from Analysis Population\*100





# Table 14.1.4.2 Demographics and Baseline Characteristics Safety Population

#### **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.1.4.3
Demographics and Baseline Characteristics
mITT Population

#### **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for CCI dosing (CCI) will only be added if Stage 4 is initiated.

Table 14.1.4.4
Demographics and Baseline Characteristics
PK Population

#### **Programming Notes:**

- Same shell as Table 14.1.4.1.
- Keep all possible values for each category even if no subject.
- A column for column for dosing (column for dosing (column for dosing (column for dosing dosing (column for dosing dosin

Final 1 2 | 04-Oct-2023 | 





Table 14.1.5.1 Osteoarthritis Characteristics Screening Population

| | Placebo | | MEDI7352 | | |
|---|---|---|---|---|---|
| Variable | | CCI | CCI | CCI | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects diagnosed with Osteoarthritis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Joint(s)/Area(s) affected: | | | | | |
| Shoulder | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Elbow | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Hip | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Knee | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Ankle | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Spine | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Hands | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Feet | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Osteoarthritis clinically significant | | | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Radiologic investigations conducted [1] | | | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Plain radiography | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| MRI | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Joint(s)/Area(s) investigated: | | | | | |
| Shoulder | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Elbow | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Hip | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Knee | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Ankle | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Spine | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Final 1 2 | 04-Oct-2023 | 





| Hands<br>Feet | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
|---|---|---|---|---|---|
| Other | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Osteoarthritis radiologically significant | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Kellgren-Lawrence score reported | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 0 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 1 | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 2 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Grade 4 | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No/Not applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Radiologic Scoring System Used? | | | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |

MRI = magnetic resonance imaging; N = number of subjects per treatment group.

### **Programming Notes:**

- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

<sup>[1]</sup> Subjects who reported more than one radiologic investigation within each category were only counted once. Reference Listing: 16.2.4.3





# Table 14.1.5.2 Osteoarthritis Characteristics Safety Population

#### **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column for column dosing (column dosing (column for column for

Table 14.1.5.3 Osteoarthritis Characteristics mITT Population

#### **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.1.5.4 Osteoarthritis Characteristics PK Population

### **Programming Notes:**

- Same shell as Table 14.1.5.1.
- Display only Joint(s)/Areas(s) affected and investigated with non-missing value.
- A column for CC dosing (CC) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.1.6 Medical History by System Organ Class and Preferred Term Safety Population

| System Organ Class | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Preferred Term | (N=xxx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xxx) |
| Any Medical History | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | | | | | ••• |
| System Organ Class n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N = number of subjects per treatment group.

Note: All medical history terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 26.0. At each level of summarization (system organ class or preferred term), subjects having more than one medical history term were counted only once. System organ class and preferred terms are sorted in descending order of frequency of Total column, and alphabetically if same frequency.

Reference Listing: 16.2.4.2

#### **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Sort SOC and PT (within SOC) in descending order of frequency in the Total column. Sort alphabetically in case of ties.
- Uncoded Medical History Events
  - When there are uncoded Medical History Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] will be sorted at the end of the table.
- A column for column for dosing (column for dosing

Final 1 2 | 04-Oct-2023 | 





Table 14.1.7 Prior Medications by ATC Class and Preferred Name Safety Population

| ATC Class [1] | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Preferred Term | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) |
| Subjects with at Least One Prior<br>Medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Level 2 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Preferred Name n | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Level 2 n | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Name 1 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Preferred Name n | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |

ATC = Anatomical Therapeutic Class; N = number of subjects per treatment group.

Note: Prior medications are defined as medications that started before first dose of study, whether they were stopped before first dose of study medication or not. All prior medications are coded using WHO drug dictionary version vMar2023. At each level of summarization (ATC Level 2 or Preferred Name), subjects who reported more than one prior medication were only counted once. ATC Level 2 and Preferred Term are sorted in descending order of frequency of total, and alphabetically if same frequency.

Reference Listing: 16.2.9.16

# **Programming Notes:**

- If uncoded ATC Level or Preferred Name, please put them as [Not Coded]
- ATC and Preferred Name texts should be in proper case in table.
- A column for column for dosing (column for dosing (column for dosing to do

Final 1.2 | 04-Oct-2023 | 

<sup>[1]</sup> ATC Class is defined as ATC Level 2.





Table 14.1.8 Protocol Deviations Safety Population

| | Placebo | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) |
| Subjects With Any Important Protocol<br>Deviation/Violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Deviation Type 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 5 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Protocol Deviation Type 6 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

N = number of subjects per treatment group.

Notes: Percentages are n/Number of subjects by treatment group\*100.

Subjects with one or more deviations within a type of protocol deviation were counted only once.

Reference Listing 16.2.2.1

# **Programming Notes:**

• A column for column for column dosing (column for column for col

Final 1 2 | 04-Oct-2023 | 





### 2. Exposure and Compliance

Table 14.1.9
Overall Study Drug Exposure
Safety Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Category/ Statistic | (N=xx) | $\frac{CCI}{(N=xx)}$ | (N=xx) | CCI<br>(N=xx) | (N=xx) |
| Maximum Number of Doses Administered [1] | | | | | |
| 1 Dose | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| 2 Doses | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| 3 Doses | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| 4 Doses | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 5 Doses | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 6 Doses | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total Duration of Exposure (days) [2] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX |
| Total (cumulative) IP volume infused (mL) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX |

n = number of subjects by treatment group with collected parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Final 1 2 | 04-Oct-2023 | 

<sup>[1]</sup> Subjects are counted once for each level of dose administered.

<sup>[2]</sup> Duration of exposure (days) = min(date of last dose of treatment + 14 days or date of death) – date of first dose of treatment + 1. Reference Listing: 16.2.5.1





# **Programming Notes:**

- Add all categories even if count is 0.
- A column for column for column dosing (column for column for col

Final 1 2 | 04-Oct-2023 | 





## 3. Primary Efficacy Analysis

Table 14.2.1.1.1
Daily Pain NRS: Summary Statistics (Observed Cases)
mITT Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| Week 2 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | xx, xx |
| Week 2 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

CFB = Change from Baseline; DPS = Daily Pain Score; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NRS = Numeric Rating Scale; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are weekly a verages of the average daily pain scores on an 11-point (0-10) NRS and CFB for the same variable. Total N for the mITT population = 106 at Week 2 as Subject CFF has < 4 days of diary pain data on that visit, completing the following visits till Week 12.

[1] Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

Reference Listing: 16.2.6.1

Final 1 2 | 04-Oct-2023 | 





# **Programming Notes:**

• Include all observed data (Not the LOCF) on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, 12 and 18.

• A column for column dosing (cc) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





# Table 14.2.1.1.2 Daily Pain NRS: Summary Statistics (LOCF) mITT Population

#### **Programming Notes:**

- Same shell as Table 14.2.1.1.1.
- Include all observed and LOCF data on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Add abbreviation in footnote: LOCF = Last Observation Carried Forward.
- Add the following note in footnote: "LOCF applied to Week 12 only".
- A column for column for dosing (column dosing (column dosing (column for column for co

Table 14.2.1.1.3
Daily Pain NRS: Summary Statistics (BOCF)
mITT Population

#### **Programming Notes:**

- Same shell as Table 14.2.1.1.1.
- Include all observed and BOCF data on weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Add abbreviation in footnote: BOCF = Baseline Observation Carried Forward.
- Add the following note in footnote: "BOCF applied to Week 12 only".
- A column for column dosing (column

Final 1 2 | 04-Oct-2023 | 





# Table 14.2.1.2.1 Daily Pain NRS: Primary MCP-Mod Analysis (LOCF) mITT Population

Primary 'MCP' step

| Model | | |
|-----------------------------|---------|------------------------------|
| Contrast [1] | t value | 1-sided adjusted P-value [2] |
| Hyperbolic E <sub>max</sub> | | |
| ED50 = 7.5 | XX.XX | 0.xxxx |
| ED50 = 15 | XX.XX | 0.xxxx |
| ED50 = 30 | XX.XX | 0.xxxx |
| ED50 = 60 | XX.XX | 0.xxxx |
| ED50 = 750 | XX.XX | 0.xxxx |

Primary Overall MCP test

CFB = Change from Baseline; LOCF = Last Observation Carried Forward; MCP = Multiple Comparisons; Procedure; NRS = Numeric rating scale.

Reference Listing: 16.2.6.1

<sup>[1]</sup> ED50 = Effective Dose giving half of the asymptotic maximum effect.

<sup>[2]</sup> Multiplicity Adjusted P-value.







Final 1 2 | 04-Oct-2023 | 





#### 'MOD' step [3] Selected Model xxxxxxxxxx

| Parameter | Estimate | 95% CI of Estimate [6] |
|---------------------------------------|----------|------------------------|
| ED50 | XX.X | [x.xx to x.xx] |
| ED90 [4] | XX.X | [x.xx to x.xx] |
| Asymptotic ED90 [5] | XX.X | [x.xx to x.xx] |
| Dose to achieve target (-1.25) effect | XX.X | [x.xx to x.xx] |
| Treatment effect at dose = CC | XX.X | [x.xx to x.xx] |

CI: Confidence Interval; LOCF = Last Observation Carried Forward; MCP = Multiple Comparisons; Procedure; MOD = Modelling; NRS = Numeric rating scale.

#### **Programming Notes:**

• The 'MOD' step will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

<sup>[3]</sup> Results from the 'MOD' step will only be available in case any of the MCP tests is statistically significant.

<sup>[4]</sup> ED90 = Effective Dose giving 90% of the effect of the maximum dose studied.

<sup>[5]</sup> Asymptotic ED90 = Effective Dose giving 90% of the asymptotic maximum effect.

<sup>[6] 2.5%</sup> and 97.5% quantiles taken from 100000 samples from the multivariate normal distribution for model fitted estimates and its covariance matrix. Reference Listing: 16.2.6.1





Table 14.2.1.2.2 Statistical Analysis of CFB to Week 12 Daily Pain NRS: Primary ANCOVA Analysis (LOCF) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjusted Asymmetric CL | | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | [x.xx to x.xx] | | |
| Co-Medication Type | | | 3 | | | | 0.xxxx |
| Baseline pain NRS | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | | |

ANCOVA = analysis of covariance; CFB = Change from Baseline;

CL = Confidence limits; LOCF = Last Observation Carried Forward; NRS = Numeric rating scale.

[1] Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

[2] P-value is derived from the following model: ANCOVA by dose using NRS baseline value and co-medication as covariates, with CFB to Week 12 (LOCF) as dependent variable.

# Least Square Means

| Treatment | Number of Subjects | LS mean [3] | 95% CI of LS mean |
|--------------|--------------------|-------------|-------------------|
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LOCF = Last Observation Carried Forward; LS = least square; NRS = Numeric rating scale.

[3] The LS mean is a model estimate using fitted group parameter and the baseline

weekly average pain NRS parameter evaluated at the grand mean over each group.

Reference Listing: 16.2.6.1





## **Programming Notes:**

• Concomitant co-medication Type indicated for Pa inful Diabetic Neuropathy: either anticonvulsant class (pregabalin or gabapentin) or antidepressant class (duloxetine, venla faxine, or amitriptyline).

• Rows for column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.2.1.3.1 Statistical Analysis of CFB Daily Pain NRS: MMRM Analysis. (Observed Cases) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | | | |
| Co-medication type | | | 3 | | | | 0.xxxx |
| Week | | | 6 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 18 | | | | 0.xxxx |
| Baseline pain NRS | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| MEDI7352 col vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | xx.xx | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM = Mixed Model for Repeated Measures; NRS = Numeric rating scale.

Note: model was fitted using an unstructured covariance structure. Estimates for difference vs Placebo at Week 12.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, NRS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: Week xxxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CC - Placebo | | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LS = least square; NRS = Numeric rating scale.

Reference Listing: 16.2.6.1

## **Programming Notes:**

- Include LSmeans and difference in LSmean with Placebo in repeated tables for the Treatment\*Week interaction.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline weekly average pain NRS parameter evaluated at the grand mean over each group.




# Table 14.2.1.3.2 Daily Pain NRS: Sensitivity of Primary MCP-Mod Analysis (BOCF) mITT Population

# **Programming Notes:**

- Same shell as Table 14.2.1.2.1, substituting "LOCF = Last Observation Carried Forward" by "BOCF = Baseline Observation Carried Forward".
- The MCP-MOD approach will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

Final 1 2 | 04-Oct-2023 | 





# 4. Secondary Efficacy Analysis

Table 14.2.2.1
Galer NPS: Summary Statistics (Observed Cases)
mITT Population

| Parameter: xxxxx | | | | | |
|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | Total |
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Week 4 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Week 4 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

• • •

Final 1 2 | 04-Oct-2023 | 



feel a single type of pain only sometimes



xx(xx.x%)

xx(xx.x%)

#### For Pain Duration Frequency

| Baselme [1] | | | | | |
|---|---|---|---|---|---|
| I feel a background pain all of the time and occasional flare-ups | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| I feel a single type of pain all the time | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

xx (xx.x%)

xx(xx.x%)

xx(xx.x%)

#### Week 4

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NPS = Neuropathic Pain Scale; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are Pain Intensity, Unpleasantness, and Descriptor scores on an 11-point (0-10) NRS, and Pain Duration/Frequency on a 3-point NRS (1-3), plus CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.6.2

#### **Programming Notes:**

- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Repeat for the Parameters: Pain intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, Surface Pain Intensity (All in an 11-point NRS), Galer NPS Total Score (ranging from 0 to 100), and Pain Duration/Frequency (in a 3-point NRS).
- A column for occurrence dosing (occurrence dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





### Table 14.2.2.2 Galer NPS: MMRM Analysis (Observed Cases) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | | XX.XXX | | | |
| Co-Medication type | | | 3 | | | | 0.xxxx |
| Week | | | 3 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 9 | | | | 0.xxxx |
| Baseline NPS | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| MEDI7352 col vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 vs Placebo | xx.xx | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; NPS = Neuropathic Pain Scale.

Note: model was fitted using an unstructured covariance structure.

Final 1 2 | 04-Oct-2023 | 

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, baseline total NPS score value, and Co-medication type as covariates, with total NPS score CFB as dependent variable.





Least Square Means: Week: xxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CC | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CC | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |

CI = Confidence interval; LS = least square; NPS = Neuropathic Pain Scale.

# **Programming Notes:**

- Include LSmeans and difference in LSmean with Placebo in repeated tables for the Treatment\*Week interaction.
- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Analysis is done for Galer NPS Total Score.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline total NPS score evaluated at the grand mean over each group. Reference Listing: 16.2.6.2





Table 14.2.3.1
DSIS: Summary Statistics (Observed Cases)
mITT Population

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | CCI<br>(N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 4 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 4 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

• • •

Reference Listing: 16.2.6.3

CFB = Change from Baseline; DSIS = Daily Sleep Interference; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are weekly averages of the average daily sleep interference scores on an 11-point (0-10) NRS and CFB for the same variable.

<sup>[1]</sup> Baseline is defined as the average of the 'non-missing' DSIS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.





# **Programming Notes:**

- Include all observed data on weekly averages of the average daily Sleep Interference score for Baseline, Week 4, 8, 12, and 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Final 1 2 | 04-Oct-2023 | 





### Table 14.2.3.2 DSIS: MMRM Analysis (Observed Cases) mITT Population

#### Model parameter estimates

| | | | | | 2-sided 95% unadjuste | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom | Standard Error | CL | [1] | P-value [2] |
| Intercept | xx.xx | XX.XX | | XX.XXX | | | |
| Co-medication type | | | 3 | | | | 0.xxxx |
| Week | | | 3 | | | | 0.xxxx |
| Treatment | | | 3 | | | | 0.xxxx |
| Treatment*Week | | | 9 | | | | 0.xxxx |
| Baseline DSIS | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 CCI vs Placebo | xx.xx | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; DSIS = Daily Sleep Interference.

Note: model was fitted using an unstructured covariance structure.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Time, Treatment, Treatment\*Time, DSIS baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: Week xxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CC | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI | XX | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [ x.xx to x.xx ] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LS = least square.

### **Programming Notes:**

- Include LS means and difference in LS mean with Placebo in repeated tables for the Treatment\*Week interaction.
- Include all observed data on weekly average DSIS for Baseline, Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline weekly average DSIS parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.3





Table 14.2.4.1 SF-36: Summary Statistics (Observed Cases) mITT Population

Parameter: xxxxx

| | Placebo | | MEDI7352 | | Total |
|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | • |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Baseline [1] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | xx, xx | xx, xx |
| Week 12 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx |
| Week 12 CFB | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |

• • •

Final 1 2 | 04-Oct-2023 | 





### When parameter is "Change in general Health"

| Baseline [1] | | | | | |
|---|---|---|---|---|---|
| Much better now than one year ago | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Somewhat better now than one year ago | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| About the same as one year ago | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Somewhat worse now than one year ago | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Much worse now than one year ago | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

#### Week 12

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NRS = numeric rating scale; SD = standard deviation; SF-36 = 36-Item Short-Form Health Survey; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are derived SF-36 scores and Change in General Health on a 5-point NRS (1-5), plus CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.6.4

#### **Programming Notes:**

- Include all observed data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Vitality (Energy/fatigue), Emotional well-being, Social functioning, Pain and General Health (from 0 to 100), Physical Health Summary, Mental Health Summary, and Change in general Health (in a 5-point NRS).
- A column for column dosing (cc) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





#### Table 14.2.4.2 SF-36: MMRM Analysis (Observed Cases) mITT Population

Model parameter estimates: xxxxxxxx

| | | | | 2-sided 95% unadjust | ed Asymmetric CL | 2-sided |
|---|---|---|---|---|---|---|
| Parameter | Estimate | t value | Degrees of freedom Standard E | rror CL | [1] | P-value [2] |
| Intercept | XX.XX | XX.XX | xx.xxx | | | |
| Co-medication type | | | 3 | | | 0.xxxx |
| <del>Week</del> | | | 1 | | | 0.xxxx |
| Treatment | | | 3 | | | 0.xxxx |
| <del>Treatment*Week</del> | | | 3 | | | 0.xxxx |
| Baseline SF-36 | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] | | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 CCI vs Placebo | XX.XX | XX.XX | 1 xx.xxx | [x.xx to x.xx] | [x.xx to x.xx] | 0.xxxx |
| Model residual standard deviation | XX.XX | | | | | |

CFB = Change from Baseline; CL = Confidence limits; MMRM: Mixed Model for Repeated Measures; SF-36 = 36-Item Short-Form Health Survey.

Note: model was fitted using an unstructured covariance structure.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: MMRM using Treatment, SF-36 baseline value, and Co-medication type as covariates, with CFB as dependent variable.





Least Square Means: xxxxxxxx

| Treatment | Number of patients | LS mean [3] | 95% CI of LS mean |
|---|---|---|---|
| Placebo | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI | XX | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |
| MEDI7352 - Placebo | | X.XX | [x.xx to x.xx] |
| MEDI7352 CCI - Placebo | | X.XX | [x.xx to x.xx] |

CI = Confidence interval; LS = least square.

#### **Programming Notes:**

- Include LSmeans and difference in LSmean with Placebo..
- Include all observed data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical Health Summary, and Mental Health Summary Add parameter name after 'Model parameter estimates:' and after 'Least Square Means:'
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 

<sup>[3]</sup> The LS mean is a model estimate using fitted group parameter and the baseline SF-36 parameter evaluated at the grand mean over each group. Reference Listing: 16.2.6.4





Table 14.2.5.1 Rescue Medication Use: Summary Statistics mITT Population

| Variable | Placebo MEDI7352 | | | | Total |
|---|---|---|---|---|---|
| | CCI CCI CCI | | | | _ |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Number of subjects taking any rescue medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of subjects taking any permitted rescue medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of days rescue<br>medication was used [1] | | | | | |
| n<br>Maan (SD) | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3<br>Min, Max | XX.X, XX.X<br>XX, XX | XX.X, XX.X<br>XX, XX | XX.X, XX.X<br>XX, XX | XX.X, XX.X<br>XX, XX | XX.X, XX.X<br>XX, XX |
| Cumulative consumption of Paracetamol Rescue Medication (mg) [2] n Mean (SD) Median Q1, Q3 Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| Paracetamol Rescue Medication<br>Average Daily Dose (mg) [3] | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Final 1 2 | 04-Oct-2023 | 





Number of subjects taking any prohibited rescue medication

xx(xx.x%)

xx (xx.x%)

xx (xx.x%)

xx (xx.x%)

xx(xx.x%)

N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

- [1] Each day on which permitted rescue medication was used at least once is counted.
- [2] Calculated as the total dose of paracetamol rescue medication (mg).
- [3] Calculated as: cumulative consumption of paracetamol rescue medication (mg)/total number of days rescue medication was used.

Reference Listing: 16.2.6.5

# **Programming Notes:**

- A column for column dosing (column dosing (column dosing (column dosing (column dosing (column dosing dosing (column dosing dosing dosing dosing dosing (column dosing d
- Refer to

Final 1 2 | 04-Oct-2023 | 





# Table 14.2.6.1.1 Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel Haenszel (Observed Cases) mITT Population

#### Cochran-Mantel-Haenszel Test

| Treatment/ Category | Number of Subjects (%) | Risk Difference [1] | 95% CI of Risk<br>Difference | 2-sided<br>P-value [2] |
|---|---|---|---|---|
| Placebo (n = xx) >=30% decrease from Baseline | xx (xx.x%) | | | |
| MEDI7352 (n = xx)<br>>=30% decrease from Baseline | xx (xx.x%) | x.xx | [ x.xx to x.xx ] | 0.xxxx |
| MEDI7352 (n = xx)<br>>=30% decrease from Baseline | xx (xx.x%) | x.xx | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 (n = xx)<br>>=30% decrease from Baseline | xx (xx.x%) | x.xx | [x.xx to x.xx] | 0.xxxx |

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

#### **Programming notes:**

• Include all observed data for Week 12.

<sup>[1]</sup> Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

<sup>[2]</sup> P-value < 0.05 indicates a significant association between number of subjects with >=30% decrease from Baseline and treatment across strata. Note: a separate CMH test is performed for each dose versus placebo at Week 12. Reference Listing: 16.2.6.1





# Table 14.2.6.1.2 Daily Pain NRS Responder Analysis (≥30%): Cochran-Mantel Haenszel (Observed Cases): All Visits mITT Population

Cochran-Mantel-Haenszel Test: MEDI7352 xxx µg/kg vs Placebo

| Visit/ | Number of | | 95% CI of Risk | 2-sided |
|---|---|---|---|---|
| Category | Patients (%) | Risk Difference [1] | Difference | P-value [2] |
| Placebo, Week 4 $(n = xx)$ | | | | |
| >=30% decrease from Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | | | | |
| >=30% decrease from Baseline | xx(xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 4 $(n = xx)$ | | | | |
| >=30% decrease from Baseline | xx(xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 8 (n = xx) | | | | |
| >=30% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 12 $(n = xx)$ | | | | |
| >=30% decrease from Baseline | xx(xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | , , | | | |
| >=30% decrease from Baseline | xx (xx.x%) | X.XX | [ x.xx to x.xx ] | 0.xxxx |

Final 1 2 | 04-Oct-2023 | 





Placebo, Week 18 (n = xx)

>=30% decrease from Baseline xx (xx.x%)

MEDI7352 xxx  $\mu$ g/kg, Week 4 (n = xx)

>=30% decrease from Baseline xx(xx.x%) x.xx [x.xx to x.xx] 0.xxxx

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

[1] Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

[2] P-value < 0.05 indicates a significant association between number of subjects with >=30% decrease from Baseline and treatment across strata. Note: a separate CMH test is performed for each dose versus placebo.

Reference Listing: 16.2.6.1

#### **Programming Notes:**



• Include all observed data for Week 4, 8, 12, and 18.

Final 1 2 | 04-Oct-2023 | 





#### Table 14.2.6.2 Daily Pain NRS Responder Analysis (≥30%): GEE Analysis (Observed Cases) mITT Population

Model parameter estimates: Week X

| Parameter | Estimate | Z value | Degrees of freedom | Standard Error | 2-sided 95% CL | 2-sided<br>P-value [2] |
|---|---|---|---|---|---|---|
| Intercept | XX.XX | XX.XX | | XX.XXX | | |
| Co-medication type | | | 3 | | | 0.xxxx |
| Week | | | 3 | | | 0.xxxx |
| Treatment | | | 3 | | | 0.xxxx |
| Treatment*Week | | | 9 | | | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | 0.xxxx |
| MEDI7352 ccl vs Placebo | XX.XX | XX.XX | 1 | XX.XXX | [x.xx to x.xx] | 0.xxxx |
| Dispersion | XX.XX | | | | | |

CL = Confidence limits; GEE: Generalized Estimation Equations; NRS = Numeric rating scale.

Note: model was fitted using a first-order autoregressive covariance structure. Estimates for MEDI7352 dose vs placebo and for 2-sided 95% CL displayed in odds ratio scale.

Reference Listing: 16.2.6.1

# **Programming notes:**

- Include all observed data for Week 4, 8, 12, and 18.
- Rows for CCI dosing (CCI) will only be added if Stage 4 is initiated.

<sup>[1]</sup> Lower limit of 1-sided 90% CL and upper limit of 1-sided 80% CL.

<sup>[2]</sup> P-value is derived from the following model: GEE using Time, Treatment, Treatment\*Time and Co-medication type as covariates, with dependent binary variable indicating whether weekly average pain NRS has >=30% decrease from Baseline.





Table 14.2.7.1.1 Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases)

#### mITT Population

#### Cochran-Mantel-Haenszel Test

| 2-sided |
|-------------|
| P-value [2] |
| 0.xxxx |
| 0 |
| 0.xxxx |
| 0.xxxx |

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

### **Programming notes:**

• Include all observed data for Week 12.

<sup>[1]</sup> Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

<sup>[2]</sup> P-value < 0.05 indicates a significant association between number of subjects with >=50% decrease from Baseline and treatment across strata. Note: a separate CMH test is performed for each dose versus placebo at Week 12. Reference Listing: 16.2.6.1





# Table 14.2.7.1.2 Daily Pain NRS Responder Analysis (≥50%): Cochran-Mantel Haenszel (Observed Cases): All Visits mITT Population

Cochran-Mantel-Haenszel Test: MEDI7352 xxx  $\mu$ g/kg vs Placebo

| Visit/ | Number of | | 95% CI of Risk | 2-sided |
|---|---|---|---|---|
| Category | Patients (%) | Risk Difference [1] | Difference | P-value [2] |
| Placebo, Week 4 $(n = xx)$ | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 4 $(n = xx)$ | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 8 (n = xx) | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 12 $(n = xx)$ | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | | | | |
| >=50% decrease from Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |

Final 1 2 | 04-Oct-2023 | 





Placebo, Week 18 (n = xx)

>=50% decrease from Baseline xx (xx.x%)

MEDI7352 xxx  $\mu$ g/kg, Week 4 (n = xx)

>=50% decrease from Baseline xx(xx.x%) x.xx [x.xx to x.xx] 0.xxxx

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

[1] Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

[2] P-value < 0.05 indicates a significant association between number of subjects with >=50% decrease from Baseline and treatment across strata. Note: a separate CMH test is performed for each dose versus placebo.

Reference Listing: 16.2.6.1

#### **Programming Notes:**



• Include all observed data for Week 4, 8, 12, and 18.

Final 1 2 | 04-Oct-2023 | 





#### Table 14.2.7.2 Daily Pain NRS Responder Analysis (≥50%): GEE Analysis (Observed Cases) mITT Population

# **Programming notes:**

- Same shell as Table 14.2.6.2. Change footnote in [2] as: "p-value is derived from the following model: GEE using Time, Treatment, Treatment\*Time and Co-medication type as covariates, with dependent binary variable indicating whether weekly average pain NRS has >=50% decrease from Baseline. Note: model was fitted using an unstructured covariance structure, with 'MEDI7352 [C] and 'MEDI7352 [C] treatment groups, together with co-medication categories (both types at the same time and none) dropped from the analysis to make the generalized Hessian matrix positive definite. Estimates for MEDI7352 dose vs placebo and for 2-sided 95% CL displayed in odds ratio scale."
- Include all observed data for Week 4, 8, 12, and 18.
- Rows for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.2.8.1
Patient Global Impression of Change: Summary Statistics mITT Population

| | Placebo | | MEDI7352 | MEDI7352 | |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | OCI<br>(N=xx) | (N=xx) | | (N=XX) |
| Week 4 | | | | | |
| Number of PGIC Responders | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Very Much Improved | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Much Improved | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Minimally Improved | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No change | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Minimally Worse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Much Worse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Very Much Worse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

Week 8

. . .

N = number of subjects per treatment group; PGIC = Patient Global Impression of Change.

Note: Percentages for Number of subjects in the different improvement categories relative to baseline are n/Number of Subjects by treatment group at each visit \*100.

Reference Listing: 16.2.6.6

# **Programming notes:**

- Include all observed data on PGIC scores for Week 4, 8, 12 and 18.
- A column for column for dosing (column to see a dead if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





# Table 14.2.8.2 Patient Global Impression of Change: Cochran-Mantel Haenszel mITT Population

Cochran-Mantel-Haenszel Test: MEDI7352 xxx µg/kg vs Placebo

| Visit/ | Number of | | 95% CI of Risk | 2-sided |
|---|---|---|---|---|
| Category | Patients (%) | Risk Difference [1] | Difference | P-value [2] |
| Placebo, Week 4 $(n = xx)$ | | | | |
| Improved relative to Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 4 $(n = xx)$ | | | | |
| Improved relative to Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 8 (n = xx) | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [x.xx to x.xx] | 0.xxxx |
| Placebo, Week 12 $(n = xx)$ | | | | |
| Improved relative to Baseline | xx (xx.x%) | | | |
| MEDI7352 xxx $\mu$ g/kg, Week 4 (n = xx) | | | | |
| Improved relative to Baseline | xx (xx.x%) | X.XX | [ x.xx to x.xx ] | 0.xxxx |

Final 1 2 | 04-Oct-2023 | 





Placebo, Week 18 (n = xx)

Improved relative to Baseline xx (xx.x%)

MEDI7352 xxx  $\mu$ g/kg, Week 4 (n = xx)

Improved relative to Baseline xx(xx.x%) x.xx [x.xx to x.xx] 0.xxxx

CI = confidence interval; CMH = Cochran-Mantel-Haenszel; NRS = numeric rating scale.

[1] Common effect for the strata (co-medication type\*median Baseline Pain NRS) specific risk difference, representing common difference in probability a cross strata of MEDI7352 dose - Placebo.

[2] P-value < 0.05 indicates a significant association between improvement relative to Baseline and treatment across strata.

Note: median Baseline Pain NRS was calculated from subjects having valid NRS data on at least one of the above four post-baseline visits. Note: a separate CMH test is performed for each dose versus placebo.

Reference Listing: 16.2.6.6

# **Programming Notes:**

• Include all observed data on PGIC scores for Week 4, 8, 12 and 18.

Final 1 2 | 04-Oct-2023 | 





# 5. Exploratory Efficacy Analyses



Final 1 2 | 04-Oct-2023 | 







Final 1 2 | 04-Oct-2023 | 





# 6. Safety and Tolerability

# 6.1. Displays of Adverse Events

Table 14.3.1.1 Summary of Overall Adverse Events Safety Population

| | Placebo | | MEDI7352 | | | |
|---|---|---|---|---|---|---|
| Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with any AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE TEAE categorized as Mild TEAE categorized as Moderate TEAE categorized as Severe | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Subjects with any SAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any SAE possibly related to IP [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE leading to Discontinuation of IP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with any TEAE related to IP<br>TEAE categorized as Mild related to IP<br>TEAE categorized as Moderate related<br>to IP<br>TEAE categorized as Severe related to<br>IP | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Subjects with any SAE leading to Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1 2 | 04-Oct-2023 | 





AE = adverse event; IP = Investigational product, N = number of subjects per treatment group; SAE = serious adverse event; TEAE = treatment emergent adverse event.

[1] Possibly related is defined as with reasonable possibility that the AE was caused by the IP, as assessed by investigator.

Note: Subjects who reported more than one adverse event within each category were only counted once. A TEAE is defined as an adverse event with an onset at the time of or following the start of treatment with IP. For TEAEs categorized by severity, subjects were counted at the maximum severity. Reference Listing: 16.2.7.1, 16.2.7.2, 16.2.7.3, 16.2.7.4

# **Programming Notes:**

• A column for column for dosing (column for dosing

Final 1 2 | 04-Oct-2023 | 





Table 14.3.1.2
Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| System Organ Class | Placebo | | M | EDI7352 | | Total |
|---|---|---|---|---|---|---|
| Preferred Term | (N=xx)<br>n (n/N * 100) m | CCI<br>(N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | All MEDI7352<br>(N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 3 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT category; N = number of subjects per treatment group; IP = investigational product; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Note: Results are n (n/N \* 100) m is number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing: 16.2.7.1





# **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table.
- A column for column for column dosing (column for column for col

Final 1 2 | 04-Oct-2023 | 





Table 14.3.1.3

Treatment Emergent Adverse Events by Severity, System Organ Class and Preferred Term Safety Population

| System Organ Class Preferred Term | Placebo MEDI7352 | | | | | |
|---|---|---|---|---|---|---|
| Severity | (N=xx) | CCI<br>(N=xx) | CCI CCI All MEDI7352 | | | |
| Subjects with at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT/Severity category; N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Note: Results are n (n/N \* 100).

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT at the maximum severity.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing 16.2.7.1

Final 1 2 | 04-Oct-2023 | 





# **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Present only severity categories with at least one subject.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A column for column for dosing (column for dosing (column for dosing dosing (column for dosing dos

Final 1 2 | 04-Oct-2023 | 





Table 14.3.1.4
Treatment Emergent Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term Safety Population

| | | Б | arety ropulation | | | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Placebo | Total | | | | |
| Relatedness | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Related [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Related [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Related [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

. . .

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT/Relatedness category; N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

[1] Related is defined as reasonable possibility that the AE was caused by investigational product, as a ssessed by the investigator. If investigator's assessment is missing the event is judged as related.

Note: Results are n (n/N \*100).

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT for the most related AE.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing 16.2.7.1





# **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Present only severity categories with at least one subject.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A column for column for dosing (column for dosing

Final 1 2 | 04-Oct-2023 | 




Table 14.3.1.5
Treatment Emergent Adverse Events by ADA Status Category, System Organ Class and Preferred Term Safety Population

Treatment: xxxxxxx

| Treatment: XXXXXXX | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | TE | TE | Post-Baseline | |
| | ADA | | | Non-TE- | Persistently | Transiently | and Baseline | Only Baseline |
| System Organ Class | Negative | ADA Positive | TE-ADA + | ADA + | ADA + | ADA + | Positive | Positive |
| D C 1.T | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term | n (n/N * 100) m | n (n/N * 100) m | n (n/N * 100) m | n (n/N * 100) m | n (n/N * 100) m | n (n/N * 100) m | n (n/N * 100) m | n (n/N * 100) m |
| C 1 | ( 0() | ( 0/) | ( 0/) | ( 0() | ( 0/) | ( 0() | ( 0() | ( 0() |
| Subjects with at Least | XX (XX.X%) XX | XX (XX.X%) XX | XX (XX.X%) XX | XX (XX.X%) XX | XX (XX.X%) XX | XX (XX.X%) XX | xx(xx.x%)xx | XX (XX.X%) XX |
| One TEAE | | | | | | | | |
| System Organ Class 1 | xx(xx.x%)xx | xx(xx.x%)xx | xx (xx.x%)xx | xx(xx.x%)xx | xx(xx.x%)xx | xx(xx.x%)xx | xx (xx.x%) xx | xx(xx.x%)xx |
| Preferred Term 1 | xx (xx.x%) xx | ` ' | | , , | | | xx (xx.x%) xx | , , |
| Preferred Term 2 | , | | | . , | | | xx (xx.x%) xx | |
| Preferred Term 3 | , | , , | , | , | , | ` / | xx (xx.x%) xx | , |
| 110101100 1011110 | ( , 0) | ( | ( | ( | ( | (, 9) | ( | (, 5) |
| System Organ Class 2 | xx (xx x%)xx | xx (xx x%)xx | xx (xx x%)xx | xx (xx x%)xx | xx (xx x%)xx | xx (xx x%)xx | xx (xx.x%) xx | xx (xx x%)xx |
| Preferred Term 1 | xx(xx.x%)xx | | | | xx(xx.x%)xx | | xx(xx.x%)xx | 1 |
| Preferred Term 2 | , | ` ' | | , , | | | xx(xx.x%)xx | ` / |
| Preferred Term 3 | , | , , | , | , | , | ` / | xx(xx.x%)xx | , |
| Tierened Tenn 5 | AA (AA.A /0) AA | AA (AA.A /0) AA | AA (AA.A / 0) AA | AA (AA.A /0) AA | AA (AA.A /0) AA | AA (AA.A /0) AA | AA (AA.A /0) AA | AA (AA.A / 0) AA |
| System Organ Class 3 | vv (vv v%)vv | vv (vv v%)vv | vv (vv v <sup>0</sup> / <sub>0</sub> )vv | vv (vv v%)vv | vv (vv v <sup>0</sup> / <sub>0</sub> )vv | vv (vv v%)vv | xx (xx.x%)xx | vv (vv v%)vv |
| Preferred Term 1 | xx(xx.x%)xx | ` / | ` / | ` / | xx(xx.x%)xx | ` / | xx(xx.x%)xx | , |
| Preferred Term 2 | , | | | . , | | | | |
| Preferred Term 3 | , | , , | , | , | , | ` / | XX (XX.X%) XX | , |
| Fierenea renn 3 | XX (XX.X 70) XX | AA (XX.X70) XX | XX (XX.X70) XX | AA (XX.X 70) XX | XX (XX.X 70) XX | AA (XX.X 70) XX | xx(xx.x%)xx | AA (XX.X 70) XX |

AE = adverse event; ADA = Anti-Drug Antibodies; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT category; N = number of subjects per ADA status category; PT = Preferred Term; SOC = System Organ Class; TE-ADA + = Treatment emergent ADA positive; TEAE = treatment-emergent adverse event.

ADA categories are defined in the Statistical Analysis Plan.

Note: Results are n (n/N \*100) m is number of events.

A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

Table is sorted by international order for SOC, and alphabetically for PT.

Reference Listing: 16.2.7.1





#### **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Repeat for Placebo. CCI and Overall.
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]", and sorted at the end of the table. SOC.
- A table for column dosing (column dosing will only be added if Stage 4 is initiated.

#### Table 14.3.1.6

Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One TEAE leading to IP discontinuation".
- Update Reference Listing to 16.2.7.2.
- A column for column for column dosing (column dosing (column for column for

#### Table 14.3.1.7

Non-Serious Adverse Events Occurring in More than 5% of Subjects by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One Non-Serious TEAEAE".
- Update footnote adding: "The 5% threshold for an AE to be displayed is taken from the Total column."
- Update Reference Listing to 16.2.7.1.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Final 1 2 | 04-Oct-2023 | 





Table 14.3.1.8

Treatment Emergent Adverse Events Occurring in More than 5% of Subjects by Preferred Term Safety Population

| | | | sarety ropulation | 11 | | |
|---|---|---|---|---|---|---|
| | Placebo | | M | EDI7352 | | Total |
| Preferred Term | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | All MEDI7352<br>(N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m |
| Subjects with at Least<br>One TEAE | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 1 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 2 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| Preferred Term 3 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| ••• | | | | | | |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each PT category;

N = number of subjects per treatment group; PT = Preferred Term; TEAE = treatment-emergent adverse event.

Note: Results are n (n/Number of subjects in the Safety population within each PT\*100) m is number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each PT.

AEs are displayed by descending frequency of PT based on 'All MEDI7352' column, and alphabetically for PT of same frequency.

The 5% threshold for a TEAE to be displayed is taken from the Total column.

Reference Listing: 16.2.7.1

#### **Programming Notes:**

- PT texts should be in proper case in table.
- In case a term is not coded (e.g., in a dry run) it will be labelled as "Not Coded [PT]" and sorted at the end of the table.
- A column for column for dosing (column for dosing





# Table 14.3.1.9 Treatment Emergent Adverse Events by Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.8.
- Display all TEAEs, not only the most common.
- PT texts should be in proper case in table.
- In case a term is not coded (e.g., in a dry run) it will be labelled as Not Coded [PT]", and sorted at the end of the table.
- A column for column for dosing (column for dosing to the second dosing

Final 1 2 | 04-Oct-2023 | 





## 6.2. Summary of Deaths and Other Serious Adverse Events

Table 14.3.2.1.1
Serious Adverse Events by System Organ Class and Preferred Term
Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One Treatment Emergent SAE", add "SAE = Serious Adverse Event" to abbreviations.
- Change footnote for "Reference Table 14.3.3.1".
- A column for column for column dosing (column dosing (column for column for

Table 14.3.2.1.2
Life-Threatening Serious Adverse Events by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One Life-Threatening SAE", add "SAE = Serious Adverse Event" to abbreviations.
- Add "Note: Life-threatening SAEs as judged by the investigator".
- Change footnote for "Reference Table 14.3.3.1".
- A column for column for column dosing (column dosing (column for column for

Final 1 2 | 04-Oct-2023 | 





## Table 14.3.2.1.3 Serious Adverse Events with Outcome Death by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Number of Subjects with at Least One SAE with Outcome Death", add "SAE = Serious Adverse Event" to abbreviations.
- Change footnote for "Reference Table 14.3.3.2".
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.3.2.1.4
Serious Adverse Events by Relationship to Study Medication, System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.4. Change first row to be "Number of subjects with at Least One Treatment Emergent SAE", add "SAE = Serious Adverse Event" to abbreviations.
- Change footnote for "Reference Table 14.3.3.1".
- A column for CC dosing (CC) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





#### Table 14.3.3.1 Listing of Serious Adverse Events Safety Population

| Subject ID/<br>Treatment Arm | AE ID<br>Numbe | 110101100 101111 | AE Start Date/Time<br>(Study Day)/<br>End Date/Time(Study Day) | Severity/<br>Relationship [1 | Outcome/<br>Action Taken with IP/<br>] Therapy taken for this AES | SAE<br>Leading<br>to Study<br>DC? | | Serious?/<br>Serious<br>?Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:M:M (X)/<br>DDMMMYYYY/HH:M<br>M (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/<br>Yes | No | No | XX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:M:M (X)/<br>DDMONYYYY/HH:<br>MM (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXXX/<br>No | Yes | XX | XX /<br>XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/HH:M:M<br>M (X)/<br>Ongoing | XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX/No | No | XX | XX /<br>XXX |

 $\overline{DC}$  = discontinuation; ID = identification; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Study Day = date of interest – date of first infusion. A TEAE is defined as an adverse event with an onset at the time of or following the start of treatment with IP.

SAEs were coded using MedDRA version 26.0

<sup>[1]</sup> Reasonable possibility AE caused by IP as assessed by the investigator.





## **Programming Notes:**

- If time missing, display "--:--".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e, no AEs occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment ID/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g.. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Final 1 2 | 04-Oct-2023 | 





Table 14.3.3.2 Listing of Deaths Safety Population

| Subject ID/<br>Treatment<br>Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time<br>(Study Day) | Severity/<br>Relationship | Outcome/<br>Action Taken/<br>Therapy? | AE<br>Leading<br>to IP DC? | TEAE? | Serious? /<br>Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>DDMMMYYYY/H<br>H:MM (X) | XXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX/<br>Yes | No | No | XX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>DDMMMYYYY/H<br>H:MM (X) | XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX/No | Yes | XX | XX / XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/H<br>H:MM (X)/<br>Ongoing | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXX/<br>No | No | XX | XX / XXX |

DC = discontinuation; ID = identification; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Study Day = date of interest – date of first infusion. A TEAE is defined as an adverse event with an onset at the time of or following the start of treat ment with IP.

AEs were coded using MedDRA version 26.0

Final 1 2 | 04-Oct-2023 | 





## **Programming Notes:**

- If time missing, display "--:--".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e, no Aes occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g., in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Final 1 2 | 04-Oct-2023 | 





## 6.3. Displays of Significant Adverse Events and Adverse Events of Special Interest

Table 14.3.2.2.1
Treatment Emergent Adverse Events Associated with Abnormal Liver by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at least One TEAE Associated with Abnormal Liver".
- Update Reference Listing to 16.2.7.3.
- A column for column for column dosing (column dosing (column for column for

Table 14.3.2.2.2
Potential joint Related Adverse Events of Special Interest by System Organ Class and Preferred Term Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at least One Potential Joint Related AESI"
- Add abbreviation for AESI = Adverse Event of Special Interest. Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.4
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





#### Table 14.3.2.2.3 Serious and/or severe Infections by System Organ Class and Preferred Term Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One SAE or Severe AE Related to Infection". Add "SAE = Serious Adverse Event" to abbreviations. Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.5.
- A column for column for dosing (column for dosing

Final 1 2 | 04-Oct-2023 | 





Table 14.3.2.2.4

Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP by System Organ Class and Preferred Term Safety Population

| | | | Safety Fopulation | .1 | | |
|---|---|---|---|---|---|---|
| System Organ Class | Placebo | | M | EDI7352 | | Total |
| Preferred Term | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m | All MEDI7352<br>(N=xx)<br>n (n/N * 100) m | (N=xx)<br>n (n/N * 100) m |
| Subjects with at Least<br>One Anaphylactic<br>Reaction,<br>Hypersensitivity or<br>Infusion-Related<br>Reactions Leading to<br>Discontinuation of IP | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1<br>Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx |
| Subjects with at Least One Anaphylactic Reaction, Hypersensitivity or Infusion-Related Reactions Not Leading to Discontinuation of IP [1] | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 Preferred Term 3 | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx | xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx<br>xx (xx.x%) xx |

AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; n = number of subjects within each SOC/PT category; N = number of subjects per treatment group; IP = investigational product; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment-emergent adverse event.

Final 1 2 | 04-Oct-2023 | 





[1] Anaphylactic reactions, hypersensitivity or infusion-related reactions not leading to discontinuation of IP were included in table as they were categorized as AE of special interest under Protocol Amendment 4 (V5.0). Definition for AE of special interest changed from Amendment 6 (V6.0) onwards, including anaphylactic reactions, hypersensitivity or infusion-related reactions leading to permanent discontinuation of IP..

Note: Results are n (n/N \* 100) m is number of events.

A TEAE is defined as AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0. Subjects are counted once for each SOC and once for each PT.

AEs are displayed by descending frequency of SOC, then descending frequency of PT within SOC, based on 'All MEDI7352' column. Table is sorted by international order for SOC of same frequency, and alphabetically for PT of same frequency.

Reference Listing: 16.2.7.6

#### **Programming Notes:**

- Same shell as Table 14.3.1.2. Change first row to be "Subjects with at Least One Anaphylactic Reaction, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of IP". Remove references to TEAEs in footnote.
- Update Reference Listing to 16.2.7.6.
- A column for column for dosing (column for dosing (column for dosing (column for dosing dosing (column for dosing dosin

Final 1.2 | 04-Oct-2023 | 





## 6.4. Laboratory Data

Table 14.3.4.1
Descriptive Summary of Clinical Chemistry
Safety Population

Parameter: xxxxx (unit)

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Low CS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Low CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Final 1 2 | 04-Oct-2023 | 





Day 1 CFB

| n | XX | XX | XX | XX | XX | XX |
|---|---|---|---|---|---|---|
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |

CFB = change from baseline; CS = clinically Significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = not clinically significant; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Reference Listing: 16.2.8.1

### **Programming Notes:**

- Present only scheduled visits.
- Sort Parameters in the following Order: Albumin, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Bicarbonate, Calcium, Chloride, Creatinine, High-Sensitivity C-Reactive Protein (hs-CRP), Estimated Glomerular Filtration Rate (eGFR by Cockcroft-Gault), Serum Glucose, Lactate Dehydrogenase (LDH), Potassium, Sodium, Total Bilirubin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

Note: Percentages are n/Number of subjects with not missing data by treatment group at each visit\*100.





Table 14.3.4.2 Shift Table of Clinical Chemistry Results Safety Population

| Parameter (Unit)/ | | | | | Baseline | Grade [1] | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | | | Placebo | | | | ME | DI7352, CCI | | |
| Post-Baseline | | | (N=xxx) | | | | | (N=xxx) | | |
| Grade | Low | Normal | High | Missing | Total | Low | Normal | High | Missing | Total |
| XXXXXX (Unit) | | | | | | | | | | |
| Week x | | | | | | | | | | |
| Low | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| High | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| Missing | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| Total | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Week x | | | | | | | | | | |
| Low | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) |
| Missing | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Total | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |

n = number of subjects within each category; N = number of subjects per treatment group.

Percentages are n/Number of subjects by treatment group at each visit for the parameter\*100.

Reference Listing 16.2.8.1

## **Programming Notes:**

- Repeat above in new pages for MEDI7352, CC MEDI7352, CC and All MEDI7352.
- Repeat the above for dosing only if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.1.

Final 1 2 | 04-Oct-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





## Table 14.3.4.3 Descriptive Summary of Hematology Safety Population

#### **Programming Notes:**

- Same shell as Table 14.3.4.1
- Present only scheduled visits.
- Sort Parameters in the following Order: Absolute basophil count, absolute eosinophil count, absolute lymphocytes count, Absolute Monocyte Count, Absolute Neutrophil Count, Basophils %, Eosinophils %, Hematocrit (HCT), Hemoglobin (HGB), hemoglobin A1C (HgbA1C), Lymphocytes %, mean corpuscular hemoglobin (MHC), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), Monocytes %, Neutrophils %, Platelets, Red blood cell count (RBC), Red Cell Distribution Width, white blood cell Count (WBC).
- Update Reference listing to 16.2.8.2.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.3.4.4 Shift Table of Hematology Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.4.2
- Repeat the shell for dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.3.
- Update Reference listing to 16.2.8.2

Final 1 2 | 04-Oct-2023 | 





## Table 14.3.4.5 Descriptive Summary of Coagulation Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.4.1
- Present only scheduled visits.
- Sort Parameters in the following Order: Activated Partial Thromboplastin Clotting Time (APTT), Fibrinogen, International normalized ratio (INR), Prothrombin Time (PT).
- Update Reference listing to 16.2.8.3.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Table 14.3.4.6 Shift Table of Coagulation Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.4.2
- Repeat for column dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.5.
- Update Reference listing to 16.2.8.3.

Final 1 2 | 04-Oct-2023 | 





Table 14.3.4.7 Descriptive Summary of Urinalysis Safety Population

Parameter: xxxxx (unit)

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Low NCS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Low CS | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High NCS | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| Low NCS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Low CS | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High NCS | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |

Final 1 2 | 04-Oct-2023 | 





..

## Repeat for all visits for Parameters: Specific Gravity and pH

| Baseline [1] | | | | | | |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Negative | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Positive | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| High NCS | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| If Positive, Specify [2] | | | | | | |
| 100 mg/dL | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| 250 mg/dL | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| 500 mg/dL | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) |
| >= 1000 mg/dL | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Negative | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Positive | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High NCS | x(xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |
| High CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) |

...

#### Repeat for all visits for Parameters: Blood, Glucose, Ketones and Protein

CFB = change from baseline; CS = clinically significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = not clinically significant; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Percentages are n/Number of subjects with not missing data by treatment group at each visit\*100.

Reference Listing: 16.2.8.4

Final 1 2 | 04-Oct-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

<sup>[2]</sup> Percentages are n/Number of Subjects with a Positive Result\*100.





## **Programming Notes:**

- Present only scheduled visits.
- Sort Parameters in the following Order: Blood Urine, Glucose, Ketones, pH, Protein, Specific Gravity.
- Categories for If Positive, Specify:
  - o Blood, Urine: Trace, Small, Moderate.
  - O Glucose: 100 mg/dL, 250 mg/dL, 500 mg/dL,  $\geq 1000 \text{ mg/dL}$ .
  - o Ketones: Trace, 15 mg/dL, 40 mg/dL.
  - o Protein: Trace, 30 mg/dL, 100 mg/dL, 300 mg/dL.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosing dosing (column dosing dos

Final 1 2 | 04-Oct-2023 | 





#### Table 14.3.4.8 Shift Table of Urinalysis Results Safety Population

## **Programming Notes:**

- Same shell as Table 14.3.4.2
- Repeat for dosing if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.4.7.
- Update Reference listing to 16.2.8.4

Final 1 2 | 04-Oct-2023 | 





Table 14.3.4.9

Maximum On-Treatment ALT and AST versus Maximum On-Treatment Total Bilirubin Safety Population

| | | | Total E | Bilirubin |
|---------|------|-----------------|-----------|-----------|
| | | | <2 x ULN | >=2 x ULN |
| Group | Nobs | | n (%) | n (%) |
| Placebo | | | | |
| N=xxx | XXX | ALT | | |
| | | <3 x ULN | x (xx.x%) | x (xx.x%) |
| | | >=3 - <5 x ULN | x (xx.x%) | x(xx.x%) |
| | | >=5 -<10 x ULN | 0 | 0 |
| | | >=10 x ULN | 0 | 0 |
| | XXX | AST | | |
| | | <3 x ULN | x (xx.x%) | x(xx.x%) |
| | | >=3 - <5 x ULN | x (xx.x%) | x(xx.x%) |
| | | >=5 -<10 x ULN | 0 | 0 |
| | | >=10 x ULN | 0 | 0 |

ALT = a lanine aminotransferase; AST = a spartate a minotransferase; IP = investigational product; n = number of subjects per category; N = number of subjects per treatment group; Nobs = number of subjects per treatment group with at least one post-baseline assessment on treatment; ULN = upper limit of normal.

Note: On-treatment assessments include assessments on or after the date of first dose of IP. Baseline is defined as the last observation recorded prior to the first dose of treatment.

Percentages are based on Nobs.

Reference Listing: 16.2.8.1





## **Programming Notes:**

• Per Protocol, the elevations of ALT or AST and Total Bilirubin do not have to occur at the same time or within a specified time frame. That is the reason why the table is presented by Subject instead of by visit. So, if for example, one subject has ALT >= 3 - <5 x ULN at Day 1, and TBL >= 2 x ULN at Week 18, n in that cell will increase by one.

• A column for dosing (CC) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





## 6.5. Other Safety Data

Final 1 2 | 04-Oct-2023 | 





#### Table 14.3.5.1 Descriptive Summary of Vital Signs Safety Population

Parameter: xxxxx

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx | xx, xx |
| Day 1: 15 Minutes Pos | st- | | | | | |
| Dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 1: 15 Minutes Pos | st- | | | | | |
| Dose CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | xx.x | xx.x | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

<sup>• • •</sup> 

Note: 'Day 1: 5 minutes after Infusion Completion' time point was only applied to subjects enrolled in Stage 1, with data collected under eCRF versions 4.0 (11DEC2018) or older.

Reference Listing: 16.2.9.1

CFB = Change from Baseline; eCRF = Electronic Case Report Form; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





### **Programming Notes:**

- Repeat for Supine Heart Rate, Supine Systolic Blood Pressure, Supine Dia stolic Blood Pressure, Respiratory Rate, Body Temperature, Standing Heart Rate, Standing Systolic Blood Pressure, Standing Dia stolic Blood Pressure.
- After Week 2 (inclusive), Supine measure are taken in sitting position. We will consider them as supine (in resting position) for calculating Change from Baseline (always at supine position).
- Include the following timepoints: Baseline, Day 1: 5 Minutes Post-Dose, Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 7 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that Body To, and standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- A column for column for dosing (column for dosing

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.2 Descriptive Summary of Digital ECG Data Safety Population

Parameter: xxxxx

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Day 1: 1 hour Post-Dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Day 1: 1 hour Post-Dose | | | | | | |
| CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Data shown are averages of the 3 replicates taken for each parameter and timepoint, and CFB for the same variables.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.9.2





## **Programming Notes:**

- Repeat for PR, QRS, QT, RR, HR (Heart Rate) and QTcF taken from external data.
- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.3
Summary of Overall Evaluation of Safety ECG Data
Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| AbnormalCS | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal NCS | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 1: 1 hour Post-Dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| AbnormalCS | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abnormal NCS | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

CS = clinically significant; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NCS = Not clinically significant.

Note: Data are taken as the most conservative from the 3 replicates taken by timepoint.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Reference Listing: 16.2.9.2

#### **Programming Notes:**

- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.4 Covid-19 Screening Safety Population

| Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| | CCI | CCI | CCI | All MEDI7352 | |
| (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| xx (xx.x%) | xx (xx.x%) | | | xx (xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | | | xx(xx.x%) |
| xx(xx.x%) | | xx(xx.x%) | | | xx (xx.x%) |
| xx(xx.x%) | | | | | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX | XX | XX | XX | XX | XX |
| xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| XX, XX | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| ` / | , , | | , , | | xx (xx.x%) |
| | ` / | , | ` / | ` , | xx (xx.x%) |
| | xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.xx) xx.x (xx.xx) xx.x (xx.xx) xx.x xx.x xx.x xx.x (xx.x%) xx (xx.x%) xx (xx.x%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.XX) XX (XX.XX) XX.X (XX.XX) XX (XX.XX) XX.X (XX.XX) XX (XX.XX) XX (XX.XXX) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (N=xx) (N=xx) (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (N=xx) (N=xx) (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.x%) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) xx (xx.xx) </td <td>(N=xx) (N=xx) (N=xx) (N=xx) (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx x xx xx xx xx xx xx xx xx xx xx xx x</td> | (N=xx) (N=xx) (N=xx) (N=xx) (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx x xx x |

Final 1 2 | 04-Oct-2023 | 





| Subjects with COVID-19 Antigen Testing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|---|
| Performed | | | | | | |
| COVID-19 Positive | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| COVID-19 Negative | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

COVID-19 = coronavirus disease 2019; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Note: Percentages for COVID-19 screened subjects are n/Number of subjects by treatment group\*100. Percentages for symptoms/test results are n/Number of subjects by treatment group at each visit without missing result\*100. Reference Listing: 16.2.8.8

### **Programming Notes:**

- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10.
- A column for column dosing (column dosing d

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.5
Summary of Sub-Scores for Total Neuropathy Score-Nurse
Safety Population

| Visit/ | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| Subjects performing TNSn | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Sensory Symptom Score | | | | | | |
| 0 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 1 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 1<br>2<br>3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Motor Symptom Score | | | | | | |
| 0 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 1 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 2 3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Autonomic Symptom Score | | | | | | |
| 0 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 1 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1<br>2<br>3<br>4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pin Sensibility Score | | | | | | |
| 0 | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| 1 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 3 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 3 | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1 2 | 04-Oct-2023 | 





| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|
| Vibration Sensibility Score | | | | | | |
| 0 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| ••• | | | | | | |

N = number of subjects per treatment group; TNSn = Total Neuropathy Score-Nurse.

Note: Percentages for subjects performing TNSn are n/Number of subjects by treatment group\*100. Percentages for each Score are n/Number of subjects by treatment group at each visit without missing score\*100.

Reference Listing: 16.2.9.5

## **Programming Notes:**

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12 and Week 18.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





Table 14.3.5.6
Descriptive Summary of Total Neuropathy Score-Nurse
Safety Population

| Score: xxxxx | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | (N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n<br>Mean (SD)<br>Median<br>Q1, Q3<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| Day 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |
| Day 1 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

TNSn = Total Neuropathy Score-Nurse; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment. Reference Listing: 16.2.9.5

## **Programming Notes:**

- Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12 and Week 18.
- Include the following scores: Sensory Symptom Score, Motor Symptom Score, Autonomic Symptom Score, Pin Sensibility Score, Vibration Sensibility Score,

Final 1 2 | 04-Oct-2023 | 




and TNSn Total.

- A column for column for dosing (column for dosing (column for dosing (column for dosing dosing (column for dosing dosin

Table 14.3.5.7.1 Summary of Motor and Sensory Nerve Conduction Studies Safety Population

Parameter: xxxxx

| Parameter, XXXXX | | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| Visit/ | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 18 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 18 CFB | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

Final 1 2 | 04-Oct-2023 | 





| Ev | aluat | ion Result |
|----|-------|------------|
| - | 4. | F47 |

| Baseline [1] | | | | | | |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Abnormal | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 18 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Abnormal | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

CFB = Change from Baseline; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Note: Percentages are number of subjects by treatment group at each visit for each category/Number of subjects with not missing data by treatment group for each visit\*100.

Reference Listing: 16.2.9.6

#### **Programming Notes:**

#### $\mathsf{CC}$

• Repeat for the following Parameters: Lower Limb - Right Side/Fibular Nerve/Motor Evaluation/Amplitude (mV), Lower Limb - Right Side/Tibial Nerve/Motor Evaluation/Amplitude (mV), Lower Limb - Left Side/Fibular Nerve/Motor Evaluation/Amplitude (mV), Lower Limb - Left Side/Sural Nerve/Motor Evaluation/Amplitude (mV), Lower Limb - Left Side/Sural Nerve/Sensory Evaluation/Amplitude (mV), Upper Limb - Right Side/Medial Nerve/Motor Evaluation/Amplitude (mV), Upper Limb - Right Side/Medial Nerve/Sensory Evaluation/Amplitude (mV), Upper Limb - Right Side/Medial Nerve/Sensory Evaluation/Amplitude (mV), Upper Limb - Right Side/Medial Nerve/Sensory Evaluation/Amplitude (mV), Upper Limb - Left Side/Medial Nerve/Motor Evaluation/Amplitude (mV), Upper Limb - Left Side/Medial Nerve/Motor Evaluation/Amplitude (mV), Upper Limb - Left Side/Medial Nerve/Sensory Evaluation/Amplitude (mV), Upper Limb - Left Side/Medial Nerve/Sensory Evaluation/Amplitude (mV), Upper Limb - Right Side/Fibular Nerve/Motor Evaluation/Conduction Velocity (msec), Lower Limb - Right Side/Tibial Nerve/Motor Evaluation/Conduction Velocity (msec), Lower Limb - Right Side/Sural Nerve/Sensory Evaluation/Conduction Velocity (msec), Lower Limb - Left Side/Fibular Nerve/Motor Evaluation/Conduction Velocity (msec), Lower Limb - Left Side/Fibular Nerve/Motor Evaluation/Conduction Velocity (msec), Upper Limb - Right Side/Medial Nerve/Sensory Evaluation/Conduction Velocity (msec), Upper Limb - Right Side/Ulnar Nerve/Motor Evaluation/Conduction Velocity (msec), Upper Limb - Right Side/Ulnar Nerve/Sensory Evaluation/Conduction Velocity (msec), Upper Limb - Left Side

Final 1.2 | 04-Oct-2023 | 





(msec), Upper Limb - Left Side/Ulnar Nerve/Sensory Evaluation/Conduction Velocity (msec), Lower Limb - Right Side/Fibular Nerve/Motor Evaluation/Duration of Action Potential (msec), Lower Limb - Right Side/Tibial Nerve/Motor Evaluation/Duration of Action Potential (msec), Lower Limb - Right Side/Sural Nerve/Sensory Evaluation/Duration of Action Potential (msec), Lower Limb - Left Side/Fibular Nerve/Motor Evaluation/Duration of Action Potential (msec), Lower Limb - Left Side/Tibial Nerve/Motor Evaluation/Duration of Action Potential (msec), Lower Limb - Left Side/Sural Nerve/Sensory Evaluation/Duration of Action Potential (msec), Upper Limb - Right Side/Medial Nerve/Motor Evaluation/Duration of Action Potential (msec), Upper Limb - Right Side/Ulnar Nerve/Motor Evaluation/Duration of Action Potential (msec), Upper Limb - Right Side/Medial Nerve/Sensory Evaluation/Duration of Action Potential (msec), Upper Limb - Right Side/Ulnar Nerve/Sensory Evaluation/Duration of Action Potential (msec), Upper Limb - Left Side/Medial Nerve/Motor Evaluation/Duration of Action Potential (msec), Upper Limb - Left Side/Ulnar Nerve/Motor Evaluation/Duration of Action Potential (msec), Upper Limb - Left Side/Medial Nerve/Sensory Evaluation/Duration of Action Potential (msec), Upper Limb - Left Side/Ulnar Nerve/Sensory Evaluation/Duration of Action Potential (msec), Lower Limb - Right Side/Fibular Nerve/Motor Evaluation/Peak Latency (msec), Lower Limb - Right Side/Tibial Nerve/Motor Evaluation/Peak Latency (msec), Lower Limb - Right Side/Sural Nerve/Sensory Evaluation/Peak Latency (msec), Lower Limb - Left Side/Fibular Nerve/Motor Evaluation/Peak Latency (msec), Lower Limb - Left Side/Tibial Nerve/Motor Evaluation/Peak Latency (msec), Lower Limb - Left Side/Sural Nerve/Sensory Evaluation/Peak Latency (msec), Upper Limb - Right Side/Medial Nerve/Motor Evaluation/Peak Latency (msec), Upper Limb - Right Side/Ulnar Nerve/Motor Evaluation/Peak Latency (msec), Upper Limb - Right Side/Medial Nerve/Sensory Evaluation/Peak Latency (msec), Upper Limb - Right Side/Ulnar Nerve/Sensory Evaluation/Peak Latency (msec), Upper Limb - Left Side/Medial Nerve/Motor Evaluation/Peak Latency (msec), Upper Limb - Left Side/Ulnar Nerve/Motor Evaluation/Peak Latency (msec), Upper Limb - Left Side/Medial Nerve/Sensory Evaluation/Peak Latency (msec), Upper Limb - Left Side/Ulnar Nerve/Sensory Evaluation/Peak Latency (msec).

• A column for column for dosing (column for dosing (column for dosing to do

Final 1.2 | 04-Oct-2023 | 





Table 14.3.5.7.2
Shift Table of Motor and Sensory Nerve Conduction Results
Safety Population

| Parameter (Unit)/ | | | | Baseline | Grade [1] | | | |
|---|---|---|---|---|---|---|---|---|
| Visit | | Plac | cebo | | | 6) | | |
| Post-Baseline | | (N= | xxx) | | | | | |
| Grade | Normal | Abnormal | Missing | Total | Normal | Abnormal | Missing | Total |
| XXXXXX (Unit) | | | | | | | | |
| Week 18 | | | | | | | | |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Abnormal | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | |
| Missing | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | |
| Total | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| XXXXXX (Unit) | | | | | | | | |
| Week 18 | | | | | | | | |
| Normal | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) |
| Abnormal | x(xx.x%) | x(xx.x%) | x (xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Missing | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Total | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x(xx.x%) | x (xx.x%) |

...

Percentages are n/Number of subjects by treatment group at each visit for the parameter\*100.

Reference Listing 16.2.9.6

## **Programming Notes:**

CCI

- Repeat above in new pages for MEDI7352, CCI MEDI7352, CCI and All MEDI7352.
- Repeat the above for old dosing only if Stage 4 is initiated.
- Repeat for every scheduled visit.
- Present parameters in the same order as in Table 14.3.5.7.1.

Final 1 2 | 04-Oct-2023 | 

n = number of subjects within each category; N = number of subjects per treatment group.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





Table 14.3.5.8 Summary of Strength and Deep Tendon Reflexes Safety Population

| Visit/ | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Variable | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | | | |
| Subjects performing SDTR assessment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ankle Dorsiflexion Strength | | | | | | |
| 0 - Normal Power | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 - Mild Weakness | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 - Moderate Weakness | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 - Severe Weakness | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 4 - Paralysis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Deep Tendon Reflexes | | | | | | |
| 0 - Normal | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 1 - Ankle reflex reduced | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| 2 - Ankle reflex absent | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 - Ankle reflex absent and knee reflex | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| reduced | | | | | | |
| 4 - All reflexes (both ankle and knee) absent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

...

Note: Percentages for subjects performing SDTR assessment are n/Number of subjects by treatment group\*100. Percentages for each Score are n/Number of subjects by treatment group at each visit\*100.

Reference Listing: 16.2.9.7

n = number of subjects by treatment group at each visit for each category; N = number of subjects per treatment group; SDTR = strength and deep tendon reflexes.

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





## **Programming Notes:**

• Include the following timepoints: Baseline, Day 1, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.

• A column for column for dosing (column to see a dead if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.9 Summary of Local Injection Site Reactions Safety Population

| Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| xx(xx.x%) | xx(xx.x%) | | xx (xx.x%) | · | xx(xx.x%) |
| , | ` , | , | ` , | ` / | xx(xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| xx(xx.x%) | | | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| | | | | | xx(xx.x%) |
| | | | | | xx (xx.x%) |
| ` / | , | | , | . , | xx(xx.x%) |
| | (N=xx) xx (xx.x%) | Placebo (N=xx) (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | MEDI7352 COI (N=xx) COI (N=xx) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | Placebo MEDI7352 CGI (N=xx) CGI (N=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | Placebo MEDI7352 Cl |

Final 1 2 | 04-Oct-2023 | 





#### Induration/ Swelling

...

| None | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|---|
| Mild | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Severe | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

n = number of subjects by treatment group at each visit for each category; N = number of subjects per treatment group.

Note: Percentages for subjects performing injection site assessment are n/Number of subjects by treatment group\*100. Percentages for each Score are n/Number of subjects by treatment group at each visit\*100. Subject PPD suffered an injection site reaction starting on 25MAR2019 and ending on 23APR2019, spanning Study visits Week 8, 10 and 12. However, injection site assessment was not performed on this subject till Week 18, existing high possibility for symptoms to have receded by then.

Reference Listing: 16.2.9.8

## **Programming Notes:**

- Include the following timepoints: Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.
- A column for column dosing column dosing column dosing column dosing column for column for column for column dosing column dos

Final 1.2 | 04-Oct-2023 | 





Table 14.3.5.10
Summary of Hypersensitivity/Anaphylactic Reactions
Safety Population

| | | Sa | tety Population | | | |
|---|---|---|---|---|---|---|
| | Placebo | | MEDI7352 | | | Total |
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with any | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Hypersensitivity/ | , | , | , | , | , | |
| Anaphylaxis | | | | | | |
| Highest Severity Grade | | | | | | |
| Mild | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Moderate | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x% |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x% |
| Type of Reaction | | | | | | |
| Urticaria | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Pruritus | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Rash | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Flushing | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Swollen Lips, Tongue, | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Uvula and/or Vulva | | | | | | |
| Dyspnoea | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Wheeze-Bronchospasm | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Stridor | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Hypoxia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Hypotension | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Crampy Abdominal Pain | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Vomiting | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Diarrhoea | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |
| Other | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x% |

• • •

N = number of subjects per treatment group.

Reference Listing: 16.2.9.9





## **Programming Notes:**

- Display only Type of reaction with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.11 Summary of Liver Diagnostic Investigations Safety Population

| | | Safety Pop | oulation | | | |
|---|---|---|---|---|---|---|
| | Placebo | • | MEDI7352 | | | Total |
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | $\overline{(N=xx)}$ | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Liver Diagnostics<br>Performed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Type of Diagnostic Investigation | | | | | | |
| Ültra sound | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| CT | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| MRI/MRCP | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Flushing | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| ERCP | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| X-Ray | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Tox Screening for | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Acetaminophen/Paracetamol | | | | | | |
| Tox Screening for Ethanol | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tox Screening, Other | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Specialist Consulted | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis A | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis B | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis C | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis D | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Hepatitis E | xx xx.x% | xx xx.x%) | xx xx.x%) | xx xx.x% | xx xx.x%) | xx xx.x%) |
| Serology for Cytomegalovirus | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Serology for Epstein Barr Virus | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Autoimmune Serology | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

CT = Computerized tomography; ERCP = Endoscopic retrograde cholangiopancreatography; MRI = Magnetic resonance imaging; MRCP = Magnetic resonance cholangiopancreatography; N = number of subjects per treatment group.

Reference Listing: 16.2.9.10

Final 1 2 | 04-Oct-2023 | 





## **Programming Notes:**

- Display only Diagnostic Investigations with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.12 Summary of Liver Risk Factors and Lifestyle Events Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| | | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category | (N=xx) | $\overline{(N=xx)}$ | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Liver Risk Factors | vv (vv v0/) | vv (vv v0/.) | vv (vv v0/) | vv (vv v0/) | vv (vv v0/) | vv (vv v0/) |
| Assessed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Assessed | | | | | | |
| Liver Risk Factor | | | | | | |
| Alcohol Abuse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Increased Alcohol Consumption | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| within 1 Month of Reported Event | | | | | | |
| IV Drug Abuse | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tattoo | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Acupuncture | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Sexually Transmitted Diseases | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Toxic/Chemical Agent Exposure | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Travel (Areas at Risk in the Last Year) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Pregnancy | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Parenteral Nutrition | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Excessive Physical Exercise | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Changes Diet/Fasting Episodes/Weight | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Loss Diet | | | | | | |
| Previous Drug Reaction | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Blood Transfusion | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Patient Exposed to Anyone with | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) |
| Jaundice in the Last Month | , | , | , | , | , | , |
| History of Hypotension | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Final 1 2 | 04-Oct-2023 | 





| Low Blood Pressure at Time of Event of Liver Injury and/or Abnormal Liver | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|
| Laboratory Value<br>History of Liver Disease<br>Other | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |

IV = intravenous; N = number of subjects per treatment group.

Reference Listing: 16.2.9.10

## **Programming Notes:**

- Display only Liver Risk Factor with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.13 Summary of Liver Signs and Symptoms Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Liver Signs/Symptoms<br>Assessed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Liver Sign/Symptom | | | | | | |
| Anorexia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Asthenia | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Pyrexia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pruritus | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Jaundice | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Arthra lgia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Abdominal Pain | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Abdominal Tenderness | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Nausea | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Vomiting | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Rash | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Mucosal Inflammation | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Purpura | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Hepatomegaly | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Splenomegaly | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) |
| Lymphadenopathy | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Ascites | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Confusional State | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Coma | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Upper Quadrant Tenderness | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x%) | xx xx.x% | xx xx.x% |
| Biliary Obstruction | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Eosinophilia | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Dark Urine | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group.

Reference Listing: 16.2.9.12

Final 1 2 | 04-Oct-2023 | 





## **Programming Notes:**

- Display only Liver Signs/Symptoms with non-missing value.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.14 Summary of Infection Diagnostic Investigations Safety Population

| | Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Infection Diagnostic<br>Investigations | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Method | (0/) | (0/) | (0/) | (0/) | (0/) | (0/) |
| Microscopy, Culture and Sensitivity<br>Serological Tests | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| Nucleic Acid Based Tests | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X-Ray | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group. Reference Listing: 16.2.9.13

## **Programming Notes:**

- Display only Methods with non-missing value.
- A column for dosing local ) will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 





Table 14.3.5.15
Summary of Infection Risk Factors and Lifestyle Events
Safety Population

| | Placebo | Safety Fopulati | MEDI7352 | | | Total |
|---|---|---|---|---|---|---|
| | Placedo | | | | A 11 N (ED) (72 52 | 10111 |
| Statistic or Category | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | (N=xx) | All MEDI7352<br>(N=xx) | (N=xx) |
| Subjects with Infection Risk Factor Occurred | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Infection risk factor | | | | | | |
| Extensive Burns within the Last Year | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Tattoo, Piercing or Acupuncture within the | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| last Year | , | , , | . , | , | , , | , |
| Sexually Transmitted Diseases | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Travel to Areas at Risk of Tuberculosis or | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tropical Diseases | , | , | · · · · · · | | , , | , , , , , |
| Infections Related to Travel | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Blood Transfusion (within the Last Year) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Exposure to Nosocomial Pathogens within the | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Last Year | , | , | , | , | , | , |
| Contact History with Infection Source | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Previous BCG Immunization | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Evidence of BCG Scar | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tuberculin Skin or Quantiferon Test Confirms | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Previous Exposure or Immunity to | , | , , | , | , , | , , | , , |
| Tuberculosis | | | | | | |

BCG = Bacillus Calmette-Guerin; N = number of subjects per treatment group. Reference Listing: 16.2.9.14

## **Programming Notes:**

- Display only infection risk factors with non-missing value.
- A column for column for dosing (column for dosing

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.16 Summary of Infection Signs and Symptoms Safety Population

| Placebo | | MEDI7352 | | | Total |
|---|---|---|---|---|---|
| | CCI | CCI | CCI | All MEDI7352 | |
| Statistic or Category (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects with Infection Sign/Symptom xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Occurred Ax (Ax.X76) | AA (AA.A.70) | AA (AA.A70) | AA (AA.A70) | AA (AA.A70) | AA (AA.A70) |
| Infection Sign/Symptoms | | | | | |
| Pyrexia xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Headache xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Confusional State xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Convulsion $xx (xx.x\%)$ | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Rhinitis $xx (xx.x\%)$ | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Oropharyngeal Pain xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Cough $xx(xx.x\%)$ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Productive Cough $xx (xx.x\%)$ | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Haemoptysis xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Wheezing $xx (xx.x\%)$ | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Dyspnoea xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Pleuritic Pain xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Vomiting $xx (xx.x\%)$ | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Diarrhoea $xx (xx.x\%)$ | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Genital Discharge xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Haematuria xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Dysuria $xx (xx.x\%)$ | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Hepatosplenomegaly $xx (xx.x\%)$ | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Jaundice xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lymphadenopathy xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Final 1 2 | 04-Oct-2023 | 





| Rash | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
|---|---|---|---|---|---|
| Petechial | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Vesicular | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Macular | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Papular | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Urticaria | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Erythema | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Blanching | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Splinter Haemorrhages | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Night sweats | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Chills | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Myalgia | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Weight Decrease | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = number of subjects per treatment group.

Reference Listing: 16.2.9.15

## **Programming Notes:**

- Display only infection Signs/Symptoms with non-missing value.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Final 1 2 | 04-Oct-2023 | 





#### Table 14.3.5.17 Summary of Concomitant Medications by ATC Level 2 and Preferred Name Safety Population

#### **Programming Notes:**

- Same shell as Table 14.1.7.
- Change footnote Note by: "Note: Concomitant medications are defined as medications continuing or starting on or after first dose of study medication. All concomitant medications are coded using WHO drug dictionary version vMar2023. At each level of summarization (ATC Level 2 or Preferred Name), subjects who reported more than one concomitant medication were only counted once. ATC Level 2 and Preferred Name are sorted in in descending order of frequency of total, and alphabetically if same frequency".
- If uncoded ATC Level or Preferred Name, please put them as [Not Coded]
- ATC and Preferred Name texts should be in proper case in table.
- A column for column for dosing (column for dosing (column for dosing (column for dosing to dos

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.18
Summary of Concomitant Procedures
Safety Population

| System Organ Class | Placebo | MEDI7352 | | Total | |
|---|---|---|---|---|---|
| Preferred Term | (N=xxx) | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| Any Concomitant Procedure | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term n | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N = number of subjects per treatment group; PT = Preferred Term; SOC = System Organ Class.

Note: All Procedure terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 26.0. At each level of summarization (system organ class or preferred term), subjects having more than one Procedure term were counted only once. System organ class and preferred terms are sorted in descending order of frequency of Total column, and alphabetically if same frequency.

When there are uncoded Procedure Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] are sorted at the end of the table.

Reference Listing: 16.2.9.18

#### **Programming Notes:**

- SOC and PT texts should be in proper case in table.
- Sort SOC and PT (within SOC) in descending order of frequency in the Total column. Sort alphabetically in case of ties.
- Uncoded Procedure events
  - o When there are uncoded Procedure Events in the database, the events will be summarized with SOC and PT set to [Not Coded]. The [Not Coded] will be sorted at the end of the table.
- A column for column dosing (column dosing (column dosing (column dosing (column dosing dosi

Final 1 2 | 04-Oct-2023 | 





Table 14.3.5.19
Anti-Drug Antibody Results and Titre Summary by Timepoint
Safety Population

| | Placebo | | MED | [7352 | |
|---|---|---|---|---|---|
| Visit/<br>Statistic | (N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | CCI<br>(N=xx) | All MEDI7352<br>(N=xx) |
| Baseline [1] | | | | | |
| n [2] | XX | XX | XX | XX | XX |
| ADA Positive: n (%) [3] | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Week 2 | | | | | |
| n [2] | XX | XX | XX | XX | XX |
| ADA Positive: n (%) [3] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

ADA = Anti-Drug Antibodies; N = number of subjects per treatment group; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

Reference Listing: 16.2.9.19

#### **Programming Notes:**

- Keep in mind that in this table 'Total' column does not include placebo.
- Repeat for all scheduled post-baseline visits.
- A column for column dosing (column dosing) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.

<sup>[2]</sup> Number of subjects with at least one ADA assessment at the specific visit.

<sup>[3]</sup> Number of subjects with a positive result at the specific visit. The denominator for all percentages is the number of subjects with an ADA result for each visit.





Table 14.3.5.20
Descriptive Summary of Anti-Drug Antibody Results and Titre by ADA Categories
Safety Population

| | y Population | | | |
|---|---|---|---|---|
| Placebo | | MED | 17352 | |
| (N=xx) | (N=xx) | (N=xx) | (N=xx) | All MEDI7352<br>(N=xx) |
| xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |
| xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| , | • | , | , , , , | , , |
| XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| | Placebo (N=xx) xx/xxx (xx.x%) xx.x xx.x, xx.x xx, xx xx, xx xx/xxx (xx.x%) xx.x xx.x, xx.x xx.x, xx.x xx.x, xx.x xx.x, xx.x xx.x, xx.x | (N=xx) CCI (N=xx) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx. | Placebo MED (N=xx) (N=xx) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx/xxx xx.x xx/xxx xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx/xxx xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x </td <td>Placebo MEDI7352 (N=xx) CGI (N=xx) xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx.x, xx.x xx.x, xx.x xx.x xx.x, xx.x xx.x, xx.x xx.x, xx.x xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x, xx.x xx.x xx.x xx.x, xx.x xx.x xx.x xx.x, xx.x xx.x xx.x xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%)</td> | Placebo MEDI7352 (N=xx) CGI (N=xx) xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx.x, xx.x xx.x, xx.x xx.x xx.x, xx.x xx.x, xx.x xx.x, xx.x xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x, xx.x xx.x xx.x xx.x, xx.x xx.x xx.x xx.x, xx.x xx.x xx.x xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx.x xx.x xx.x xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) |

Final 1 2 | 04-Oct-2023 | 





| Treatment-Boosted ADA Positive n/Nobs (%) [1] [3] Maximum ADA Titre | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
|---|---|---|---|---|---|
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Non-TE-ADA Positive [6] | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | XX, XX | XX, XX |
| Both baseline and post-baseline positive | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Only baseline positive | | | | | |
| n/Nobs (%) [1] [4] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | , , | , , | , | , , | , , , |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| TE-persistently ADA positive [7] | | | | | |
| n/Nobs (%) [1] [3] | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) | xx/xxx(xx.x%) |
| Maximum ADA Titre | | | | | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |

Final 1 2 | 04-Oct-2023 | 





TE-transiently ADA positive [8]
n/Nobs (%) [1] [3]
Maximum ADA Titre
Median
Q1, Q3
Min, Max

| xx/xxx ( $xx.x%$ ) | xx/xxx ( $xx.x%$ ) | xx/xxx(xx.x%) | xx/xxx ( $xx.x%$ ) | xx/xxx (xx.x%) |
|---|---|---|---|---|
| XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |

ADA = Anti-Drug Antibodies; N=number of subjects per treatment group; TE-ADA = Treatment Emergent ADA; SD = standard deviation; Q1 = first quartile; Q3 = third quartile.

- [1] n represents the number of subjects satisfying the conditions of the specified ADA category
- [2] Nobs represents the number of subjects with any ADA result at baseline and/or post-baseline.
- [3] Nobs represents the number of subjects with an ADA result at baseline and at least one post-baseline ADA assessment.
- [4] Nobs represents the number of subjects with an ADA result at baseline.
- [5] TE-ADA positive is defined as either ADA negative at baseline and post-baseline ADA positive (Treatment Induced ADA Positive), or as ADA positive at baseline with pre-existing titre boosted by 4-fold or greater during the study period (Treatment-boosted ADA Positive). ADA incidence is the proportion of TE-ADA+ subjects in a population.
- [6] ADA post-baseline positive but not fulfilling the conditions for TE-ADA+
- [7] ADA negative at baseline and having at least 2 post-baseline ADA positive measurements with ≥16 weeks (112 days) between first and last positive, or an ADA positive result at the last available post-baseline assessment.
- [8] ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.

Reference Listing: 16.2.9.19

## **Programming Notes:**

- If a participant has more than 1 non-missing titre during the study, the maximum titre for each participant is summarized.
- Only present summary statistics if titre is available.
- If no positive results for a particular block of the table, then the summary statistics for the titres for that particular block would not appear.
- It is assumed that participants with a missing baseline ADA result are ADA negative at baseline.
- A column for column dosing (column dosing will only be added if Stage 4 is initiated.





## 7. Pharmacokinetic/Pharmacodynamic Data

Table 14.4.1 Summary of Serum MEDI7352 Concentrations PK Population

ADA Status: xxxxxxxxxx

| | | MEDI7352 | |
|---|---|---|---|
| Visit/ | CCI | CCI | CCI |
| Statistic | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean $[gMean \pm gSD]$ | x.xx [x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] |
| gCV% | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Week 2 | | | |
| $n (n \le LLOQ)$ | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean $[gMean \pm gSD]$ | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] |
| gCV% | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Week 4 | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean [gMean $\pm$ gSD] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] |
| gCV% | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX |

gCV% = Geometric Coefficient of Variation (%); gMean = Geometric Mean; gSD = Geometric SD; LLOQ = Lower Limit of Quantification; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; NC = not calculable; NQ = not quantifiable. [1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Note: serum MEDI7352 concentration units = ng/mL

Reference Listing: 16.2.10.1

Final 1 2 | 04-Oct-2023 | 





## **Programming Notes:**

- Include the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours/ Pre-Dose, Week 11/ Pre-Dose, Week 10 + 14 Days/Pre-Dose; Week 18.
- Repeat the table for 'ADA Positive', 'ADA Negative' and 'Overall'.
- Any values reported as NRR (not reportable) or NS (missing) will be excluded from the summary tables.
- At a time point where less than or equal to 50% of the concentration values are NQ (below LLOQ), all NQ values will be set to the LLOQ, and all descriptive statistics will be calculated accordingly.
- At a time point where more than 50% (but not all) of the values are NQ, the gmean, gmean  $\pm$  gSD and gCV% will be set to NC. The maximum value will be reported from the individual data, and the minimum and median will be set to NQ.
- If all concentrations are NQ at a time point, no descriptive statistics will be calculated for that time point. The gmean, minimum, median and maximum will be reported as NQ and the gCV% and gmean ± gSD as NC.

Final 1.2 | 04-Oct-2023 | 





#### Table 14.4.2 Summary of Serum total NGF Concentrations Safety Population

ADA Status: xxxxxxxxxx

| | Placebo | | MEDI7352 | |
|---|---|---|---|---|
| Visit/ | | CCI | CCI | CCI |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline [1] | | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean $[gMean \pm gSD]$ | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] | ` ′ |
| gCV% | XX.X | XX.X | xx.x | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx |
| Week 2 | | | | |
| n (n < LLOQ) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean [gMean $\pm$ gSD] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | x.xx[x.xx to x.xx] | , , |
| gCV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx |
| Week 4 | | | | |
| $n (n \le LLOQ)$ | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| gMean [gMean $\pm$ gSD] | x.xx[x.xx to x.xx] | x.xx [x.xx to x.xx] | x.xx [x.xx to x.xx] | , , |
| gCV% | XX.X | xx.x | XX.X | XX.X |
| Median | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX |

gCV% = Geometric Coefficient of Variation (%); gMean = Geometric Mean; gSD = Geometric SD; LLOQ = Lower Limit of Quantification; n = number of subjects by treatment group at each visit for the parameter; N = number of subjects per treatment group; ; NC = not calculable; NGF = Nerve-Growth Factor; NQ = not quantifiable.

Note: serum total NGF concentration units = pg/mL

Reference Listing: 16.2.10.2

<sup>[1]</sup> Baseline is defined as the last observation recorded prior to the first dose of treatment.





## **Programming Notes:**

- Repeat for ADA Status: "ADA Positive", "ADA Negative" and "Overall".
- Include the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.
- A column for column for dosing (column for dosing

Final 1 2 | 04-Oct-2023 | 





## **Planned Listing Descriptions and Shells**

| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| Listing 16.2.1.1 - Subject Disposition - Screening Population | U |
| Listing 16.2.1.2 - Assignment to Analysis Populations - Screening Population | U |
| Listing 16.2.1.3 - Reason for IP Discontinuation and Withdrawal from the Study - Safety Population | U |
| Listing 16.2.1.4 - List of Reasons for Screening Failure - Screen Failure Population | U |
| Listing 16.2.1.5 - Subject Visits and COVID-19 Impact - Screening Population | U |
| Listing 16.2.2.1 - Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria - Screening Population | U |
| Listing 16.2.2.2-Protocol Deviations - Sa fety Population | found.Error! U |
| Listing 16.2.3 - Randomization and Treatment Group - Sa fety Population | |
| Listing 16.2.4.1 - Demographic and Baseline Characteristics - Screening Population | U |
| Listing 16.2.4.2 - Medical History - Safety Population | U |
| Listing 16.2.4.3 - Osteoarthritis Characteristics - Screening Population | U |
| Listing 16.2.5.1 - Study Drug Administration: Individual Doses - Safety Population | U |
| Listing 16.2.6.1 - Daily Pain NRS - mITT Population | U |
| Listing 16.2.6.2 - Galer NPS - mITT Population | U |
| Listing 16.2.6.3 - DSIS - mITT Population | U |
| Listing 16.2.6.4 - SF-36 - mITT Population | U |
| Listing 16.2.6.5 - Rescue Medication Usage - mITT Population | R |
| Listing 16.2.6.6 - Patient Global Impression of Change - mITT Population | U |

Final 1 2 | 04-Oct-2023 | 





| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| CCI CCI | U |
| Listing 16.2.7.1 - Adverse Events - Safety Population | U |
| Listing 16.2.7.2 - Treatment Emergent Adverse Events Leading to Study Drug Discontinuation Sa fety Population | |
| Listing 16.2.7.3 - Treatment Emergent Adverse Events Associated with Abnormal Liver - Safety Population | R |
| Listing 16.2.7.4 - Joint Related Adverse Events of Special Interest - Safety Population | R |
| Listing 16.2.7.5 - Serious and/or Severe Infections - Safety Population | R |
| Listing 16.2.7.6 - Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of Study Drug - Safety Population | R |
| Listing 16.2.8.1 - Clinical Chemistry Laboratory Evaluations - Safety Population | U |
| Listing 16.2.8.2 - Hematology Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.3 - Coagulation Laboratory Evaluations - Safety Population | R |
| Listing 16.2.8.4 - Urinalysis Laboratory Evaluations - Safety Population | |
| Listing 16.2.8.5 - Serology Laboratory Evaluations - Safety Population | |
| Listing 16.2.8.6 - Pregnancy Test Results - Safety Population | |
| Listing 16.2.8.7 - Drug Test Results - Safety Population | U |
| Listing 16.2.8.8 - COVID-19 Screening and Vaccination - Safety Population | U |
| Listing 16.2.9.1 - Vital Signs Measurements - Safety Population | U |
| Listing 16.2.9.2.1 - 12-Lead Digital ECG Results - Safety Population | U |
| Listing 16.2.9.2.2 - 12-Lead Safety ECG Results - Safety Population | U |
| Listing 16.2.9.3 - Physical Examination Results - Safety Population | U |
| Listing 16.2.9.4 - Neurological Examination Results - Safety Population | U |
| Listing 16.2.9.5 - Total Neuropathy Score-Nurse - Safety Population | U |

Final 1 2 | 04-Oct-2023 | 





| Number Title Population | Unique (U)<br>or Repeated<br>(R) |
|---|---|
| Listing 16.2.9.6 - Motor and Sensory Nerve Conduction Studies - Safety Population | U |
| Listing 16.2.9.7 - Strength and Deep Tendon Reflexes - Safety Population | |
| Listing 16.2.9.8 - Injection Site Reactions - Safety Population | U |
| Listing 16.2.9.9 - Hypersensitivity/Anaphylactic Reactions - Safety Population | U |
| Listing 16.2.9.10 - Liver Diagnostic Investigations - Safety Population | |
| Listing 16.2.9.11 - Liver Risk Factors and Lifestyle Events - Safety Population | |
| Listing 16.2.9.12 - Liver Signs and Symptoms - Safety Population | |
| Listing 16.2.9.13 - Infection Diagnostic Investigations - Safety Population | |
| Listing 16.2.9.14 - Infection Risk Factors and Lifestyle Events - Safety Population | |
| Listing 16.2.9.15 - Infection Signs and Symptoms - Safety Population | |
| Listing 16.2.9.16 - Prior and Concomitant Medications - Safety Population | |
| Listing 16.2.9.17 - Prohibited Concomitant Medications - Safety Population | |
| Listing 16.2.9.18 - Concomitant Procedures - Safety Population | |
| Listing 16.2.9.19 - Anti-drug Antibody Test Results - Safety Population | |
| Listing 16.2.10.1 - Serum MEDI7352 Concentrations - PK Population | |
| Listing 16.2.10.2 - Serum total NGF Concentrations - PD Population | U |

Final 1 2 | 04-Oct-2023 | 





## **Listing Change Log:**

| Output<br>Number | Date of<br>Change | Change<br>Made By<br>(initials) | Description/Rationale |
|---|---|---|---|

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.1.1 Subject Disposition Screening Population

| Subject<br>ID | Re-screened?/<br>Previous<br>Subject ID | Treatment<br>Arm | Re-consent/ Date/Time of Initial IC/ Initial Protocol Version | Date/Time of<br>Informed Consent | Protocol<br>Version at<br>consent/<br>Re-consent | Consent for Colsample? /Date of Consent | Consent for<br>COVID-19 Sa fety<br>Mea sures / Date of<br>Consent | Current<br>Protocol<br>version |
|---|---|---|---|---|---|---|---|---|
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | Yes/ XXXX | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXXXX |
| XXXX | No | XXXX | Yes /<br>DDMMMYYYY/hh:mm<br>/ XXXX | DDMMMYYYY/<br>hh:mm | XXXX | Yes/<br>DDMMMYYYY | No | XXXXX |
| XXXX | No | XXXX | No | DDMMMYYYY/<br>hh:mm | XXXX | No | No | XXXXX |

COVID-19 = corona virus disease 2019; IC = Informed Consent;

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.1.2 Assignment to Analysis Populations Screening Population

| SubjectID | Treatment<br>Arm | Screened [1] | Randomized | SAF [2] | mITT[3] | PK [4] | Reason to Exclude from<br>Safety [5] | Reason to Exclude from mITT [6] |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Yes | No | No | No | No | | |
| XXXXXX | XXXX | Yes | Yes | Yes | Yes | Yes | | |
| XXXXXX | XXXX | Yes | Yes | No | No | No | XXX | |
| XXXXXX | XXXX | Yes | Yes | Yes | Yes | Yes | | |
| XXXXXX | XXXX | Yes | Yes | Yes | No | No | XXX/ XXX | XXX/ XXX |

mITT = Modified Intent-To-Treat Population Set; NRS = numeric rating scale; PK = pharmacokinetics; SAF = Safety Population Set.

## **Programming Notes:**

- If there is more than one major deviation, please concatenate with "/"
- Sort by Treatment Arm/ Subject ID.

Final 1 2 | 04-Oct-2023 | 

<sup>[1]</sup> The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments.

<sup>[2]</sup> The Safety Population includes all subjects who receive at least 1 dose of double-blind study medication.

<sup>[3]</sup> The mITT Population includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.

<sup>[4]</sup> The PK Population includes all subjects for who a pharmacokinetic sample was obtained and analysed.

<sup>[5]</sup> Major deviation reason/s to exclude from Safety Population for randomized subject.

<sup>[6]</sup> Major deviation reason/s to exclude from mITT Population for randomized subject.




## Listing 16.2.1.3 Reason for IP Discontinuation and Withdrawal from the Study Safety Population

| Subject ID/<br>Treatment<br>Arm | IP<br>Discontinuation<br>[1]/ Study<br>Withdrawal | Completion/<br>Discontinuation<br>Date (Study Day) | Date of Last Dose | Number of doses | Primary<br>Reason for<br>DC/<br>Withdrawal | Blind Broken? /<br>Date/Time /<br>Reason | Reason for<br>breaking<br>the Blind | Study<br>Duratio<br>n |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXX | IP<br>Discontinuation | DDMMMYYYY(XX) | DDMMMYYYY | XX | XXXXXX<br>X | Yes /<br>DDMMMYYYY/<br>hh:mm | XXXXXX | XX |
| XXXXXX/<br>XXXX | IP<br>Discontinuation | DDMMMYYYY (XX) | DDMMMYYYY | XX | XXXXXX<br>X | No | | XX |
| XXXXXX/<br>XXXX | Study<br>Withdrawal | DDMMMYYYY (XX) | DDMMMYYYY | XX | Other:<br>XXXXXX<br>X | No | | XX |

DC = Discontinuation; IP = Investigational product.

Note: Study Day is calculated relative to the date of first dose. Study Duration = Reference end date – date of first dose of treatment + 1.

## **Programming Notes:**

- If reason for non-completion is Other, concatenate the specify text as follows: "Other: XXXXXXXXX".
- If reason for non-completion is adverse event, concatenate with AE line number as follows: "Adverse event number X".
- For Physician decision, screen-fail and withdrawal by subject, please provide explanation if presented on the logic "Physician decision: XXX".
- Do not include subjects who completed the study.
- Sort by Treatment Arm/ Subject ID.

<sup>[1]</sup> Any withdrawal from the study before last IP dose (Week 10) is considered an IP discontinuation.





### Listing 16.2.1.4 List of Reasons for Screening Failure Screen Failure Population

| Subject ID | Treatment Arm | Screen failure Date | Primary Reason for Screen Failure |
|---|---|---|---|
| XXXXXX | Screen Failure | DDMMMYYYY | XXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY | XXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY | |
| XXXXXX | Screen Failure | DDMMMYYYY | Other: XXXXXXXXX |
| XXXXXX | Screen Failure | DDMMMYYYY | |

## **Programming Notes:**

- If reason for non-completion is Other, concatenate the "Primary Reason for Screen Failure" text as follows: "Other: XXXXXXXXX".
- Sort by Subject ID.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.1.5 Visits List and COVID-19 Impact Screening Population

| Subject ID/<br>Treatment<br>Arm | Visit<br>Name | Visit Date<br>(Study<br>Day) | Is COVID-<br>19<br>Pandemic<br>Ongoing? | Impacted<br>by<br>COVID-19 | Was visit<br>performed?/<br>Visit Type | Visit<br>Performe<br>d Via | VS Data<br>provided? /<br>Assessments<br>Missed? | IP dosing<br>missed due to<br>COVID-19 /<br>Details | End of<br>Treatment<br>linked to<br>COVID-19 | Subject<br>discontinued<br>due to<br>COVID-19?/<br>Details |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | Yes | Yes | Yes/<br>Delayed | On site | Y/<br>Efficacy | Y/ XXXX | Other: XXXX | Y/ XXXX |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | Yes | No | Yes | | N/ Safety | | | |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | No | Yes | Yes | Video | N/<br>Efficacy,<br>Safety | Y/ Other:<br>XXXX | | |
| xxxxx/<br>xxxx | Visit<br>X | DDMMM<br>YYYY<br>(XX) | No | No | No / Missed | | | | | |

COVID-19 = corona virus disea se 2019; IP = Investigational Product; VS = Vital Signs.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Visit Type: Missed, Abbreviated, Delayed.
- Visit Performed Via: Video, Phone, On Site Other: xxxxxx.
- Details on IP dosing missed: Treatment on hold due to Sponsor Decision, Subject infected with COVID-19, Subject decision, Other: xxxxxx.
- End of treatment, reason if due to COVID: Subject infected with COVID-19, Subject decision, Travel restrictions, Site closed, Study delayed/cancelled, Other: xxxxxx.
- Details on Subjects discontinuing due to COVID-19: Subject infected with COVID-19, Subject decision, End of Treatment due to Sponsor, Other: xxxxxx.
- Sort by Treatment Arm/ Subject ID/ Visit Date.

Final 1 2 | 04-Oct-2023 | 





Listing 16.2.2.1
Subjects Not Meeting All Inclusion Criteria or Meeting any Exclusion Criteria
Screening Population

| SubjectID | Treatment Arm | Enrolled | Randomized | Inclusion or<br>Exclusion | Criteria<br>Number | Criteria Label |
|---|---|---|---|---|---|---|
| XXXXXX | Screen Failure | Yes | No | Inclusion | XX | XXXXXXXXXXXXXXXXX |
| | | Yes | No | Exclusion | XX | XXXXXXXXXXXXXXXXX |

## **Programming Notes:**

• Sort by Subject ID.

Final 1 2 | 04-Oct-2023 | 





### Listing 16.2.2.2 Protocol Deviations Safety Population

| SubjectIDTr | eatment Ar | m Analysis Population Event Date (Study Day) | ) Event Tyne | Description | Category | Covid-<br>19<br>Related? |
|---|---|---|---|---|---|---|
| Sasjeetib II | Cu tillollt / til | Trinary 515 Topumator Event Date (Study Day) | , Event Type | Description | cutegory | iciated: |
| XXXXXX | XXXX | Screened\RND\SAF\DDMMMYYYY (XX) mITT | XXXXXXXXXX | XXXXXXX | Non-<br>important | Y |
| | 12221 | | XXXXXXXXXXXX | XXXXXXXXXXXXX | - | |
| XXXXXX | XXXX | DDMMMYYYY (XX) | XXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX | |
| | | | XXXXXXXXXXXXXX | XXXXXXXXXX | XXXXX | |
| XXXXXX | XXXX | DDMMMYYYY (XX) | XXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX | |

COVID-19 = Corona virus disease 2019; mITT = Modified Intent-To-Treat Population; RND = Randomized Subjects; SAF = Safety Population. Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- The structure of this listing may change depending on the information in the protocol deviations file. In the analysis population column, include only the analysis population where subject is included in.
- o Sort by Treatment Arm/ Subject ID. If date is present in file, add a column for date of event and sort by date. If no date is present, sort by category with non-important first and then important.
- Event Type: Inclusion Criteria, Exclusion Criteria, Study Drug, Assessment Safety, Assessment Efficacy, Lab/endpoint data, Visit Window, Informed Consent, Prohibited Co-Medication, Overdose/Misuse, Other.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.3 Randomization and Treatment group Safety Population

| Subject ID | Treatment Arm | Randomization Stage | Randomization Treatment | Randomization Date / Time<br>(Study Day) | Randomization<br>Number |
|---|---|---|---|---|---|
| XXXXXX | XXXX | Stage 1 | Active | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 3 | Active CC | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 2 | Placebo | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 2 | Active <b>CC</b> | DDMMMYYYY/hh:mm (-X) | XXXX |
| XXXXXX | XXXX | Stage 3 | Placebo | DDMMMYYYY/hh:mm (-X) | XXXX |

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID.

Final 1 2 | 04-Oct-2023 | 





## Listing 16.2.4.1 Demographic and Baseline Characteristics Screening Population

| Subject<br>ID | Treatment<br>Arm | Birth Date | Age<br>(years) | Sex | Surgically sterile?/ Postmenopausal? [2] | Ethnicity | Race | Weight (kg) | Height | BMI (kg/m²) | Fully<br>vaccinated<br>for COVID-<br>19? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | DDMMMYYY | XX | XX | Tostinenopausur. [2] | XXXXX | XXXX | XX.X | XX.X | XX.X | Y |
| XXX | XXX | MMMYYY | XX | XX | No/ Yes | XXXXX | XXXX | XX.X | XX.X | XX.X | N |

COVID-19 = Corona virus disease 2019.

Note: Height and weight are the values at Screening.

[1] Age was calculated as age at time of consent.

[2] For Female Subject Only.

## **Programming Notes:**

o Sort by Treatment Arm/ Subject ID

Final 1 2 | 04-Oct-2023 | 





Listing 16.2.4.2 Medical History Safety Population

| Subject ID | Treatment Arm | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day)/ |
|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |
| | | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXX | MMMYYYY (X)/<br>Ongoing |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>Ongoing |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |

MedDRA = Medical Dictionary for Regulatory Activities. Note: Study Day is calculated relative to the date of first dose. Medical History were coded using MedDRA version 26.0. Only subjects with medical history recorded are listed.

## **Programming Notes:**

- SOC & PT text should be in proper case in listing.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date of medical event.

Final 1 2 | 04-Oct-2023 | 





## Listing 16.2.4.3 Osteoarthritis Characteristics Screening Population

| Subject ID | Treatment<br>Arm | Subject with OA? / Joint/<br>Area affected | Is OA<br>considered<br>CS? | Radiological<br>Investigations<br>Conducted? / Details | Joint Area<br>Investigated | Is OA<br>considered<br>RS? | K-L Score<br>Reported | Radiologic Scoring<br>System / Details/<br>Result |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Y / Shoulder | Y | Y/ Other: XXXXXX | Shoulder | Y | Grade 3 | XXXXXX/<br>XXXXXX/<br>XX |
| XXXXXX | XXXX | Y / Ankle | N | Y/MRI | Ankle | N | N | N |

CS = Clinically Significant; K-L = Kellgren-Lawrence; OA = Osteoarthritis; RS = Radiologically Significant.

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID

Final 1 2 | 04-Oct-2023 | 





## Listing 16.2.5.1 Study Drug Administration: Individual Doses Safety Population

| | | Start<br>Date/ | End<br>Date/ | Was<br>Infusion<br>Performed?/<br>Infusion<br>Volume | Actually | If<br>Difference<br>between | Any | Any | Infusion | | Reason<br>for |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID/ | <b>3</b> 7, | Time | Time | (mL)[1]/ | Administered | [1] and [2] | Injection | Infusion | Rate | D | Infusion |
| Treatment<br>Arm | Visit<br>Name | (Study<br>Day) | (Study<br>Day) | Reason not Performed | Volume (mL) [2] | Volume,<br>Reason | Site<br>Reactions? | Related<br>Reactions | (mL/<br>hour) | Rate Change Justification | Rate<br>Change |
| XXXX/<br>XXXX | XXX | DDMM<br>MYYYY<br>/hh:mm<br>(X) | DDMM<br>MYYYY<br>/hh:mm<br>(X) | Y/<br>XX | XX | | | | xx.x | | |
| XXXX/<br>XXXX | XXX | DDMM<br>MYYYY<br>/hh:mm<br>(X) | DDMM<br>MYYYY<br>/hh:mm<br>(X) | Y/<br>XX | XX | XXXXX | Y | Y | xx.x | XXXXX | XXXXX<br>XX |
| XXXX/<br>XXXX | XXX | | | N/<br>XXXXXX | | | | | | | |

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / End Date.
- Rate Change Justification: Increased, Decreased, Interrupted.

Final 1 2 | 04-Oct-2023 | 





Listing 16.2.6.1 Daily Pain NRS mITT Population

| Subject ID | Treatment Arm | Study Visit [1] | Subject Diary (ePRO) Date / Study Day | Baseline Flag [2] | DPS |
|---|---|---|---|---|---|
| XXXXXX | XXXX | Baseline | DDMMMYYYY/ (-7) | Y | X |
| | | Baseline | DDMMMYYYY/ (-6) | Y | XX |
| | | ••• | ••• | ••• | ••• |
| | | Baseline | DDMMMYYYY/ (-2) | Y | XX |
| | | Baseline | DDMMMYYYY/ (-1) | Y | XX |
| | | ••• | | | |
| | | Week 2 | DDMMMYYYY/ (13) | | XX |
| | | Week 2 | DDMMMYYYY/ (14) | | XX |
| | | ••• | | | |
| | | Week X | DDMMMYYYY/ (X) | | XX |
| | | ••• | ••• | | |
| XXXXXX | XXXX | Baseline | DDMMMYYYY/ (-7) | Y | XX |
| DDG D 1 D | | | | ••• | ••• |

DPS = Daily Pain Score; ePRO = Electronic Patient-Reported Outcome; NRS = Numeric Rating Scale.

Note: Data shown in column 'DPS' are average daily pain scores on an 11-point (0-10) NRS. Study Day is calculated relative to the date of first dose. [1] Study Visit is defined as the 7-day period ending within the protocol window Day  $\pm 3$ , where at least 4 days out of 7 have recorded diary pain scores.

Final 1 2 | 04-Oct-2023 | 

<sup>[2]</sup> Baseline is defined as the 7-day period prior to randomization i.e., Day -7 to Day -1, inclusive. A subject is considered to have an evaluable baseline pain score if there are at least 4 days of recorded diary pain scores in the 7-day period.





## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Subject Diary Date.
- Display all measurement per Subject, starting on the Study Day = -7.
- Display Study Visit for days involved in weekly averages of the average daily pain scores for Baseline, Week 2, 4, 6, 8, 10, and 12
- Flag Baseline records only when there is at least 5 days of recorded diary pain scores in the 7-day Baseline period

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.6.2 Galer NPS mITT Population

| Subject ID | Treatment Arm | Parameter | Study Visit | Collection Date / Study<br>Day | Baseline Flag [1] | NPS |
|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Pain intensity | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | | Week 4 | DDMMMYYYY/(X) | | XX |
| | | | Week 8 | DDMMMYYYY/ (X) | | XX |
| | | | | ••• | | XX |
| | | | Week X | DDMMMYYYY/ (X) | | XX |
| | | | | ••• | | XX |
| | | XXXX | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | ••• | ••• | | | <b></b> |
| XXXXXX | XXXX | Pain intensity | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | | ••• | ••• | | <b></b> |
| | | XXXX | Week X | DDMMMYYYY/ (X) | | XX |
| | | ••• | ••• | | | |

NPS = Neuropathic Pain Scale; NRS = Numeric Rating Scale.

Note: Data shown in column 'NPS' are Pain Intensity, Unpleasantness, and Descriptor scores on an 11-point (0-10) NRS, and Pain Duration/Frequency on a 3-point NRS (1-3).

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Final 1 2 | 04-Oct-2023 | 





## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter / Collection Date.
- Keep Parameter sorting from the last bullet point in this programming notes.
- Include all observed data on Galer NPS scores for Baseline, Week 4, 8, 12, and 18.
- Repeat for the Parameters: Pain intensity, Pain Unpleasantness, Pain Sharpness, Pain Hotness, Pain Dullness, Pain Coldness, Pain Sensitivity, Pain Itching, Deep Pain Intensity, Surface Pain Intensity (All in an 11-point NRS), and Pain Duration/Frequency (in a 3-point NRS).

Final 1 2 | 04-Oct-2023 | 





Listing 16.2.6.3
DSIS
mITT Population

#### **Programming Notes:**

- Same shell as Listing 16.2.6.1.
- Update footnote as:
  - DSIS = Daily Sleep Interference Scale; ePRO = Electronic Patient-Reported Outcome; NRS = Numeric Rating Scale. Note: Data shown in column 'DSIS' are daily Sleep Interference scores on an 11-point (0-10) NRS. Study Day is calculated relative to the date of the day of first dose.
  - [1] Study Visit is defined as the seven-day period ending within the protocol window Day  $\pm 3$ .
  - [2] Baseline is defined as the seven-day period prior to randomization i.e., Day -7 to Day -1,.
- Sort by Treatment Arm/ Subject ID / Subject Diary Date.
- Display all measurement per Subject, starting on the Study Day = -7.
- Display Study Visit for days involved in weekly averages of the average Sleep interference scores for Baseline, Week 4, 8, 12, and 18.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.6.4 SF-36 mITT Population

| Subject ID | Treatment<br>Arm | Parameter | Item<br>Number | Item name | Study Visit | Collection Date / Study<br>Day | Baseline<br>Flag[1] | SF-36 |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Physical functioning | 3 | Vigorous<br>Activities | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | | | | Week 12 | DDMMMYYYY/ (X) | | XX |
| | | | 4 | Moderate<br>Activities | Baseline | DDMMMYYYY/ (X) | Y | XX |
| | | ••• | ••• | ••• | ••• | | | |
| | | | - | Total | Baseline | DDMMMYYYY/ (X) | Y | |
| | | | | | Week 12 | DDMMMYYYY/ (X) | | XX |
| XXXXXX | XXXX | Role<br>limitations<br>due to<br>physical | | Cut Amount<br>of Time<br>Spent on<br>Work/Act | Baseline | | | |
| | | health | 13 | WOIK/ACt | | DDMMMYYYY/(X) | Y | XX |
| | | | | | Week 12 | DDMMMYYYY/ (X) | | XX |
| | | | ••• | | ••• | ••• | | ••• |
| | | ••• | | | ••• | | ••• | |

SF-36 = 36-Item Short-Form Health Survey; NRS = Numeric Rating Scale.

Note: Data shown in column 'SF-36' are derived SF-36 scores and Change in General Health on a 5-point NRS (1-5).

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

Final 1 2 | 04-Oct-2023 | 





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter / Item / Collection Date.
- Keep Parameter sorting from the last bullet point in this programming notes.
- Include all data on SF-36 scores for Baseline and Week 12.
- Repeat for the Parameters: Physical functioning (items 3, 4, 5, 6, 7, 8, 9, 10, 11, 12), Role limitations due to physical health (items: 13, 14, 15, 16), Role limitations due to emotional problems (items: 17, 18, 19), Vitality (Energy/fatigue) (items: 23, 27, 29, 31), Emotional well-being (items: 24, 25, 26, 28, 30), Social functioning (20, 32), Pain (items: 21, 22) and General Health (items: 1, 33, 34, 35, 36), all with values ranging from 0 to 100. Change in general Health (in a 5-point NRS, item: 2).

Final 1 2 | 04-Oct-2023 | 





## Listing 16.2.6.5 Rescue Medication Usage mITT Population

| Subject<br>ID | Treatment Arm | ATC Class (Level 2)/<br>Preferred Name/<br>Verbatim Term | Primary<br>Indication | Start Date (Study Day)/<br>End Date (Study Day) | Dose<br>(unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | MMMYYYY (-XX)/<br>DDMMMYYYY (-X) | XXXX<br>unit | XXXXXXXX | XXXXX |
| | XXXX | XXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | MMMYYYY (-X)/<br>Ongoing | XXXX<br>unit | XXXXXXXX | XXXXX |
| | XXXX | XXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXX | Painful<br>Diabetic<br>Neuropathy | DDMMMYYYY (X)/<br>DDMMMYYYY<br>(XX) | XXXX<br>unit | XXXXXXXX | XXXXX |

ATC = anatomical therapeutic chemical.

Note: Study Day is calculated relative to the date of first dose.

Medications were coded using WHO drug dictionary version vMar2023.

### **Programming Notes:**

- ATC & Preferred Name text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name.
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX") but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications

Final 1 2 | 04-Oct-2023 | 





## Listing 16.2.6.6 Patient Global Impression of Change mITT Population

| Subject ID | Treatment Arm | Study Visit | Collection Date / Study Day | PGIC |
|---|---|---|---|---|
| XXXXXX | XXXX | Week 4 | DDMMMYYYY/(X) | XXXXXXXX |
| | | Week 8 | DDMMMYYYY/(X) | XXXXXXXX |
| | | Week 12 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 18 | DDMMMYYYY/(X) | XXXXXXX |
| XXXXXX | XXXX | Week 4 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 8 | DDMMMYYYY/(X) | XXXXXXX |
| | | Week 12 | DDMMMYYYY/(X) | XXXXXXXX |
| | | Week 18 | DDMMMYYYY/(X) | XXXXXXXX |
| | | ••• | ••• | ••• |

PGIC =Patient Global Impression of Change.

Note: Data shown in column 'PGIC' are Subjects ratings about overall improvement in health status.

Study Day is calculated relative to the date of first dose.

[1] Baseline is defined as the last observation recorded prior to the first dose of treatment.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include all observed data on PGIC scores for Week 4, 8, 12, and 18.

Final 1 2 | 04-Oct-2023 | 







Final 1 2 | 04-Oct-2023 | 







Final 1 2 | 04-Oct-2023 | 





Listing 16.2.7.1 Adverse Events Safety Population

| Subject ID/<br>Treatment<br>Arm | AE ID<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | AE Start Date/Time<br>(Study Day)/<br>End Date/Time<br>(Study Day) | Severity/<br>Relationship<br>[1] | Outcome/ Action Taken with IP/ Therapy taken for this AE | AE Leading<br>to Study DC | ?<br>TEAE | Serious? /<br>Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMMMYYYY/HH<br>MM (X)/<br>X DDMMMYYYY/HH<br>MM (X) | XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>Yes | No | Yes | No |
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMMMYYYY/HH<br>MM (X)/<br>X DDMONYYYY/HH:<br>MM (X) | XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>No | Yes | No | Yes / XXX |
| XXXXX/<br>XXXX | X | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXX | DDMONYYYY/HH:<br>MM (X)/<br>X Ongoing | XXXXXX/<br>XXXXXX | XXXXXXXX/<br>XXXXXXX/<br>No | No | No | Yes / XXX |

AE = adverse event; DC = discontinuation; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Study Day is calculated relative to the date of first dose. A TEAE is defined as an AE with an onset at the time of or following the start of treatment with IP.

AEs were coded using MedDRA version 26.0

<sup>[1]</sup> Reasonable possibility AE caused by IP as assessed by the investigator .





## **Programming Notes:**

- If time missing, display "--:--".
- AE ID number represents Record position within Subject.
- If no events meet the criteria for display (i.e, no AEs occur in the study), present "No events are reported.".
- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically by SOC /PT if same date for two events).

In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Listing 16.2.7.2
Treatment Emergent Adverse Events Leading to Study Drug Discontinuation
Safety Population

#### **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update listing deleting seventh and eight columns

Listing 16.2.7.3
Treatment Emergent Adverse Events Associated with Abnormal Liver
Safety Population

## **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update listing deleting 8<sup>th</sup> column.

Final 1 2 | 04-Oct-2023 | 





## Listing 16.2.7.4 Joint Related Adverse Events of Special Interest Safety Population

### **Programming Notes:**

• Same shell as Listing 16.2.7.1.

Listing 16.2.7.5 Serious and/or Severe Infections Safety Population

#### **Programming Notes:**

• Same shell as Listing 16.2.7.1.

Listing 16.2.7.6

Anaphylactic Reactions, Hypersensitivity or Infusion-Related Reactions Leading to Discontinuation of Study Drug Safety Population

### **Programming Notes:**

- Same shell as Listing 16.2.7.1.
- Update footnote: Anaphylactic reactions, hypersensitivity or infusion-related reactions not leading to discontinuation of IP were included in listing as they were categorized as AE of special interest under Protocol Amendment 4 (V5.0). Definition for AE of special interest changed from Amendment 6 (V6.0) onwards, including anaphylactic reactions, hypersensitivity or infusion-related reactions leading to permanent discontinuation of IP.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.8.1 Clinical Chemistry Laboratory Evaluations Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Parameter | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Original<br>Result<br>(Unit) | Standard<br>Results<br>(unit) | Reference<br>Range<br>[1] | Baseline<br>Flag | CFB | Results<br>Assessment<br>/ Reason<br>CS | Lab ID<br>Number | Fasting<br>Status | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXXX | Chemistry panel | XXXXXX | | | | | | | ND: xxx | | | |
| XXXXX/<br>XXXX | Albumin | XXXXXX<br>XXXXXX<br>XXXXXX<br>XXXXXX | DDMMMYYYY/ HH:MM (X) DDMMMYYYY/ HH:MM (X) DDMMMYYYY/ HH:MM (X) DDMMMYYYY/ HH:MM (X) | XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX) | XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX)<br>XX<br>(XX) | XX - YY XX - YY XX - YY XX - YY | Y | XX.X<br>XX.X<br>XX.X | H-CS /<br>XXX<br>H-NCS | XXXXXXX<br>XXXXXXX<br>XXXXXXX<br>XXXXXXX | Y<br>Y<br>Y<br>N | XXXX |

CFB = change from baseline; CS = clinically significant; H = High; L = Low; NCS = not clinically significant; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

[1] Reference range is used to identify potentially clinically significant laboratory values.

#### **Programming Notes:**

- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Chemistry panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Albumin, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Bicarbonate, Calcium, Chloride, Creatinine, High-Sensitivity C-Reactive Protein (hs-CRP), Estimated Glomerular Filtration Rate (eGFR by Cockcroft-Gault), Serum Glucose, Lactate Dehydrogenase (LDH), Potassium, Sodium, Total Bilirubin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.8.2 Hematology Laboratory Evaluations Safety Population

### **Programming Notes:**

- Same shell as Listing 16.2.8.1.
- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Hematology panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Absolute basophil count, a bsolute eosinophil count, a bsolute lymphocytes count, Absolute Monocyte Count, Absolute Neutrophil Count, Basophils %, Eosinophils %, Hematocrit (HCT), Hemoglobin (HGB), hemoglobin A1C (HgbA1C), Lymphocytes %, mean corpuscular hemoglobin (MHC), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), Monocytes %, Neutrophils %, Platelets, Red blood cell count (RBC), Red Cell Distribution Width, white blood cell Count (WBC).

Listing 16.2.8.3 Coagulation Laboratory Evaluations Safety Population

### **Programming Notes:**

- Same shell as Listing 16.2.8.1.
- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Coagulation panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Activated Partial Thromboplastin Clotting Time (APTT), Fibrinogen, International normalized ratio (INR), Prothrombin Time (PT).

Final 1.2 | 04-Oct-2023 | 





## Listing 16.2.8.4 Urinalysis Laboratory Evaluations Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Parameter | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Original<br>Result<br>(Unit) | Standard<br>Results<br>(unit) | Reference<br>Range<br>[1] | Baseline<br>Flag | CFB | Results<br>Assessment<br>/ Reason<br>CS | Lab ID<br>Number | Fasting<br>Status | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Urinalysis<br>panel | XXXXXX | | | | | | | ND: xxx | | | |
| XXXXX | pH/<br>Specific<br>Gravity | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX<br>(XX) | XX<br>(XX) | XX - YY | Y | | | XXXXXXX | Y | |
| | Glavity | XXXXXX | DDMMMYYYY/ | XX | XX | XX - YY | | XX.X | H-CS/ | XXXXXXX | Y | XXXX |
| | | XXXXXX | HH:MM (X)<br>DDMMMYYYY/ | (XX)<br>XX | (XX)<br>XX | XX - YY | | XX.X | XXX | XXXXXXX | Y | |
| | | XXXXXX | HH:MM (X)<br>DDMMMYYYY/<br>HH:MM (X) | (XX)<br>XX<br>(XX) | (XX)<br>XX<br>(XX) | XX - YY | | XX.X | H-NCS | XXXXXXX | N | |
| | Blood<br>Urine/<br>Glucose/<br>Ketones/<br>Protein | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Trace | | | Y | | H-NCS | XXXXXXX | Y | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | 100<br>(mg/dL) | 100<br>(mg/dL) | | | | H-CS /<br>XXX | XXXXXXX | Y | XXXX |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Negative | | | | | | XXXXXXX | N | |

Final 1 2 | 04-Oct-2023 | 





CFB = change from baseline; CS = clinically significant; H = High; L = Low; NCS = not clinically significant; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

[1] Reference range is used to identify potentially clinically significant laboratory values.

### **Programming Notes:**

- Keep parameter sorting from the last bullet point below.
- For results assessment, do not populate column if result is normal.
- Sort by Treatment Arm/ Subject ID / Parameter / Date time of collection.
- If the whole panel is not done at a visit, present the information on first row of the subject under 'Urinalysis panel' parameter and don't present the 'not done' information for each parameter. Display "ND: reason why" in the result assessment column.
- Sort Parameters in the following Order: Blood Urine, Glucose, Ketones, pH, Protein, Specific Gravity.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.8.5 Serology Laboratory Evaluations Safety Population

| Subject<br>ID | Treatment<br>Arm | Was<br>Serology<br>Test<br>Collected? | Date/Time of<br>Collection<br>(Study Day) | Test (Unit) [1] | Result | Lab ID<br>Number | Fasting<br>Status | Reason not collected | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXX | Yes | DDMMMYYY<br>Y/HH:MM (X) | Hepatitis B Ag | Negative | XXXX | Y | | XXXXXXXX |
| | | | | Hepatitis C Ab | Positive | XXXX | Y | | |
| | | | | HIV-1/ -2 Ag | Not Done | XXXX | Y | XXXXXXX | |
| | | | | Quantiferon<br>Gold Plus NIL | X.XX (IU/mL) | XXXX | Y | | |

Ab = antibody; Ag = antigen; HIV = human immunodeficiency virus; TB = tuberculosis.

Note: Study Day is calculated relative to the date of first dose.

[1] if Applicable

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date of collection / Test.
- Keep parameter sorting from the last bullet point below
- Sort Parameters in the following Order: Hepatitis B Antigen, Hepatitis C Virus Antigen, Hepatitis C Virus Antibody, HIV-1/-2 Antigen, Quantiferon Gold Plus NIL, Quantiferon Gold Plus TB, Quantiferon Gold Plus Mitogen minus NIL, Quantiferon Gold Plus TB1 minus NIL, Quantiferon Gold Plus TB2 minus NIL

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.8.6 Pregnancy Test Results Safety Population

| Subject ID | Treatment<br>Arm | Visit | Was a Urine pregnancy test performed? | Date/Time Performed (Study Day) | If not, Reason | Result |
|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxx | Xxxx | Ddmmmyyyy/ hh:mm (XX) | xxxx | XXXX |
| | | xxxxx | Xxxx | Ddmmmyyyy/ hh:mm (XX) | Other: xxxx | XXXX |

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment.

Final 1 2 | 04-Oct-2023 | 





Listing 16.2.8.7 Drug Test Results Safety Population

| Subject ID | Treatment<br>Arm | Was Drug Test<br>Performed? | Date/ Time Assessment<br>(Study Day) | Result | Findings | Reason Test<br>not Performed |
|---|---|---|---|---|---|---|
| XXXXXX | XXXX | Yes | DDMMMYYYY/ HH:MM<br>(XX) | Negative | Negative | |
| XXXXXX | XXXX | Yes | DDMMMYYYY/ HH:MM<br>(XX) | Positive | Cocaine /<br>Opiates | |

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Concatenate all findings by "/"
- Sort by Treatment Arm/ Subject ID / Date of assessment.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.8.8 COVID-19 Screening Safety Population

| | | | | | • | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID/ | | COVID-19 Sx<br>Screening?/Date | | Body T <sup>o</sup><br>Check?/Date/ | | COVID-19<br>swab?/ Date/ | | COVID-19 Ab testing?/ Date/ | Ab | COVID-19<br>Ag testing?/ | Ag |
| Treatment | | / Time (Study | | Time (Study | Body T <sup>o</sup> | Time (Study | Swab | Time (Study | testing | Date/ Time | testing |
| Arm | Visit | Day) | Sx | Day) | (Unit) | Day) | result | Day) | results | (Study Day) | results |
| xxxxx/ | | Yes/ | XXX/ | Yes/ | | Yes/ | | Yes/ | | Yes/ | |
| | XXXX | Ddmmmyyyy/ | XXX | Ddmmmyyyy/ | | Ddmmmyyyy/ | Xxxx | Ddmmmyyyy/ | Xxxx | Ddmmmyyyy | Xxxx |
| XXXX | | hh:mm (XX) | | hh:mm (XX) | XX(XX) | hh:mm (XX) | | hh:mm (XX) | | / hh:mm(XX) | |
| | | Yes/ | XXX | Yes/ | | Yes/ | | Yes/ | | Yes/ | |
| | XXXX | Ddmmmyyyy/<br>hh:mm (XX) | | Ddmmmyyyy/<br>hh:mm (XX) | XX (XX) | Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Ddmmmyyyy/<br>hh:mm (XX) | Xxxx | Ddmmmyyyy<br>/ hh:mm(XX) | Xxxx |
| | | IIII.IIIII (2 <b>22</b> ) | | IIII.IIIII (2 <b>22</b> ) | 222 (222) | 1111.111111 (2020) | | 1111.111111 (2020) | | / IIII.IIIII (2 <b>22</b> ) | |

Ab = Antibody; Ag = Antigen; COVID-19 = Corona virus disease 2019; Sx = Symptoms; T° = Temperature.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Concatenate all Symptoms by "/"
- Sort by Treatment Arm/ Subject ID / Date of assessment

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.9.1 Vital Signs Measurements Safety Population

| Subject<br>ID | Treatment<br>Arm | Parameter | Study<br>Visit | Position [1] /<br>T <sup>o</sup> Method | Date/Time of<br>Collection<br>(Study Day) | Original Result<br>(Unit) | Baseline Flag | CFB |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Temperature | | XXXX | DDMMMYYYY/<br>HH:MM (X) | XX (XX) | Y | |
| | | <b>F</b> | XXXXXX | XXXX | DDMMMYYYY/<br>HH:MM (X) | XX (XX) | | XX |
| | | Resting<br>Heat Rate | Screening | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | | |
| | | | Day 1:<br>Pre-Dose | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | Y | XX |
| | | | XXXXXX | Supine | DDMMMYYYY/<br>HH:MM (X) | XX | | XX |
| | | | XXXXXX<br>XXXXXX | Sitting<br>Sitting | DDMMMYYYY/<br>HH:MM (X) | ND<br>XX | | XX |

CFB = change from baseline; eCRF = Electronic Case Report Form; ND = not done.

Note: Study Day is calculated relative to the date of first dose.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

'Day 1:5 minutes after Infusion Completion' time point was only applied to subjects enrolled in Stage 1, with data collected under eCRF versions 4.0 (11DEC2018) or older.

[1] Resting position measurements encompass Sitting and Supine position measurements.

Final 1 2 | 04-Oct-2023 | 





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Parameter (Order in the second bullet point)/ Date time of collection.
- Repeat for Resting Heart Rate, Resting Systolic Blood Pressure, Resting Dia stolic Blood Pressure, Respiratory Rate, Body Temperature, Standing Heart Rate, Standing Systolic Blood Pressure, Standing Dia stolic Blood Pressure.
- After Week 2 (inclusive), Supine measure are taken in sitting position. We will consider them as supine (in resting position) for calculating Change from Baseline (always at supine position).
- Include the following timepoints: Screening, Baseline (Day 1: Pre-Dose), Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: Pre-Dose, Week 10: 5 minutes after Infusion Completion, Week 11, Week 12, Week 18.
- Note that Body T<sup>o</sup>, and standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.9.2.1 12-Lead Digital ECG Results Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Visit | ECG Date / Time<br>(Study Day) | Tra cin | PR Interval (msec) | QRS<br>duration<br>(msec) | QT<br>Interval<br>(msec) | RR<br>interval<br>(bpm) | Heart Rate (beats/min) | QTcF<br>Interval<br>(msec) | Findings | Reason<br>Not<br>Done |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Day 1:<br>Pre-Dose | DDMMMYYYY<br>/ HH:MM (XX) | 1 | XX | XX | xx | XX | XX | XX | xx:<br>xxxxx | |
| | | | 2 | XX | XX | XX | XX | XX | XX | | |
| | | | 3 | XX | XX | XX | XX | XX | XX | xx:<br>xxxxx | |
| XXXXX | XXXX | DDMMMYYYY/<br>HH:MM (XX) | 1 | xx | XX | XX | XX | XX | XX | xx:<br>xxxxx | |
| | | | 2 | XX | XX | XX | XX | XX | XX | | |
| | | | 3 | XX | XX | XX | XX | XX | XX | | |

CS = clinically significant; ECG = electrocardiogram; NCS = Not clinically significant

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date time of collection / Tracing.
- For Findings, concatenate test name with test result for category "FINDINGS".
- Include the following timepoints: Day 1: Pre-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.

Final 1 2 | 04-Oct-2023 | 





#### 00Listing 16.2.9.2.2 12-Lead Safety ECG Results Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit | ECG Date / Time<br>(Study Day) | Tracing | ECG Result/<br>Comment | PR Interval (msec) | QRS duration (msec) | QTcF<br>Interval<br>(msec) | Reason<br>Not Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | Day 1: Pre-<br>Dose | DDMMMYYYY /<br>HH:MM (XX) | 1 | Abnormal CS/ xxxx | XX | XX | xx | |
| | | | 2 | Abnormal CS/xxxx | XX | XX | XX | |
| | | | 3 | Abnormal NCS/<br>xxxx | XX | XX | XX | |
| XXXXX | XXXX | DDMMMYYYY/<br>HH:MM (XX) | 1 | Normal | XX | XX | XX | |
| | | | 2 | Normal | XX | XX | XX | |
| | | | 3 | Normal | XX | XX | XX | |

CS = clinically significant; ECG = electrocardiogram; NCS = Not clinically significant

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Date time of collection / Tracing.
- Include the following timepoints: Screening, Day 1: Pre-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 4, Week, 8, Week 12, and Week 18.

Final 1 2 | 04-Oct-2023 | 




# Listing 16.2.9.3 Physical Examination Results Safety Population

| Subject ID | Treatment<br>Arm | Visit | Examination<br>Type | Exam Date/ Time<br>(Study Day) | Body System | Result / Change<br>from previous<br>assessment [1] | If Abnormal,<br>findings /<br>Specify<br>Changes [2] | Reason Not<br>Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Screening | Complete | DDMMMYYYY<br>/ HH:MM (XX) | Head, Neck and<br>Thyroid<br>Ears, Eyes, Nose<br>and Throat | Normal<br>Abnormal CS | XXXXXXX | |
| | | Day 1 | Targeted | DDMMMYYYY<br>/ HH:MM (XX) | Ears, Eyes, Nose<br>and Throat | XXXXXXXXX | xxxxxxx | |

CS = Clinically Significant, NCS = Not Clinically Significant

Note: Study Day is calculated relative to the date of first dose.

[1] For targeted examination type: Change from previous assessment.

[2] For targeted examination type: Specify Changes.

#### **Programming Notes:**

- Keep sorting from eCRF: Head, Neck and Thyroid/Ears, Eyes, Nose and Throat/ Chest (including breasts)/ Lungs/Heart/LymphNodes/Abdomen/Hepatic/Gastrointestinal/Anorectal/Genitourinary/Skin/Musculoskeletal/Extremities/Neurological/Other.
- Complete Physical examination only at Screening, Week 12, 18 (it can also be unscheduled).
- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Body system

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.9.4 Neurological Examination Results Safety Population

| Subject ID | Treatment<br>Arm | Visit | Exam Date/ Time<br>(Study Day) | Body System | Result | If Abnormal,<br>findings | Reason Not<br>Done |
|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Screening | DDMMMYYYY /<br>HH:MM (XX) | Mental Status Cranial Nerves | Normal AbnormalCS | XXXXXXX | Bone |
| | | Day 1 | DDMMMYYYY /<br>HH:MM (XX) | Cranial Nerves | XXXXXXXXX | XXXXXXXX | |

CS = Clinically Significant, NCS = Not Clinically Significant

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Keep sorting from eCRF: Mental status/ Cranial Nerves/ Motor Function/ Reflexes / Sensation and Propioception / Coordination / Other.
- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Body system

Final 1 2 | 04-Oct-2023 | 





Listing 16.2.9.5
Total Neuropathy Score-Nurse
Safety Population

| | | | | ~ | ery repulsion | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | | Sensory | Motor | | Pin | Vibration | | _ |
| ID/ | | Date/ Time of | Symptom | Symptom | Autonomic | Sensibility | Sensibility | | |
| Treatment | | collection | Score | Score | Symptom | Score | Score | TNSn Total | |
| Arm | Visit | (Study Day) | (0-4) | (0-4) | Score (0-4) | (0-4) | (0-4) | (0-20) | Reason Not Done |
| XXXXX/<br>XXXX | Screening | DDMMMYYYY<br>/ HH:MM (XX) | XX | XX | XX | XX | XX | XX | |
| | Day 1 | DDMMMYYYY<br>/ HH:MM (XX) | XX | XX | XX | XX | XX | XX | |
| | Week 2 | DDMMMYYYY<br>/ HH:MM (XX) | ND | ND | ND | ND | ND | ND | XXXXXXXXXXXX |

ND = Not Done; TNSn = Total Neuropathy Score-Nurse.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.6 Motor and Sensory Nerve Conduction Studies Safety Population

| Subject ID/<br>Treatment<br>Arm | Visit | Date/Time of<br>Collection<br>(Study Day) | Location /<br>Evaluation | Was<br>Evaluation<br>Preformed<br>?/Nerve | Amplitude<br>(Motor =<br>mV; sensory<br>= microV)/<br>Range | Peak<br>Latency<br>(msec)/<br>Range | Conduction<br>velocity<br>(msec) /<br>Range | Duration<br>of action<br>potential<br>(msec)/<br>Range | Evaluation<br>Result | If<br>Abnomal,<br>Specify/<br>Reason<br>Not Done | Significant Changes from Baseline?/ if Yes, Specify |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX/<br>XXXX | Screening | DDMMMYY<br>YY / HH:MM<br>(XX) | Lower Limb - Right Side/ | Y/<br>XXXXXX<br>Y/<br>XXXXXX<br>N | xx [x.xx to x.xx] xx [x.xx to x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx to x.xx ] | xx [x.xx to x.xx] xx [x.xx to x.xx] | xx [x.xx to x.xx] xx [x.xx to x.xx to | Abnormal<br>Normal | XXXXX | NA<br>NA |
| | Week 18 | DDMMMYY<br>YY/ HH:MM<br>(XX) | XXXXXX/<br>XXXXXX/<br>XXXXXX/<br>XXXXXX/<br>XXXXXX/ | Y/<br>XXXXXX<br>Y/<br>XXXXXX<br>Y/<br>XXXXXX | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx]<br>xx<br>[x.xx to<br>x.xx] | Abnormal Normal Abnormal | XXXXX | N<br>N<br>Y/<br>XXXXXXX |

NA = Not Applicable
Note: Study Day is calculated relative to the date of first dose.





### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment / Location Evaluation
- Keep sorting from eCRF: Lower Limb right side/Motor evaluation, Lower Limb right side/Sensory evaluation, Lower Limb left side/ Motor evaluation, Upper Limb right side/ Sensory evaluation, Upper Limb left side/ Motor evaluation, Upper Limb left side/ Motor evaluation, Upper Limb left side/ Sensory evaluation.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.7 Strength and Deep Tendon Reflexes Safety Population

| Subject ID | Treatment<br>Arm | Visit | Date/ Time of<br>collection<br>(Study Day) | Ankle Dorsiflexion<br>Strength | Deep Tendon Reflexes | Reason Not Done |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | Screening | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | |
| | | Day 1 | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | |
| | | Week 2 | DDMMMYYYY /<br>HH:MM (XX) | ND | ND | XXXXXXXXXXXX |

ND = Not Done.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

• Sort by Treatment Arm/ Subject ID / Visit / Date of assessment

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.8 Injection Site Reactions Safety Population

| Subject<br>ID | Treatment<br>Arm | Visit | Date/Time of Assessment<br>(Study Day) | Pain | Tenderness | Erythema/redness | Induration/<br>swelling | Reason Not Done |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | Day 1: 15<br>Minutes<br>after Start of<br>Infusion | DDMMMYYYY /<br>HH:MM (XX) | XXXX | XXXX | XXXX | XXXX | |
| | | Day 1: 30<br>Minutes<br>after Start of<br>Infusion | DDMMMYYYY /<br>HH:MM (XX) | XX | XX | XX | XX | |
| | | Week 18 | DDMMMYYYY /<br>HH:MM (XX) | ND | ND | ND | ND | XXXXXXXXXXXX |

ND = Not Done.

Note: Study Day is calculated relative to the date of first dose.

# **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Visit / Date of assessment
- Include the following timepoints: Day 1: 15 Minutes after Start of Infusion, Day 1: 30 Minutes after Start of Infusion, Day 1: 45 Minutes after Start of Infusion, Day 1: 60 Minutes after Start of Infusion, Day 1: 4 hours after Start of Infusion, Week 2, Week 4, Week 6, Week, 8, Week 10, Week 12, and Week 18.

Final 1 2 | 04-Oct-2023 | 





Listing 16.2.9.9
Hypersensitivity/Anaphylactic Reactions
Safety Population

| Subject<br>ID | Treatment<br>Arm | AE ID<br>Number | Onset Date/Time (Study Day)/<br>Resolution Date/Time (Study<br>Day) | Type of<br>Reaction | Severity grade for<br>the Symptom<br>with Highest<br>Severity | Onset Time<br>for Highest<br>Severity | Leading to IP Discontinuation? |
|---|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXX | XXXX | /HH:MM | Yes |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXX | | | No |
| | | ••• | | | | | |
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXX | XXXX | /HH:MM | No |

AE = Adverse Event.

Note: Study Day is calculated relative to the date of first dose.

## **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Onset Date/Time / Resolution Date/Time / Reaction Type.
- Keep sorting from eCRF: Urticaria, Pruritus, Rash, Flushing, Swollen lips, tongue, uvula and/or vulva, Dyspnoea, Wheeze-bronchospasm, Stridor, Hypoxia, Hypotension, Crampy abdominal pain, Vomiting, Diarrhoea, Other.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.10 Liver Diagnostic Investigations Safety Population

| Subject ID | Treatment<br>Arm | Potential Hy's<br>Law Case<br>Number | Liver Diagnostic Investigation<br>Date (Study Day) | Liver Diagnostic<br>Investigation | Liver Dia gnostic<br>Investigation<br>Results | Comments |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY (X) | XXXX | XXXX | XXXXX |
| | | X | DDMMMYYYY (X) | XXXXX | XXXXX | |
| XXXXX | XXXX | X | DDMMMYYYY (X) | XXXXX | XXXXX | |

CT = Computerized tomography; ERCP = Endoscopic retrograde cholangiopancreatography; MRI = Magnetic resonance imaging; MRCP = Magnetic resonance cholangiopancreatography.

Note: Study Day is calculated relative to the date of first dose.

#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Diagnostic Date / Liver Diagnostic Investigation.
- Keep sorting from eCRF: Ultra sound, CT, MRI/MRCP, ERCP, Liver Biopsy, X-Ray, Tox Screening for Acetaminophen/Paracetamol, Tox Screening for Ethanol, Tox Screening, Other, Specialist (e.g. Hepatologist) Consulted, Serology for Hepatitis A, Serology for Hepatitis B, Serology for Hepatitis C, Serology for Hepatitis D, Serology for Hepatitis E, for Cytomegalovirus (CMV), Serology for Epstein Barr Virus (EBV), Autoimmune Serology, Other.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.11 Liver Risk Factors and Lifestyle Events Safety Population

| | | Potential | | Liver Risk Factor Start Date | Liver Risk | | |
|---|---|---|---|---|---|---|---|
| | | Hy's Law | Assessment Date | (Study Day)/ | Factor/ | | |
| | Treatment | Case | (Study Day) | Liver Risk Factor Stop Date | Reference | Liver Risk | |
| Subject ID | Arm | Number | | (Study Day) | Period | Factor Details | Comments |
| XXXXX | XXXX | | DDMMMYYYY | DDMMMYYYY (X)/ | XXXX/ | | |
| $\mathcal{M}\mathcal{M}$ | $\Lambda \Lambda \Lambda \Lambda$ | X | | ` / | | vvvv | vvvvv |
| | | | (X) | DDMMMYYYY (X) | XXX | XXXX | XXXXX |
| | | 37 | DDMMMYYYY | DDMMMYYYY (X)/ | XXXXX/ | | |
| | | X | (X) | DDMMMYYYY (X) | XXX | XXXXX | |
| | | ••• | | | | | |
| XXXXX | XXXX | | DDMMMYYYY | DDMMMYYYY (X)/ | XXXXX/ | | |
| $\mathcal{M}\mathcal{M}$ | ΛΛΛΛ | X | (X) | Ongoing | XXXX | XXXXX | |
| | | | (11) | Oligonia | 2000 | | |

Note: Study Day is calculated relative to the date of first dose.

#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Assessment Date / Liver Risk Factor Start Date / Stop Date / Liver Risk Factor.
- Keep sorting from eCRF: Alcohol Abuse, Increased Alcohol Consumption within 1 Month of Reported Event, IV Drug Abuse, Tattoo, Acupuncture, Sexually Transmitted Diseases, Toxic/Chemical Agent Exposure, Travel (Areas at Risk in the Last Year), Pregnancy, Parenteral Nutrition, Excessive Physical Exercise, Changes Diet/Fasting Episodes/Weight Loss Diet, Previous Drug Reaction (Associated with an Elevation of Liver Tests), Blood Transfusion, Subject Exposed to Anyone with Jaundice in the Last Month, History of Hypotension, Low Blood Pressure at Time of Event of Liver Injury and/or Abnormal Liver Laboratory Value, History of Liver Disease, Other.
- Concatenate comments with "/".

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.9.12 Liver Signs and Symptoms Safety Population

| Subject ID | Treatment Arm | Potential Hy's<br>Law Case Number | Start Date (Study Day)/<br>Stop Date (Study Day) | Liver Sign/<br>Symptom | Intermittent |
|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXX | N |
| | | X | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXX | N |
| XXXXX | XXXX | <br>X | DDMMMYYYY (X)/<br>Ongoing | XXXXX | Y |

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Liver Sign/Symptom.
- Keep sorting from eCRF: Anorexia, Asthenia, Pyrexia, Pruritus, Jaundice, Arthralgia, Abdominal Pain, Abdominal Tenderness, Nausea, Vomiting, Rash, Mucosal Inflammation, Purpura, Hepatomegaly, Splenomegaly, Lymphadenopathy, Ascites, Confusional State, Coma, Upper Quadrant Tenderness, Biliary Obstruction, Eosinophilia, Dark Urine, Other.
- If Rash, Lymphadenopathy or Other, Concatenate Symptom with Commentas: "Rash: xxxxxx". "Lymphadenopathy: xxxxxx", "Other: xxxxxxxx"

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.13 Infection Diagnostic Investigations Safety Population

| | | AE ID | Start Date/ Time (Study Day)/ | | Examination | |
|---|---|---|---|---|---|---|
| Subject ID | Treatment Arm | Number | Stop Date/ Time (Study Day) | Method | performed | Test Result |
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXX | Y | XXXXX |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X)) | XXXXX | Y | XXXXX |
| | | ••• | | | | |
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXX | N | XXXXX |

AE = adverse event.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Method.
- Keep sorting from eCRF: Microscopy, Culture and Sensitivity, Serological Tests, Nucleic Acid Based Tests, X-Ray, Other.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.14 Infection Risk Factors and Lifestyle Events Safety Population

| Subject ID | Treatment<br>Arm | AE ID<br>Number | Start Date/ Time (Study Day)/<br>Stop Date/ Time (Study Day) | Infection Risk<br>Factor | Infection Risk<br>Occurrence | Comments |
|---|---|---|---|---|---|---|
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXX | Y | XXXXX |
| | | X | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X)) | XXXXX | Y | XXXXX |
| | | ••• | | | | |
| XXXXX | XXXX | X | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXX | N | Ongoing |

AE = adverse event; BCG = Bacillus Calmette-Guérin.

Note: Study Day is calculated relative to the date of first dose.

#### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Infection Risk Factor.
- Keep sorting from eCRF: Extensive Burns within the Last Year (Thermal Burn), Tattoo, Piercing or Acupuncture within the Last Year, Sexually Transmitted Diseases, Travel to Areas at Risk of Tuberculosis or Tropical Diseases, Infections Related to Travel (e.g. Tuberculosis and Tropical Diseases), Blood Transfusion (within the Last Year), Exposure to Nosocomial Pathogens within the Last Year, Contact History with Infection Source, Previous BCG Immunization, Evidence of BCG Scar, Tuberculin Skin or Quantiferon Test Confirms Previous Exposure or Immunity to Tuberculosis.
- Fill Comment column if Infection risk factor test = Unknown Previous BCG Immunization, not done, known Sexually Transmitted Disease reference Period, or Infection risk factor specifications.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.15 Infection Signs and Symptoms Safety Population

| | _ | | System Organ Class/ | Surety Topulation | | Infection | |
|---|---|---|---|---|---|---|---|
| | Treatment | AE ID | Preferred Term/ | Start Date/ Time (Study Day)/ | Clinical | Sign/Symptom | |
| Subject ID | Arm | Number | Verbatim Term | Stop Date/ Time (Study Day) | Event | Occurrence | Comments |
| XXXXX | XXXX | V | XXXXXXXXXX/ | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM | | | |
| | | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (X) | XXXXX | Y | XXXXX |
| | | V | XXXXXXXXXX/ | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM | | | |
| | | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (X)) | XXXXX | Y | XXXXX |
| | | ••• | | | | | |
| XXXXX | XXXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>Ongoing | | N | |
| | | | XXXXXXXXXXX | | XXXXX | 11 | Ongoing |

AE = adverse event.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Start Date / Stop Date / Clinical Event.
- Keep sorting from eCRF: Pyrexia, Headache, Confusional State, Convulsion, Rhinitis, Oropharyngeal Pain, Cough, Productive Cough, Haemoptysis, Wheezing, Dyspnoea, Pleuritic Pain, Vomiting, Diarrhoea, Genital Discharge, Haematuria, Dysuria, Hepatosplenomegaly, Jaundice, Lymphadenopathy, Rash, Night sweats, Chills, Myalgia, Weight Decrease.
- Fill Comment column if Maximum To (Unit) available for Pyrexia, or if site for Rash or Lymphadenopathy is known.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.16 Prior and Concomitant Medications Safety Population

| Subject<br>ID/<br>Treatment<br>Arm | Prior/<br>Concomitant<br>[1] | ATC Class (Level 2)/<br>Preferred Name/<br>Verbatim Term | Given<br>for/as | Primary<br>Indication | Start Date (Study<br>Day)/<br>End Date (Study<br>Day) | Dose (unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|---|
| XXXXXX<br>/ XXXX | Prior | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXX | Medical<br>History | XXXXXXX | MMMYYYY<br>(-XX)/<br>DDMMMYYYY<br>(-X) | XXXX unit | XXXXXX<br>XXX | XXXXX |
| | Both | XXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXX | Prophylaxis | XXXXXXX | MMMYYYY<br>(-X)/<br>Ongoing | XXXX unit | XXXXXX<br>XXX | XXXXX |
| | Concomitant | XXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXXX | Adverse<br>event | XXXXXXX | DDMMMYYYY<br>(X)/<br>DDMMMYYYY<br>(XX) | XXXX unit | XXXXXX<br>XXX | XXXXX |

ATC = anatomical therapeutic chemical; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

Note: Study Day is calculated relative to the date of first dose.

Medications were coded using WHO-DDE version vMar2023.

[1] Prior medications are defined as medications that started before first dose of study, whether they were stopped before first dose of study medication or not. Concomitant medications are defined as medications starting on or after first dose of study medication Both indicates medication that was started before the day of first dose and continued after.





## **Programming Notes:**

- ATC & Preferred Name text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name.
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX") but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by Treatment ID/ Subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications)

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.17 Prohibited Concomitant Medications Safety Population

#### **Programming Notes:**

- Same Shell as Listing 16.2.9.16.
- Display prohibited prior and concomitant medications provided by the Medical Coder:
- Prohibited concomitant medications:
  - $\circ$  NSAIDs analgesic therapies (with acetylsalicylic acid with doses  $\geq 325$  mg/day).
  - o COX-2 analgesic therapies.
  - o Immunotherapeutics.
  - o Live viral or attenuated bacterial vaccines.
  - o Oral, IV, intramuscular, or any other parenteral (other than oral) steroids (inhaled or topical steroids are permitted).
  - o Biologic therapeutic agents.
- Prohibited prior and/or concomitant medications:
  - o Anti-NGF therapies.
  - o Anti-TNF therapies.
- ATC & PN text should be in proper case in table.
- Ensure proper WHO-DDE version is printed in footnote.
- Sort by subject, start date/time, end date/time, ATC level 2 & Preferred Name.
- If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXX").
- Adjust footnotes for frequency and routes as needed.
- Sort by subject ID / Start Date / End Date (alphabetically for ATC Class Level 2 if same date for two medications)

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.9.18 Concomitant Procedures Safety Population

| | | | Surety 10 | 5 <b>4714</b> 410 11 | | |
|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Arm | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day) | Reason for Procedur | Reason (derived verbati | m If Reason is Other,<br>Specify |
| XXXXX | XXXX | XXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX | |
| XXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX | |
| XXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>Ongoing | OTHER | OTHER | XXXXXXXXXX |

MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study Day is calculated relative to the date of first dose. All Procedure terms were coded using the MedDRA version 26.0. Concomitant Procedures are defined as medications continuing or starting on or after first dose of study medication.

## **Programming Notes:**

- SOC & PT text should be in proper case in table.
- Sort by Treatment Arm/ Subject ID / Start Date / End Date (alphabetically for SOC if same date for two events).
- In case a term is not coded (e.g. in a dry run) it will be labelled as "Not Coded [SOC]" and "Not Coded [PT]". SOC and PT abbreviations should be added in this case in footnote.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.9.19 Anti-drug Antibody Test Results Safety Population

| Subject<br>ID | Treatment<br>Arm | Study<br>Visit | Date/Time of<br>Collection<br>(Study Day) | Screening<br>Status Result | Confirmatory<br>Status result | ADA Titer | Lab ID<br>Number | Comments |
|---|---|---|---|---|---|---|---|---|
| | 1 2212 | , 1510 | (Stady Bay) | 200000100000 | 20000010000 | 112111111 | 110111001 | |
| XXXXX | XXXX | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Positive | Positive | XX | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Positive | Positive | XX | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Negative | Negative | XX | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | Missing | Not<br>Reportable<br>Result | NRR | XXXXXXX | XXXX |

ADA = Anti-Drug Antibodies; NA = Not Applicable; NRR = Not Reportable Result; QNS = Quantity Not Sufficient. Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- ADA titre reported as <30 (below the minimum required dilution) is a negative result for the presence of ADA.
- Include Following timepoints: Screening, Weeks 2, 4, 8, 10, 12, 18.

Final 1 2 | 04-Oct-2023 | 





# Listing 16.2.10.1 Serum MEDI7352 Concentrations PK Population

| Subject | Treatment | Study | PK Blood<br>Sample<br>Collected? /<br>Reason Not | Date/Time of<br>Collection | MEDI7352<br>Concentration | | |
|---|---|---|---|---|---|---|---|
| ID <sup>°</sup> | Arm | Visit | Collected | (Study Day) | (ng/mL) | Lab ID Number | Comments |
| XXXXX | XXXX | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | NRR | XXXXXXX | XXXX |
| | | XXXXXX | No /<br>XXXXXX | , | | | |

NA = Not Applicable; NRR = Not Reportable Result.

Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours a fter Infusion, Week 10 + 24 hours: a fter Week 10/ Pre-Dose, Week 11: after Week 10/ Pre-Dose, Week 10 + 14 Days: after Week 10/ Pre-Dose, Week 18.

Final 1 2 | 04-Oct-2023 | 





#### Listing 16.2.10.2 Serum total NGF Concentrations Safety Population

| | | | PD Blood Sample | Surety Topular | | | |
|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Arm | Study<br>Visit | Collected? /<br>Reason Not<br>Collected | Date/Time of<br>Collection<br>(Study Day) | Total NGF<br>Concentration<br>(pg/mL) | Lab ID Number | Comments |
| XXXXX | XXXX | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | XX | XXXXXXX | |
| | | XXXXXX | Yes | DDMMMYYYY/<br>HH:MM (X) | NS | XXXXXXX | XXXX |
| | | XXXXXX | No /<br>XXXXXX | (-) | | | |

BLLOQ = Below the Lowest Limit of Quantitation; NA = Not Applicable; ND = Not Detected; NS = No Value due to Insufficient Volume or No Sample Received; PD: Pharmacodynamic; SAT = Greater than the Top of the Standard Curve; tNGF = total Nerve-Growth Factor. Note: Study Day is calculated relative to the date of first dose.

### **Programming Notes:**

- Sort by Treatment Arm/ Subject ID / Collection Date.
- Include the following timepoints: Day 1, Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.

Final 1 2 | 04-Oct-2023 | 





## **Planned Figure Descriptions and Shells**

| Number Title Population | Unique (U) or<br>Repeated (R) |
|---|---|
| Figure 14.2.1.1 - Daily Pain NRS: MCP-Mod Dose Response Model - mITT Population | U |
| Figure 14.2.1.2 - Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Missing Data Handling - mITT Population | U |
| Figure 14.2.1.3.1 - Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup - mITT Population | R |
| Figure 14.2.1.3.2 - Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup, Including Opioids mITT Population | CCI |
| Figure 14.2.1.4 - Daily Pain NRS: MMRMLS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases) mITT Population | U |
| Figure 14.3.6.1.1 - Vital Sign Profiles: Mean (±SD) Systolic Blood Pressure over time - Safety Population | U |
| Figure 14.3.6.1.2 - Vital Sign Profiles: Mean (±SD) Diastolic Blood Pressure over time - Safety Population | |
| Figure 14.3.6.1.3 - Vital Sign Profiles: Mean (±SD) Heart Rate over time - Safety Population | |
| Figure 14.3.6.1.4 - Vital Sign Profiles: Mean (±SD) Respiratory Rate over time - Safety Population | R |
| Figure 14.3.6.1.5 - Vital Sign Profiles: Mean (±SD) Temperature over time - Safety Population | R |
| Figure 14.4.1.1 - Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 over time - PK Population | R |
| Figure 14.4.1.2 - Pharmacokinetics: Individual Plot of Serum MEDI7352 Concentrations over time - PK Population | U |
| Figure 14.4.2.1 - Pharmacodynamics: Line Plot of Geometric Mean (with and without gSD) total NGF over time - Safety Population | R |
| Figure 14.4.2.2 - Pharmacodynamics: Individual Plot of Serum total NGF over time - Safety Population | R |

Final 1 2 | 04-Oct-2023 | 





# **Figures Change Log**

| Output<br>Number | Date of<br>Change | Change<br>Made By<br>(initials) | Description/Rationale |
|---|---|---|---|

Final 1 2 | 04-Oct-2023 | 





Figure 14.2.1.1
Daily Pain NRS: MCP-Mod Dose Response Model mITT Population

#### Weekly Average to Week 12 Daily Pain NRS CFB, Emax dose-response model



CI = Confidence Interval; CFB = Change from Baseline; DPS = Daily Pain Score; NRS = Numeric Rating Scale.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e.,

Day -7 to Day -1, inclusive. Envelope depicts 95% CI of mean dose-response. Added dots are actual doses ± 95% CI.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment.

Reference Listing: 16.2.6.1

Final 1 2 | 04-Oct-2023 | 





### **Programming Notes:**

- Insert the following text as legend: "Weekly Average to Week 12 Daily Pa in NRS CFB, xxxx dose-response model", with 'xxxx' as the selected dose-response model (e.g., Hyperbolic E<sub>max</sub>).
- Dose (μg/kg) in x axis and Daily Pain NRS CFB in y axis.
- Add model parameter values as an inset plot. For e.g., Sigmoid  $E_{max}$ ;  $E_0 = xxx$ ,  $E_{max} = xxx$ , ED50 = xxx,  $\lambda = xxx$ .
- The MCP-MOD approach will only be performed if stage 4 is initiated, otherwise there would be insufficient dosing data to fit the non-linear models.

Final 1 2 | 04-Oct-2023 | 





Figure 14.2.1.2
Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Missing Data Handling mITT Population

# Weekly Average CFB to Week 12 Daily Pain NRS 0 Daily Pain NRS CFB Data OBS LOCF BOCF -6 0 5 150 450 Dose (µg/kg)

BOCF = Baseline Observation Carried Forward; CFB = Change from Baseline; DPS = Daily Pain Score; LOCF = Last Observation Carried Forward; NRS = Numeric Rating Scale; OBS = Observed Cases.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1





### **Programming Notes:**

- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS".
- Dose (μg/kg) and Observed/LOCF/BOCF in x axis and Daily Pain NRS CFB in y axis.
- A level for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





# Figure 14.2.1.3.1 Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup mITT Population

CFB = Change from Baseline; DPS = Daily Pain Score; NRS = Numeric Rating Scale. Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.2
- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS".
- Dose (μg/kg) in x axis, Anticonvulsant/ Antidepressant/ Both/ None in right side Co-medication labels, and Daily Pain NRS CFB in y axis.
- A level for column dosing column dosing column will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





# Figure 14.2.1.3.2 Daily Pain NRS CFB: Boxplots at Week 12 by Treatment Group and Co-Medication Subgroup, Including Opioids mITT Population

BOTH = Anticonvulsant and Antidepressant; CFB = Change from Baseline; DPS = Daily Pain Score; NRS = Numeric Rating Scale. Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

### **Programming Notes:**

#### CCI

- Same shell as Figure 14.2.1.2
- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS".
- Dose (μg/kg) in x axis, Anticonvulsant/Antidepressant/Both/Opioid/None in right side Co-medication labels, and Daily Pain NRS CFB in y axis.
- A level for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





Figure 14.2.1.4
Daily Pain NRS: MMRM LS Means (95% Confidence Interval) over 12-weeks by Treatment Group (Observed Cases) mITT Population

#### Weekly Average CFB to Week 12 Daily Pain NRS ± 95% CI



CFB = Change from Baseline; CI = Confidence Interval; DPS = Daily Pain Score; LS = Least Square; MMRM = Mixed Model for Repeated Measures; NRS = Numeric Rating Scale.

Baseline is defined as the average of the 'non-missing' DPS within the seven-day period prior to randomization i.e., Day -7 to Day -1, inclusive.

Final 1 2 | 04-Oct-2023 | 





mITT Population = includes all subjects in the Safety Population who have at least 1 daily NRS assessment while receiving double-blind treatment. Reference Listing: 16.2.6.1

### **Programming Notes:**

- Insert the following text as legend: "Weekly Average CFB to Week 12 Daily Pain NRS  $\pm$  95% CI".
- Week in x axis and Daily Pain NRS CFB in y axis.
- Include a profile for each dose treatment group.
- Include the following timepoints: Week 2, 4, 6, 8, 10, and 12.
- Extract data for this figure from the MMRM of CFB Daily Pain NRS with Observed Cases.
- A profile for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





#### Figure 14.3.6.1.1 Vital Sign Profiles: Mean (±SD) Systolic Blood Pressure over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes a fter Infusion Completion; BASE = Baseline; D1 = Day 1; SBP = Systolic Blood Pressure; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average SBP  $\pm$  Standard Deviation".
- Study Visit in x axis and Systolic Blood Pressure (mmHg) in y axis.
- Include a profile for Resting SBP and another for Standing SBP.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1: 30 Minutes Post-Dose, Day 1: 45 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes a fter Infusion Completion, Week 10: Pre-Dose, Week 10: 5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing ) will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 





#### Figure 14.3.6.1.2 Vital Sign Profiles: Mean (±SD) Diastolic Blood Pressure over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes a fter Infusion Completion; BASE = Baseline; D1 = Day 1; DBP = Diastolic Blood Pressure; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11: W12 = Week 12: W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average DBP ± Standard Deviation".
- Study Visit in x axis and Diastolic Blood Pressure (mmHg) in y axis.
- Include a profile for Resting DBP and another for Standing DBP.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1:30 Minutes Post-Dose, Day 1:45 Minutes Post-Dose, Day 1:1 hour Post-Dose, Day 1:2 hours Post-Dose, Day 1:4 hours Post-Dose, Week 2: Pre-Dose, Week 2:5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4:5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6:5 minutes a fter Infusion Completion, Week 8: Pre-Dose, Week 8:5 minutes a fter Infusion Completion, Week 10: Pre-Dose, Week 10:5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for column dosing (column dosing (column dosing (column)) will only be added if Stage 4 is initiated)

Final 1.2 | 04-Oct-2023 | 





#### Figure 14.3.6.1.3 Vital Sign Profiles: Mean (±SD) Heart Rate over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 30M PD = 30 Minutes Post-Dose; 4H PD = 4 hours Post-Dose; 45M PD = 45 Minutes Post-Dose; 5M PD = 5 minutes a fter Infusion Completion; BASE = Baseline; D1 = Day 1; HR = Heart Rate; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average HR  $\pm$  Standard Deviation".
- Study Visit in x axis and Heart Rate (Beats/min) in y axis.
- Include a profile for Resting HR and another for Standing HR.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1:30 Minutes Post-Dose, Day 1:45 Minutes Post-Dose, Day 1:1 hour Post-Dose, Day 1:2 hours Post-Dose, Day 1:4 hours Post-Dose, Week 2: Pre-Dose, Week 2:5 minutes a fter Infusion Completion, Week 4: Pre-Dose, Week 4:5 minutes a fter Infusion Completion, Week 6: Pre-Dose, Week 6:5 minutes a fter Infusion Completion, Week 8: Pre-Dose, Week 8:5 minutes a fter Infusion Completion, Week 10: Pre-Dose, Week 10:5 minutes after Infusion Completion, Week 11, Week 12, Week 18. (Do not include Screening records).
- Note that standing measures are not taken on Day 1, at 15, 30 and 45 minutes post-dose.
- Make one plot for each dose treatment group, for a total of 4 plots with two profiles each.
- A plot for CC dosing (CC) will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 





#### Figure 14.3.6.1.4 Vital Sign Profiles: Mean (±SD) Respiratory Rate over time Safety Population

1H PD = 1 Hour Post-Dose; 15M PD = 15 Minutes Post-Dose; 2H PD = 2 Hours Post-Dose; 4H PD = 4 hours Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average Respiratory Rate ± Standard Deviation".
- Study Visit in x axis and Respiratory Rate (Breaths/min) in y axis.
- Include the following timepoints: Baseline, Day 1: 15 Minutes Post-Dose, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 5 minutes after Infusion Completion, Week 10 + 24 hours, Week 11, Week 12, Week 18. (Do not include Screening records).
- Make one plot with 4 profiles (one for each treatment group).
- A profile for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 





Figure 14.3.6.1.5
Vital Sign Profiles: Mean (±SD) Temperature over time
Safety Population

1H PD = 1 Hour Post-Dose; 2H PD = 2 Hours Post-Dose; 4H PD = 4 hours Post-Dose; 5M PD = 5 minutes after Infusion Completion; BASE = Baseline; D1 = Day 1; T° = Temperature; W2 = Week 2; W4 = Week 4; W6 = Week 6; W8 = Week 8; W10 = Week 10; W11 = Week 11; W12 = Week 12; W18 = Week 18.

Baseline is defined as the last observation recorded prior to the first dose of treatment.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

Reference Listing: 16.2.9.1

#### **Programming Notes:**

- Same shell as Figure 14.2.1.4
- Insert the following text as legend: "Average Body To ± Standard Deviation".
- Study Visit in x axis and Body Temperature (°C) in y axis.
- Include the following timepoints: Baseline, Day 1: 1 hour Post-Dose, Day 1: 2 hours Post-Dose, Day 1: 4 hours Post-Dose, Week 2: Pre-Dose, Week 2: 5 minutes after Infusion Completion, Week 4: Pre-Dose, Week 4: 5 minutes after Infusion Completion, Week 6: Pre-Dose, Week 6: 5 minutes after Infusion Completion, Week 8: Pre-Dose, Week 8: 5 minutes after Infusion Completion, Week 10: 5 minutes after Infusion Completion, Week 10: 4 hours, Week 11, Week 12, Week 18. (Do not include Screening records).
- Make one plot with 4 profiles (one for each treatment group).
- A plot for column dosing (cc) will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 



Figure 14.4.1.1
Pharmacokinetics: Line Plot of Geometric Mean (with and without gSD) Serum MEDI7352 Concentrations over Time PK Population



ADA = Antidrug Antibodies; gSD = Geometric Standard Deviation; LLOQ = Lower Limit of Quantification.

Final 1 2 | 04-Oct-2023 | 





PK Population = includes all subjects for who a pharmacokinetic sample was obtained and analyzed. ADA positive represents number of participants with at least one positive ADA result. ADA negative represents number of participants with only negative ADA results (no positive). Reference Listing: 16.2.10.1

### **Programming Notes:**

- Insert the following text as upper legend: "Geometric Mean serum MEDI7352 ± Geometric Standard Deviation (Linear Scale)" for the linear plot, and "Geometric Mean serum MEDI7352 (Semi-Logarithmic Scale)" for the semi-log plot. Below legend, add legend for ADA status: "Overall", "ADA Positive", "ADA Negative".
- Insert legend with different point symbols and colors for each treatment group (CCI) for the Overall plot, and a legend with different point symbols and colors for each ADA status (ADA+, ADA-) for each treatment group plot by ADA status.
- Study Day in x axis and Serum MEDI7352 concentration (ng/mL) in y axis (in linear and log<sub>10</sub> scale, for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10: Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 10 + 14 days, Week 18.
- Make one overall plot by treatment group, and a plot for each treatment group by ADA status for a total of 4 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (1.00 ng/mL)".
- A line for column dosing (column dosing (column dosing (column)) will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 





Figure 14.4.1.2
Pharmacokinetics: Individual Plot of Serum MEDI7352 Concentrations over time PK Population



ADA = Antidrug Antibodies; LLOQ = Lower Limit of Quantification.

PK Population = includes all subjects for who a pharmacokinetic sample was obtained and analyzed.

ADA positive represents number of participants with at least one positive ADA result.

ADA negative represents number of participants with only negative ADA results (no positive).

Reference Listing: 16.2.10.1

Final 1 2 | 04-Oct-2023 | 





#### **Programming Notes:**

- Insert the following text as upper legend: "MEDI7352 Concentration by Subject, Treatment group, and ADA status" followed by "(Linear Scale)" or "(Semi-Logarithmic Scale)" depending on the plot (linear or semi-log). Below legend, add legend for Treatment Group:
- Insert legend with different colors for each ADA status (Positive/ Negative).
- Time (days) in x axis and Serum MEDI7352 concentration (ng/mL) in y axis (in linear and log<sub>10</sub> scale, for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 10 + 14 days, Week 18.
- Make one plot for each Treatment group (CC), for a total of 3 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (1.00 ng/mL)".
- Plots for column dosing (cc) will only be added if Stage 4 is initiated.

Final 1 2 | 04-Oct-2023 | 





# Figure 14.4.2.1 Pharmacodynamics Line Plot of Geometric Mean (with and without gSD) Serum total NGF over time Safety Population

ADA = Antidrug Antibodies; gSD = Geometric Standard Deviation; LLOQ = Lower Limit of Quantification, NGF = Nerve-Growth Factor.

Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication.

ADA positive represents number of participants with at least one positive ADA result.

ADA negative represents number of participants with only negative ADA results (no positive).

Reference Listing: 16.2.10.3

#### **Programming Notes:**

- Same shell as Figure 14.4.1.1
- Insert the following text as upper legend: "Geometric Mean Serum Concentration of tNGF ± Geometric Standard Deviation (Linear Scale)" for the linear plot, and "Geometric Mean Serum Concentration of tNGF (Semi-Logarithmic Scale)" for the semi-log plot. Below legend, add legend for ADA status: "Overall", "ADA Positive", "ADA Negative".
- Insert legend with different point symbols and colors for each treatment group (Placebo, Colors for the Overall plot, and a legend with different point symbols and colors for each ADA status (ADA+, ADA-) for each treatment group plot by ADA status.
- Study Day in x axis and Serum tNGF Concentration (pg/mL) in y axis (in linear and log<sub>10</sub> scale for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10: Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12, Week 18.
- Make one overall plot by treatment group, and a plot for each treatment group by ADA status for a total of 5 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (10.00 pg/mL)".
- A plot for column dosing (column dosing will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 





# Figure 14.4.2.2 Pharmacodynamics: Individual Plot of Serum total NGF over time Safety Population

ADA = Antidrug Antibodies; LLOQ = Lower Limit of Quantification; NGF = Nerve-Growth Factor. Safety Population = includes all subjects who receive at least 1 dose of double-blind study medication. ADA positive represents number of participants with at least one positive ADA result. ADA negative represents number of participants with only negative ADA results (no positive). Reference Listing: 16.2.10.3

### **Programming Notes:**

- Same shell as Figure 14.4.1.2
- Insert the following text as legend: "Total NGF by Subject, Treatment group, and ADA status" followed by "(Linear Scale)" or "(Semi-Logarithmic Scale)" depending on the plot (linear or semi-log). Below legend, add legend for Treatment Group:
- Insert legend with different colors for each ADA status (Positive/ Negative).
- Time (days) in x axis and Serum tNGF concentration (pg/mL) in y axis (in linear and log<sub>10</sub> scale for each plot).
- Include data from the following timepoints: Baseline (Day 1), Week 2, Week 4, Week 6, Week 8, Week 10: Pre-Dose, Week 10; Before End of Infusion, Week 10: 8 Hours after Infusion, Week 10 + 24 hours, Week 11, Week 12; Week 18.
- Make one plot for each Treatment group (CC) Placebo), for a total of 4 plots.
- Include a marker for LLOQ, and an inset within the plot with "LLOQ (10.00 pg/mL)".
- Plots for column dosing (CC) will only be added if Stage 4 is initiated.

Final 1.2 | 04-Oct-2023 | 